## **Statistical Analysis Plan**

**Study ID:** 207966

**Official Title of Study:** A Phase IIIb, Randomized, Multicenter, Parallel-group, Non-inferiority, Open-label Study Evaluating the Efficacy, Safety, and Tolerability of Longacting Cabotegravir Plus Long-acting Rilpivirine Administered Every 8 Weeks or Every 4 Weeks in HIV-1-infected Adults who are Virologically Suppressed (ATLAS-2M), further referred to as A2M.

**NCTID:** NCT03299049

**Sub-study Protocol Amendment Title:** Sub-sudy to the A2M study to Evaluate the Pharmacokinetics, Tolerability and Efficacy of Cabotegravir and Rilpivirine Long-Acting Injections Following Intramuscular Administration in the Vastus Lateralis Muscle (thigh) in HIV-infected Adult Participants who have Received at Least Three Years of Gluteal Injections in the A2M Study.

**NCTID:** NCT05896761

**Date of Document:** 23 September 2022

The sub-study was added to the protocol of the main study via an amendment. Details of the sub-study can be found in the protocol section 11.13 Appendix 13: Vastus Lateralis Muscle (Thigh) PK sub-study Amendment. A separate record has been created on ClinicalTrials.gov for the sub-study.

## The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for Protocol 207966: Study<br>Evaluating the Efficacy, Safety, and Tolerability of Long-<br>acting Cabotegravir Plus Long-acting Rilpivirine<br>administered every 8 weeks in Virologically Suppressed<br>HIV-1-infected Adults |
| Compound Number | : | GSK1265744 |
| Effective Date | : | 08-Sep-2022 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Thigh PK Sub-study Clinical Study Report for Protocol 207966. Reporting details pertaining to the primary Week 48 and the earlier analyses (Week 24 IDMC, Week 24, Week 96 and Week 152) have been retained for completeness.
- This version of the RAP includes amendments to the originally approved RAP.

# Author(s)

| Author | Date |
|--------------------------------------------|-------------|
| Lead | |
| PPD | 08-Sep-2022 |
| Statistics Leader (Dev Biostats Stats Dev) | 00-SCp-2022 |

Copyright 2022 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Review Confirmations**

(Method: E-mail)

| Reviewer | Date |
|---|---|
| Clinical Development Lead, CAB Treatment (ViiV Healthcare) | 16-Sep-2022 |
| PPD (ViiV Healthcare) | 15-Sep-2022 |
| Principal Programmer (Infectious Diseases, Biostatistics Programming) | 14-Sep-2022 |
| PPD (CMO GCSP SERM) | 19-Sep-2022 |
| PPD Clinical Pharmacology Modelling and Simulation (CPMS) | 23-Sep-2022 |
| Clinical Development Manager (Translational Medicine, ViiV<br>Sci Med Office) | 16-Sep-2022 |
| PPD (ViiV Healthcare) | 9-Sep-2022 |
| PPD Cabotegravir Global Health Outcomes | 19-Sep-2022 |

# **Clinical Statistics and Clinical Programming Line Approvals:**

(Method: Veeva Vault TMF eSignature)



# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 8 |
| | 1.1. | RAP Amendments | |
| 2. | SUMN | MARY OF KEY PROTOCOL INFORMATION | 12 |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | | 2.2.1. Thigh PK Sub-study Objectives and Endpoints | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | PLAN | NED ANALYSES | 19 |
| | 3.1. | IDMC Analyses | 19 |
| | 3.2. | Final Analyses | 20 |
| 4. | ANAL | YSIS POPULATIONS | 21 |
| | 4.1. | Protocol Deviations | 23 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | /ENTIONS | 24 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | 24 |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | 25 |
| | | 5.4.1. Covariates and Other Strata | |
| | | 5.4.2. Examination of Subgroups | |
| | 5.5. | Multiple Comparisons and Multiplicity | |
| | | 5.5.1. Primary Comparison of Interest | |
| | | 5.5.2. Other Comparisons of Interest | 29 |
| | 5.6. | Other Considerations for Data Analyses and Data Handling Conventions | 30 |
| 6. | | POPULATION ANALYSES | |
| | 6.1. | Overview of Planned Study Population Analyses | |
| | 6.2. | Prior and Concomitant Medications | 32 |
| 7. | | CACY ANALYSES | |
| | 7.1. | Primary Efficacy Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.1.5. Statistical Analyses / Methods | 35 |
| | 7.6 | 7.1.5.1. Statistical Methodology Specification | |
| | 7.2. | Secondary Efficacy Analyses | |
| | | 7.2.1. Endpoints | |
| | | 7.2.2. Summary Measure | |
| | | 7.2.3. Population of Interest | |
| | | 7.2.4. Strategy for Intercurrent (Post-Randomization) Events | 39 |

| | | | Statistical Analyses / Methods | |
|---|---|---|---|---|
| | 7.3. | | 7.2.5.1. Statistical Methodology Specificationry Efficacy Analyses | |
| | | | ,,,, | |
| 8. | SAFET | Y ANALY | SES | .44 |
| | 8.1. | | Events Analyses | .44 |
| | | 8.1.1. | Analyses for Injection Site Reaction Adverse Events from | |
| | | | Study Drug Injection | |
| | 8.2. | | Events of Special Interest Analyses | |
| | 8.3. | | aboratory Analyses | |
| | 8.4. | Other Saf | ety Analyses | .46 |
| 9. | | | ETIC ANALYSES | |
| | 9.1. | | / Variables | |
| | 0.0 | | Drug Concentration Measures | |
| | 9.2. | | of Planned Analyses | |
| | 9.3. | Statistical | Analyses / Methods | .48 |
| 10 | DODLII | ATION DI | HARMACOKINETIC ANALYSES | E0 |
| 10. | POPUI | -ATION PI | TARMACURINETIC ANALYSES | .50 |
| 11 | PHARI | MACOKINI | ETIC / PHARMACODYNAMIC ANALYSES | 50 |
| 11. | 11.1. | | of Planned Analyses | |
| | 11.2. | | Analyses / Methods | |
| | 11.2. | Otatiotioai | 7 thaty 300 7 thickhoud | .02 |
| 12. | HEALT | H OUTCO | DMES ANALYSES | .53 |
| | 12.1. | | / Variables | |
| | | • | Main Study | |
| | | | Sub-study | |
| | 12.2. | | Measure | |
| | 12.3. | | n of Interest | |
| | 12.4. | Analysis o | of Reason for switch will be based on a subset of Intent-to- | |
| | | | osed population who either were randomized to SOC arm | |
| | | in ATLAS | or did not participate in ATLAS study (i.e. SOC | |
| | | population | n).Strategy for Intercurrent (Post-Randomization) Events | .54 |
| | 12.5. | | Analyses / Methods | |
| | | 12.5.1. | Statistical Methodology Specification | .54 |
| 13. | VIROL | OGY | | .57 |
| 14. | REFE | RENCES | | .59 |
| 4- | 4.0054 | IDIOEO | | 00 |
| 15. | | | 4. Desta and Destation Management and Destation of an Des | .60 |
| | 15.1. | | 1: Protocol Deviation Management and Definitions for Per | 00 |
| | | | Population | |
| | 15.0 | | Exclusions from Per Protocol Population | |
| | 15.2. | | 2: Schedule of Activities Protocol Defined Schedule of Events for Q4W Arm in Main | .03 |
| | | | | 64 |
| | | | Study Protocol Defined Schedule of Events for Q8W Arm in Main | .04 |
| | | | Study | 72 |
| | | | Protocol Defined Schedule of Events for Q4W Arm in Sub- | . 1 2 |
| | | | study | 79 |
| | | • | ouay | |

| | 15.2.4. | Protocol Defined Schedule of Events for Q8W Arm in Sub- | |
|---|---|---|---|
| | | study | |
| 15.3. | | 3: Assessment Windows | |
| | 15.3.1. | Definitions of Assessment Windows for Analyses | 88 |
| | 15.3.2. | Definitions of Assessment Windows for Analyses other | |
| | | than Health Outcome and PK | 89 |
| | 15.3.3. | Assessment Window for Phase Conclusion | 95 |
| | 15.3.4. | Assessment Window for Health Outcome Data | 95 |
| | | 15.3.4.1. PIN / HAT-QoL / HIVTSQs / HIVTSQc / | |
| | | ACCEPT / Preference in Main Study | 95 |
| | | 15.3.4.2. Reasons for Continuation/Switch in Main Study | 97 |
| | | 15.3.4.3. HIVTSQs/HIVTSQc/Preference in Sub-study | 97 |
| | | 15.3.4.4. Tolerability of Injections (NRS) in Sub-study | |
| | 15.3.5. | Assessment Window for PK Concentration Data | |
| | | 15.3.5.1. Maintenance and Extension Phase | |
| | | Assessments | 98 |
| | | 15.3.5.2. Long-term Follow-up Phase Assessments | |
| | | 15.3.5.3. Sub-study Assessments | 99 |
| | 15.3.6. | Multiple Assessments within an Assessment Window | |
| 15.4. | | 4: Study Phases and Treatment State | |
| 10.1. | 15.4.1. | Study Phases | |
| | 15.4.2. | Treatment State | |
| | 10.1.2. | 15.4.2.1. Treatment States for AE Data | |
| | 15.4.3. | Study Period | |
| 15.5. | | stady Forlidastady Forlida Standards & Handling Conventions | |
| 10.0. | 15.5.1. | Reporting Process | |
| | 15.5.1. | Reporting Standards | |
| | 15.5.2. | Reporting Standards for Pharmacokinetic | |
| 15.6. | | (6: Derived and Transformed Data | |
| 15.0. | 15.6.1. | General | |
| | 15.6.1. | Study Population | |
| | 15.6.2.<br>15.6.3. | | |
| | | Efficacy | |
| | 15.6.4. | Safety | |
| | 15.6.5. | Pharmacokinetic | |
| | 15.6.6. | Health Outcomes | |
| 45.7 | | Virology | |
| 15.7. | | 7: Reporting Standards for Missing Data | |
| | | Premature Withdrawals | |
| | 15.7.2. | | |
| | | 15.7.2.1. Handling of Missing and Partial Dates | |
| | | 15.7.2.2. Handling of Missing data for Statistical Analysis | |
| 15.8. | | 8: Values of Potential Clinical Importance | |
| 15.9. | | (9: Snapshot Algorithm Details | |
| | | ( 10: Variables Defined for Time to Event Analysis | |
| | | 11: Identification of Adverse Events of Special Interest | |
| | | c 12: Identification of COVID-19 Adverse Events | |
| 15.13. | | ( 13: IDMC | |
| | 15.13.1. | Adhoc CVF IDMC Analyses | 179 |
| | | Week 24 IDMC Analyses | |
| 15.14. | Appendix | ( 14: Abbreviations & Trademarks | 180 |
| | | Abbreviations | |
| | 15.14.2. | Trademarks | 182 |

| 15.15. | Appendix | x 15: List of Data Displays | 183 |
|---|---|---|---|
| | 15.15.1. | Data Display Numbering | 183 |
| | | Mock Example Shell Referencing | |
| | 15.15.3. | Deliverables | 184 |
| | | List of Data Displays for Week 24 IDMC and Week 24 | |
| | | Planned Analyses | 184 |
| | | 15.15.4.1. Study Population Tables | 185 |
| | | 15.15.4.2. Efficacy Tables | |
| | | 15.15.4.3. Efficacy Figures | |
| | | 15.15.4.4. Safety Tables | |
| | | 15.15.4.5. Safety Figures | |
| | | 15.15.4.6. Pharmacokinetic Tables | 102 |
| | | 15.15.4.7. Pharmacokinetic Figures | |
| | | 15.15.4.8. Virology Tables | |
| | | 15.15.4.9. ICH Listings | |
| | 15 15 5 | 15.15.4.10. Non-ICH Listings | 190 |
| | 15.15.5. | List of Data Displays for Week 48/96/End-of-Study | 204 |
| | | Planned Analyses | |
| | | 15.15.5.1. Study Population Tables | |
| | | 15.15.5.2. Efficacy Tables | |
| | | 15.15.5.3. Efficacy Figures | |
| | | 15.15.5.4. Safety Tables | |
| | | 15.15.5.5. Safety Figures | 232 |
| | | 15.15.5.6. Pharmacokinetic Tables | |
| | | 15.15.5.7. Pharmacokinetic Figures | 238 |
| | | 15.15.5.8. Pharmacokinetic / Pharmacodynamic Tables | |
| | | 15.15.5.9. Pharmacokinetic / Pharmacodynamic Figures | |
| | | 15.15.5.10. Health Outcomes Tables | |
| | | 15.15.5.11. Health Outcomes Figures | |
| | | 15.15.5.12. Virology Tables | |
| | | 15.15.5.13. ICH Listings | |
| | 45.45.0 | 15.15.5.14. Non-ICH Listings | |
| | 15.15.6. | List of Data Displays for Week 152 Planned Analyses | |
| | | 15.15.6.1. Study Population Tables | |
| | | 15.15.6.2. Efficacy Tables | |
| | | 15.15.6.3. Efficacy Figures | |
| | | 15.15.6.4. Safety Tables | |
| | | 15.15.6.5. Safety Figures | 288 |
| | | 15.15.6.6. Pharmacokinetic Tables | |
| | | 15.15.6.7. Pharmacokinetic Figures | |
| | | 15.15.6.8. Pharmacokinetic / Pharmacodynamic Figures | |
| | | 15.15.6.9. Health Outcomes Tables | |
| | | 15.15.6.10. Health Outcomes Figures | 302 |
| | | 15.15.6.11. Virology Tables | |
| | | 15.15.6.12. ICH Listings | |
| | | 15.15.6.13. Non-ICH Listings | |
| | 15.15.7. | List of Data Displays for Sub-study Analysis | |
| | | 15.15.7.1. Study Population Tables | |
| | | 15.15.7.2. Efficacy Tables | |
| | | 15.15.7.3. Efficacy Figures | |
| | | 15.15.7.4. Safety Tables | 319<br>327 |
| | | TO TO A SOLOTY FIGURAGE | 377 |

| | 207966 |
|----------------------------------------------------------|--------|
| 15.15.7.6. Pharmacokinetic Tables | 328 |
| 15.15.7.7. Pharmacokinetic Figures | 330 |
| 15.15.7.8. Health Outcomes Tables | |
| 15.15.7.9. Virology Tables | 335 |
| 15.15.7.10. ICH Listings | |
| 15.15.7.11. Non-ICH Listings | |
| 15.16 Appendix 16: Example Mock Shells for Data Displays | |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronolog | gy: | |
|---|---|---|
| 2017N326521_00 | 17-JUL-2017 | Original |
| 2017N326521_01 | 14-SEP-2017 | The primary purpose of protocol amendment # 1 is to revise the study sample size to randomize approximately 1020 participants including 510 participants per arm based on a non-inferiority margin of 4% between the CAB LA + RPV LA Q8W and Q4W arms. |
| 2017N326521_02 | 03-Jul-2018 | The primary reasons for amendment #2 are to: |
| | | <ul> <li>Add the additional interim analysis of data when all<br/>subjects have completed the Week 24 visit, with the<br/>intent of expediting the submission of study results<br/>to Health Authorities;</li> </ul> |
| | | <ul> <li>Change the objective for assessing the preference<br/>for CAB LA + RPV LA every 8 weeks or CAB LA +<br/>RPV LA every 4 weeks LA compared to oral<br/>antiretroviral (ARV) and the preference for CAB<br/>LA+ RPV LA every 8 weeks compared to CAB LA +<br/>RPV LA every 4 weeks from an exploratory<br/>objective to a secondary objective. A change to the<br/>supporting version of the Preference questionnaire<br/>administered to participants at Week 48 (or<br/>withdrawal) is also acknowledged;</li> </ul> |
| | | <ul> <li>Add revisions and clarifications for the<br/>administration of health outcomes questionnaires;</li> </ul> |
| | | <ul> <li>Extend exclusion criterion #28 to also exclude<br/>hereditary coagulation and platelet disorders such<br/>as haemophilia or Von Willebrand Disease;</li> </ul> |
| | | <ul> <li>Update exclusion criterion #11 to indicate that<br/>CD4+ counts &lt;200 cells/µL are not exclusionary;</li> </ul> |
| | | <ul> <li>Offer clarification that withdrawal assessments will<br/>be performed for any participant who withdraws<br/>prematurely from the Maintenance or Extension<br/>Phase. Additional guidance for participants<br/>withdrawing at Week 52 or Week 100 has been<br/>added;</li> </ul> |
| | | <ul> <li>Offer guidance to monitor medications that are<br/>dependent on OAT1 and OAT3 transport upon<br/>concomitant exposure with CAB;</li> </ul> |
| | | <ul> <li>Specify that 2-hour post-dose ECG should be<br/>performed at Day 1 and Week 48 only for<br/>participants receiving CAB LA + RPV LA as it is not<br/>required to perform 2-hour post-dose ECG for<br/>those receiving oral CAB + RPV at Day 1;</li> </ul> |

| Revision Chronology: | | |
|---|---|---|
| 3, | | <ul> <li>Exclude language that previously indicated hormonal contraception may be susceptible to interaction with the study drugs. The lack of a demonstrated interaction with a representative contraceptive supports use of CAB and RPV across a broad range of estrogen and progestin or progestin only hormonal contraceptives;</li> <li>Add minor clarifications and corrections to typographical errors/formatting to protocol text.</li> </ul> |
| 2017N326521_03 | 21-May-2020 | The primary reason for protocol amendment 03 is to include information on Covid-19 specific guidance for clinical trial continuity (participant and study management) during the pandemic. This information is included within Appendix 10: COVID-19 Pandemic and Clinical Trial Continuity. |
| 2017N326521_04 | 05-Aug-2020 | The primary reasons for protocol amendment 04 are to add a formal efficacy and safety secondary analysis at Week 152, allowing participants to continue treatment with randomized study medication through at minimum the Week 152 timepoint. The study endpoints and additional assessments in support of the planned secondary analyses have been updated for Week 152. Health outcomes assessments including the HIV-TSQs, Accept, and PIN questionnaires are included at Week 152 to gain further insight into participant's long-term treatment experience with Long-acting Cabotegravir Plus Long-acting Rilpivirine. The Preference questionnaire will also be administered at Week 152 only to participants who received oral bridging during the Maintenance and/or Extension Phases. Additional minor clarifications to protocol language have also been incorporated. |
| TMF-11797977 | 16-Apr-2021 | <ul> <li>To allow participants who become pregnant to remain in the study and not be withdrawn due to pregnancy. Allowing pregnant participants to continue in the study will negate any additional and subsequent fetal exposures to new antiretrovirals agents that would occur if the pregnant participant was withdrawn from the study and placed on an oral SOC regimen. An Appendix, "Information and Guidance for Managing Pregnant Participants" was inserted as Appendix 11, and all subsequent appendices were renumbered accordingly.</li> <li>Contraceptive methods have been updated to permit the use of progestogen-only implantable and injectable contraceptives without the requirement of a second highly effective method.</li> <li>Removal of the optional collection of cord blood and/or breast milk after delivery.</li> </ul> |

| : | |
|---|---|
| | <ul> <li>Removal of the option for study treatment rechallenge following suspected druginduced liver injury (DILI)</li> <li>Clarification of which participants enter the LTFU phase when CAB+RPV LA marketed product is locally available.</li> </ul> |
| | Clarification added: The Reason for Oral Bridgingand Preference questionnaire will also be administered at Withdrawal if it occurred at or before Week 152 only to participants who received oral bridging during the Maintenance and/or Extension Phases. |
| | <ul> <li>Medical Device reporting requirement added</li> <li>Co-enrolment (Only applicable for South African participants)</li> </ul> |
| | <ul> <li>Clinical and safety references updated</li> <li>Removal of the reference to "randomized study treatment" in Overall design sections for alignment with CAB program studies and transition to marketed product plan.</li> </ul> |
| 11-Aug-2021 | <ul> <li>The primary purposes of this amendment are: <ul> <li>Included Thigh Injection Sub-study appendix</li> </ul> </li> <li>Added safety and PK laboratory assessments during pregnancy for subjects who become pregnant during the study and decide to continue receiving IM treatment in the study.</li> <li>Medical device deficiencies reporting requirements updated to be aligned with GSK reporting processes.</li> <li>Updated safety information</li> <li>Other minor clarifications added</li> </ul> |
| | 11-Aug-2021 |

# 1.1. RAP Amendments

# **Revision Chronology:**

| RAP Section | Amendment Details |
|---|---|
| Reporting and Analysis Pl | Reporting and Analysis Plan_Study207966_Final_V1 [17-JAN-2019] |
| Reporting and Analysis Plan_Study207966_Amendment_Final_V1 [23-JUN-2020] | |
| Reporting and Analysis Plan_Study207966_Amendment_2_Final_V1 [28-JUN-2020] | |
| Reporting and Analysis Plan_Study207966_Amendment_3_Final_V1 | |
| Data Handling and Data<br>Displays for Sub-study | <ul> <li>Updated visit/phase slotting algorithms to handle the newly added assessments and time points in the protocol.</li> <li>Added new analysis populations for sub-study analysis.</li> </ul> |

| | Defined a separate list of displays for sub-study analysis. |
|---|---|
| Safety Analysis | <ul> <li>Added calculation methods for extent of exposure in sub-study.</li> <li>Extended lipid LOCF approach to include both Thigh Injection and Return to Gluteal Injection phases in sub-study.</li> <li>Updated the display shells for summaries of COVID-19 assessments to accommodate possible scenarios of multiple COVID-19 case diagnosis per participant.</li> </ul> |
| Added analysis methods for PK parameters derived from sub-sconcentration-time data. Extended evaluability criteria to include sub-study PK concentration. | |
| Study Population Analysis | <ul> <li>Added windows for evaluating concomitant ART/non-ART medications in sub-study.</li> <li>Added a listing for data collected from the Transition to CAB + RPV LA Marketed Product Status eCRF form.</li> </ul> |
| Health Outcomes Analysis Added analysis for the newly added Preference Thigh Injection questionnaire. | |
| General Updates | <ul> <li>Added sub-study Schedule of Activities per new protocol.</li> <li>Added additional minor clarifications and corrections to typographical errors/formatting to RAP text.</li> </ul> |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 6 [(Dated: 11/AUG/2021)].

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To demonstrate the non-inferior<br>antiviral activity of CAB LA + RPV LA<br>every 8 weeks (every two months)<br>compared to CAB LA + RPV LA every<br>4 weeks (monthly) over 48 weeks in<br>suppressed HIV-1 infected<br>antiretroviral therapy (ART)-<br>experienced participants | Proportion of participants with plasma HIV-RNA greater than or equal to 50 copies/mL as per Food and Drug Administration (FDA) Snapshot algorithm at Week 48 (Intent-to-Treat Exposed [ITT-E] population) |
| Secondary Objectives | Secondary Endpoints |
| To demonstrate the antiviral and immunologic activity of CAB LA + RPV LA every 8 weeks compared to CAB LA + RPV LA every 4 weeks | <ul> <li>Proportion of participants with plasma HIV-1 RNA &lt;50 c/mL (c/mL) at Week 24, Week 48, Week 96 and Week 152 using the FDA Snapshot algorithm (Intent-to-Treat Exposed [ITT-E] population)</li> <li>Proportion of participants with protocol-defined confirmed virologic failure (CVF) through Week 24, Week 48, Week 96 and Week 152</li> <li>Proportion of participants with HIV-RNA greater than or equal to 50 c/mL as per FDA Snapshot algorithm at Week 24, Week 96 and Week 152</li> <li>Absolute values and changes from Baseline in viral load and CD4+ cell counts over time including Week 48 and Week 96 and Week 152</li> </ul> |
| To evaluate the safety and tolerability<br>of CAB LA + RPV LA every 8 weeks<br>compared to CAB LA + RPV LA every<br>4 weeks | <ul> <li>Incidence and severity of AEs and laboratory abnormalities over time including Week 24, Week 48, Week 96 and Week 152</li> <li>Proportion of participants who discontinue treatment due to AEs over time including Week 24, Week 48, Week 96 and Week 152</li> <li>Change from Baseline in laboratory parameters over time including Week 48, Week 96 and Week 152</li> </ul> |
| To assess viral resistance in<br>participants experiencing protocol-<br>defined confirmed virologic failure | Incidence of treatment emergent genotypic and phenotypic resistance to CAB, RPV through Week 24, Week 48, Week 96 and Week 152 |
| To characterize CAB and RPV concentrations and population pharmacokinetics and identify important determinants of variability | <ul> <li>Plasma PK parameters for CAB LA and RPV LA (when evaluable, Ctrough, concentrations post dose [~Cmax], and area under the curve [AUC])</li> <li>Demographic parameters including, but not limited to, age, sex, race, body weight, body mass index, and relevant laboratory parameters will be evaluated as</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | potential predictors of inter- and intra-participant variability for pharmacokinetic parameters |
| <ul> <li>To assess preference for CAB LA + RPV LA every 8 weeks or CAB LA + RPV LA every 4 weeks LA compared to oral antiretroviral (ARV)</li> <li>To assess preference for CAB LA+ RPV LA every 8 weeks compared to CAB LA + RPV LA every 4 weeks</li> </ul> | Preference for CAB LA + RPV LA every 8 weeks and CAB LA + RPV LA every 4 weeks compared to oral ARV and preference for CAB LA + RPV LA every 8 weeks compared to CAB LA + RPV LA every 4 weeks will be assessed using a preference questionnaire at week 48 (or Withdrawal). |
| To assess patient reported health-related quality of life, treatment satisfaction, injection tolerability, and treatment acceptance. | <ul> <li>Change from Baseline (Day 1) in HRQoL at Week 24, and Week 48 (or Withdrawal)</li> <li>Change from baseline (Day 1) in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) at Week 24, 48 and 152 (or Withdrawal)</li> <li>Change in treatment satisfaction over time using the HIV Treatment Satisfaction Change Questionnaire HIVTSQc at Week 48 (or Withdrawal).</li> <li>Change from Week 8 in Dimension scores ("Bother of ISRs", "Leg movement", "Sleep", and "Injection Acceptance") and individual item scores assessing pain during injection, anxiety before and after injection, willingness to be injected in the future and overall satisfaction with mode of administration over time will be assessed using the Perception of Injection questionnaire (PIN) at Weeks 24, 48 and 152 (or Withdrawal)</li> <li>Change from Baseline (Day 1) in treatment acceptance at Week 24, Week 48 and 152 (or Withdrawal) will be assessed using the "General acceptance" dimension of the Chronic Treatment Acceptance (ACCEPT)</li> </ul> |
| Exploratory Objectives | questionnaire |
| To evaluate the antiviral and immunologic effects, safety and tolerability, and viral resistance of CAB LA + RPV LA for all participants in the Extension Phase. | <ul> <li>Proportion of participants with plasma HIV-1 RNA &lt;50 c/mL over time</li> <li>Proportion of participants with confirmed virologic failure over time</li> <li>Incidence of treatment emergent genotypic and phenotypic resistance to CAB and RPV over time</li> <li>Incidence and severity of AEs and laboratory abnormalities over time</li> <li>Proportion of participants who discontinue treatment due to AEs over time</li> <li>Absolute values and changes in laboratory parameters over time</li> <li>Incidence of disease progression (HIV-associated conditions, acquired immunodeficiency syndrome [AIDS] and death)</li> </ul> |
| To explore the effect of patient<br>characteristics on virologic and<br>immunologic responses to CAB LA+ | <ul> <li>Proportion of participants by patient subgroup(s) (e.g., by<br/>age, gender, BMI, race, HIV-1 subtype, Baseline CD4+,<br/>type of oral treatment [NNRTI, PI, or INSTI], duration prior</li> </ul> |

| Objectives | Endpoints |
|---|---|
| RPV LA every 8 weeks compared to CAB LA + RPV LA every 4 weeks | CAB LA and RPV LA exposure [0 weeks, 1-24 weeks, > 24 weeks]) with HIV-RNA greater than or equal to 50 c/mL, and with protocol-defined confirmed virologic failure over time including Week 48, Week 96 and Week 152 using the Snapshot algorithm for the ITT-E population Change from Baseline in CD4+ cell counts by subgroups at Week 48, Week 96 and Week 152 |
| To explore relationship(s) between<br>plasma concentrations of CAB and<br>RPV and pharmacodynamic<br>endpoints. | Relationship between plasma CAB and RPV concentrations and virologic, immunologic responses, and/or occurrence of adverse events [AEs] over time. |
| <ul> <li>To assess reason for switching using<br/>a single question.</li> <li>To assess reason for continuation</li> </ul> | For patients randomized from oral SOC, the reasons for willingness to switch ART at baseline (Day 1) will be assessed |
| using a single question | <ul> <li>For patients randomized from CAB LA + RPV LA every 4 weeks in ATLAS, the reasons for willingness to continue long-acting ART at baseline (Day 1) will be assessed</li> </ul> |
| To assess preference for CAB LA + RPV LA every 8 weeks or every 4 weeks compared to daily oral for participants receiving oral bridging during the Maintenance and/or Extension phases | Preference for CAB LA + RPV LA every 8 weeks or every<br>4 weeks compared to daily oral for participants receiving<br>oral bridging during the Maintenance and/or Extension<br>phases will be assessed using a preference questionnaire<br>at week 152 |

# 2.2.1. Thigh PK Sub-study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the PK of monthly and<br>every two months dosing of CAB LA<br>and RPV LA injections following<br>intramuscular administration in the<br>vastus lateralis (thigh) muscle<br>(compared to gluteal injections) in<br>HIV-1 infected participants currently<br>enrolled in the A2M sub-study | <ul> <li>Plasma PK parameters for CAB LA and RPV LA (Ctau,<br/>concentrations post dose [~Cmax], and area under the<br/>curve [AUC (0-tau)]) for thigh injections during the thigh<br/>injection phase compared with similar PK parameters for<br/>gluteal injections.</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To assess safety and tolerability of monthly and every two months dosing of CAB LA and RPV LA following intramuscular injections in the vastus lateral (thigh) muscle in HIV-1 infected participants currently enrolled in the A2M sub-study. | <ul> <li>Incidence and severity of ISRs and AEs of special interest during the thigh injection phase.</li> <li>Proportion of participants who discontinue treatment due to ISRs and AEs of special interest during the thigh injection phase.</li> </ul> |
| To assess the ability to maintain<br>virologic suppression (HIV-RNA < 50<br>copies/mL) in subjects who transition<br>to thigh administrations of CAB and | <ul> <li>Proportion of participants with plasma HIV-1 RNA &lt;50 c/mL over time (including at Week 16) during the thigh injection phase using the FDA Snapshot algorithm.</li> <li>Proportion of participants with plasma HIV-RNA ≥50 c/mL over time (including at Week 16) as per Food and Drug</li> </ul> |

| Objectives | Endpoints |
|---|---|
| RPV after receiving at least 3 years of gluteal injections. | Administration (FDA) Snapshot algorithm during the thigh injection phase. Proportion of participants with protocol-defined confirmed virologic failure (CVF) during the thigh injection phase. |
| To assess viral resistance in participants experiencing protocoldefined confirmed virologic failure. | <ul> <li>Incidence of treatment emergent genotypic and<br/>phenotypic resistance to CAB, RPV during the thigh<br/>injection phase.</li> </ul> |
| To assess patient reported outcomes during the thigh injection phase by administering the following health outcome measurements: Numerical Rating Scale (NRS) and HIVTSQ. To assess participant's preference of thigh injections during the thigh injection phase compared to gluteal injections. | <ul> <li>Numerical Rating Scale (NRS): To assess the tolerability of injections during both the Thigh and Gluteal Injection Phase</li> <li>HIVTSQ (both s and c versions): To measure levels of satisfaction and detect change in satisfaction when switching from gluteal to thigh injections in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Questionnaire (HIVTSQ) during the Thigh Injection Phase as well as the change from thigh during the Return to Gluteal Phase.</li> <li>Preference Questionnaire: To assess patient's preference, and reasons for preference, for injections received during the Thigh Injection Phase compared with prior gluteal injections as well as for injections received</li> </ul> |
| | during the Return to Gluteal phase compared with prior thigh injections. |
| Exploratory Objectives | Exploratory Endpoints |
| To assess additional safety events including other AEs, SAEs, and safety labs of monthly and every two months dosing of CAB LA and RPV LA following intramuscular injections in the vastus lateral (thigh) muscle in HIV-1 infected participants currently enrolled in the A2M sub-study. | Incidence of other AEs not of special interest, SAEs and change in laboratory and change in laboratory parameters from the last gluteal injection (prior to the Thigh Injection Phase). |

# 2.3. Study Design



N=1020, randomized 1:1 to each arm and stratified by prior CAB+RPV Exposure # SOC Patients not transitioning from the ATLAS study must be on uninterrupted current regimen (either the initial or second cART regimen) for at least 6 months prior to Screening. Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL in the 12 months prior to Screening: one within the 6 to 12 month window, and one within 6 months prior to Screening. No history of virologic failure. No evidence of viral resistance based on the presence of any resistance-associated major INI, or NNRTI mutation (except K103N) from prior genotype assay results. No current or prior history of etravirine use.

†Optional Extension Phase to continue randomized CAB LA + RPV LA Q4W or Q8W at Wk 100 ¥Participants who withdraw from IM arm must go into 52 week long term follow up phase if randomized regimen is not yet locally approved and commercially available.





Note: All injection visits during the sub-study should be kept to the same projected visit schedule as in the main study.

| Overview of S | tudy Design and Key Features |
|---|---|
| Design | Study 207966 (Antiretroviral Therapy as Long Acting Suppression every 2 Months- |
| Features | ATLAS-2M) is a Phase IIIb, randomized, open-label, active-controlled, multicenter, |
| | parallel-group, non-inferiority study designed to assess the antiviral activity and safety of CAB LA + RPV LA administered every 4 weeks compared CAB LA + RPV |
| | LA administered every 8 weeks in approximately 1020 adult HIV-1 infected patients. |
| | The ATLAS-2M main study comprises a Screening Phase (up to 35 days), and a |
| | Maintenance Phase (Day 1 to Week 100), followed by an Extension Phase (post |
| | Week 96). Additionally, any participant who receives at least a single dose of CAB |
| | LA and/or RPV LA and discontinues the CAB LA + RPV LA regimen will enter the |
| | Long-term Follow-up Phase and will initiate highly active antiretroviral therapy |
| | (HAART) for 52 weeks after the last dose of CAB LA and/or RPV LA, or until the |
| | assigned CAB LA + RPV LA regimen is locally approved and commercially |
| | available. |
| | Two groups of patients who fulfill eligibility requirements will be randomized (1:1) at |
| | Day 1 in the main study to receive CAB LA + RPV LA Q4W, or CAB LA + RPV LA |
| | Q8W regimen for at least 100 weeks: |
| | <ul> <li>Group 1: Patients randomized from current ART Standard of Care (SOC)<br/>therapy</li> </ul> |
| | Group 2: Patients currently receiving CAB LA + RPV LA Q4W |
| | After a minimum of 152 weeks on the ATLAS-2M main study, approximately 82 (41) |
| | per treatment arm) eligible participants will be enrolled in the sub-study. The |
| | enrolled sub-study participants will receive the study treatment on the same |
| | frequency as their randomized treatment, for example, participants randomized to the Q8W treatment in the main study will continue receiving the study treatment in |
| | every 8 weeks in the sub-study. |
| | The ATLAS-2M sub-study will consist of three phases including a Screening Phase |
| | (1 injection interval: 4 weeks for Q4W participants and 8 weeks for Q8W |
| | participants), a Thigh Injection Phase with 16 weeks of thigh injections (4 injection |
| | intervals for Q4W participants and 2 injection intervals for Q8W participants) and a |
| | Return to Gluteal Injection Phase with 8 weeks of gluteal injections for both Q4W |
| | and Q8W participants. At the conclusion of the sub-study, participants will have the |
| | option to continue on the A2M main study or if commercial access treatment is |
| | available, the participants can transition off the sub-study and withdraw from |
| Daaina | ATLAS-2M and proceed directly to CAB/RPV LA. |
| Dosing | • Group 1: oral therapy with CAB 30 mg + RPV 25 mg once daily at main study Day 1 |
| | for 28 days (±3 days) to determine individual safety and tolerability, followed by |
| | CAB LA + RPV LA Q4W or CAB LA + RPV LA Q8W (as randomized at main study Day 1) |
| | Group 2: CAB LA + RPV LA Q4W or CAB LA + RPV LA Q8W (as randomized at |
| | main study Day 1) |
| Time & | Refer to Appendix 2: Schedule of Activities |
| Events Treatment | Pandamized (1:1) at Day 1 to receive CARTA - RRVI A CAMA or CARTA - RRVI |
| Assignment | <ul> <li>Randomized (1:1) at Day 1 to receive CAB LA + RPV LA Q4W or CAB LA + RPV<br/>LA Q8W</li> </ul> |
| , toolgilliont | GSK RandAll NG used to generate randomization schedules |
| | <ul> <li>Stratified Randomization by prior CAB+RPV exposure (0 weeks, 1 to 24 weeks, &gt;24</li> </ul> |
| | weeks) |
| Interim | Futility analysis at (approx.) 50% of subjects completing Week 24 |
| Analysis | Continuous time monitoring of confirmed virologic failure (CVF) in the Q8W |
| | randomized arm until all participants complete Week 24 visit |

## **Overview of Study Design and Key Features**

- The main analysis will be conducted to evaluate the primary objective of the protocol at Week 48.
- Preliminary analyses at Week 24 and analyses at Week 96 and Week 152
- Sub-study analysis
- Further data cuts and analyses may be conducted as necessary in order to support regulatory submissions and publications.

# 2.4. Statistical Hypotheses / Statistical Analyses

The study is designed to demonstrate that the antiviral effect of Q8W dosing with CAB LA + RPV LA is non-inferior to Q4W dosing CAB LA + RPV LA in subjects stably suppressed on an oral SOC regimen or Q4W CAB LA + RPV LA regimen prior to randomization. Non-inferiority in the proportion of participants with HIV-1 RNA  $\geq$ 50 c/mL at Week 48 (defined by the US FDA snapshot algorithm) can be concluded if the upper bound of a two-sided 95% confidence interval for the difference between the two treatment arms (Q8W – Q4W) is less than 4%.

If  $f_{Q8W}$  is the snapshot failure rate for Q8W CAB LA + RPV LA, and  $f_{Q4W}$  is the snapshot failure rate for Q4W CAB LA + RPV LA then the null (H<sub>0</sub>) and alternative (Ha) hypotheses can be written as follows:

$$H_o$$
:  $f_{O8W} - f_{O4W} \ge 4\% \text{ vs } H_a$ :  $f_{O8W} - f_{O4W} < 4\%$ 

# 3. PLANNED ANALYSES

Analyses will be conducted to support Independent Data Monitoring Committee (IDMC) review of study data. At least four analyses in main study will be conducted to evaluate the objectives of the protocol after all subjects have completed their visits at Week 24, Week 48, Week 96 and Week 152, respectively. Prior to Week 48 analysis complete, the Week 24 results will be restricted to only those study team members and GSK/ViiV Healthcare senior management who need to be involved in the analysis and interpretation of the results for reporting to regulatory authorities. Details on protection against operation bias for Week 48 analysis are documented in the Blinded Team Operating Principles for this study. There is no planned hypothesis testing on the treatment difference at Week 24 and no decisions will be made based on the Week 24 results. Details of the planned displays for Week 24 analyses are provided in Section 15.15.4. Further data cuts and analyses may be conducted as necessary in order to support regulatory submissions and publications (first publication at Week 48). The Week 48 analysis will be primary and no results will be shared publicly until Week 48 analysis is complete. Additional analysis will be conducted to evaluate the objectives of the substudy after all subjects have completed their visits at Sub-study Week 24. A final End-of-Study analysis will be conducted when all subjects have completed the study.

# 3.1. IDMC Analyses

An IDMC will be instituted to ensure external objective medical and/or statistical review of efficacy and safety to protect the ethical interests and well-being of subjects and to protect the scientific validity of this study.

The IDMC will evaluate accumulating efficacy, tolerability, safety and PK of CAB LA + RPV LA Q8W during the study. An interim futility analysis will be performed for the IDMC to evaluate the efficacy of CAB LA + RPV LA Q8W prior to the final analyses.

The interim futility analysis will be performed with the intent of having approximately 50% of participants reaching Week 24 and providing sufficient lead time to allow the IDMC to review the data prior to any participants reaching the Week 48 visit. A futility rule based on Bayesian posterior predictive probability approach will be applied to assess the probability that the CAB LA + RPV LA Q8W injectable regimen demonstrates non-inferiority to the CAB LA + RPV LA Q4W regimen at Week 24, given the partial data set. The sponsor will remain blinded to this analysis.

In addition, the IDMC may also monitor the incidence of participants meeting Confirmed Virologic Failure (CVF) criteria before all subjects have completed Week 24 to ensure that subjects are not being sub-optimally treated in the CAB LA + RPV LA Q8W arm.

Full details of the analyses, estimated timing, and the decision criteria that will be used to determine regimen performance will be pre-specified in the IDMC Charter.

A list of outputs required for each IDMC analysis will be provided in the IDMC Charter. Data handing methods and derived data definitions will be the same as detailed in this RAP, unless otherwise stated.

# 3.2. Final Analyses

The primary analysis will be conducted to evaluate the primary objective of the protocol at Week 48. These analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed Week 48 and had a re-test for HIV-1 RNA if necessary.
- 2. All required database cleaning activities have been completed and database release (DBR) and database freeze (DBF) or database lock (DBL) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to Ramos NG procedures.

Three secondary analyses in main study will be conducted at Week 24, Week 96 and Week 152, sub-study analysis, and a final End-of-Study analysis will be conducted when all subjects have completed the study as defined in the protocol.

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | <ul> <li>Comprised of all subjects screened for inclusion in the study.</li> <li>Subjects may be re-screened once, for which they will receive a new subject number.</li> <li>For disposition displays, except for the listing of subjects who were rescreened, only the latest re-screening data will be included. All screening data will be summarized or listed for other displays.</li> </ul> | Study Population |
| Randomized | <ul> <li>All subjects who were randomly assigned to treatment in the study.</li> <li>In this study, the randomized population includes all enrolled participants, i.e. the randomized population is equivalent to the enrolled population.</li> <li>This population will be based on the treatment the participant was randomized to.</li> </ul> | Study Population |
| Safety | <ul> <li>All randomized subjects who received at least one dose of study treatment.</li> <li>Participants will be assessed according to actual treatment received.</li> </ul> | Safety |
| Intent-to-Treat<br>Exposed (ITT-E) | <ul> <li>All randomized subjects who received at least one dose of study treatment.</li> <li>Subjects will be assessed according to their randomized treatment, regardless of the treatment they received.</li> </ul> | <ul><li>Study Population</li><li>Efficacy</li><li>Health Outcomes</li></ul> |
| Per-Protocol<br>(PP) | <ul> <li>All subjects in the ITT-E population with the exception of major protocol violators.</li> <li>Protocol deviations that would exclude participants from the PP population are defined in Section 4.1 (Protocol Deviations) and Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).</li> </ul> | Efficacy (Sensitivity Analysis) |
| Pharmacokinetic<br>(PK) | All subjects who received CAB and / or RPV and underwent PK sampling during the study and provide at least 1 non-missing CAB and / or RPV plasma concentration value (Non-quantifiable [NQ] values will be considered as non-missing values). | • PK |
| Confirmed<br>Virologic Failure<br>(CVF) | All subjects in the ITT-E population who met Confirmed Virologic Failure (CVF) criteria. | <ul><li>Virology</li><li>Efficacy</li></ul> |
| Long-term Follow-<br>up (LTFU) | All subjects receiving at least one dose of CAB LA and/or RPV LA who have discontinued the CAB LA + RPV LA regimen and have either at least one Long-term Follow-up phase clinic visit (i.e. have at least one long-term follow-up visit shown in the study database, LTFU month 1, LTFU month 3, etc) or have filled out the LTFU phase conclusion form or have indicated the continuation to LTFU phase in the subject continuation form. | <ul><li>Safety</li><li>Study Population</li></ul> |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Week 24 Futility | All subjects in the ITT-E population who started study treatment at least 168 days prior to the IDMC cut-off date (in order to account for subjects who withdrew early but would have reached Week 24) | IDMC Futility Analysis (i.e. IDMC Week 24 Analyses) |
| | The IDMC cut-off date is the predicted Week 24 visit date (Last Subject Last Visit) corresponding to the time at which approximately 50% of subjects have completed Week 24. | |
| Oral Lead-in | All subjects who received at least one dose of study treatment during the oral lead-in period in ATLAS-2M study. | <ul><li>Safety</li><li>Study Population</li><li>Efficacy</li></ul> |
| Q4W ATLAS | All subjects in the ITT-E population who were randomized to Q4W arm in ATLAS. | Health Outcomes |
| SOC | All subjects in the ITT-E population who either were randomized to SOC arm in ATLAS or did not participate in ATLAS. | Health Outcomes |
| Oral Bridging | All subjects in the ITT-E population who received the oral bridging during the Maintenance and/or Extension phases. | Health Outcomes |
| Sub-study<br>Screened | <ul> <li>Comprised of all subjects screened for inclusion in the sub-study.</li> <li>All screened subjects will continue using their subject numbers received in the main study.</li> </ul> | Study Population |
| Sub-study Safety | <ul> <li>All randomized subjects who received at least one CAB and/or RPV thigh injection.</li> <li>Subjects will be assessed according to actual treatment received.</li> </ul> | <ul><li>Safety</li><li>Virology</li></ul> |
| Sub-study ITT-E | <ul> <li>All randomized subjects who received at least one CAB and/or RPV thigh injection.</li> <li>Subjects will be assessed according to their randomized treatment, regardless of the treatment they received.</li> </ul> | <ul><li>Study Population</li><li>Efficacy</li><li>Health Outcomes</li></ul> |
| Sub-study PK<br>Concentration | All subjects who received at least one CAB and/or RPV thigh injection and provided at least one non-missing CAB and/or RPV plasma concentration value (non-quantifiable values will be considered as non-missing values) during the sub-study. | • PK |
| Sub-study PK<br>Parameter | All subjects who received at least one CAB and/or RPV thigh injection and had at least one evaluable PK parameter estimate during the sub-study. | • PK |
| Sub-study CVF | All subjects receiving at least one CAB and/or RPV thigh injection who met Confirmed Virologic Failure (CVF) criteria in the sub-study. | Virology Efficacy |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Sub-study LTFU | All subjects receiving at least one CAB and/or RPV thigh injection who have discontinued the CAB LA + RPV LA regimen and have either at least one Long-term Follow-up phase clinic visit (i.e. have at least one long-term follow-up visit shown in the study database, LTFU month 1, LTFU month 3, etc) or have filled out the LTFU phase conclusion form or have indicated the continuation to LTFU phase in the subject continuation form. | Study Population |

Refer to Section 15.15: List of Data Displays which details the population used for each display.

## 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG Randomization System Data Displays for Reporting | | Reporting | |
| Code Description Description Order in | | Order in TLF | |
| Α | Q8W | Q8W | 1 |
| В | Q4W | Q4W | 2 |
| C/A | Oral followed by Q8W | Q8W | 1 |
| C/B | Oral followed by Q4W | Q4W | 2 |

#### Notes:

Unless stated otherwise, data displays will present two treatment group columns (Q8W and Q4W), where
treatment sequence C/A is pooled with sequence A and treatment sequence C/B is pooled with sequence B. The
detailed treatment sequence descriptors (i.e. C/A and C/B) may be used in selected data listings. Treatment C
refers to oral CAB + oral RPV, used for oral lead-in for subjects entering the study with no prior CAB+RPV
exposure.

Treatment comparisons will be displayed as follows using the descriptors as specified:

1. Q8W vs Q4W

# 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-treatment (see Table 8) assessment with a non-missing value, including those from unscheduled visits. 'Pre-treatment' in main study refers to prior to the study treatment (i.e. CAB and/or RPV) in this study, and 'pre-treatment' in sub-study refers to prior to the first CAB and/or RPV thigh injection.

Electrocardiograms (ECGs) are to be performed in triplicate on main study Day 1 visit. The baseline value for an ECG parameter will be the mean of the last pre-treatment set of assessments from the same date, so long as at least one of the triplicate assessments is available.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

## 5.3. Multicentre Studies

Data will be summarized for all centres combined. Country will be treated as an exploratory subgroup for analyses of the primary efficacy endpoint as described in Section 7.1.5.1 and secondary efficacy endpoint (HIV-1 RNA <50 c/mL) as described in Section 7.2.5.1. Some countries may be combined for exploratory subgroup analyses with consideration due to the number of participants enrolled.

# 5.4. Examination of Covariates, Other Strata and Subgroups

## 5.4.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|---|---|
| Strata | Randomization Strata: |
| | For the proportion of participants with plasma HIV-1 RNA ≥ 50 c/mL per FDA Snapshot algorithm at Week 48 (primary endpoint), a stratified analysis with Cochran-Mantel Haenszel weights will be used to adjust the primary treatment comparison for the randomization strata corresponding to prior exposure to CAB+RPV (0 weeks, 1-24 weeks, >24 weeks). A similar approach will be used to adjust the analysis of the proportion of participants with HIV-1 RNA <50 c/mL (per the FDA's Snapshot algorithm) at Week 48 (key secondary endpoint) and repeat analyses of these endpoints at Week 96 and Week 152. |
| | See Section 7.1.5.1 for additional details on the statistical analysis methodology. |
| Other Subgroups / Covariates | See details in Section 5.4.2 |

# 5.4.2. Examination of Subgroups

The following is a list of subgroups that may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be combined prior to un-blinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.
- For subgroup analysis, per European Medicines Agency Guideline on the investigation of subgroups in confirmatory clinical trials (EMA, 2014), factors defining a subgroup population may be put in three categories:

EMA Subgroup Category 1: Factors with strong reason to expect a heterogeneous response to treatment. In this case separate trials should usually be planned. There are no factors falling into this category in this study.

EMA Subgroup Category 2: Factors with at least some biological plausibility or external evidence such that a heterogeneous response might be hypothesized. In this study, stratified randomization strata, key demographic factors, Baseline CD4, CDC stage will be fall into this category. For these factors, subgroup analyses will be performed but

likely underpowered so that a formal proof of efficacy will not be available individually in all subgroups. If consistent findings across multiple comparisons were observed then these analyses would still be suggestive of a generalizable finding from the overall population.

EMA Subgroup Guideline Category 3: Factor with good argumentation why homogeneity of response to treatment is plausible. The impact of factors falling into this category will be explored.

• Additional covariates of clinical interest may also be considered.

| Category | Covariates and / or Subgroups |
|---|---|
| EMA Subgroup Category 2: | |
| Randomization Strata | Prior exposure to CAB+RPV (0 weeks, 1-24 weeks, >24 weeks) For analysis purposes, randomization strata will be rederived using eCRF data, even if this differs from the strata captured in RAMOS NG. |
| | All statistical analyses will adjust for the above randomization strata, unless stated otherwise. Treatment-by-Strata interactions will be assessed as specified in the analysis sections. |
| Demographic and Baseline<br>Characteristic Subgroups | <ul> <li>Age: <ul> <li>35, 35 - &lt; 50, ≥ 50</li> <li>For the statistical modelling, '&lt; 35' and '35 - &lt; 50' will be consolidated i.e. the following age group will be used:</li> <li>50, ≥ 50</li> <li>For the summary of demographic characteristics, the following age groups will also be presented:</li> <li>≤ 18, 19 - 64, ≥ 65 (FDAAA requirement)</li> <li>18 - 64, 65 - 84, ≥ 85 (EMA requirement)</li> </ul> </li> <li>Race: <ul> <li>White, Non-White</li> <li>Black/African American, Non-Black/African American For the statistical modelling, only White vs Non-White is considered.</li> </ul> </li> <li>Sex at birth: <ul> <li>Female</li> <li>Male</li> </ul> </li> <li>Country (not used for statistical modelling) <ul> <li>Argentina</li> <li>Australia</li> <li>Canada</li> <li>France</li> <li>Germany</li> <li>Italy</li> <li>Korea, Republic of</li> <li>Mexico</li> </ul> </li> </ul> |

| Category | Covariates and / or Subgroups |
|---|---|
| | Russian Federation |
| | <ul> <li>South Africa</li> </ul> |
| | <ul> <li>Spain</li> </ul> |
| | <ul> <li>Sweden</li> </ul> |
| | <ul> <li>United States</li> </ul> |
| | <ul> <li>Baseline CD4+ cell count (cells/mm³):</li> </ul> |
| | o <b>&lt;</b> 350 |
| | o 350 - < 500 |
| | o ≥ 500 |
| | Baseline HIV-1 RNA (c/mL): |
| | o <b>&lt;50</b> |
| | o ≥ 50 |
| | <ul> <li>Derived Baseline Centers for Disease Control and Prevention (CDC) category: <ul> <li>Stage I</li> </ul> </li> </ul> |
| | Stage III Print Forester to CAR, RRV |
| | Prior Exposure to CAB+RPV: Output Outpu |
| | <ul><li>0 weeks</li><li>≥ 1 weeks</li></ul> |
| | This subgroup will be used in efficacy analysis, in addition to the redrived randomization strata (prior exposure to CAB+RPV: 0, 1-24, and >24 weeks). It will also be used in health outcomes analysis. In other types of analysis, only the rederived randomization strata will be used. |
| | Baseline BMI (kg/m²) |
| | o <b>&lt;30</b> |
| | o ≥30 |
| | Baseline Third Agent Class: |
| | <ul> <li>CAB+RPV (for subjects with prior exposure to CAB+RPV in ATLAS, i.e. subjects transitioning from ATLAS who received CAB+RPV in ATLAS before entering ATLAS-2M)</li> <li>NNRTI</li> </ul> |
| | o INI |
| | o Pl |
| | <ul> <li>Baseline Genotypic Subgroup Variables: The Baseline genotypic data became available for most of the subjects after the Week 48 analysis data cut, the following subgroups will be used in post-Week 48 analyses as appropriate. The baseline genotypic data for subjects transitioning from ATLAS comes from ATLAS PBMC samples collected at Baseline and the baseline genotypic data for new subjects comes from ATLAS-2M PBMC samples collected at Baseline. Different types of mutation are defined in Section 15.6.7. Baseline HIV-1 Subtype: A, A1, AG Combined </li> </ul> |
| | ■ B |

| Category | Covariates and / or Subgroups |
|---|---|
| | • C |
| | ■ Other |
| | <ul> <li>Baseline L74I (Non-mixture) INSTI Mutation:</li> </ul> |
| | ■ Present |
| | <ul><li>Not Present</li></ul> |
| | <ul> <li>Baseline Pre-specified INSTI Mutation (Excluding L74I</li> </ul> |
| | Non-mixture): |
| | ■ Present |
| | <ul><li>Not Present</li></ul> |
| | <ul> <li>Baseline RPV RAM:</li> </ul> |
| | <ul><li>Present</li></ul> |
| | <ul><li>Not Present</li></ul> |
| | <ul> <li>Baseline NNRTI RAM (Excluding RPV RAM):</li> </ul> |
| | ■ Present |
| | <ul><li>Not Present</li></ul> |
| EMA Subgroup Category 3: | |
| Additional subgroup/covariates for | PK/PD efficacy analysis will be performed for participants without prior |
| PK/PD efficacy analysis | exposure to CAB + RPV. |
| | Mook 9 CAP/DDV Trough DV concentration (i.e. pro doce DV |
| | <ul> <li>Week 8 CAB/RPV Trough PK concentration (i.e. pre-dose PK concentration at nominal visit of Week 8)</li> </ul> |
| | concentration at nonlinar visit of week of |
| | The above covariate will be dichotomized into two subgroup factors |
| | as follows: |
| | <ul> <li>≤ first Quartile vs &gt; first quartile,</li> </ul> |
| | The concentration will also be treated as continuous variable in |
| | logistic regression modelling analysis (i.e. the concentration data will |
| | be log <sub>2</sub> transformed in this analysis so that, for assessing the effect, one unit increase of the point estimate of log2 PK concentration is |
| | equivalent to 'doubling the concentration' in the original value). |
| | equivalent to doubling the concentration in the original value). |
| | <ul> <li>Length of First CAB/RPV Injection Needle (&lt;2, ≥2 inches)</li> </ul> |
| Additional subgroup/covariates for | Last CAB/RPV trough PK concentration |
| PK/PD safety analysis | Last OnDitt V Hought It concentration |
| Tivi D saicty analysis | For the plot of Maximum Change from Baseline (CFB) in ALT/Total |
| | Bilirubin versus Last Trough CAB/RPV PK Concentrations, Last |
| | CAB/RPV Trough PK Concentration is the most recent trough PK |
| | concentration prior or equal to the date of the lab assessment with |
| | maximum CFB during the maintenance phase. |
| | For the Diet of Mayingura Taylaity Condens of Mark Francisch |
| | For the Plot of Maximum Toxicity Grades of Most Frequently Penerted Study Drug ISB adverse events (AEs) versus Last Trough |
| | Reported Study Drug ISR adverse events (AEs) versus Last Trough CAB/RPV PK Concentrations, Last CAB/RPV Trough PK |
| | Concentration is the most recent trough PK concentration prior or |
| | equal to the earliest onset date of the most frequently reported Study |
| | Drug ISR AE with maximum toxicity grade, during the maintenance |
| | phase. If a participant has no Study Drug ISR AE most commonly |

| Category | Covariates and / or Subgroups |
|---|---|
| | reported, then the last trough value during the maintenance phase will be used for the plot. |
| Additional subgroup for common drug-related study drug injection site reaction (ISR) with maximum toxicity grade | For each preferred term of the common drug-related study drug ISR with maximum toxicity grade (pain, induration, nodules and any other study drug ISR with >=5% subjects in either treatment arm) during the maintenance phase: • Needle Length for Last CAB Injection prior to and including the onset date of the earliest corresponding drug-related CAB ISR with maximum toxicity grade during the maintenance phase: ≤1.5, >1.5 to <2, ≥2 inches • Needle Length for Last RPV Injection prior to and including the onset date of the earliest corresponding drug-related RPV ISR with maximum toxicity grade during the Maintenance Phase: ≤1.5, >1.5 to <2, ≥2 inches |
| | Note: If there is no ISR of interest reported during the period of interest for a subject, the needle length of last injection during that period will be used in the summary. |

# 5.5. Multiple Comparisons and Multiplicity

# 5.5.1. Primary Comparison of Interest

The primary analysis will be based on the ITT-E population. The primary comparison will be made at a one-sided 2.5% level of significance. Treatment with Q8W will be declared non-inferior to Q4W if the upper end of a two-sided 95% confidence interval for the difference between the two groups (Q8W – Q4W) in the proportion of participants with HIV-1 RNA  $\geq$ 50 c/mL at Week 48 (defined by the US FDA snapshot algorithm) lies below 4%.

The primary comparison of interest is the comparison between Q8W (CAB LA + RPV LA Q8W) and Q4W (CAB LA + RPV LA Q4W) for the primary endpoint in the ITT-E population. This analysis will be adjusted for by the re-derived randomization strata based on eCRF data.

## 5.5.2. Other Comparisons of Interest

If the primary comparison of interest (Section 5.5.1) using the ITT-E population demonstrates non-inferiority of Q8W compared to Q4W then the following key secondary comparisons will be tested:

• Treatment with Q8W will be declared non-inferior to Q4W with respect to the proportion of participants with HIV-1 RNA < 50 c/mL at Week 48 (defined by the US FDA snapshot algorithm) if the lower end of a two-sided 95% confidence interval for the difference between in rates (Q8W – Q4W) lies above -10% using the ITT-E population

 Superiority of Q8W compared to Q4Wwith respect to change from baseline HIVTSQs total score at Week 48 using the ITT-E population and a two-sided 5% level of significance. Refer to Section 12.5.1 for details.

For the primary endpoint treatment comparison at Week 48, no multiple comparison adjustment is necessary for testing non-inferiority followed by superiority (conditional on achieving a significant test for non-inferiority) since testing follows a pre-specified sequence of hypothesis such that if the first hypothesis tested is not significant, all subsequent tests will not be performed. This fixed sequence procedure controls the type I error rate at the nominal level. The primary endpoint treatment comparison at Week 48 will also be performed using the PP population and the results will be compared for consistency with the results from the ITT-E population.

In addition to the primary and the key secondary comparisons, the comparisons between two treatment arms for ACCEPT (general acceptance score), PIN (Domain scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness)), HAT-QoL (Life satisfaction, HIV medications, disclosure worries) and HIVTSQc (Treatment Satisfaction score) at timepoints through Week 48 will also be performed as supportive analyses.

Lastly, for the IDMC interim analyses, since the statistical stopping guidelines will not result in early stopping for positive efficacy findings, these interim treatment comparisons will not inflate the Type I error rate for the primary treatment comparison.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|-------------------------------------------------------------------|
| 15.2.3 | Error! Not a valid result for table.: Assessment Windows |
| 15.4 | Appendix 4: Study Phases and Treatment State |
| 15.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 15.6 | Appendix 6: Derived and Transformed Data |
| 15.7 | Appendix 7: Reporting Standards for Missing Data |
| 15.8 | Appendix 8: Values of Potential Clinical Importance |
| 15.9 | Appendix 9: Snapshot Algorithm Details |
| 15.10 | Appendix 10: Variables Defined for Time to Event Analysis |
| 15.11 | Appendix 11: Identification of Adverse Events of Special Interest |
| 15.12 | Appendix 12: Identification of COVID-19 Adverse Events |
| 15.13 | Appendix 13: IDMC |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and oral study treatment accountability will be based on GSK Core Data Standards.

Table 1 provides an overview of the planned study population analyses, with details of the planned displays are presented in Appendix 15: List of Data Displays.

Table 1 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | |
|---|---|---|
| | Table | Listing |
| Randomization | | |
| Randomization [1] | | <b>Y</b> [2] |
| Subject Disposition | | |
| Study Populations [3] | Y | |
| Study Recruitment [3] | Y | |
| Reasons for Screening Failures [3] | Y | Υ |
| Rescreened Subjects [3] | | Υ |
| Age Ranges | Y | |
| Subject Disposition | <b>Y</b> [4][5] | |
| Reasons for Withdrawal | <b>Y</b> [4][5] | Υ |
| IP Discontinuation | Y | Υ |
| Important Protocol Deviations | Y | Υ |
| Deviations leading to exclusion from PP | Y | Υ |
| Inclusion and Exclusion Criteria Deviations | Y | Υ |
| Demography and Baseline | | |
| Demographics Characteristics [6] | Y | Υ |
| Race & Racial Combinations [7] | Y | Υ |
| Hepatitis Status at Entry | Y | |
| Baseline CDC Classification of HIV infection (2014) | Y | |
| Baseline Cardiovascular Risk Assessments | Y | |
| Distribution of CD4+ Cell Counts at Screening and Baseline | Y | |
| Prior Exposure to CAB+RPV | Y | |
| HIV-1 Risk Factors | Y | |

| Display Type Data Displays Genera | | olays Generated |
|---|---|---|
| | Table | Listing |
| Medical Conditions, Concomitant Medications & Antiretrov | viral Therapy | |
| Medical Conditions (Current/Past) [8] | Υ | |
| Medical Conditions: Sub-conditions (Current/Past) [9, 10] | Υ | |
| Concomitant Medications (non-ART) | Υ[10] | |
| Prior ART Medications | Y | Υ |
| Concomitant ART Medications during Maintenance Phase | | Υ |
| ART Medications Received during LTFU Phase | | Y |
| Lipid Modifying Agents (Baseline and during Maintenance Phase) | Υ | |
| Substance use at Entry | Υ | |
| Medical History of Seizure | | Y |
| Other | | |
| Oral Study Treatment Accountability [11] | | Y |
| Transition to CAB+RPV LA Marketed Product | | Υ |

#### NOTES:

- T = Tables, L = Listings, Y = Display Generated,
- 1. Base on Randomized population.
- One listing of participants randomized but not treated, and one listing of randomized and actual strata and treatment assignment.
- 3. All Subjects screened population.
- 4. Participants who have not been recorded as either completing or withdrawing from the study will be categorized as "Ongoing at time of the analysis" for summary purposes.
- Analysis of subject disposition will be performed for each Study Phase separately, as well as for overall study conclusion.
- 6. Age and ethnicity collected at Screening; weight and height collected at Baseline.
- 7. The five high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high level categories which exist in the data. The nine race categories collected will be summarised along with categories for mixed race. A by-subject listing of race will also be produced.
- 8. Medical conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).
- 9. Sub conditions are Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous System Conditions.
- 10. summarised by, Ingredient combinations.
- 11. Dispensation information (dates and number of tablets dispensed and returned).

## 6.2. Prior and Concomitant Medications

Non-ART and/or ART Medications will be classified by categories shown in Table 2. The same medication may be classified by more than one category. For example, if the medication was started after the maintenance treatment start date and was stopped at nominal Week 104 visit while subject was still receiving study treatment, this medication would be considered both 'concomitant during maintenance' and 'concomitant during extension'.

# Table 2 Derived Data for Non-ART Medications/ART Medications

| | Definition |
|---|---|
| Prior | Medication Taken < Maintenance Treatment Start Date |
| Concomitant<br>during<br>Maintenance | For subjects continuing into Extension Phase: Maintenance Treatment Start Date <sup>[a]</sup> ≤ Medication Taken < Date of Nominal Week 100 Visit |
| | For subjects not continuing into Extension Phase: For participants continuing into LTFU Phase: Maintenance Treatment Start Date <sup>[a]</sup> ≤ Medication Taken < LTFU ART Start Date <sup>[b]</sup> |
| Concomitant during Extension | For subjects continuing into Extension Phase and not entering the sub-study: If subjects continued into LTFU Phase after the Extension phase: Date of Nominal Week 100 Visit <sup>[c]</sup> ≤ Medication Taken < LTFU ART Start Date If subjects transitioned to marketed product/alternative HAART and did not withdraw study due to safety related reason, then Date of Nominal Week 100 Visit <sup>[c]</sup> ≤ Medication Taken < Date of end of study +35 days (Q4W) or +63 days (Q8W) For subjects continuing into Extension Phase, entering the sub-study but not returning to Extension Phase: Date of Nominal Week 100 Visit <sup>[c]</sup> ≤ Medication Taken < Date of First Sub-study Record For subjects continuing into Extension Phase, entering the sub-study and returning to Extension Phase: Before the sub-study: Date of Nominal Week 100 Visit <sup>[c]</sup> ≤ Medication Taken < Date of First Sub-study Record After the sub-study: For participants continuing into LTFU Phase after return to extension phase: End of Sub-study Date <sup>[c]</sup> < Medication Taken < LTFU ART Start Date <sup>[b]</sup> For participants transitioned to marketed product/alternative HAART and did not withdraw study due to safety related reason: End of Sub-study Date <sup>[c]</sup> < Medication Taken < Date of end of study +35 days (Q4W) or +63 days (Q8W) |
| Concomitant<br>during Sub-study<br>Screening | For subjects entering the sub-study and not receiving any thigh injection: If participants continued into LTFU Phase after the sub-study, then Date of First sub-study record ≤ Medication Taken < LTFU ART Start Date <sup>[b]</sup> If participants transitioned to marketed product/alternative HAART and did not withdraw study due to safety related reason, then Date of First sub-study record ≤ Medication Taken < Date of end of study +35 days (Q4W) or +63 days (Q8W) If participants continued into Extension Phase after the sub-study, then Date of First sub-study record ≤ Medication Taken ≤ End of Sub-study Date <sup>[c]</sup> For participants entering the sub-study and receiving thigh injection(s): Date of First sub-study record ≤ Medication Taken < Date of First Thigh Injection |

| Concomitant | For participants continuing into Return to Gluteal Injection Phase: |
|---|---|
| during Thigh | Date of First Thigh Injection [d] ≤ Medication Taken < Date of Nominal Sub-study Week |
| Injection | 16 Visit <sup>[c]</sup> |
| , | For participants not continuing into Return to Gluteal Injection Phase: |
| | If participants continued into LTFU Phase after the sub-study, then |
| | Date of First Thigh Injection ≤ Medication Taken < LTFU ART Start Date[b] |
| | If participants continued into Extension Phase after the sub-study, then |
| | Date of First Thigh Injection ≤ Medication Taken ≤ End of Sub-study Date[c] |
| | If participants transitioned to marketed product/alternative HAART and did not |
| | withdraw study due to safety related reason, then |
| | Date of First Thigh Injection ≤ Medication Taken ≤ Date of end of study +35 days |
| | (Q4W) or + 63 days (Q8W) |
| Concomitant | For participants continuing into Extension Phase after the sub-study: |
| during Return to | Date of Nominal Sub-study Week 16 Visit <sup>[c]</sup> ≤ Medication Taken ≤ End of Sub-study |
| Gluteal Injection | Date <sup>[c]</sup> |
| | For participants continuing into LTFU Phase after the sub-study: |
| | Date of Nominal Sub-study Week 16 Visit <sup>[c]</sup> ≤ Medication Taken < LTFU ART Start |
| | Date <sup>[b]</sup> |
| | For participants transitioned to marketed product/alternative HAART and did |
| | not withdraw study due to safety related reason: |
| | Date of Nominal Sub-study Week 16 Visit <sup>[c]</sup> ≤ Medication Taken ≤ Date of end of |
| | study +35 days (Q4W) or + 63 days (Q8W) |
| Received during | For subjects Who received at least one CAB and/or RPV injection and have |
| Long-term Follow- | started LTFU ART: |
| up | Medication Taken ≥ LTFU ART Start Date |

## NOTES:

- Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for medications. Use the rules in this table if medication date is completely missing.
- [a] The ART medication stopped on start date of Maintenance treatment will be considered a prior
  medication and will not be considered concomitant during the Maintenance phase. If the stop date
  of ART medication is completely missing and this medication is recorded in eCRF as prior (e.g.
  prior ART or prior ATLAS ART forms), it will be considered a prior medication and will not be
  considered concomitant during the Maintenance phase.
- [b] If subjects have missing LFTU ART start date, only the lower bound will be considered in the derivation.
- [c] Refer to Section 15.6.1 for the definition.

## 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Analyses

# 7.1.1. Endpoint / Variables

Proportion of participants with plasma HIV-1 RNA ≥50 c/mL as per Food and Drug Administration (FDA) Snapshot algorithm at Week 48 (Intent-to-Treat Exposed [ITT-E] population); see Section 15.9 for additional details.

# 7.1.2. Summary Measure

Difference in the proportion of participants with HIV-1 RNA  $\geq$ 50 c/mL at Week 48 (defined by the US FDA snapshot algorithm) between each treatment group (Q8W – Q4W).

## 7.1.3. Population of Interest

The primary efficacy analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

# 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

As defined by the Snapshot algorithm, HIV-1 RNA  $\geq$  50 c/mL is determined by the last available HIV-1 RNA measurement while the participant is on treatment within the analysis visit window of interest.

Participants without on-treatment HIV-1 RNA data for the visit of interest and who discontinue treatment for reasons not related to adverse event while having HIV-1 RNA  $\geq 50$  c/mL at time of discontinuation or who change study treatment not permitted per protocol before the analysis window are classified as having HIV-1 RNA  $\geq 50$  c/mL.

# 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 15: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.1.5.1. Statistical Methodology Specification

## **Endpoint**

Proportion of Participants with plasma HIV-1 RNA ≥ 50 c/mL at Week 48 using the Snapshot algorithm for the ITT-E population. Subjects with 'HIV-1 RNA ≥ 50 c/mL' per Snapshot algorithm include those who had plasma HIV-1 RNA ≥ 50 c/mL at Week 48, who discontinued for lack of efficacy, who discontinued for other reasons while not <50 c/mL, or who changed ART.</li>
#### **Snapshot Dataset**

- Virologic outcome ('HIV-1 RNA <50 c/mL' or 'HIV-1 RNA ≥ 50 c/mL') per Snapshot algorithm is determined by the last available on-treatment HIV-1 RNA measurement within the analysis visit window of interest (please refer to analysis window defined in Table 10). In addition, subjects who discontinue for reasons not related to adverse event with on-treatment HIV-1 RNA result at the time of discontinuation ≥ 50 c/mL or who change study treatment not permitted per protocol during maintenance phase before the analysis visit are classified as 'HIV-1 RNA ≥ 50 c/mL'.</p>
- Full details of the Snapshot algorithm are provided in Section 15.9.

## **Model Specification**

- The primary efficacy endpoint will be analysed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights, adjusting for the rederived randomization strata corresponding to prior exposure to CAB+RPV (0 weeks, 1-24 weeks, >24 weeks)
- The CMH estimate of the adjusted treatment difference will be calculated as a weighted average of strata-specific estimates of the treatment difference calculated within each stratum as follows:
  - o If  $n_k$  is the number of Q8W treated participants,  $m_k$  is the number of Q4W arm treated participants, and  $N_k = n_k + m_k$  is the total number of participants in the kth stratum, then the CMH estimate is given by

$$\hat{d}_{cmh} = \frac{\sum W_k \hat{d}_k}{\sum W_k}$$

where

$$W_k = \frac{n_k m_k}{N_k}$$

are CMH weights and  $\hat{d}_k$  are estimates of the differences in proportions between the two treatment arms, f<sub>Q8W</sub>-f<sub>Q4W</sub>, for the *kth* stratum.

• The corresponding two-sided 95% CI will be calculated as

$$\hat{d}_{cmh} \pm 1.96 \times \sqrt{\widehat{var}(\hat{d}_{cmh})}$$

where the variance estimator [Sato, 1989] is consistent in both sparse data and large strata and is given below:

$$\operatorname{var}(\hat{d}_{cmh}) = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum n_k m_k / N_k\right)^2} = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum W_k\right)^2}$$

where

$$P_k = \frac{n_k^2 y_k - m_k^2 x_k + n_k m_k (m_k - n_k)/2}{N_k^2}$$

$$Q_k = \frac{x_k (m_k - y_k) / N_k + y_k (n_k - x_k) / N_k}{2}$$

with  $x_k$  and  $y_k$  corresponding to the number of participants with Plasma HIV-1 RNA  $\geq$  50 c/mL at Week 48 per FDA Snapshot for Q8W and Q4W, respectively, for the *kth* stratum.

#### **Model Results Presentation**

- Adjusted CMH estimate of the difference in the proportion of subjects with Plasma HIV-1 ≥ 50 c/mL between each treatment group (Q8W Q4W) and corresponding 95% confidence interval.
- Non-inferiority will be concluded if the upper bound of the two-sided 95% confidence interval for the CMH adjusted treatment difference (Q8W – Q4W) is less than 4%.
- If this analysis shows non-inferiority, then a superiority hypothesis will be tested at the two-sided 5% level of significance. Superiority favoring Q8W will be declared if the upper bound of the confidence interval is below 0% for the ITT-E population analysis. If superiority is declared, the p-value for superiority will also be calculated.

#### **Subgroup Analyses**

- 1. Treatment Heterogeneity across rederived randomization strata [prior exposure to CAB+RPV (0 weeks, 1-24 weeks, >24 weeks)]:
  - The weighted least squares chi-squared statistic [Fleiss, 1981] will be used to test for oneway homogeneity across the levels of each categorical variable, with each categorical variable considered separately.
  - Following Lui and Kelly [Lui, 2000] ½ will be added to each cell in any strata for which the stratum-specific rate estimates of either f<sub>Q8W</sub> or f<sub>Q4W</sub> are zero or one, and tests will be onesided.
  - Any heterogeneity found to be statistically significant will be explored and if necessary
    results will be reported for each level of the categorical variable. Investigation of
    heterogeneity will be confined to the primary endpoint. Tests of homogeneity will be
    assessed at the one-sided 10% level of significance.
- 2. Stratum-specific analyses for two groups of participants: (Group 1) those currently receiving Standard of Care antiretroviral therapy at Baseline (i.e. no prior exposure to CAB+RPV), (Group 2) those receiving Q4W CAB LA + RPV LA therapy in the ongoing ATLAS study (i.e. have prior exposure to CAB+RPV). For each stratum (Group 1 and Group 2), the following will be presented:
  - Proportion of subjects with plasma HIV-1 RNA ≥ 50 c/mL at Week 48 by treatment group.
  - Unadjusted difference in proportions between treatment groups and corresponding twosided 95% CI.
  - Summary of study outcomes (i.e. HIV-1 RNA < 50 c/mL, HIV-1 RNA ≥50 c/mL and reason for no data in the window)

For Group 2, a stratum-adjusted analysis will also be provided, with adjustment for prior CAB+RPV exposure (1 to 24 weeks vs. >24 weeks) using Cochran-Mantel Haenszel (CMH) weights, as described in the model specification above for the overall primary analysis.

#### 3. Exploration of Subgroups

- An analysis for subgroups listed in Section 5.4.2 will be performed. This will show the
  proportion of subjects with plasma HIV-1 RNA ≥50 c/mL at the time of analysis (Week 48)
  based on the Snapshot algorithm and will be presented by treatment group.
- Unadjusted difference in proportions between treatment groups and corresponding two-sided 95% CI will also be presented by subgroups. The confidence interval will be calculated using an unconditional exact method [Chan, 1999] with two inverted one-sided tests based on the score statistic. These results will also be presented graphically.
- Summary of study outcomes (i.e. HIV-1 RNA < 50 c/mL, HIV-1 RNA ≥50 c/mL or reason for no data in the window) by subgroup will be produced.

Note: These subgroup analyses will be exploratory and likely underpowered so that interpretation may therefore focus on point estimates as well as the upper bounds of 95% CIs for the treatment differences and response rates. Additionally, multiple comparisons are being made which inflates the risk of false positive findings. Therefore, if consistent findings across the multiple comparisons were observed then these analyses would still be suggestive of a generalizable finding of non-inferiority.

#### **Sensitivity and Supportive Analyses**

- 1. Per-protocol population analysis:
  - To assess the impact of important protocol deviations, statistical analysis will be repeated using the Per-protocol population and compared for consistency with the results from the primary ITT-E population analysis.

# 7.2. Secondary Efficacy Analyses

#### 7.2.1. Endpoints

The key secondary efficacy endpoint is the proportion of participants with plasma HIV-1 RNA < 50 c/mL at Week 48 using the FDA Snapshot algorithm (Intent-to-Treat Exposed [ITT-E] population).

Other secondary efficacy endpoints for the study are listed below:

- Proportion of participants with plasma HIV-1 RNA < 50 c/mL at Week 24, Week</li>
   96 and Week 152 using the FDA Snapshot algorithm (ITT-E population)
- Proportion of participants with plasma HIV-1 RNA < 50 c/mL over time (including at Sub-study Week 16) using the FDA Snapshot algorithm during the Sub-study Thigh Injection phase (Sub-study ITT-E population)
- Proportion of participants with protocol-defined confirmed virologic failure (CVF) through Week 24, Week 48, Week 96 and Week 152
- Proportion of participants with protocol-defined confirmed virologic failure (CVF) through the Sub-study Thigh Injection phase

- Proportion of participants with HIV-1 RNA ≥50 c/mL as per FDA Snapshot algorithm at Week 24, Week 96 and Week 152
- Proportion of participants with plasma HIV-1 RNA ≥ 50 c/mL over time (including at Sub-study Week 16) using the FDA Snapshot algorithm during the Sub-study Thigh Injection phase
- Absolute values and changes from Baseline in viral load and CD4+ cell counts over time including Week 48, Week 96 and Week 152

# 7.2.2. Summary Measure

Difference in the proportion of participants with HIV-1 RNA < 50 c/mL at Week 24, Week 48, Week 96 and Week 152 (defined by the US FDA snapshot algorithm) between each treatment group (Q8W – Q4W).

Difference in the proportion of participants with HIV-1 RNA  $\geq$  50 c/mL at Week 24, Week 96 and Week 152 (defined by the US FDA snapshot algorithm) between each treatment group (Q8W – Q4W).

#### 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

# 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

As defined by the snapshot algorithm, participants with last available HIV-1 RNA measurement less than 50 c/mL while the participant is on treatment within the analysis visit window of interest are classified as HIV-1 RNA < 50 c/mL.

Participants without on-treatment HIV-1 RNA data for the visit of interest and who discontinue treatment for reasons not related to adverse event while having HIV-1 RNA  $\geq 50$  c/mL at time of discontinuation or who change study treatment not permitted per protocol before the analysis window are classified as having HIV-1 RNA  $\geq 50$  c/mL.

### 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 15: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.2.5.1. Statistical Methodology Specification

#### **Key Secondary Statistical Analysis**

### **Endpoint**

 Proportion of participants with plasma HIV-1 RNA <50 c/mL at Week 48 using the FDA Snapshot algorithm (Intent-to-Treat Exposed [ITT-E] population)


207966

# **Key Secondary Statistical Analysis**

# **Snapshot Dataset**

• As Section 7.1.5.1 and Section 15.9

# Model Specification

• As specified in Section 7.1.5.1 but with 'HIV-1 RNA <50 c/mL' replacing HIV-1 ≥ 50 c/mL

## **Key Secondary Statistical Analysis**

#### **Model Results Presentation**

- Adjusted CMH estimate of the difference in the proportion of participants with HIV-1 RNA < 50 c/mL at Week 48 between each treatment group (Q8W Q4W) and corresponding 95% confidence interval.</li>
- Non-inferiority will be concluded if the lower bound of the two-sided 95% confidence interval for the CMH adjusted treatment difference (Q8W Q4W) is greater than -10%.

## **Subgroup Analyses**

As specified in Section 7.1.5.1 but with HIV-1 RNA < 50 c/mL replacing 'HIV-1 RNA ≥ 50 c/mL.</li>

## **Sensitivity and Supportive Analyses**

- 1. Per-protocol population analysis:
  - To assess the impact of important protocol deviations, statistical analysis will be repeated using the Per-protocol population and compared for consistency with the results from the primary ITT-E population analysis.

# 7.3. Exploratory Efficacy Analyses

Table 3 provides an overview of the planned exploratory efficacy analyses. Details of the planned displays are provided in Appendix 15: List of Data Displays and will be based on GSK data standards and statistical principles. The exploratory efficacy analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

Table 3 Overview of Exploratory Efficacy Analyses

| Endpoints | | | A | bsolu | ite | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | mary | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Indiv | /idual |
| | Т | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| Proportion of participal discontinuation (TRDF) | | | | - | | | | • | | or tr | eatme | nt-rela | ited | |
| Kaplan-Meier estimate | | | | Υ | | | | | | | | | | |
| Proportion of participal<br>Snapshot | nts wi | th pla | sma l | HIV-1 | RNA≥ | ≥50 c/r | nL ov | er tim | e (Ma | inten | ance F | Phase) | - | |
| by visit | | | | Υ | <b>Y</b> [1] | | | | | | | | | |
| By visit and subgroup | | | | Υ | <b>Y</b> [2] | | | | | | | | | |
| Proportion of participants with plasma HIV-1 RNA <50 c/mL over time (Maintenance Phase) - Snapshot | | | | | | | | | | | | | | |
| by visit | | | | Υ | <b>Y</b> [3] | | | | | | | | | |
| By visit and subgroup | | | | Υ | <b>Y</b> [2] | | | | | | | | | |
| Proportion of participal<br>Snapshot | nts wi | th pla | sma | HIV-1 | RNA ≥ | ≥200 c | /mL o | ver tir | ne (M | aintei | nance | Phase | e) - | |
| by visit | | | | <b>Y</b> [4] | <b>Y</b> [5] | | | | | | | | | |
| Proportion of participal Snapshot | nts wi | th pla | sma l | HIV-1 | RNA < | (200 c | /mL ov | ver tir | ne (M | ainter | nance | Phase | e) - | |
| by visit | | | | <b>Y</b> [4] | <b>Y</b> [5] | | | | | | | | | |
| Proportion of participal in IP injection - Snapsh | | th pla | sma l | HIV-1 | RNA ≥ | ≥50 c/r | nL at | Week | 48/W | eek 9 | 6/Wee | k 152 | by de | lay |
| by delay in IP injection [6] | | | | Υ | | | | | | | | | | |
| Proportion of participa | nts wi | th pla | sma | HIV-1 | RNA < | 2 c/m | L ove | r time | (Mair | itenar | nce Ph | nase) | | |
| by visit | | | | Υ | | | | | | | | | | |
| Plasma HIV-1 RNA ove | r time | | | | | | | | | | | | | |
| by visit | | | | <b>Y</b> [7] | | <b>Y</b> [8] | <b>Y</b> [9] | | | | | | | <b>Y</b> [9] |
| Target Detected vs<br>Target Not Detected by<br>visit [10] | | | | Υ | | | <b>Y</b> [11] | | | | | | | |
| Confirmed Virologic Fa | ilure | (CVF) | | | | | | | | | | | | |
| CVF overall | | | | Υ | | | | | | | | | | |
| CVF by visit | | | | Υ | | | Υ | | | | | | | |

| Endpoints | | | A | bsolu | ite | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | mary | Individual | | Stat | s Ana | lysis | Sum | mary | Indiv | idual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Plasma HIV-1 RNA at<br>time of suspected and<br>confirmed virologic<br>failure | | | | Y | | | | | | | | | | |
| CD4+ & CD8+ Cell Cour | nts Ov | er Ti | me | | | | | | | | | | | |
| CD4+ observed [12] | | | | Υ | | | | | | | Υ | | | |
| CD8+ observed [12] | | | | Υ | | | | | | | Υ | | | |
| CD4+/CD8+ ratio observed [12] | | | | Y | | | | | | | | | | |
| HIV-1 Conditions and D | iseas | e Pro | gress | ion | | | | | | | | | | |
| HIV Conditions including/excluding Recurrences as recorded in eCRF | | | | Y | | | Y | | | | | | | |
| HIV Disease<br>Progressions [13] | | | | Υ | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of data.
- Individual = Represents FL related to any displays of individual participant's data.
- 1. Line plots, with 95% confidence intervals (Cls), for the proportion of participants with HIV-1 RNA ≥50 c/mL by treatment group at each visit. The 95% Cls will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation.
- 2. Plot of the unadjusted treatment difference and its 95% confidence intervals (Snapshot algorithm) overall and by subgroup at Week 48/Week 96/Week 152.
- 3. Line plots, with 95% confidence intervals, for the proportion of participants with HIV-1 RNA<50 c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 100%; otherwise, they are derived using the normal approximation.
- 4. Study outcomes (i.e., HIV-1 RNA <200 c/mL, HIV-1 RNA ≥200 c/mL, or reason for no data in the window) based on the snapshot algorithm at Week 48 will also be produced.
- 5. Line plots, with 95% confidence intervals, for the proportion of participants with HIV-1 RNA <200 c/mL and ≥200 c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0% or 100%; otherwise, they are derived using the normal approximation.</p>
- 6. Delay in IP injection (days) is defined in Section 15.6.3.
- 7. Using log10 transformed values.
- 8. Individual plasma HIV-1 RNA only for participants who are in the category of 'viral load ≥50 c/mL' at Week 48 per Snapshot algorithm or who are CVF participants. The figures will display all HIV-1 RNA values collected.
- 9. For CVF participants, participants with viral load ≥ 50 c/mL during the Maintenance Phase, and participants with viral load ≥ 50 c/mL during the Maintenance oral lead-in period.
- 10. See Section 15.6.3 for definition of "Target Detected" and "Target Not Detected", and for the specification of corresponding summary table.
- 11. Target Detected" and "Target Not Detected" are included in the listing for plasma HIV-1 RNA by visit.
- 12. Using available data without imputation for missing values.
- 13. See Section 15.6.3 for HIV disease progressions.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs), COVID-19 AEs and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Section 15.15: List of Data Displays.

# 8.1.1. Analyses for Injection Site Reaction Adverse Events from Study Drug Injection

Injection Site Reaction (ISR) adverse events of interest are those from study drug injections. For the summary of study drug ISR adverse events by visit and maximum severity (overall and by common ISRs): ISRs will be assigned based on onset date to the most recent planned IM injection visit prior or equal to the AE onset date.

Maximum grade at each visit will be derived as the maximum grade among ISRs assigned to the particular visit, with consideration for whether the summary applies to a particular preferred term (vs. across preferred terms), drug-related associated to CAB and/or RPV, or stratification by subgroup (such as needle length, refer to Section 5.4.2).

Drug-related ISRs (based on investigator discretion) from study drug injections will be attributed to the causal agent (CAB vs. RPV) when this can be determined specifically based on the side of injection administration and the side of the reported ISR (as collected in the eCRF). If we are unable to determine the causal agent in those cases where both drugs are given on one side and the ISR is reported non-specifically, then the attribution to a specific causal agent will remain unknown.

Common study drug ISR adverse events are defined by MedDRA preferred terms including injection site pain, injection site induration, injection site nodules and preferred terms of any other ISR with ≥5% participants in either treatment arm, coming from study drug injections. The same set of common terms will be applied to 'overall' (CAB and/or RPV), CAB alone, RPV alone.

Study drug ISRs will be attributed to the needle length ( $\leq 1.5$ , > 1.5 to < 2,  $\geq 2$  inches) specifically based on the side of injection administration and the side of the reported ISR (as collected in the eCRF). If we are unable to determine the needle length for events where both drugs are given on one side and their needle lengths are different, then the attribution to a needle length will remain unknown.

# 8.2. Adverse Events of Special Interest Analyses

Adverse events of special interest (AESI) are determined for CAB and/or RPV based on pre-clinical and clinical experience, along with information for the Integrase Inhibitor class of HIV medications and RPV safety profile. Table 4 shows the currently identified AESI, drug(s) of Interest and the reasons for inclusion. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting, and/or

emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of AESIs may change at the time of reporting.

A summary by system organ class and preferred term will be provided for each of AESI. The characteristics of event occurrences will be summarized in main study for common AESI which have at least 20 participants in either treatment arm, and will be summarized in sub-study for common AESI which have at least five participants in either treatment arm. For Depression, anxiety and suicidal ideation/behaviour AESI, a summary by system organ class, maximum DAVIDS toxicity grade and prior history of suicidal ideation will be provided. The details of the planned grouping and planned displays are provided in Section 15.11 and Appendix 15: List of Data Displays.

Table 4 Adverse Events of Special Interest

| Adverse Events of Special Interest | Drug(s) of<br>Interest | Reason for Inclusion |
|---|---|---|
| Hepatic Safety Profile: Assessment of Risk of hepatoxicity | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Hypersensitivity Reactions (HSR) | CAB | Class, Regulatory Interest,<br>Occurs in HIV population |
| Rash | RPV | Class, Regulatory Interest,<br>Occurs in HIV population |
| Prolongation of the Corrected QT Interval of the ECG in Supratherapeutic Doses | RPV | Non-clinical, Clinical,<br>Regulatory Interest |
| Suicidal Ideation/Behaviour | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Depression | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Bipolar Disorder | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Psychosis | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Mood Disorders | CAB+RPV | Clinical, Class, Regulatory<br>Interest |
| Anxiety | CAB+RPV | Clinical, Class, Regulatory<br>Interest |
| Sleep Disorders | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |

| Adverse Events of Special Interest | Drug(s) of<br>Interest | Reason for Inclusion |
|---|---|---|
| Injection Site Reactions (ISR) from Study Drug Injections [1] | CAB+RPV | Clinical |
| Seizures and Seizure-like Events | CAB | Clinical, Regulatory Interest |
| Weight Gain | CAB | Clinical, Class |
| Rhabdomyolysis | CAB | Clinical, Class |
| Pancreatitis | CAB | Clinical, Therapeutic Area,<br>More prevalent in HIV<br>population |
| Impact on Creatinine | CAB+RPV | Regulatory Interest,<br>Therapeutic Area, More<br>prevalent in HIV population |
| Safety in Pregnancy | CAB | Regulatory Interest, Class |
| Hyperglycaemia | CAB | Class, Regulatory Interest |
| NOTE: | | 1 |

[1] A separate analysis will be performed for ISRs from study drug injections as described in Section 8.1.1.

# 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analysis of results of Chemistry laboratory tests, Haematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 15: List of Data Displays.

# 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 15: List of Data Displays.

ECG values of potential clinical importance are defined as a QTc of > 500 msec or increase from baseline in QTc  $\geq$  60 msec.

#### 9. PHARMACOKINETIC ANALYSES

The GSK Division of Clinical Pharmacology Modelling and Simulation (CPMS) will be responsible for the PK analysis of CAB. The Division of Clinical Pharmacology and Pharmacometrics at Janssen Research and Development will be responsible for conduct or oversight of the PK analysis for RPV.

# 9.1. Endpoint / Variables

## 9.1.1. Drug Concentration Measures

Refer to Appendix 5 Data Display Standards & Handling Conventions (Section 15.5.3 Reporting Standards for Pharmacokinetic)

# 9.2. Overview of Planned Analyses

Table 5 provides an overview of the planned analyses with full details being presented in Appendix 15: List of Data Displays. All PK displays will be based on the PK Population, unless otherwise specified.

Table 5 Overview of Planned Pharmacokinetic Analyses

| | Stat | s Analy | /sis | Sun | nmary | Indiv | /idual |
|---|---|---|---|---|---|---|---|
| | T | F | L | T | F | F | L |
| Pharmacokinetic [5] | | | | | | | |
| Plasma CAB concentration by visit | | | | <b>Y</b> [1][2] | <b>Y</b> [1][3][4] | <b>Y</b> [3] | Y |
| Plasma RPV concentration by visit | | | | <b>Y</b> [1][2] | <b>Y</b> [1][3][4] | <b>Y</b> [3] | Y |
| Steady state concentration | Y | | | | | | |
| Plasma CAB parameters by dosing interval | Y | Υ | | Y | | | Υ |
| Plasma RPV parameters by dosing interval | Y | Υ | | Y | | | Y |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- Unless otherwise specified, all displays for evaluable concentrations except for individual displays will be presented by both overall and the rederived randomization strata.
- For both 'all' concentration and the 'evaluable' concentration. The evaluable concentration is derived from samples collected within pre-specified Time window (Section 15.6.5)
- 2. For both 'untransformed' and 'log-transformed' statistics.
- 3. The plots will be produced for the untransformed scale (i.e., a linear plot) and the log transformed scale (i.e., log-linear plot), separately.
- 4. Separate plots will be produced for Mean (SD) and Median concentration.
- 5. Standard summary statistics for concentration data will be calculated (i.e., mean, standard deviation, coefficient of variation, median, minimum and maximum). For Logarithmically transformed data, the summary statistics (i.e. geometric mean, between subject coefficient of variation, 95% confidence interval for the geometric mean and standard deviation) will also be calculated.

# 9.3. Statistical Analyses / Methods

#### Planned PK statistical analysis

# **Steady State Concentration**

#### **Endpoints**

 log<sub>e</sub>-transformation of the Trough/Pre-dose evaluable plasma concentrations (CAB/RPV) on Week 16-48 (i.e. Weeks 16, 24, 32, 40 and 48) for participants receiving Q8W study treatment

#### **Covariates**

Study Week

### **Data Handling**

All data remains as is (observed).

#### **Model Specification**

A mixed effects ANOVA model will be fitted for each rederived randomization stratum [prior exposure to CAB+RPV (0 weeks, 1-24 weeks, >24 weeks)] with Study Week (continuous variable) as a fixed effect and subject as a random effect for each analysis separately. The Kenward & Roger (KR) degrees of freedom approach will be used. The coefficient for the slope of the week effect on the loge-scale will be used to evaluate steady state for each drug (CAB/RPV). The 90% confidence intervals for the slope for each treatment will be calculated. If it does not appear that steady-state has been demonstrated, early weeks (e.g. Week 16, 24, etc...) results will be dropped and the analysis repeated.

#### Model Checking & Diagnostics

 The steady state will be claimed (the coefficient for the slope of the week effect on the (natural) log scale was close to 0 or the 90% CI for the slope estimate included zero. If steady-state is not demonstrated, concentrations from early weeks (e.g. Week 16, 20, 24, etc...) dropped in sequence and the analysis repeated until either steady state is shown or only two timepoints remain.

#### **Model Results Presentation**

• The coefficient for the slope of the week effect on the log<sub>e</sub>-scale, its standard error and 90% interval will be presented for each rederived randomization stratum.

#### **PK Parameters**

#### **Endpoints**

 As data permit, Log<sub>e</sub>-transformation of the PK parameters (Ctau, Cmax and AUC(0-tau) for each sub-study dosing interval (refer to Section 15.6.5 for definition of the dosing interval) for participants enrolled in the sub-study

## **Model Specification**

Following Loge-transformation, PK parameters will be separately analyzed by treatment arm
and analyte using a mixed effects model with dosing interval (gluteal injection, first thigh
injection and last thigh injection) as fixed effects and subject as random effects. In each
model, only subjects with evaluable PK parameter estimates in both dosing intervals are
included. For example, in the model for comparing Cmax estimated from the first CAB thigh

injection interval with Cmax estimated from the gluteal injection interval among Q8W subjects, only the Q8W subjects with evaluable Cmax estimates from both first CAB thigh injection interval and gluteal injection interval are included.

## **Model Checking & Diagnostics**

 Model assumptions will be applied, but appropriate adjustments may be made based on the data.

#### **Model Results Presentation**

 The estimated difference and 90% CI obtained on the log<sub>e</sub> scale will be exponentiated to provide an estimate of geometric mean ratio and its associated 90% CI. The estimate of within-subject variability (%CVw) will also be provided.

#### 10. POPULATION PHARMACOKINETIC ANALYSES

The Population PK analyses will be described under a separate Population-PK Reporting and Analysis Plans for CAB LA and RPV LA

# 11. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

The primary goal of this analysis is to characterize the pharmacokinetic / pharmacodynamic relationship of CAB/RPV administered in participants with HIV-1-infection who are virologically suppressed. The influence of subject demographics and baseline characteristics and additional subgroups/covariates in this population will be investigated.

## 11.1. Overview of Planned Analyses

Table 6 provides an overview of the planned analyses with full details being presented in Appendix 15: List of Data Displays. All PK displays will be based on the PK Population, unless otherwise specified.

Table 6 Overview of Planned Pharmacokinetic / Pharmacodynamic Analyses

| | Stat | s Analy | /sis | Sun | nmary | Indiv | /idual |
|---|---|---|---|---|---|---|---|
| | T | F | L | Т | F | F | L |
| CAB/RPV Week 8 concentrations by snapshot 'HIV-1 RNA ≥50 c/mL' (Yes vs. No) at Week 48 for participants without prior exposure to CAB+RPV | | | | Y | Y | | |
| Analysis of snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 by Week 8 trough concentration, and subgroup [¹¹] – univariable analysis /multivariable analysis for participants without prior exposure to CAB+RPV | Y | | | | | | |
| Individual CAB/RPV concentration-time profiles for participants with snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 or 96 or 152 | | | | | Y | | |
| Maximum change from baseline in ALT/Total Bilirubin versus last trough CAB/RPV concentrations for Week 48 and Week 152 analyses <sup>[2]</sup> | | | | | Y | | |
| Change from baseline in pre-dose QTcF versus CAB/RPV concentrations at Week 48 or 152 | | | | | Y | | |
| Maximum toxicity grades of most frequently reported study drug ISR AEs <sup>[3]</sup> versus last trough CAB/RPV PK concentrations for Week 48 analysis <sup>[2]</sup> | | | | | Y | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. Refer to Section 11.2.
- 2. Display by rederived randomization strata, i.e. prior exposure to CAB+RPV (0, 1-24, >24 weeks) derived based on eCRF.
- 3. Most frequently reported study drug ISR AEs are those top 5 in incidence in either treatment arm (i.e. Q8W or Q4W arm).

# 11.2. Statistical Analyses / Methods

## PK/PD Efficacy Analysis for Participants without Prior Exposure to CAB+RPV

#### **Endpoints**

Snapshot 'HIV-1 RNA≥50 c/mL' at Week 48

#### **Covariates**

 Treatment, demographic and baseline characteristics except for country and Prior Exposure to CAB+RPV (0, ≥1 weeks), and additional subgroup/covariates for PK/PD efficacy analysis see derivation details in Section 5.4.2.

## **Data Handling**

All data remains as is (observed).

## **Model Specification**

 Logistic regression will be used to exam the correlation between the endpoint (Snapshot 'HIV-1 RNA≥50 c/mL') at Week 48 and the covariates/subgroups. This logistic regression analysis will be performed for each covariate or subgroup, separately (univariable analysis), and will also be performed with one multivariable analysis using Backward stepwise selection approach to identify the covariates/subgroups potentially affecting virologic response.

#### **Model Checking & Diagnostics**

- For the multivariable analysis, a logistic regression model that best predicts the dependent variable (i.e. snapshot 'HIV-1 RNA≥50 c/mL') from the independent variables (i.e. covariates/factors with P <0.15 from univariable analysis) will be determined using the backward stepwise selecting approach. Week 8 trough PK concentration will be logarithmically transformed with base of 2 (i.e. one-unit increase of the point estimate of log2 PK concentration is equivalent to 'doubling the concentration' in the original value). The analysis will start with all covariates in the model and remove a covariate with the largest p-value (i.e. the least statistically significant) each time and continue until the stopping rule is reached when all remaining covariates have p-value <15%.
- If problems with model convergence occur due to zero event counts or complete/quasicomplete separation, then alternative methods such as exact logistic regression may be used.

#### **Model Results Presentation**

The odds ratio, 95% confidence interval, and p-value will be presented.

## 12. HEALTH OUTCOMES ANALYSES

# 12.1. Endpoint / Variables

# **12.1.1. Main Study**

- Preference between injections of LA HIV treatment and daily oral HIV treatment at Week 48
- Preference between LA injection every 8 weeks and LA injection every 4 weeks at Week 48 (Q8W arm only)
- Change from baseline in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) at Weeks 24, 48 and 152
- Change from baseline in life satisfaction, HIV medication, and disclosure worries using HIV/AIDS Targeted Quality of Life (HAT-QoL) at Weeks 24 and 48
- Change in treatment satisfaction over time using the HIV Treatment Satisfaction Change (HIVTSQc) questionnaire at Week 48
- Change from Week 8 in Dimension Scores and individual item scores assessing pain during injection, anxiety before and after injection, willingness to be injected in the future and overall satisfaction with mode of administration over time using Perception of Injection (PIN) questionnaire at Weeks 24, 48 and 152
- Change from baseline in treatment acceptance using ACCEPT at Weeks 24, 48 and 152
- Reasons for continuation of receiving injectable HIV treatment at Baseline (Day 1) visit. This is an exploratory endpoint.
- Reasons for switching to injectable HIV treatment at Baseline (Day 1) visit. This is an exploratory endpoint.
- Preference for CAB LA + RPV LA injection compared to daily oral for participants receiving oral bridging during the Maintenance and/or Extension phases at Week 152. This is an exploratory endpoint.

# 12.1.2. Sub-study

- Change from gluteal to thigh in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) during the Thigh Injection phase as well as the change from thigh to gluteal during the Return to Gluteal Injection phase
- Change from gluteal to thigh using the HIV Treatment Satisfaction Change (HIVTSQc) questionnaire at Sub-study Week 16
- Changes in the tolerability of injections (NRS) over time during the sub-study
- Preference for thigh injections compared with prior gluteal injections and the injections received during the Return to Gluteal Injection phase respectively.

# 12.2. Summary Measure

For main study, mean treatment difference (Q8W – Q4W) at visits of interest, except for Preference between LA injection every 8 weeks and LA injection every 4 weeks at Week 48.

For sub-study, mean difference between thigh injections and gluteal injections from visits of interest, except for the Preference between thigh injections and gluteal injections.

# 12.3. Population of Interest

The health outcomes analyses will mainly be based on the Intent-to-Treat Exposed population, unless otherwise specified.

Analysis of Reason for continuation will be based on a subset of the Intent-to-Treat Exposed population who were randomized to Q4W arm in ATLAS (i.e. ATLAS Q4W population).

12.4. Analysis of Reason for switch will be based on a subset of Intent-to-Treat Exposed population who either were randomized to SOC arm in ATLAS or did not participate in ATLAS study (i.e. SOC population). Strategy for Intercurrent (Post-Randomization) Events

If a participant discontinues treatment prior to the timepoint of interest such that there is no evaluable assessment for the timepoint of interest, the data will be computed or imputed (see Section 15.6.6).

# 12.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 15: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 12.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 12.5.1. Statistical Methodology Specification

#### Statistical Analyses

#### **Endpoints**

- Change from Baseline in
  - HIVTSQs total treatment satisfaction score at Weeks 24,48 and 152
  - ACCEPT general acceptance score at Weeks 24, 48 and 152
  - HAT-QoL (Life satisfaction, HIV medications, disclosure worries) at Weeks 24 and 48
- Change from Week 8 in PIN Domain Scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness) at Weeks 24, 48 and 152

#### **Statistical Analyses**

### **Model Specification**

- The analysis for HIVTSQs, ACCEPT and HAT-QoL will be performed for subjects with and without prior exposure to CAB+RPV separately.
  - For subjects without prior exposure to CAB+RPV, an analysis of covariance (ANCOVA) model will be used at each visit during the maintenance phase with covariates: treatment, age (<50, ≥ 50 years old), sex at birth, race (i.e. white, nonwhite) and baseline score value for other endpoints (as a continuous variable).
  - For subjects with prior exposure to CAB+RPV, an analysis of covariance (ANCOVA) model will be used at each visit during the maintenance phase with covariates: treatment, age (<50, ≥ 50 years old), prior exposure to CAB+RPV (i.e. 1 to 24 weeks, >24 weeks), sex at birth, race (i.e. white, non-white) and baseline score value (as a continuous variable).
- For PIN, an analysis of covariance (ANCOVA) model will be used at each visit during the
  maintenance phase with covariates: treatment, age (<50, ≥ 50 years old), prior exposure to
  CAB+RPV (i.e. 0 weeks, 1 to 24 weeks, >24 weeks), sex at birth, race (i.e. white, non-white),
  and Week 8 score value (as a continuous variable).
- Adjusted point estimates will be derived as LSMEANS using the observed margins (OM) option within PROC MIXED in SAS.
- The superiority testing of Q8W compared to Q4W with respect to change from baseline in HIVTSQs total score at Week 48 will be performed using the fixed sequence procedure to control for the type I error rate at the nominal level of 5%. If the superiority testing within subjects without prior exposure to CAB+RPV demonstrates Q8W is superior to Q4W in change from baseline in HIVTSQs total score at Week 48 at two-sided 5% level of significance, the superiority testing at the same level of significance (i.e. two-sided 5%) within subjects with prior exposure to CAB+RPV will be followed. No adjustment for multiplicity will be applied for other tests as they will be considered supportive.
- Interactions between treatment and each of the covariates will not be assessed unless the exploratory subgroup analyses on the primary endpoint highlights significant interactions. In this situation, the interaction(s) of interest will be assessed and, if necessary, results will be reported in the clinical study report. Interactions between treatment and the baseline score will be investigated but not included in the model. If interactions are found to be significant (p<0.10), results may be presented separately by subgroup.

#### **Dataset**

LOCF dataset will be used.

#### **Model Results Presentation**

- Adjusted treatment difference (Q8W Q4W), its 95% CI and the associated p-value. The
  interaction between treatment and the baseline score will be included in a footnote.
- Plots of adjusted mean change from baseline (95% CI) for each treatment group, and the adjusted mean difference (95%CI) between the two treatment arms from the model will be generated across visit.

#### **Statistical Analyses**

#### **HIVTSQc**

• Total Treatment Satisfaction Score (Change) at Week 48

#### **Model Specification**

- An analysis of variance (ANOVA) model will be used with covariates: treatment, age (<50, ≥ 50 years old), prior exposure to CAB+RPV (i.e. 0 weeks, 1 to 24 weeks, >24 weeks), sex at birth and race (i.e. white, non-white).
- Adjusted point estimates will be derived as LSMEANS using the observed margins (OM) option within PROC MIXED in SAS.
- Interactions between treatment and each of the covariates will not be assessed unless the exploratory subgroup analyses on the primary endpoint highlights significant interactions. In this situation, the interaction(s) of interest will be assessed and, if necessary, results will be reported in the clinical study report. If interactions are found to be significant (p<0.10), results may be presented separately by subgroup.
- No adjustment for multiplicity will be applied as these analyses will be considered supportive.

#### **Dataset**

The observed case (OC) dataset uses only the data that is available at Week 48, with no imputation for missing values.

#### **Model Results Presentation**

Adjusted means, 95% CI, and associated p-value will be presented for the treatment difference (Q8W – Q4W).

#### **Statistical Analyses**

#### PIN/HIVTSQs

- Change from Week 8 in the PIN acceptance score at Week 24, Week 48 and Week 152
- Change from Sub-study Baseline in the HIVTSQs total treatment satisfaction score at Substudy Week 16, Sub-study Week 24 (for Q8W arm) or Sub-study Week 20 (for Q4W arm).

#### **Statistical Test**

• The Wilcoxon Signed-Rank Test will be used to evaluate:

For PIN, whether the change from Week 8 to each post Week 8 main study visit, is statistically different from zero based on a two-sided p<0.05.

For HIVTSQs, whether the change from Sub-study Baseline to each post-baseline sub-study visit is statistically different from zero based on a two-sided p<0.05.

#### **Dataset**

- For PIN, LOCF dataset will be used.
- For HIVTSQs, observed dataset will be used.

#### **Results Presentation**

- For PIN, summary statistics at each timepoint (Week 8, Week 24, Week 48 and Week 152) and p-value for each comparison between scores at Week 24/48/152 with scores at Week 8.
- For HIVTSQs, summary statistics at Sub-study Baseline, Sub-study Week 16, Sub-study Week 24 (for Q8W arm) or Sub-study Week 20 (for Q4W arm), and p-value for the comparison between scores at each post-baseline sub-study visit with scores at Sub-study Baseline.

#### 13. VIROLOGY

The virology analyses will mainly use genotype and phenotype data based on plasma sample for CVF population, unless otherwise specified. Additional analyses for HIV-1 resistance may be carried out on peripheral blood mononuclear (PBMC) samples collected at Day 1, Week 48, Week 96, Week 152 or Withdrawal if prior to Week 152, Sub-study Day 1.

If pre-treatment genotypic/phenotypic results are available from both the central laboratory and Monogram Biosciences, then Baseline genotype/phenotype will be determined based only upon the data provided by Monogram assays.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 15: List of Data Displays.

Table 7 Overview of Planned Virology Analyses

| Endpoint | Absolute | | | |
|---|---|---|---|---|
| | Sum | nmary | Indivi | dual |
| | T | F | F | L |
| Genotypic resistance at time of CVF <sup>[1]</sup> | | | | T |
| Prevalence of Resistance Mutations | <b>Y</b> [2] | | | Y |
| Prevalence of Genotypic Susceptibility | Y | | | |
| Phenotypic resistance at time of CVF <sup>[1]</sup> | | | | |
| Prevalence of Phenotype | <b>Y</b> [3] | | | Y |
| Fold Change to CAB and RPV | Y | | | <b>Y</b> [4] |
| IN, PR/RT Replication Capacity | | | | Υ |
| Other | | | | • |
| Viral load, Genotypic and Phenotypic data for<br>Participants with genotype and/or phenotype<br>data for CVF and non-CVF participants | | | | <b>Y</b> [4] |
| Net Assessment | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. For the CVF as indicated by two consecutive plasma HIV-1 RNA levels ≥200 c/mL after prior suppression to <200 c/mL, the first visit of these two consecutive visits is defined as 'the suspected visit', and the 2nd one is the confirmed visit. Sample used for resistance testing is taken at the suspected visit, and only tested once a participant confirms virological failure at a subsequent visit. If the test fails with the sample at the suspected visit, we will just report it as 'no data'. The sample from the confirmed visit may be used for exploratory analyses.
- No. and percentage of participants with IN resistance mutations or major mutations in the classes of NNRTI, NRTI, PI, respectively, as defined in Section 15.6.7.
- 3. Separate outputs by phenotypic susceptibility and by number of drugs to which participants are phenotypic resistant or partial sensitive or sensitive.


207966

| Endpoint | | Abs | solute | |
|----------|-----|-------|------------|---|
| | Sum | ımary | Individual | |
| | T | F | F | Ĺ |

<sup>4.</sup> Fold change to CAB and RPV will be included in the listing for viral load, genotypic and phenotypic data for participants with genotype and/or phenotype data for CVF and non-CVF participants.

#### 14. REFERENCES

Chan, I. S. F. and Zhang, Z. (1999), "Test-Based Exact Confidence Intervals for the Difference of Two Binomial Proportions," Biometrics, 55, 1202–1209.

Chevat C, Viala-Danten M, Dias-Barbosa C, Nguyen VH. Development and psychometric validation of a self-administered questionnaire assessing the acceptance of influenza vaccination: the Vaccinees' Perception of Injection questionnaire. Health Qual Life Outcomes. 2008 mar 4; 7:21

D'Agostino RB, Vasan RS, Pencina MJ, et al. General Cardiovascular Risk Profile for Use in Primary Care (The Framingham Heart Study). Circulation 2008; 117: 743-753.

EMA/CHMP/539146/2013, Guideline on the investigation of subgroups in 4 confirmatory clinical trials, 23 January 2014

Fleiss J.L. Statistical Methods for Rates and Proportions. 2nd ed. New York: John Wiley; 1981.

Gilet H, Arnould B. Acceptance by the patients of their treatment (ACCEPT) Questionnaire, 2014.

Grundy S.M., et al. Executive summary of the third report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). JAMA. 2001; 285 (19): 2486-2497.

HIVTSQ user guidelines, Health Psychology Research Unit, Royal Holloway, University of London, 2016

Holmes WC, HIV/AIDS-Targeted Quality of Life Instrument 1999.

Kalbfleisch J.D., Prentice R.L. *The Statistical Analysis of Failure Time Data*. 1st ed. New York: John Wiley & Sons; 1980.

Levey AI, Christopher HS, Hocine T, John HE, Harold IF, Tom G, et al. Esitmating Glomerular Filtration Rate from Serum Creatinine and Cystatin C. N Engl J Med 2012, 367: 20-29.

Lui K.J., Kelly C. A Revisit on Tests for Homogeneity of the Risk Difference, Biometrics, 2000; 56:309-315.

Nilsson ME, Suryawanshi S, Gassmann-Mayer C et al, Columbia–Suicide Severity Rating Scale, Scoring and Data Analysis Guide, 2013.

Sato T. On the variance estimator for the Mantel-Haenszel risk difference. *Biometrics*. 1989; 42:311-323.

Wensing AM et al. Update of the Drug Resistance Mutations in HIV-1 Volume 27 Issue 3 July/August 2019

#### 15. APPENDICES

# 15.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

#### 15.1.1. Exclusions from Per Protocol Population

Important protocol deviations leading to exclusion from the Per Protocol population are those deviations which may

- directly impact the efficacy endpoint of HIV-1 RNA; or
- lead to permanent discontinuation of IP/withdrawal and hence indirectly impact the efficacy endpoint by causing data to be missing.

The following criteria define the important protocol deviations which, if they occur prior to an analysis timepoint of interest (e.g. Week 48/96/152), will lead to exclusion of a participant from the Per-Protocol population for that analysis. Potential protocol deviations leading to exclusion from PP population will be reviewed by the study team to confirm that they meet these criteria. A final review will occur before the clinical database has been frozen for analysis.

A participant meeting any of the following criteria will be excluded from the Per Protocol population based on case-by-case clinical determination:

| Number | Exclusion Description |
|---|---|
| 01 | Participant deviates from any inclusion or exclusion criteria that may significantly affect exposure, response to therapy or participant safety or that are fundamentally inconsistent with the intended study population, as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |
| 02 | Participant has maintenance phase non-compliance (including IM dosing errors) with investigational product up to an analysis timepoint of interest, meeting one of the following 3 conditions. For Week 48 analysis, the analysis timepoint of interest is the date of last ontreatment viral load up to Study Day 378 during maintenance phase, where Study Day 378 is the upper bound of snapshot window for Week 48 visit. For Week 96 analysis, the analysis timepoint of interest is the date of last on-treatment viral load up to Study Day 714 during the maintenance phase, where Study Day 714 is the upper bound of snapshot window for Week 96 visit. For Week 152 analysis, the analysis timepoint of interest is the date of last ontreatment viral load up to Study Day 1106 during the maintenance and extension phase, where Study Day 1106 is the upper bound of snapshot window for Week 152 visit. |
| 02 | <ul> <li>Week 48 analysis only: <ul> <li>Two or more injection intervals affected by over dosage deviations, for example</li> <li>Extra injection or excessive volume administered.</li> <li>For Q8W participants requiring oral lead-in: length of time between Week 4B injection and Week 8 injection less than 3 weeks, or between injections post Week 8 less than 7 weeks, excluding split doses.</li> <li>For Q8W participants not requiring oral lead-in: length of time between injections less than 7 weeks, excluding split doses.</li> </ul> </li> </ul> |

| Number Exclusion Description |
|---|
| <ul> <li>For Q8W participants requiring reloading injections: length of time<br/>between the reloading injection and the injection after reloading less<br/>than 3 weeks, excluding split doses.</li> </ul> |
| <ul> <li>For Q4W participants: length of time between injections less than 3<br/>weeks, excluding split doses.</li> </ul> |
| 2. Week 96 analysis only: |
| <ul> <li>For participants who permanently discontinued study treatment on/before the<br/>analysis timepoint of interest for Week 48 analysis (i.e. the date of last on-<br/>treatment viral load up to Study Day 378): two or more injection intervals<br/>affected by over dosage deviations.</li> </ul> |
| For participants who received injections beyond the analysis timepoint of interest for Week 48 analysis (i.e. the date of last on-treatment viral load up to Study Day 378): three or more injection intervals affected by over dosage deviations. |
| 3. Week 152 analysis only: |
| <ul> <li>For participants who permanently discontinued study treatment on/before the analysis timepoint of interest for Week 48 analysis (i.e. the date of last on- treatment viral load up to Study Day 378): two or more injection intervals affected by over dosage deviations.</li> </ul> |
| <ul> <li>For participants who received injections beyond the analysis timepoint of interest<br/>for Week 48 analysis (i.e. the date of last on-treatment viral load up to Study<br/>Day 378): five or more injection intervals affected by over dosage deviations.</li> </ul> |
| 4. ≥ 10% of total time on-treatment with under dosing deviations. The percentage of total time on-treatment with under dosing deviations will be calculated by (the total number of non-compliant dosing days / the total number of intended exposure days) * 100%. |
| Number of Intended Exposure Days = Date of Last Viral Load – Start Date of Study Treatment + 1, |
| where the last viral load refers to the last on-treatment viral load up to Study Day 378 during maintenance phase for Week 48 analysis, the last on-treatment viral load up to Study Day 714 during maintenance phase for Week 96 analysis, the last on-treatment viral load up to Study Day 1106 during maintenance and extension phase for Week 152 analysis. |
| The total number of non-compliant dosing days up to the analysis timepoint visit (or date of IP discontinuation/ withdrawal, whichever is earlier), is derived as follows ( <u>summing across all instances</u> ): |
| <ul> <li>For Q4W arm participants requiring oral lead-in:</li> </ul> |
| <ul> <li>Length of time (in days) until next injection from date of dosage<br/>deviation (e.g. 2 mL administered instead of 3mL for Week 4B injection,<br/>1ml administered instead of 2 mL for post Week 4B injections).</li> </ul> |
| <ul> <li>Length of time (in days) in excess beyond 35 days between injections post Week 12 and in excess beyond 28 days for Week 8 and Week 12 (e.g. missed or late injection visit).</li> </ul> |
| <ul> <li>Length of time (in days) in excess beyond 35 days from last injection<br/>until start of oral bridging post Week 12 and in excess beyond 28 days<br/>for Week 8 and Week 12.</li> </ul> |
| For Q4W arm participants not requiring oral lead-in: |

| Number | Exclusion Description |
|---|---|
| | <ul> <li>Length of time (in days) until next injection from date of dosage deviation (e.g. 1 mL administered instead of 2 mL).</li> <li>Length of time (in days) in excess beyond 35 days between injections.</li> <li>Length of time (in days) in excess beyond 35 days from last injection until start of oral bridging.</li> <li>For Q8W arm participants requiring oral lead-in: <ul> <li>Length of time (in days) until next injection from date of dosage deviation (e.g. 2 mL administered instead of 3mL).</li> <li>Length of time (in days) in excess beyond 63 days between injections post Week 16 and in excess beyond 28 days for Week 8 and 56 days for Week 16 (e.g. missed or late injection visit). The similar calculation of the length of time in excess will be used for the period after the reloading dose injection visit.</li> <li>Length of time (in days) in excess beyond 63 days from last injection until start of oral bridging post Week 16 and in excess beyond 28 days for Week 8 and 56 days for Week 16.</li> </ul> </li> </ul> |
| | <ul> <li>For Q8W arm participants not requiring oral lead-in: <ul> <li>Length of time (in days) until next injection from date of dosage deviation (e.g. 2 mL administered instead of 3 mL).</li> <li>Length of time (in days) in excess beyond 63 days between injections.</li> <li>Length of time (in days) in excess beyond 63 days from last injection until start of oral bridging.</li> </ul> </li> <li>For subjects requiring reloading injections, the number of non-compliant days for the first and second injection visits after the reloading will be calculated similarly to that for Week 8 and Week 12 for subjects on the same treatment arm requiring oral lead-in.</li> <li>Interrupted days in oral study treatment (oral lead-in or oral bridging) if the oral dose has been interrupted for 3 or more consecutive days and the primary interruption reason is not adverse event or laboratory abnormality (based on the eCRF Exposure forms). 3 days will be assumed if such interrupted days are not available in the database.</li> </ul> |
| 03 | Prohibited medications: receiving ART medication other than that prescribed/allowed by the study (excluding permanent changes in ART regimen; such cases will be retained as 'HIV1-RNA ≥50 c/mL' in the per protocol snapshot analysis) or receiving prohibited concomitant medication that would impact exposure or response to therapy with duration and route of administration taken into consideration, as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |
| 04 | Permanent discontinuation of IP/withdrawal due to a reason of "Protocol Deviation" (as recorded in the eCRF). |
| 05 | Other important protocol deviations that exclude Participant from per protocol population as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). The participants who has taken SOC oral bridging at/prior to the analysis timepoint due to COVID-19 may be excluded from per protocol population for the analysis and will be evaluated based on case-by-case clinical determination. |

# 15.2. Appendix 2: Schedule of Activities

While some assessments included in the Time and Events Table are conducted less frequently following the primary endpoint (Week 48), IM injections for participants during the Extension Phase will continue to be administered Q4W or Q8W based on original study randomization assignment.

All patients will be randomized at Day 1 to initiate either Q4 weekly or Q8 weekly administration of IM CAB LA + RPV LA. Only participants randomized from oral SOC treatment will participate in the Day 1 to Week 4 Oral CAB + Oral RPV lead-in treatment.

# 15.2.1. Protocol Defined Schedule of Events for Q4W Arm in Main Study

| | | | | | | | | | | Maint | tenanc | | | | | | | | | | Exte<br>Phas | nsion<br>se | | ıts.y | × |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| re | /isit a | | | Week | | | | | | | | | | | | | | | | | dn-w | | | | |
| Procedure<br>Screening Vis | Screening Visit | Day 1 | Week 4A (Oral<br>Lead-in Only) <sup>b</sup> | Week 4B | ∞ | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 4 | 48 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W After<br>Week 100 | Q8W After<br>Week 96 | 152 | Withdrawal Assessments. <sup>y</sup> | Long-Term Follow-up <sup>z</sup> |
| Written<br>informed<br>consent | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Eligibility<br>Verification<br>(Inclusion/Ex<br>clusion<br>Criteria) | X | | X | | | | | | | | | | | | | | | | X <sup>e</sup> | | | | | | |
| Randomization | W | X | | | | | | | | | | | | | | | | | | | | | | | |
| Demography<br>Medical<br>History <sup>d</sup> | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Cardiovascular<br>risk assessment <sup>d</sup> | X | X | | | | | | | | | | | | | | | | | | | | | | | |
| Medication<br>History/ Prior<br>ART history | X | | | | | | | | | | | | | | | | | | | | | | | | |
| Syphilis<br>serology +<br>Reflex Rapid<br>Plasma<br>Reagin<br>(RPR) | X | X | | | | | | | | | | | | | | | | | | | | | | | |

| | | | | | | | | | | Main | tenanc | e Phas | e | | | | | | | | Exte<br>Phas | nsion<br>se | | ts.y | 2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <u> -</u> | 'isit " | | | | | | | | | | | | Week | | | | | | | | | | | ssmen | m-w |
| Procedure | Screening Visit | Day 1 | Week 4A (Oral<br>Lead-in Only) <sup>b</sup> | Week 4B | ∞ | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W After<br>Week 100 | Q8W After<br>Week 96 | 152 | Withdrawal Assessments. <sup>y</sup> | Long-Term Follow-up <sup>z</sup> |
| Symptom<br>Directed<br>Physical<br>Exam and<br>Medical<br>Assessment <sup>e</sup> | х | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | X | Х | X | Х | Х |
| Weight,<br>Height and<br>BMI <sup>f</sup> | | X | | | | | | | | | | | | | Х | | | | Х | | | | Х | х | |
| Vital Signs:<br>BP, HR,<br>Temperature) <sup>g</sup> | Х | X | | | | | | | | | | | | | X | | | | X | | | | Х | Х | |
| 12-lead ECG<br>h<br>(triplicate at Day<br>1 pre-dose) | Х | Х | | | | | | | | | | | | | х | | | | Х | | | | Х | Х | |
| CDC HIV-1<br>stage | Х | X | | | | | | | | | | | | | | | | | | | | | | | |
| HIV<br>Associated<br>Conditions | | X | Х | X | X | X | X | X | Х | X | X | X | X | X | X | X | X | X | X | X | Х | Х | X | X | X |
| AEs, SAEs,<br>Concomitant<br>Medications | Х | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | Х | X | X | Х | X |

| | | | | | | | | | | Maint | enanc | e Phas | e | | | | | | | | Exte<br>Phas | nsion<br>se | | ts.y | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ē. | 'isit a | | | | | | | | | | | | Week | | | | | | | | | | | ssmen | , dn-w |
| Procedure | Screening Visit a | Day 1 | Week 4A (Oral<br>Lead-in Only) <sup>b</sup> | Week 4B | ∞ | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W After<br>Week 100 | Q8W After<br>Week 96 | 152 | Withdrawal Assessments. <sup>y</sup> | Long-Term Follow-up <sup>z</sup> |
| ISR<br>Assessment<br>for IM<br>injections | | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Columbia<br>Suicide<br>Severity<br>Rating Scale<br>(eC-SSRS) <sup>j</sup> | X | X | | X | X | | X | | X | | X | | X | | X | | | X | X | | | | | X | |
| Clinical<br>chemistry<br>and<br>Hematology | х | X | Х | X | Х | | X | | X | | X | | X | | X | | | X | X | X | | Х | X | Х | X |
| Pregnancy<br>Testing <sup>k</sup> | S | U | S | U | S | U | S | U | S | U | S | U | S | U | S | S | U | S | S | S | U | S | S | S | S |
| HIV-1 RNA<br>and sample<br>for storage<br>(S) <sup>1</sup> | Х | X | Х | Х | Х | | Х | | Х | | х | | Х | | Х | S | | Х | Х | S | | Х | Х | Х | Х |
| CD4+ cell<br>count | Х | X | | X | X | | X | | Х | | Х | | X | | X | | | X | X | | | Х | X | Х | Х |
| CD8+ cell<br>count | | X | | | | | | | X | | | | | | X | | | | X | | | | X | X | |
| Urinalysis <sup>m</sup> | | X | X | | | | | | X | | | | | | X | | | | X | | | | X | X | |

| | | | | | | | | | | Maint | enanc | e Phas | e | | | | | | | | Exte<br>Phas | nsion<br>se | | ts.y | <b>N</b> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ī. | /isit a | | | | | | | | | | | | Week | | | | | | | | | | | ssmen | w-up |
| Procedure | Screening Visit a | Day 1 | Week 4A (Oral<br>Lead-in Only) <sup>b</sup> | Week 4B | ∞ | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W After<br>Week 100 | Q8W After<br>Week 96 | 152 | Withdrawal Assessments.y | Long-Term Follow-up <sup>z</sup> |
| Fasting Lab Assessment: Glucose, Cholesterol (Total, HDL and LDL) and Triglycerides <sup>n</sup> | | Х | | | | | | | | | | | | | X | | | | Х | | | | Х | X | |
| Hepatitis B (HBsAg), Anti-HBc, and Anti- HBsAG, Hepatitis C (anti-HCV Ab) PT/PTT/INR | X | X | | | | | | | | | | | | | | | | | | | | | | | |
| PBMCs <sup>p</sup> | Λ | X | | | | | | | | | | | | | X | | | | X | | | | X | X | |
| Genetics<br>sample <sup>q</sup> | | Х | | | | | | | | | | | | | | | | | | | | | | | |
| PK sampling <sup>r</sup> (S)=Storage only | | | | Х | Х | S | Х | S | Х | S | Х | S | Х | S | X | s | S | S | X | S | | | Х | Х | s |

| | | | | | | | | | | Main | tenanc | e Phas | | | | | | | | | Exte<br>Phas | nsion<br>se | | ts.y | z |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <u> 5</u> | 'isit a | | | | | | | | | | | | Week | | | | | | | | | | | ssmen | dn-w |
| Procedure | Screening Visit a | Day 1 | Week 4A (Oral<br>Lead-in Only) <sup>b</sup> | Week 4B | ∞ | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W After<br>Week 100 | Q8W After<br>Week 96 | 152 | Withdrawal Assessments. <sup>y</sup> | Long-Term Follow-up z |
| Oral CAB<br>and Oral<br>RPV<br>Dispensation <sup>8</sup> | | X | Х | | | | | | | | | | | | | | | | | | | | | | |
| IP<br>accountability<br>(Pill Counts) <sup>S</sup> | | | Х | Х | | | | | | | | | | | | | | | | | | | | | |
| IM treatment<br>administratio<br>n when<br>transitioning<br>from SOC <sup>t</sup> | | | | X | х | X | X | X | X | x | X | x | X | X | Х | Х | Х | Х | Х | X | Х | X | X | | |
| IM treatment<br>administration<br>when<br>transitioning<br>from CAB +<br>RPV LA Q4W | | X | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х | Х | Х | Х | Х | Х | Х | Х | | |
| | | | | | | - | - | - | | Pat | ient R | eporte | d Out | comes | u | - | | | | - | - | - | - | | |
| HAT-QoL<br>(short-form) | | X | | | | | | | X | | | | | | X | | | | | | | | | X | |
| HIV TSQs<br>HIV TSQc v | | X | | | | | | | X | | | | | | X | | | | | | | | X | X | |
| ACCEPT | | X | | | | | | | X | | | | | | X | | | | | | | | X | X | |

| | | | | | | | | | | Maint | enanc | e Phas | | | | | | | | | Exte<br>Phas | nsion<br>se | | its.y | z |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| re | Visit a | | | | | | | | | | | | Week | | | | | | | | | | | Assessments. | |
| Procedure | Screening \ | Day 1 | Week 4A (Oral<br>Lead-in Only) <sup>b</sup> | Week 4B | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W After<br>Week 100 | Q8W After<br>Week 96 | 152 | Withdrawal Asse | Long-Term Follow-up |
| Reason for<br>Switch or<br>Reason for<br>continuation w | | Х | | | | | | | | | | | | | | | | | | | | | | | |
| Preference<br>Questionnaires | | | | | | | | | | | | | | | Xx | | | | | | | | Xaa | X | |
| PIN | | | | | X | | | | X | | | | | | X | | | | | | | | X | X | |

- a. Complete all Screening assessments within 35 days. Participants may begin the Maintenance Phase as soon as all Screening assessments are complete. Participants may be rescreened once and will be assigned a new participant number. Participants transitioning from the 201585 (ATLAS) study must reach ATLAS Week 48 (at minimum) prior to initiating Screening procedures for ATLAS-2M and must reach ATLAS Week 52 (at minimum) prior to randomization in ATLAS-2M.
- b. Visits Week 4a is part of the CAB + RPV Oral Lead-in period and is required only for participants transitioning from current SOC to CAB LA + RPV LA.
- c. Confirmation of eligibility to continue the Maintenance Phase and eligibility to enter the Extension Phase.

AEs or lab abnormalities at the last on-study visit. This visit may be conducted by telephone.

- d. Collect full routine medical history plus (report at Baseline visit): HIV risk factors (may be collected at a later study visit), cardiovascular risk factors (assessments include smoking status and history, family history of cardiac events), recent [≤6 months] illicit drug use, intravenous drug use, gastrointestinal disease, metabolic, psychiatric, renal, bone, and neurologic disorders.
- e. Physical exams should be conducted as part of normal routine clinical care. Medical assessments include any decisions the study staff must make for participants management and/or care of participant.
- f. Height collected at Baseline Day 1 only.
- g. Measure vital signs after about 5 minutes of rest in a semi-supine position.
- h. A 12-lead ECG will be performed after resting in a semi-supine position for at least 5 minutes. ECGs will be performed pre-dose. For participants transitioning from ATLAS, the pre-dose Week 48 ECG can also serve as the ATLAS-2M Screening ECG. ECG pre-dose will be performed in triplicate at

- Day 1. A 2-hour post-dose ECG will also be performed at Days 1 and Week 48 for participants receiving CAB LA + RPV LA with an allowable window of ±30 minutes.
- i. Only SAEs related to study participation or to a concomitantly administered ViiV/GSK product will be collected between obtaining informed consent and administration of study drug at Day 1.
- j. On Day 1, the eC-SSRS is to be administered prior to randomization. The eC-SSRS will preferably be completed at the beginning of the visit following administration of other PROs required prior to injections. The eC-SSRS is not required during the Withdrawal visit if withdrawal occurs during the Extension Phase.
- k. Women of childbearing potential only. SR=serum, UR=urine. Pregnancy events will be captured starting at Day 1 following initial exposure to study drug. Urine pregnancy test performed at Day 1 prior to administration of study drug, at Week 4B, and at study visits when other blood draws are not required in order to limit needle sticks. Serum pregnancy test can substitute for urine pregnancy test if locally required but must be appropriately timed to confirm pregnancy status prior to randomization and first IM administration.
- l. Week 48, Week 96 and Week 152 HIV-1 RNA retest (within 4 weeks) for results > 50 c/mL will be captured as unscheduled visit. Plasma for storage samples will be used for possible future analyses.
- m. A morning specimen is preferred. To assess biomarkers: urine albumin/creatinine ratio; urine protein/creatinine ratio; and urine phosphate. Urine phosphate results from visit 4a are not required by protocol to inform the safety review at visit 4b prior to receipt of initial CAB LA + RPV LA injections.
- n. An overnight fast is preferred; however, a minimum of a 6-hour fast is acceptable.
- o. Only collect if the Withdrawal visit occurs at Week 48, Week 96 or Week 152.
- p. Whole blood/PBMC collection samples may be used for virologic analyses. PBMCs will be collected at baseline Day 1, Week 48, Week 96, Week 152 or Withdrawal if prior to Week 152.
- q. Genetics sample should be collected only for patients who did not participate in the 201585(ATLAS) study (sample was previously collected and stored). Informed consent for genetic research must be obtained before sample collection. Sample may be collected at any visit after signing informed consent, but preferably at the Day 1 visit.
- r. One blood sample for CAB and RPV each to be collected at each PK timepoint. At Day 1, for participants from the ATLAS Q4W arm, PK samples are to be collected pre-dose relative to IM administration. At Week 4B, for participants randomized from SOC, Pre dose PK samples are to be collected: AFTER review of the PK diary to ensure that the samples are taken 20/28 hours after previous oral dose (diaries to be given at *Day 1 or W4a*); PRIOR to the final oral dose of CAB + RPV; PRIOR to the first IM injection.
- s. Only for Participants entering CAB + RPV Oral Treatment
- t. Participants switching to CAB LA + RPV LA will take final dose of oral lead-in regimen in the clinic at the Week 4B visit and begin injections. If possible, injections should be spaced approximately 2 cm from one another and from the site of any previous injection and or any injection site reaction. Bring RPV LA to approximately room temperature prior to injecting. Time and location of injection (right or left) as well as needle length used will be collected in the eCRF. The first injection can be performed as soon as central lab results become available and safety parameters are reviewed.

- u. All Patient Report Questionnaires/Surveys will be administered via paper instrument at the beginning of the visit before any other assessments are conducted and prior to administration of the eC-CSSRS. Conduct questionnaires/surveys at Withdrawal only if occurring at or prior to Week 152.
- v. The HIV-TSQc is to be administered to all participants transitioning from ATLAS and new participants transitioning from oral SOC. For participants transitioning from ATLAS, the version of the HIV-TSQc instrument to be administered will be based on the initial randomization arm at ATLAS Day 1.
- w. For patients randomized to oral SOC at Day 1 in ATLAS or new patients on SOC, the reasons for willingness to switch ART will be assessed at Day 1. For patients randomized to CAB LA + RPV LA Q4W in ATLAS, the reasons for willingness to continue long-acting ART in ATLAS-2M will be assessed at Day 1.
- x. Preference Questionnaire will be administered to all participants.
- y. Refer to Section 5.5 of the protocol for additional information on performing withdrawal assessments. HIV-1 RNA will be collected as Storage sample only if withdrawal assessments coincide with Week 52 or Week 100 or Week 156 (as per Section 5.5)
- z. Participants receiving one or more injections with CAB LA and/or RPV LA will be assessed with clinic visits at months 3, 6, 9 and 12 during the Long-Term Follow-Up Phase
- aa. Preference at Week 152 will be administered only to participants who received oral bridging during the Maintenance and/or Extension Phases

Note: BP – Blood pressure, HR – Heart Rate, HDL – High Density Lipoprotein, LDL – Low Density Lipoprotein, PT Prothrombin Time, PTT Partial Thromboplastin Time, INR International normalized ratio
## 15.2.2. Protocol Defined Schedule of Events for Q8W Arm in Main Study

| | æ | | | | | | | | Ma | intena | nce Pl | hase | | | | | | | | Exter<br>Phas | nsion<br>e | | dn-w |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| lure | Visit | | | | | | | | | | W | eek | | | | | | | | | | | Follor |
| Procedure | Screening Visit | Day 1 | Week 4A<br>Oral lead-in | Week 4B<br>(Oral lead-in<br>ONLY) b | × | 6 | 16 | 24 | 32 | 40 | 41 | 48 | 99 | 64 | 72 | 80 | 88 | 96 | 100 | Q8W After<br>Week 96 | 152 | Withdrawal | Long-Term Follow-up |
| Written<br>informed<br>consent | X | | | | | | | | | | | | | | | | | | | | | | |
| Eligibility<br>Verification<br>(Inclusion/<br>Exclusion<br>Criteria) | X | | xc | | | | | | | | | | | | | | | xc | | | | | |
| Randomization | | X | | | | | | | | | | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | | | | | | | | | | |
| Medical<br>History <sup>d</sup> | X | | | | | | | | | | | | | | | | | | | | | | |
| Cardiovascular<br>risk assessment <sup>d</sup> | X | X | | | | | | | | | | | | | | | | | | | | | |
| Medication<br>History/ Prior<br>ART history | X | | | | | | | | | | | | | | | | | | | | | | |
| Syphilis<br>serology +<br>reflex Rapid<br>Plasma Reagin<br>(RPR) | X | X | | | | | | | | | | | | | | | | | | | | | |
| Symptom<br>Directed<br>Physical Exam<br>and Medical<br>Assessment <sup>c</sup> | X | X | X | X | Х | х | х | х | х | х | X | X | X | X | Х | Х | X | X | х | Х | X | X | х |

| | e , | | | | | | | | Ma | intena | nce P | hase | | | | | | | | Exte<br>Phas | nsion<br>e | | dn-w |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| lure | Visi | | | | | | | | | | w | eek | | | | | | | | | | <b>.</b> | Follo |
| Procedure | Screening Visit | Day 1 | Week 4A<br>(Oral lead-in | Week 4B<br>(Oral lead-in<br>ONLY) b | ∞ | 6 | 16 | 24 | 32 | 40 | 41 | 48 | 99 | 64 | 72 | 80 | 88 | 96 | 100 | Q8W After<br>Week 96 | 152 | Withdrawal | Long-Term Follow-up |
| Weight, Height<br>and BMI <sup>f</sup> | | X | | | | | | | | | | X | | | | | | Х | | | X | Х | |
| Vital Signs<br>(BP, HR,<br>Temperature) <sup>g</sup> | X | X | | | | | | | | | | X | | | | | | Х | | | X | X | |
| 12-lead ECG h<br>(triplicate at Day 1<br>pre-dose) | Х | X | | | | | | | | | | X | | | | | | Х | | | Х | Х | |
| CDC HIV-1<br>stage | X | X | | | | | | | | | | | | | | | | | | | | | |
| HIV Associated<br>Conditions | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| AEs, SAEs,<br>Concomitant<br>Medications | xi | X | X | X | X | X | X | X | X | X | X | X | Х | Х | Х | X | X | X | X | X | X | X | x |
| ISR Assessment<br>for IM injection | | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Columbia<br>Suicide Severity<br>Rating Scale<br>(eC-SSRS) <sup>j</sup> | Х | Х | | X | х | | х | Х | Х | Х | | Х | Х | X | Х | Х | X | Х | | | | Х | |
| Clinical<br>chemistry and<br>Hematology | X | X | X | X | X | | X | X | X | X | | X | X | Х | X | X | X | X | X | X | X | X | X |
| Pregnancy<br>Testing <sup>k</sup> | S | U | S | U | S | | S | S | S | S | | S | S | S | S | S | S | S | S | S | S | S | S |

| | æ | | | | | | | | Ma | intena | ınce Pl | hase | | | | | | | | Exter<br>Phas | nsion<br>e | | dn-w |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| dure | y Visit | | | | | | | | | | W | eek | | | | | | | | | | ν. | Follo |
| Procedure | Screening Visit | Day 1 | Week 4A<br>Oral lead-in | Week 4B<br>(Oral lead-in<br>ONLY) b | ∞ | 6 | 16 | 24 | 32 | 40 | 41 | 48 | 99 | 64 | 72 | 80 | 88 | 96 | 100 | Q8W After<br>Week 96 | 152 | Withdrawal | Long-Term Follow-up |
| HIV-1 RNA and<br>sample for<br>storage (S) <sup>1</sup> | X | X | | X | X | | X | X | X | X | | X | X | X | X | X | X | X | S | X | X | X | X |
| CD4+ cell count | X | X | | X | X | | X | X | X | X | | X | X | X | X | X | X | X | X | X | X | X | X |
| CD8+ cell count | | X | | | | | | X | | | | X | | | | | | X | | | X | X | |
| Urinalysis <sup>m</sup> | | X | X | | | | | X | | | | X | | | | | | X | | | X | X | |
| Fasting Labs<br>Glucose,<br>Cholesterol<br>(Total, HDL<br>and LDL) and<br>Triglycerides <sup>n</sup> | | Х | | | | | | | | | | X | | | | | | X | | | X | Xº | |
| Hepatitis B<br>(HBsAg), Anti-<br>HBc, and Anti-<br>HBsAG,<br>Hepatitis C<br>(anti-HCV Ab) | Х | | | | | | | | | | | | | | | | | | | | | | |
| PT/PTT/INR | X | X | | | | | | | | | | | | | | | | | | | | | |
| PBMCs <sup>p</sup> | | X | | | | | | | | | | X | | | | | | X | | | X | X | |
| Genetics sample | | X | | | | | | | | | | | | | | | | | | | | | |

| | e 1 | | | | | | | | Ma | intena | ınce P | hase | | | | | | | | Exte<br>Phas | nsion<br>e | | dn-w |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| lure | Visi | | | | | | | | | | W | eek | | | | | | | | | | >. | Follo |
| Procedure | Screening Visit | Day 1 | Week 4A<br>Oral lead-in | Week 4B<br>(Oral lead-in<br>ONLY) b | œ | 6 | 16 | 24 | 32 | 40 | 41 | 48 | 99 | 64 | 72 | 80 | 88 | 96 | 100 | Q8W After<br>Week 96 | 152 | Withdrawal | Long-Term Follow-up |
| PK sampling<br>when<br>transitioning | | | | Х | X | X | X | X | Х | X | X | X | S | S | S | S | S | X | S | | Х | X | S |
| from SOC r<br>(S)=Storage<br>only | | | | | | | | | | | | | | | | | | | | | | | |
| PK sampling<br>when<br>transitioning<br>from CAB +<br>RPV Q4W <sup>r</sup><br>(S)=Storage<br>only | | X | | | X | х | х | Х | х | х | х | х | S | S | S | S | S | Х | S | | х | X | s |
| Oral CAB and<br>Oral RPV<br>Dispensation <sup>8</sup> | | X | Х | | | | | | | | | | | | | | | | | | | | |
| IP<br>accountability<br>(Pill Counts) | | | X | X | | | | | | | | | | | | | | | | | | | |
| IM treatment<br>administration<br>when<br>transitioning<br>from SOC <sup>t</sup> | | | | Х | X | | X | X | X | X | | X | X | X | X | X | X | X | | X | Х | | |

| | e , | | | | | | | | Ma | ainten: | mce P | hase | | | | | | | | Phas | nsion<br>e | | OII-M |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| dure | y Visi | | | | | | | | | | W | eek | | | | | | | | | | <b>&gt;</b> , | Follo |
| Procedure | Screening Visit | Day 1 | Week 4A<br>(Oral lead-in | Week 4B<br>(Oral lead-in<br>ONLY) b | * | 6 | 16 | 24 | 32 | 40 | 41 | 48 | 99 | 64 | 72 | 80 | 88 | 96 | 100 | Q8W After<br>Week 96 | 152 | Withdrawal | Long-Term Follow-up |
| IM treatment<br>administration<br>when<br>transitioning<br>from CAB +<br>RPV Q4W | | х | | | х | | х | х | х | х | | х | х | х | х | х | х | х | | х | х | | |
| | | | | | | | | | Pati | ent Re | porte | 1 Oute | omes t | | | | | | | | | | _ |
| HAT-QoL<br>(short-form) | | X | | | | | | Х | | | | X | | | | | | | | | | X | |
| HIV TSQs | | X | | | | | | X | | | | X | | | | | | | | | X | X | |
| HIV TSQc V | | | | | | | | | | | | X | | | | | | | | | | X | |
| ACCEPT | | Х | | | | | | Х | | | | Х | | | | | | | | | Х | Х | П |
| Reason for<br>Switch or<br>Reason for<br>continuation W | | x | | | | | | | | | | | | | | | | | | | | | |
| Preference<br>Questionnaires | | | | | | | | | | | | Xx | | | | | | | | | Xaa | X | Ī |
| PIN | | | | | Х | | | Х | | | | Х | | | | | | | | | X | X | |

Safety Follow Up Visit: Conduct approximately 4 weeks after the last dose of IP. Required only if the participant has ongoing AEs or lab abnormalities at the last on-study visit. This visit may be conducted by telephone.

- a. Participants may be rescreened once and will be assigned a new participant number. Participants transitioning from the 201585 (ATLAS) study must reach ATLAS Week 48 (at minimum) prior to initiating Screening procedures for ATLAS-2M and must reach ATLAS Week 52 (at minimum) prior to randomization in ATLAS-2M.
- b. Visits Weeks 4A and 4B are part of the CAB + RPV Oral Lead-in period and are required only for participants transitioning from current SOC to CAB LA + RPV LA.
- c. Confirmation of eligibility to continue the Maintenance Phase, and eligibility to enter the Extension Phase.

- d. Collect full routine medical history plus (report at Baseline visit): HIV risk factors (may be collected at a later study visit), cardiovascular risk factors (assessments include smoking status and history, family history of cardiac events), recent [≤6 months] illicit drug use, intravenous drug use, gastrointestinal disease, metabolic, psychiatric, renal, bone, and neurologic disorders.
- e. Physical exams should be conducted as part of normal routine clinical care. Medical assessments include any decisions the study staff must make for participants management and/or care of participant.
- f. Height collected at Baseline Day 1 only.
- g. Measure vital signs after about 5 minutes of rest in a semi-supine position.
- h. A 12-lead ECG will be performed after resting in a semi-supine position for at least 5 minutes. ECGs will be performed pre-dose. For participants transitioning from ATLAS, the pre-dose Week 48 ECG can also serve as the ATLAS-2M Screening ECG. ECG pre-dose will be performed in triplicate at Day 1. A 2-hour post-dose ECG will also be performed at Days 1 and Week 48 for participants receiving CAB LA + RPV LA with an allowable window of ± 30 minutes.
- i. Only SAEs related to study participation or to a concomitantly administered ViiV/GSK product will be collected between obtaining informed consent and administration of study drug at Day 1.
- j. On Day 1, the eC-SSRS is to be administered prior to randomization. The eC-SSRS will preferably be completed at the beginning of the visit following administration of other PROs required prior to injections. The eC-SSRS is not required during the Withdrawal visit if withdrawal occurs during the Extension Phase.
- k. Women of childbearing potential only. SR=serum, UR=urine. Pregnancy events will be captured starting at Day 1 following initial exposure to study drug. Serum pregnancy test can substitute for urine pregnancy test if locally required but must be appropriately timed to confirm pregnancy status prior to randomization and first IM administration.
- l. Week 48, Week 96 and Week 152 HIV-1 RNA retest (within 4 weeks) for results > 50 c/mL will be captured as unscheduled visit. Plasma for storage samples will be used for possible future analyses.
- m. A morning specimen is preferred. To assess biomarkers: urine albumin/creatinine ratio; urine protein/creatinine ratio; and urine phosphate. Urine phosphate results from visit 4a are not required by protocol to inform the safety review at visit 4b prior to receipt of initial CAB LA + RPV LA injections.
- n. An overnight fast is preferred; however, a minimum of a 6-hour fast is acceptable.
- o. Only collect if the Withdrawal visit occurs at Week 48, Week 96 or Week 152.
- p. Whole blood/PBMC collection samples may be used for virologic analyses. PBMCs will be collected at baseline Day 1, Week 48, Week 96, Week 152 or Withdrawal if prior to Week 152.
- q. Genetics sample should be collected only for patients who did not participate in the 201585(ATLAS) study (sample was previously collected and stored). Informed consent for genetic research must be obtained before sample collection. Sample may be collected at any visit after signing informed consent, but preferably at the Day 1 visit.
- r. One blood sample for CAB and RPV each to be collected at each PK timepoint. At Day 1, for participant from the ATLAS Q4W arm, PK samples are to be collected pre-dose relative to IM administration. injection. At Week 4B, for participants randomized from SOC, Pre dose PK samples are to be collected: AFTER review of the PK diary to ensure that the samples are taken 20/28 hours after previous oral dose (diaries to be given at Day 1 or W4a); PRIOR to the final oral dose of CAB + RPV; and PRIOR to the first IM injection. At Week 9 and 41, the PK samples should be collected 3 to 10 days after the Week 8 and Week 40 visits, respectively.
- s. Only for Participants entering CAB + RPV Oral Treatment

- t. Participants switching to CAB LA + RPV LA will take final dose of oral lead-in regimen in the clinic at the Week 4B visit and begin injections. If possible, injections should be spaced approximately 2 cm from one another and from the site of any previous injection and or any injection site reaction. Bring RPV LA to approximately room temperature prior to injecting. Time and location of injection (right or left) as well as needle length used will be collected in the eCRF. The first injection can be performed as soon as central lab results become available and safety parameters are reviewed.
- u. All Patient Report Questionnaires/Surveys will be administered via paper instrument at the beginning of the visit before any other assessments are conducted and prior to administration of the eC-CSSRS. Conduct questionnaires/surveys upon Withdrawal only if occurring at or prior to Week 48
- v. The HIVTSQc is to be administered to all participants transitioning from ATLAS and new participants transitioning from oral SOC. For participants transitioning from ATLAS, the version of the HIV-TSQc instrument to be administered will be based on the initial randomization arm at ATLAS Day 1
- w. For patients randomized to oral SOC at Day 1 in ATLAS or new patients on SOC, the reasons for willingness to switch ART will be assessed at Day 1. For patients randomized to CAB LA + RPV LA Q4W in ATLAS, the reasons for willingness to continue long-acting ART in ATLAS-2M will be assessed at Day 1.
- x. Preference Questionnaire will be administered to all participants
- y. Refer to Section 5.5 of the protocol for additional information on performing withdrawal assessments. HIV-1 RNA will be collected as Storage sample only if withdrawal assessments coincide with Week 52 or Week 100 (as per Section 5.5)
- z. Participants receiving one or more injections with CAB LA and/or RPV LA will be assessed with clinic visits at months 3, 6, 9 and 12 during the Long-Term Follow-Up Phase
- aa. Preference at Week 152 will be administered only to participants who received oral bridging during the Maintenance and/or Extension Phases

Note: BP – Blood pressure, HR – Heart Rate, HDL – High Density Lipoprotein, LDL – Low Density Lipoprotein, PT Prothrombin Time, PTT Partial Thromboplastin Time, INR International normalized ratio

## 15.2.3. Protocol Defined Schedule of Events for Q4W Arm in Sub-study

| Procedure | <u>Gl</u> ı | ng Phase <sup>d</sup><br>ateal<br>astration | | Q4 | Thigh Injec | ction Phase <sup>d</sup><br>h administrat | tion_ | | | rn to Glu<br>Pha<br>Weekly <u>gl</u> | se <sup>d</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>(Week<br>-4) | Week -3 | Day1 | Week<br>1 | Week 4 | Week 8 | Week 12 | Week<br>13 | Week<br>16 | Week<br>17 | Week<br>20 | Week<br>24 |
| IM treatment administration <sup>i</sup> | X | | X | | X | X | X | | X | | X | |
| Written Inform<br>consent | x | | | | | | | | | | | |
| Eligibility Verification (Inclusion/Exclusio n criteria) | X | | | | | | | | | | | |
| Symptom directed<br>physical exam and<br>Medical<br>assessment <sup>a</sup> | x | | X | | X | X | X | | X | | X | x |
| Weight and BMI | | | X | | | | | | X | | | |

| Procedure | Glı | ng Phase <sup>d</sup><br>uteal<br>istration | | Q4 | Thigh Injed<br>Weekly <u>thig</u> | ction Phase <sup>d</sup><br>h administra | <u>tion</u> | | | rn to Glu<br>Pha<br>Weekly <u>g</u> l | sed | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>(Week | Week -3 | Day1 | Week<br>1 | Week 4 | Week 8 | Week 12 | Week<br>13 | Week<br>16 | Week<br>17 | Week<br>20 | Week<br>24 |
| | -4) | | | | | | | | | | | |
| Vital Signs, BP,<br>HR, temp <sup>b</sup> | X | | X | | | | | | X | | | |
| Smoking status | X | | | | | | | | | | | |
| 12-lead ECG <sup>c</sup> | X | | X | | | | | | X | | | |
| HIV associated conditions | X | X | X | X | X | X | X | X | X | X | X | X |
| AEs, SAEs,<br>concomitant<br>medications | х | X | X | X | X | X | X | X | X | X | X | X |
| ISR assessments<br>for IM injections | X | X | X | X | X | X | X | X | X | X | X | X |
| Clinical Chemistry<br>and Hematology | X | | X | | X | X | X | | X | | | X |
| Pregnancy Testing,<br>SERUM <sup>e</sup> | s | | s | | s | s | s | | s | | U | S |

| Procedure | Glı | ng Phase <sup>d</sup><br>uteal<br>istration | | Q4 | Thigh Injec | ction Phase <sup>d</sup><br>h administrat | tion_ | | | rn to Glu<br>Pha<br>Weekly <u>gl</u> | se <sup>d</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>(Week<br>-4) | Week -3 | Day1 | Week<br>1 | Week 4 | Week 8 | Week 12 | Week<br>13 | Week<br>16 | Week<br>17 | Week<br>20 | Week<br>24 |
| HIV-1 RNA and<br>sample for storage<br>(S) | X | | X | | X | X | X | | X | | | X |
| CD4+ cell count | X | | X | | X | X | X | | X | | | X |
| CD8+ cell count | | | X | | | | | | X | | | |
| Urinalysis <sup>f</sup> | | | X | | | | | | X | | | |
| Fasting lab assessments: Glucose, Cholesterol (Total, HDL and LDL) and triglyceridesg | | | X | | | | | | х | | | |
| PBMC for storage | | | X | | | | | | | | | |

| Procedure | Glu | ng Phase <sup>d</sup><br>uteal<br>istration | | Q4 | Thigh Injec | ction Phase <sup>d</sup><br>h administra | <u>tion</u> | | | rn to Glu<br>Pha<br>Weekly <u>g</u> l | se <sup>d</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>(Week<br>-4) | Week -3 | Day1 | Week<br>1 | Week 4 | Week 8 | Week 12 | Week<br>13 | Week<br>16 | Week<br>17 | Week<br>20 | Week<br>24 |
| | | | | PK | Sample colle | ection <sup>j</sup> | | | | | | |
| Pre dose PK<br>sampling | X | | X | | X | X | X | | X | | | |
| 2h Post dose PK sampling | | | X | | X | X | X | | | | | |
| Post dose PK<br>sampling (~Cmax) | | X | | X | | | | X | | X | | |
| | | | | | PROsl | | | | | | | |
| HIVTSQc | | | | | | | | | X <sup>k</sup> | | | |
| HIVTSQs | | | X | | | | | | Xk | | х | |
| NRSh | X | X | X | X | | | X | X | X | X | | |
| Preference Thigh inj. vs Gluteal inj. | | | | | | | X | | | | х | |

- a. Physical exams should be conducted as part of normal routine clinical care. Medical assessments include any decisions the study staff must make for participants management and/or care of participant.
- b. Measure vital signs after about 5 minutes of rest in a semi-supine position.
- c. A 12-lead ECG will be performed after resting in a semi-supine position for at least 5 minutes. ECGs will be performed pre-dose. A 2-hour post dose ECG will also be performed at sub-study Day1 visit.
- d. All injection visits during the sub-study should kept to the same projected visit schedule as in the parent study.
- e. Women of childbearing potential only. SR=serum, UR=urine. Urine pregnancy test can be performed at study visits when other blood draws are not required in order to limit needle sticks.
- f. A morning specimen is preferred.
- g. An overnight fast is preferred; however, a minimum of a 6-hour fast is acceptable.
- h. Should be collected 30 to 60 minutes post injection
- Week 24 IM administration will not be considered part of the sub-study assessments. The IM administration at W24 and any assessments completed after IM administration at this visit will be considered part of the parent study.
- j. PK window allowed for sample collection: For 1-week post dose sample (3 to 10 days post dose), for 4-week post dose sample (+-7 days) and for 2-hours post dose samples (±1 hour)
- k. At Week 16, HIVTSQs should be administered before HIVTSQc.
- All Patient Report Questionnaires/Surveys except NRS will be administered via paper instrument (in exceptional circumstances the questionnaires could be completed via telephonic interview, please refer to COVID19 appendix for additional details) at the beginning of the visit before any other assessments are conducted.

Note: There is a typo in the schedule of events table where weight and BMI will be collected at Week -4 visit instead of Day 1 visit.

### 15.2.4. Protocol Defined Schedule of Events for Q8W Arm in Sub-study

| Procedure | | ning Phas | | | | | tion phase <sup>d</sup><br>administratio | on_ | | | Gluteal Inje<br>ekly <u>glutea</u> | ection Phase <sup>d</sup><br>l admin. |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>(Week -8) | Week<br>-7 | Week<br>-4 | Day1 | Week<br>1 | Week<br>4 | Week 8 | Week<br>9 | Week<br>12 | Week 16 | Week<br>17 | Week 24 |
| IM treatment<br>administration <sup>i</sup> | X | | | X | | | X | | | X | | |
| Written Inform<br>consent | X | | | | | | | | | | | |
| Eligibility<br>Verification<br>(Inclusion/Exclusion<br>criteria) | X | | | | | | | | | | | |
| Symptom directed<br>physical exam and<br>Medical assessment <sup>a</sup> | X | | | X | | | X | | | X | | X |
| Weight and BMI | X | | | | | | | | | X | | |
| Vital Signs, BP, HR,<br>temp <sup>b</sup> | X | | | X | | | | | | X | | |
| Smoking status | X | | | | | | | | | | | |
| 12-lead ECG <sup>c</sup> | X | | | X | | | | | | X | | |

| Procedure | | ning Phas<br>administra | | | | | tion phased<br>administration | on_ | | | Gluteal Inje<br>ekly <u>glutea</u> | ection Phased<br>l admin. |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>(Week -8) | Week<br>-7 | Week<br>-4 | Day1 | Week<br>1 | Week<br>4 | Week 8 | Week<br>9 | Week<br>12 | Week 16 | Week<br>17 | Week 24 |
| HIV associated conditions | x | x | x | x | X | X | X | x | X | X | X | X |
| AEs, SAEs,<br>concomitant<br>medications | X | X | х | X | x | X | X | х | х | X | X | X |
| ISR assessments for IM injections | X | X | X | X | X | X | X | X | X | X | X | X |
| Clinical Chemistry<br>and Hematology | X | | | X | | | X | | | X | | X |
| Pregnancy Testing,<br>SERUM <sup>e</sup> | s | | | s | | | s | | | s | | s |
| HIV-1 RNA and<br>sample for storage (S) | X | | | X | | X | X | | Х | X | | X |
| CD4+ cell count | X | | | X | | | X | | | X | | X |
| CD8+ cell count | X | | | X | | | | | | X | | |
| Urinalysis <sup>f</sup> | X | | | X | | | | | | X | | |
| Fasting lab<br>assessments: Glucose,<br>Cholesterol (Total, | X | | | X | | | | | | X | | |

| Procedure | | ning Phas | | | | | tion phased<br>administratio | <u>on</u> | | | Gluteal Inje<br>ekly <u>glutea</u> | ection Phased<br>l admin. |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>(Week -8) | Week<br>-7 | Week<br>-4 | Day1 | Week<br>1 | Week<br>4 | Week 8 | Week<br>9 | Week<br>12 | Week 16 | Week<br>17 | Week 24 |
| HDL and LDL) and triglycerides <sup>g</sup> | | | | | | | | | | | | |
| PBMC for storage | | | | X | | | | | | | | |
| | | | | | PK s | samples <sup>j</sup> | | | | | | |
| Pre dose PK sampling | X | | | X | | | X | | | X | | |
| 2h Post dose PK sampling | | | | X | | | X | | | | | |
| Post dose PK<br>sampling (~Cmax) | | X | X | | X | X | | X | X | | X | |
| | | | | | P | ROsl | | • | | | | |
| HIVTSQc | | | | | | | | | | $\mathbf{X}^{\mathbf{k}}$ | | |
| HIVTSQs | | | | X | | | | | | $X^k$ | | X |
| NRSh | X | X | | X | X | | X | X | | X | X | |
| Preference Thigh inj.<br>vs Gluteal inj. | | | | | | | X | | | | | X |

- a. Physical exams should be conducted as part of normal routine clinical care. Medical assessments include any decisions the study staff must make for participants management and/or care of participant.
- Measure vital signs after about 5 minutes of rest in a semi-supine position.
- c. A 12-lead ECG will be performed after resting in a semi-supine position for at least 5 minutes. ECGs will be performed pre-dose. A 2-hour post dose ECG will also be performed at sub-study Day1 visit.
- All injection visits during the sub-study should kept to the same projected visit schedule as in the parent study.
- Women of childbearing potential only. SR=serum, UR=urine. Urine pregnancy test can be performed at study visits when other blood draws are not required
  in order to limit needle sticks.
- A morning specimen is preferred.
- g. An overnight fast is preferred; however, a minimum of a 6-hour fast is acceptable.
- Should be collected 30 to 60 minutes post injection
- Week 24 IM administration will not be considered part of the sub-study assessments. The IM administration at W24 and any assessments completed after IM administration at this visit will be considered part of the parent study.
- j. PK window allowed for sample collection: For 1-week post dose sample (3 to 10 days post dose), for 4-week post dose sample (+-7 days) and for 2-hours post dose samples (±1 hour)
- At Week 16, HIVTSQs should be administered before HIVTSQc.
- All Patient Report Questionnaires/Surveys except NRS will be administered via paper instrument (in exceptional circumstances the questionnaires could be completed via telephonic interview, please refer to COVID19 appendix for additional details) at the beginning of the visit before any other assessments are conducted.

#### 15.3. Appendix 3: Assessment Windows

#### 15.3.1. Definitions of Assessment Windows for Analyses

Laboratory data, vital signs, ECGs, health outcomes assessments, and genotypic/phenotypic data will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database.

In most cases the window around an assessment will include all dates from the midpoints between the target day and that of the previous and the proceeding visits. In general, the nominal target study day for week w is (7\*w)+1.

For parameters which are not scheduled to be assessed at particular visits, the all-inclusive assessment windows will still be used; however, data summaries will only report scheduled visits. Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

Prior to visit slotting, assessments are first assigned to a study phase (screening, maintenance, extension, sub-study screening, thigh injection, return to gluteal injection or long-term follow-up) based on the Tables in Section 15.4.1 and treatment state based on Section 15.4.2.

Maintenance phase assessments other than health outcome and PK are assigned based on the Study Day as shown in Table 8. Table 8 also includes visiting slotting for screening assessments. The analysis visits from Week 4 to Week 100 should be only applied to the assessments that are already assigned to Maintenance phase (on-treatment). Extension phase assessments other than health outcome and PK are assigned based on the Study Day as shown in Table 9. The analysis visits from Week 104 (except for Follow-up) in the Extension phase should be only applied to the assessments that are already assigned to Extension phase (on-treatment). The snapshot visits up to Week 152 during the Maintenance or Extension phase are assigned based on Study Day as shown in Table 10.

The sub-study assessments other than health outcome, PK and HIV-1 RNA are assigned analysis visits based on Study Day as shown in Table 11. The assessment visit windows for HIV-1 RNA data are defined in Table 12, and the snapshot windows for visits up to Sub-study Week 16 are defined in Table 13.

Long-term Follow-up phase assessments are assigned based on the LTFU study day as shown in **** The analysis visits in LTFU should be only applied to the assessments that are already assigned to LTFU phase regardless of treatment state. See Section 15.6.1, for derivation of Study Day and LTFU Study Day.

# 15.3.2. Definitions of Assessment Windows for Analyses other than Health Outcome and PK

 Table 8
 Assessment Windows for Screening and Maintenance Phase Data

| All Parameters | | | |
|---|---|---|---|
| except for where | Tarrest Official a David | A sealers to Matter doors | Analysis |
| noted <sup>[c]</sup> | Target Study Day | Analysis Window | Timepoint |
| | The study day of first record | Study Day ≤ 1 | Screening |
| | 1 | Last available recorded value up to<br>and including the Maintenance<br>treatment start date, excluding<br>post-dose ECG taken on the<br>Maintenance treatment start date | Baseline |
| ECG | 1 | Value taken post-dose on the<br>Maintenance treatment start date | Day 1 (Post Dose) |
| Urinalysis <sup>[a]</sup> | 29 | 2 ≤ Study Day ≤ 70 | Week 4 |
| | 29 | 2 ≤ Study Day ≤ 42 | Week 4 |
| | 57 | 43 ≤ Study Day ≤ 84 | Week 8 |
| | 113 | 85 ≤ Study Day ≤ 140 | Week 16 |
| Urinalysis <sup>[a]</sup> , CD8,<br>CD4/CD8 ratio | 169 | 141 ≤ Study Day ≤ 210 | Week 24 |
| | | 141 ≤ Study Day ≤ 196 | |
| | 225 | 197 ≤ Study Day ≤ 252 | Week 32 |
| | 281 | 253 ≤ Study Day ≤ 308 | Week 40 |
| Urinalysis <sup>[a]</sup> , fasting glucose, lipids <sup>[b]</sup> , CD8, CD4/CD8 ratio, weight, vital signs, ECG | 337 | 309 ≤ Study Day ≤ 378 | Week 48 |
| | | 309 ≤ Study Day ≤ 364 | |
| | 393 | 365 ≤ Study Day ≤ 420 | Week 56 |
| | 449 | 421 ≤ Study Day ≤ 476 | Week 64 |
| | 505 | 477 ≤ Study Day ≤ 532 | Week 72 |
| | 561 | 533 ≤ Study Day ≤ 588 | Week 80 |
| | 617 | 589 ≤ Study Day ≤ 644 | Week 88 |
| Urinalysis <sup>[a]</sup> , fasting<br>glucose, lipids <sup>[b]</sup> , CD8,<br>CD4/CD8 ratio, weight,<br>vital signs, ECG | se, lipids <sup>[b]</sup> , CD8, CD8 ratio, weight, al signs, ECG $645 \le Stu$ | | Week 96 |
| | | 645 ≤ Study Day ≤ min (Study Day of Nominal Week100 Visit -1, 700) | |

| All Parameters<br>except for where<br>noted <sup>[c]</sup> | Target Study Day | Analysis Window | Analysis<br>Timepoint |
|---|---|---|---|
| | 701 | min (Study Day of Nominal Week<br>100 Visit, 701) ≤ Study Day ≤<br>(Study Day of Nominal Week 100<br>Visit) | Week 100 |
| If a | participant permane | ently discontinued study treatment: | |
| | | For Participants on Q8W Arm: Date > max (Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1, Date of Last Injection + 63) | |
| | | For Participants on Q4W Arm: | Follow-up |
| NOTES | | Date > max (Date of Last Dose of<br>Oral Study Treatment (CAB+RPV<br>or SOC Bridging) + 1, Date of Last<br>Injection + 35) | |

- The nominal Week 100 visit refers to the Week 100 visit per eCRF.
- Follow-up will be derived only for participants who permanently discontinued study treatment.

  [a] **Urinalysis:** All parameters provided by the central laboratory under the category of urinalysis, including Urine Albumin/Creatinine, Urine Creatinine, Urine pH, Urine Protein/Creatinine, Urine Erythrocytes, Urine Specific Gravity, Urine Leukocytes, Urine Retinol Binding Protein, Urine Phosphate, Urine Creatinine.

  [b] **Lipids:** Cholesterol, HDL Cholesterol Direct, LDL Cholesterol Calculation, LDL Cholesterol Direct, Total

Cholesterol/HDL Cholesterol Ratio, Triglycerides [c] Analysis windows for parameters with sparse collection are noted.

Table 9 Assessment Windows for Extension Phase Data

| All Parameters except for where noted <sup>[d]</sup> | Target<br>Study Day | Analysis Window | Analysis Timepoint |
|---|---|---|---|
| | 729 | (Study Day of Nominal Week 100 Visit + 1) ≤ Study Day ≤ 756 | Week 104 <sup>[a]</sup> |
| | 785 | 757 ≤ Study Day ≤ 812 | Week 112 |
| | 841 | 813 ≤ Study Day ≤ 868 | Week 120 |
| | 897 | 869 ≤ Study Day ≤ 924 | Week 128 |
| | 953 | 925 ≤ Study Day ≤ 980 | Week 136 |
| | 1009 | 981 ≤ Study Day ≤ 1036 | Week 144 |
| Urinalysis <sup>[b]</sup> , fasting glucose, lipids <sup>[c]</sup> , CD8, CD4/CD8 ratio, weight, vital signs, ECG | 1065 | 1037 ≤ Study Day ≤ 1106 | Week 152 |
| | | 1037 ≤ Study Day ≤ 1092 | |

| All Parameters except for where noted[d] | Target<br>Study Day | Analysis Window | Analysis Timepoint |
|---|---|---|---|
| | 7*w + 1 | (7*w - 27) | Week w |
| | | ≤ Study Day ≤ (7*w + 28) | w = 160, 168, |
| | If a particip | pant permanently discontinued study trea | atment: |
| | | For participants on Q8W Arm: Date > max (Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1, Date of Last Injection + 63) | Follow up |
| | | For participants on Q4W Arm: Date > max (Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1, Date of Last Injection + 35) | Follow-up |

- The nominal Week 100 visit refers to the Week 100 visit per eCRF.
- Follow-up will be derived only for participants who permanently discontinued study treatment.
   [a] Assessments taken after Week 100 injection at the nominal Week 100 visit will be assigned to Week 104.
   Adverse events started on the same day as nominal Week 100 visit date will also be assigned to Week 104.
   [b] Urinalysis: All parameters provided by the central laboratory under the category of urinalysis, including Urine Albumin/Creatinine, Urine Creatinine, Urine PH, Urine Protein/Creatinine, Urine Erythrocytes, Urine Specific Gravity, Urine Leukocytes, Urine Retinol Binding Protein, Urine Phosphate, Urine Creatinine.
   [c] Lipids: Cholesterol, HDL Cholesterol Direct, LDL Cholesterol Calculation, LDL Cholesterol Direct, Total Cholesterol/HDL Cholesterol Ratio, Triglycerides
- [d] Analysis windows for parameters with sparse collection are noted.

Table 10 Assessment Windows for Summary of Snapshot Data Up to Week 152— Data Assigned to Maintenance or Extension Phase

| Snapshot Anal | | |
|---|---|---|
| (If no on-treatment viral load data in de | Analysis | |
| Default | Default Expanded +6 Week Upper Window <sup>a</sup> | |
| Last available recorded value up to and including the date of first Maintenance Phase dose of IP | Last available recorded value up to and including the date of first Maintenance Phase dose of IP | Baseline |
| 2 ≤ Study Day ≤ 42 | 2 ≤ Study Day ≤ 70 | Week 4 |
| $43 \le \text{Study Day} \le 84$ | 43 ≤ Study Day ≤ 98 | Week 8 |
| 85 ≤ Study Day ≤ 140 | 85 ≤ Study Day ≤ 154 | Week 16 |
| 141 ≤ Study Day ≤ 196 | 141 ≤ Study Day ≤ 210 | Week 24 |
| 197 ≤ Study Day ≤ 252 | 197 ≤ Study Day ≤ 266 | Week 32 |
| 253 ≤ Study Day ≤ 308 | 253 ≤ Study Day ≤ 322 | Week 40 |
| 295 ≤ Study Day ≤ 378 | 295 ≤ Study Day ≤ 378 | Week 48 |
| 365 ≤ Study Day ≤ 420 | 365 ≤ Study Day ≤ 434 | Week 56 |
| 421 ≤ Study Day ≤ 476 | 421 ≤ Study Day ≤ 490 | Week 64 |
| 477 ≤ Study Day ≤ 532 | 477 ≤ Study Day ≤ 546 | Week 72 |
| 533 ≤ Study Day ≤ 588 | 533 ≤ Study Day ≤ 602 | Week 80 |
| 589 ≤ Study Day ≤ 644 | 589 ≤ Study Day ≤ 658 | Week 88 |
| 631 ≤ Study Day ≤ 714 | 631 ≤ Study Day ≤ 714 | Week 96 |
| (Study Day of Nominal Week 100 Visit + 1) $\leq$ Study Day $\leq$ 756 | (Study Day of Nominal Week 100 Visit + 1) $\leq$ Study Day $\leq$ 770 | Week 104 |
| 757 ≤ Study Day ≤ 812 | 757 ≤ Study Day ≤ 826 | Week 112 |
| 813 ≤ Study Day ≤ 868 | 813 ≤ Study Day ≤ 882 | Week 120 |
| 869 ≤ Study Day ≤ 924 | 869 ≤ Study Day ≤ 938 | Week 128 |
| 925 ≤ Study Day ≤ 980 | 925 ≤ Study Day ≤ 994 | Week 136 |
| 981 ≤ Study Day ≤ 1036 | 981 ≤ Study Day ≤ 1050 | Week 144 |
| 1023 ≤ Study Day ≤ 1106 | 1023 ≤ Study Day ≤ 1106 | Week 152 |

- For post-baseline visits (i.e. Week 4 and afterwards), apply Snapshot analysis windows only to viral load data that is on-treatment (per Table 20) within the Maintenance Phase (per Table 18).
- An on-treatment viral load assessment may be assigned to more than one snapshot analysis window, e.g. on-treatment assessment taken on Study Day 300 will be in both Week 40 and Week 48.
- a. ± 6 Week window is always used at key analysis timepoints (Week 48, Week 96 and Week 152). For analysis timepoint of Week 24, if no viral load data in default window, expand to ± 6 Week window, i.e. (127 ≤ Study Day ≤ 210) in Week 24 IDMC and Week 24 Analyses, and expand upper bound to +6 weeks in all other analyses.

Table 11 Assessment Windows for Sub-study Baseline, Thigh Injection Phase and Return to Gluteal Injection Phase Data (Excluding HIV-1 RNA Data)

| All Parameters<br>except for where<br>noted <sup>[c]</sup> | Target Study<br>Day | Analysis Window | Analysis Timepoint |
|---|---|---|---|
| | 7*w + 1 | Last available recorded value up to<br>and including the date of first thigh<br>injection, excluding post-dose ECG<br>taken on the date of first thigh injection | Sub-study<br>Baseline <sup>[d]</sup> |

| All Parameters<br>except for where<br>noted <sup>[c]</sup> | Target Study<br>Day | Analysis Window | Analysis Timepoint |
|---|---|---|---|
| ECG | 7*w + 1 | Value taken post-dose on the date of first thigh injection | Sub-study Day 1<br>(Post Dose) |
| Injection Site Reaction | 7*w + 1 | First thigh injection date≤Study Day≤ max (7*w + 1, First thigh injection date +1) | Sub-study Day 1 |
| | 7*(w+8) + 1 | Min $(7*w + 2$ , first thigh injection date+1) $\leq$ Study Day $\leq$ 7*(w+12) | Sub-study Week 8 |
| Urinalysis <sup>[a]</sup> , fasting glucose, lipids <sup>[b]</sup> , CD8, CD4/CD8 ratio, weight, vital signs, ECG | 7*(w+16) + 1 | $7*(w+12) + 1 \le Study Day \le 7*(w+22)$ | Sub-study Week 16 |
| | | $7*(w+12) + 1 \le Study Day \le 7*(w+20)$ | |
| | 7*(w+24) + 1 | $7*(w+20) + 1 \le Study Day \le 7*(w+28)$ | Sub-study Week 24 |
| If a | participant per | manently discontinued study treatment | |
| | | For Participants on Q8W Arm: Date > max (Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1, Date of Last Injection + 63) | Fall |
| | | For Participants on Q4W Arm: | Follow-up |
| | | Date > max (Date of Last Dose of Oral<br>Study Treatment (CAB+RPV or SOC<br>Bridging) + 1, Date of Last Injection +<br>35) | |

- The "w" in the target study day calculation refers to the corresponding week number in Extension for the planned Sub-study Day 1 visit. For example, if a participant's last planned Extension phase visit before entering the Sub-study is Week 192, the "w" would be 200 if the participant is on Q4W arm and would be 208 if the participant is on Q8W arm.
- Follow-up will be derived only for participants who permanently discontinued study treatment.
- Sub-study Day 1 (Post Dose), Sub-study Week 8 and Sub-study Week 16 visits are Thigh Injection phase visits, Sub-study Week 24 is Return to Gluteal Injection phase visit.
- [a] **Urinalysis:** All parameters provided by the central laboratory under the category of urinalysis, including Urine Albumin/Creatinine, Urine Creatinine, Urine pH, Urine Protein/Creatinine, Urine Erythrocytes, Urine Specific Gravity, Urine Leukocytes, Urine Retinol Binding Protein, Urine Phosphate, Urine Creatinine.
- [b] **Lipids**: Cholesterol, HDL Cholesterol Direct, LDL Cholesterol Calculation, LDL Cholesterol Direct, Total Cholesterol/HDL Cholesterol Ratio, Triglycerides
- [c] Analysis windows for parameters with sparse collection are noted.
- [d] The values considered for deriving Sub-study Baseline value include both Extension phase and sub-study data.

Table 12 Assessment Windows for Sub-study Baseline, Thigh Injection Phase and Return to Gluteal Injection Phase HIV-1 RNA Data

| Phase | Target Study<br>Day | Analysis Window | Analysis Timepoint |
|---|---|---|---|
| Sub-study Screening | 7*w + 1 | Last available recorded value up to<br>and including the date of first thigh<br>injection | Sub-study<br>Baseline <sup>[a]</sup> |
| | 7*(w+4) + 1 | Min $(7*w + 2$ , first thigh injection date $+1) \le $ Study Day $\le 7*(w+6)$ | Sub-study Week 4 |
| Thigh Injection | 7*(w+8) + 1 | $7*(w+6) + 1 \le Study Day \le 7*(w+10)$ | Sub-study Week 8 |
| | 7*(w+12) + 1 | $7*(w+10) + 1 \le Study Day \le 7*(w+14)$ | Sub-study Week 12 |
| | 7*(w+16) + 1 | $7*(w+14) + 1 \le Study Day \le 7*(w+20)$ | Sub-study Week 16 |
| Return to Gluteal<br>Injection | 7*(w+24) + 1 | $7*(w+20) + 1 \le Study Day \le 7*(w+28)$ | Sub-study Week 24 |
| If a participant permanently discontinued study treatment: | | | |
| | | For Participants on Q8W Arm: Date > max (Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1, Date of Last Injection + 63) | Follow-up |
| | | For Participants on Q4W Arm: | i ollow-up |
| | Date > max (Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1, Date of Last Injection + 35) | | |

- The "w" in the target study day calculation refers to the corresponding week number in Extension for the planned Sub-study Day 1 visit. For example, if a participant's last planned Extension phase visit before entering the Sub-study is Week 192, the "w" would be 200 if the participant is on Q4W arm and would be 208 if the participant is on Q8W arm.
- Follow-up will be derived only for participants who permanently discontinued study treatment.

  [a] The values considered for deriving Sub-study Baseline value include both Extension phase and sub-study data.

Table 13 Assessment Windows for Summary of Snapshot Data Up to Week 16 in Sub-study— Data Assigned to Thigh Injection Phase

| Snapshot A (If no on-treatment viral load da w | | |
|---|---|---|
| Default | Analysis Timepoint | |
| Last available recorded value up to and including the date of first thigh injection Last available recorded value up to and including the date of first thigh injection | | Sub-study Baseline <sup>[a]</sup> |
| $Min(7^*w + 2, first thigh injection date+1) \le Study Day \le 7^*(w+6)$ $Min(7^*w + 2, first thigh injection date+1) \le Study Day \le 7^*(w+10)$ | | Sub-study Week 4 |
| $7*(w+6) + 1 \le Study Day \le 7*(w+10)$ | $7*(w+6) + 1 \le Study Day \le 7*(w+14)$ | Sub-study Week 8 |
| $7^*(w+10) + 1 \le Study Day \le 7^*(w+14)$ $7^*(w+10) + 1 \le Study Day \le 7^*(w+16)$ | | Sub-study Week 12 |
| $7*(w+10) + 1 \le Study Day \le 7*(w+22)$ | $7*(w+10) + 1 \le Study Day \le 7*(w+22)$ | Sub-study Week 16 |

#### NOTES

• The "w" in the target study day calculation refers to the corresponding week number in Extension for the planned Sub-study Day 1 visit. For example, if a participant's last planned Extension phase visit before entering

- the Sub-study is Week 192, the "w" would be 200 if the participant is on Q4W arm and would be 208 if the participant is on Q8W arm.
- For post-baseline visits (i.e. Week 4 and afterwards), apply Snapshot analysis windows only to viral load data that is on-treatment (per Table 20) within the Thigh Injection Phase (per Table 18).
- An on-treatment viral load assessment may be assigned to more than one snapshot analysis window, e.g. ontreatment assessment taken on 7\*(w+14) will be in both Sub-study Week 12 and Sub-study Week 16 visits.
- ± 6 Week window is always used at the key analysis timepoint, Sub-study Week 16 visit.
- [a] The values considered for deriving Sub-study Baseline value include both Extension phase and sub-study data.

Table 14 Assessment Windows for Summaries of Long-Term Follow Up
Phase Data for Participants Who Received At Least One Injection of
CAB+RPV and Permanently Discontinued Study Treatment

| Analysis Window | Analysis Timepoint | Target Study<br>Day of Window |
|---|---|---|
| 1 ≤ LTFU Study Day ≤ 63 | LTFU Month 1/WD[a] | 30 |
| 64 ≤ LTFU Study Day ≤ 135 | LTFU Month 3 | 90 |
| 136 ≤ LTFU Study Day ≤ 225 | LTFU Month 6 | 180 |
| 226 ≤ LTFU Study Day ≤ 315 | LTFU Month 9 | 270 |
| 316 ≤ LTFU Study Day ≤ 405 | LTFU Month 12 | 360 |
| $(30*m - 44) \le LTFU \text{ Study Day} \le (30*m + 45)$ | LTFU Month m | 30*m |
| | m = 15, 18,21, | |

• An assessment may be assigned to both LTFU and maintenance/extension phases.

a. For participants who receives at least one injection of CAB+RPV and permanently discontinues study treatment, they will not complete withdrawal visit, will instead move directly into the LTFU and have LTFU Month 1 visit as the first planned LTFU visit per protocol amendment 1; however, per protocol amendment 2, they will complete withdrawal visit and then have LTFU Month 3 visit as the first planned LTFU visit. Data have been collected either per protocol amendment 1 or per protocol amendment 2 and are included in the database. The analysis timepoint of LTFU Month 1/WD is intended for slotting data mainly collected from either LTFU Month 1 visit per protocol amendment 1 or withdrawal visit per protocol amendment 2 if the date of assessments or onset date of event falls within the specified analysis window.

#### 15.3.3. Assessment Window for Phase Conclusion

The 'Phase Conclusion' records in disposition data will be slotted based on Table 8 (for Maintenance Phase conclusion records), Table 9 (for Extension Phase conclusion records), and Table 12 (for Thigh Injection Phase and Return to Gluteal Injection Phase conclusion records). However, if the discontinuation date is post-treatment per Table 20, the record will be slotted to the last on-treatment visit within the same phase rather than follow up.

#### 15.3.4. Assessment Window for Health Outcome Data

## 15.3.4.1. PIN / HAT-QoL / HIVTSQs / HIVTSQc / ACCEPT / Preference in Main Study

PIN, HAT-QoL, HIVTSQs, HIVTSQc, ACCEPT, Preference, reasons for oral bridging and preference questionnaire assessments will be assigned to analysis visits as follows:

- 1. Baseline will be defined as last available recorded value up to and including the Maintenance treatment start date (expected to be collected at Day 1). Baseline is not applicable for PIN, HIVTSQc and Preference assessments.
- 2. For post-baseline visits, if the nominal visit identifier as captured in the source dataset corresponds to a scheduled collection per the Time and Events Schedule (see Section 15.2 and Table 15) and the assessment is collected in the Maintenance or Extension Phase (per Table 18), then the nominal visit identifier will be kept as the analysis visit.
- 3. For post-baseline visits, if the nominal visit identifier is unscheduled or withdrawal, then the following procedure will be used:
  - a) Assign the assessment to a study phase according to Table 18. Proceed to step b if the assessment is assigned to the Maintenance or Extension Phase.
  - b) Identify the 'last nominal visit' with the HO assessment performed prior to the unscheduled/withdrawal visit to be slotted in the same phase.
  - c) The unscheduled/withdrawal visit will be slotted to the planned nominal visit subsequent to the 'last nominal visit' in the same phase. If the 'last nominal visits' does not exist (e.g. no records originate from a planned nominal visit), then the unscheduled/withdrawal visit will be slotted to the first planned nominal visit after Day 1 in the same phase. If the planned nominal visit subsequent to the 'last nominal visit' is not available, then the unscheduled/withdrawal visit will be slotted to the last planned nominal visit after Day 1 in the same phase.

Example 1, for HATQoL, the planned nominal visits are Day 1, Week 24, and 48. If a participant has the 'last nominal visit' (with HATQoL assessment) at Week 24 prior to withdrawal at Week 36, the withdrawal assessment will be slotted to the subsequent planned nominal visit of Week 48.

Example 2, for HATQoL, if there is unscheduled visit between Week 24 and Week 48. This unscheduled visit will be slotted to Week 48 per the rule. In this case, there are two assessments with analysis visit equal to Week 48 (i.e. the slotted value and the value at original nominal week 48 visit). The original nominal value will be selected for summary per the rule below for multiple records—see Section 15.3.5.1.

Table 15 Planned Nominal Visit of Health Outcome Data in Main Study

| Questionnaire | Day 1 | Week 8 | Week 24 | Week 48 | Week 152 |
|---|---|---|---|---|---|
| PIN | | Х | Х | Х | Х |
| HAT-QoL | Х | | Х | Х | |
| HIVTSQs | Х | | Х | Х | Х |
| HIVTSQc | | | | Х | |
| ACCEPT | Х | | Х | Х | Х |
| Preference | | | | Х | |
| Reasons for Oral Bridging and | | | | | Х |
| Preference | | | | | |
| NOTES: | | | | | |
| Day 1 visits are recorded as "Baseline" visits in the database. | | | | | |

#### 15.3.4.2. Reasons for Continuation/Switch in Main Study

Reasons for Continuation/Switch assessments are planned to be taken at nominal Baseline (Day 1) visit only. The assessments taken within  $\pm$  2 weeks window from maintenance phase treatment start date will be regarded as evaluable. The assessments taken outside this window will be excluded from the summary.

#### 15.3.4.3. HIVTSQs/HIVTSQc/Preference in Sub-study

HIVTSQs, HIVTSQc, Preference Thigh Injection vs Gluteal Injection questionnaire assessments will be assigned to analysis visits as follows:

- Sub-study Baseline will be defined as last available recorded value up to and
  including the date of first thigh injection. Baseline is not applicable for HIVTSQc
  and Preference Thigh Injection vs Gluteal Injection assessments as they are not
  planned to be collected during the Sub-study Baseline. In Sub-study Baseline
  value derivation for HIVTSQs, the assessments conducted in the main study will
  also be considered.
- 2. For post-baseline visits, if the nominal visit identifier as captured in the source dataset corresponds to a scheduled collection per the Time and Events Schedule (see Section 15.2) and the assessment is collected in the planned phase (per Table 18, visits at/before Sub-study Week 16 belong to Thigh Injection phase, and visits after Sub-study Week 16 belong to Return to Gluteal Injection phase), then the nominal visit identifier will be kept as the analysis visit.
- 3. For post-baseline visits, if the nominal visit identifier is unscheduled or it is scheduled however not conducted in the planned phase (e.g. the sub-study Week 16 HIVTSQs assessment is conducted after the Week 16 gluteal injection and therefore belong to Return to Gluteal Injection phase), then this visit will be assigned to the planned visit in the same phase.

#### 15.3.4.4. Tolerability of Injections (NRS) in Sub-study

After assigning the phases per Table 18, the NRS assessments will be slotted to analysis visits per Table 16.

Table 16 Assessment Window for NRS Data

| Phase | Assessment Window | Visit |
|---|---|---|
| Sub-study | Q8W: post-dose and on the Week -8 injection date | Q8W: Sub-study Week -8 |
| Screening | Q4W: post-dose and on the Week -4 injection date | Q4W: Sub-study Week -4 |
| | Q8W: (Week -8 injection date+1, Week -8 injection | Q8W: Sub-study Week -7 |
| | date+14), inclusive | Q4W: Sub-study Week -3 |
| | Q4W: (Week -4 injection date+1, Week -4 injection | |
| | date+14), inclusive | |
| Thigh | Post-dose and on the Day 1 injection date | Sub-study Day 1 |
| Injection | (Day 1 injection date+1, Day 1 injection date+14), | Sub-study Week 1 |
| | inclusive | |
| | Q8W: post-dose and on the Week 8 injection date | Q8W: Sub-study Week 8 |
| | Q4W: post-dose and on the Week 12 injection date | |

| | | Q4W: Sub-study Week<br>12 |
|---|---|---|
| | Q8W: (Week 8 injection date+1, Week 8 injection date+14), inclusive Q4W: (Week 12 injection date+1, Week 12 injection date+14), inclusive | Q8W: Sub-study Week 9<br>Q4W: Sub-study Week<br>13 |
| Return to | Post-dose and on the Week 16 injection date | Sub-study Week 16 |
| Gluteal | (Week 16 injection date+1, Week 16 injection | Sub-study Week 17 |
| | date+14), inclusive | |

#### 15.3.5. Assessment Window for PK Concentration Data

#### 15.3.5.1. Maintenance and Extension Phase Assessments

For PK concentration data at the withdrawal/unscheduled/LTFU Month 1visits during the maintenance and extension phase (after assignment to study phase per Table 18), the visit will be slotted to the analysis visit per the following steps:

- Identify the 'last nominal visit' with the planned PK pre-dose assessment prior to the visit to be slotted during the same study phase
- Identify the nominal visit corresponding to the next planned pre-dose PK assessment visit (excluding visits with storage PK collection), that is subsequent to the 'last nominal visit' with PK pre-dose assessment during the same study phase. If the 'last nominal visit' during the maintenance phase does not exist, the first planned pre-dose PK assessment visit for the participant during the maintenance phase will be considered the nominal visit corresponding to the next planned pre-dose PK assessment. If the 'last nominal visit' during the extension phase does not exist, slot the PK assessment to the nominal visit of the next planned injection occurring on or after the date of the PK assessment during the extension phase.
- If the nominal visit corresponding to next planned pre-dose PK assessment visit is prior to/at Week 48 visit, the PK assessment at the unscheduled/withdrawal/LTFU Month 1 visit will be slotted to this nominal visit corresponding to next planned pre-dose PK assessment visit.
- Otherwise, the PK assessment at the unscheduled/withdrawal/LTFU Month1 visit will be slotted to the earliest nominal visit from the following:
  - Nominal visit corresponding to the next planned pre-dose PK assessment visit
  - The nominal visit of the next planned injection occurring on or after the date of the PK assessment during the same study phase. If both the next planned pre-dose PK assessment visit and the next planned injection visit during the same study phase are not available, for example, withdrawal PK assessment taken after Week 96 for participants on Q8W arm, the PK assessment will be slotted to Week 100 visit.

During the maintenance and extension phase, the planned nominal visits for PK Pre-dose are Week 4B, 8, 16, 24, 32, 40, 48, 96, 152 for Q4W arm; and are Day 1, Week 4B, 8, 16, 24, 32, 40, 48, 96, 152 for Q8W arm while Day 1 is required only for those transitioning from ATLAS on Q4W injections and Week 4B is required only for participants transitioning from oral SOC and requiring oral CAB+RPV lead-in. In addition, the participants on Q8W arm have planned nominal visits at Week 9 and 41 for 1-week post-dose.

For participants requiring oral CAB+RPV lead-in, the planned injection visits are Week 4B, Week 8, continuing every 4 weeks for Q4W arm and continuing every 8 weeks for Q8W arm. For participants not requiring oral CAB+RPV lead-in, the planned injection visits are every 4 weeks starting from Day 1 for Q4W arm and every 8 weeks starting from Day 1 for Q8W arm.

Example 1: If a participant on Q8W arm has the 'last nominal visit' (with PK pre-dose assessment) at Week 24 and then withdraws around Week 28, with the last injection at Week 24 and a Maintenance Phase PK assessment labelled at 'LTFU Month 1'., This PK assessment labelled as 'LTFU Month 1' will be slotted to the subsequent planned nominal visit of Week 32.

Example 2: If a participant on Q4W arm has the 'last nominal visit' (with PK pre-dose assessment) at Week 48 and then have an unscheduled Maintenance Phase PK assessment around Week 74. This assessment will be slotted to the next planned injection visit, Week 76.

There will be no slotting for planned nominal visits (i.e. analysis visit =visit).

#### 15.3.5.2. Long-term Follow-up Phase Assessments

PK concentration data at nominal visits other than withdrawal/LTFU Month 1/LTFU Month 3/LTFU Month 6/LTFU Month 9/LTFU Month 12/Liver Event which have been assigned to the LTFU phase (according to according to Table 18) will be slotting to analysis visits per the following steps:

- Identify the 'last nominal PK visit' with the PK assessment performed prior to the visit to be slotted during the LTFU phase
- The PK assessments will be slotted to the nominal visit corresponding to the next planned LTFU PK assessment visit that is subsequent to the 'last nominal PK visit' during the LTFU phase. If the 'last nominal visit' does not exist, the PK assessment will be slotted per .

There will be no slotting for planned PK nominal visits (i.e. analysis visit =visit): LTFU Month 1 or withdrawal, LTFU Month 3, LTFU Month 6, LTFU Month 9 and LTFU Month 12.

#### 15.3.5.3. Sub-study Assessments

Unscheduled sub-study assessments will not be slotted to any analysis visit. There will be no slotting for planned nominal visits (i.e. analysis visit=visit).

#### 15.3.6. Multiple Assessments within an Assessment Window

If after window assignment there are multiple valid assessments of a parameter within the same window, then the following hierarchy will be used to determine the value to be used for summary statistics of observed values:

For data other than health outcome/PK concentration:

- 1. the assessment closest to the window target Study Day;
- 2. if there are multiple assessments equidistant from the target Study Day, then the mean of these values will be used. For HIV-1 RNA, the geometric mean of the number of copies will be used as opposed to the arithmetic mean. For post-dose ECG, the assessment closest to the two-hour post injection will be used.

For Health outcome and PK concentration data, the following hierarchy will be used to determine the value to be used for summary statistics of observed values:

- 1. If there are multiple on-treatment assessments assigned to the same analysis visit, the assessment from the planned nominal visit will be used for summary statistics.
- 2. If there are multiple on-treatment assessments assigned to the same analysis visit and none originates from a planned nominal visit (e.g. two unscheduled/withdrawal nominal visits), then
  - a. the assessment closest to the window target Study Day will be used;
  - b. if there are multiple assessments equidistant from the target Study Day, then the earliest assessment will be used.

Assessments not chosen for use in summary statistics by this algorithm will still appear in the associated listings. Also, all applicable valid assessments, irrespective of proximity to the target study day, will be used when categorizing values across visits, such as 'maximum grade' or 'at any time', and for any algorithm that has specific rules for which observation to use (e.g. snapshot algorithm, LOCF or CVF identification).

#### 15.4. Appendix 4: Study Phases and Treatment State

#### 15.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the Treatment Start Date defined in Section 15.6.1.

AEs will be assigned to study phases as defined in Table 17. For example, adverse events on/after start of maintenance phase IP and prior to start of Extension phase IP/LTFU ART will be assigned to the Maintenance Phase.

Laboratory data (efficacy, safety, PK and virology), HIV associated Conditions, health outcomes assessments, vital signs, and ECGs will be assigned to study phases as defined as in Table 18. For example, assessments/events occurring after start of maintenance phase IP and up to and including start of extension phase IP/LTFU ART will be assigned to the Maintenance Phase.

Assessments/events are assigned to study phases sequentially, starting from the top of each table, except for the assessments/events occurring after returning to Extension phase from the sub-study participation. No study phases will be assigned to medications.

Table 17 Assignment of Study Phases for AEs

| Study Phase | Definition |
|---|---|
| Screening | Date < Maintenance Treatment Start Date |
| Maintenance | For participants continuing into Extension Phase: |
| | Maintenance Treatment Start Date ≤ Date < Date of Nominal Week 100 Visit |
| | For participants <u>not</u> continuing into Extension Phase: For participants continuing into LTFU Phase: Maintenance Treatment Start Date ≤ Date < LTFU ART Start Date <sup>[a]</sup> |

| Extension | For participants continuing into Extension Phase and not entering the sub- |
|---|---|
| LAGIOOII | study: |
| | If participants continued into LTFU Phase after the Extension phase:Date of Nominal Week 100 Visit ≤ Date < LTFU ART Start Date <sup>[a]</sup> |
| | If participants transitioned to marketed product/alternative HAART and did not |
| | withdraw study due to safety related reason, then |
| | Date of Nominal Week 100 Visit <sup>[a]</sup> ≤ Date < Date of end of study +35 days (Q4W) or + 63 days (Q8W) |
| | For participants continuing into Extension Phase, entering the sub-study be not returning to Extension Phase: |
| | Date of Nominal Week 100 Visit ≤ Date < Date of First Sub-study Record |
| | For participants continuing into Extension Phase, entering the sub-study and |
| | returning to Extension Phase: |
| | Before the sub-study: Date of Nominal Week 100 Visit ≤ Date < Date of First Substudy Record |
| | After the sub-study: |
| | For participants continuing into LTFU Phase after return to extension phase:<br>End of Sub-study Date <sup>[b]</sup> < Date < LTFU ART Start Date <sup>[a]</sup> |
| | For participants transitioned to marketed product/alternative HAART and did not |
| | withdraw study due to safety related reason: |
| | End of Sub-study Date <sup>[b]</sup> < Date < Date of end of study +35 days (Q4W) or + 63 days (Q8W) |
| Sub-study | For participants entering the sub-study and not receiving any thigh injection: |
| Screening | If participants continued into LTFU Phase after the sub-study, then |
| | Date of First sub-study record ≤ Date < LTFU ART Start Date <sup>[a]</sup> |
| | If participants transitioned to marketed product/alternative HAART and did not |
| | withdraw study due to safety related reason, then |
| | Date of First sub-study record ≤ Date < Date of end of study +35 days (Q4W) or +63 days (Q8W) |
| | If participants continued into Extension Phase after the sub-study, then |
| | Date of First sub-study record ≤ Date ≤ End of Sub-study Date <sup>[b]</sup> |
| | For participants entering the sub-study and receiving thigh injection(s): |
| | Date of First sub-study record ≤ Date < Date of First Thigh Injection |
| Thigh Injection | For participants continuing into Return to Gluteal Injection Phase: |
| J , | Date of First Thigh Injection ≤ Date < Date of Nominal Sub-study Week 16 Visit <sup>[c]</sup> |
| | For participants not continuing into Return to Gluteal Injection Phase: |
| | If participants continued into LTFU Phase after the sub-study, then |
| | Date of First Thigh Injection ≤ Date < LTFU ART Start Date[a] |
| | If participants continued into Extension Phase after the sub-study, then |
| | Date of First Thigh Injection ≤ Date ≤ End of Sub-study Date <sup>[b]</sup> |
| | If participants transitioned to marketed product/alternative HAART and did not |
| | withdraw study due to safety related reason, then |
| | Date of First Thigh Injection ≤ Date < Date of end of study +35 days (Q4W) or +63 days (Q8W) |


207966

| Return to Gluteal | For participants continuing into Extension Phase after the sub-study: |
|---|---|
| Injection | Date of Nominal Sub-study Week 16 Visit[c] ≤ Date ≤ End of Sub-study Date[b] |
| | For participants continuing into LTFU Phase after the sub-study: |
| | Date of Nominal Sub-study Week 16 Visit <sup>[c]</sup> ≤ Date < LTFU ART Start Date <sup>[a]</sup> |
| | For participants transitioned to marketed product/alternative HAART and did not |
| | withdraw study due to safety related reason: |
| | Date of Nominal Sub-study Week 16 Visit[c] ≤ Date < Date of end of study +35 days |
| | (Q4W) or + 63 days (Q8W) |

- Date = AE Start date
- For AEs started on the End of Sub-study Date, if participants received injection belonging to the Extension Phase on End of Sub-study Date, Extension Phase will be assigned to these AEs.
- [a] If participants have missing LFTU ART start date, only the lower bound will be considered in the derivation. For AEs leading to withdrawal and started on the same date as LTFU ART Start Date, appropriate study treatment associated phase (e.g. Maintenance, Extension, Sub-study Screening, Thigh Injection, Return to Gluteal Injection), instead of Long-term Follow-up phase, will be assigned.
- [b] End of Sub-study Date is defined in Section 15.6.1.
- [c] Nominal Sub-study Week 16 Visit Date is defined in Section 15.6.1.

Table 18 Assignment of Study Phases for Lab Assessments (including PK and Virology), ECG, Protocol Deviations, Vital Sign, Health Outcomes, HIV Associated Conditions

| Study Phase | Definition |
|---|---|
| Screening | Date ≤ Maintenance Treatment Start Date |
| C | Note: 2-hour post-dose ECG taken on the Maintenance Treatment Start Date will be excluded. |
| Maintenance | For participants continuing into Extension Phase: Maintenance Treatment Start Date < Date ≤Date of Nominal Week 100 Visit <sup>[a]</sup> Note: 2-hour post-dose ECG taken on the Maintenance Treatment Start Date will be included. |
| | For participants not continuing into Extension Phase: For participants continuing into LTFU Phase: Maintenance Treatment Start Date < Date ≤ LTFU ART Start Date <sup>[b]</sup> For participants transitioned to marketed product/alternative HAART and did not withdraw study due to safety related reason: Maintenance Treatment Start Date < Date ≤ Date of end of study +35 days |
| | (Q4W) or + 63 days (Q8W) Note: 2-hour post-dose ECG taken on the Maintenance Treatment Start Date will be included. |
| Extension | For participants continuing into Extension Phase and not entering the sub-study: If participants continued into LTFU Phase after the Extension phase: Date of Nominal Week 100 Visit <sup>[a]</sup> < Date ≤ LTFU ART Start Date <sup>[b]</sup> If participants transitioned to marketed product/alternative HAART and did not withdraw study due to safety related reason, then Date of Nominal Week 100 Visit <sup>[a]</sup> < Date ≤ Date of end of study +35 days (Q4W) or + 63 days (Q8W)For participants continuing into Extension Phase, entering the sub-study but not returning to Extension Phase: Date of Nominal Week 100 Visit <sup>[a]</sup> < Date < Date of First Sub-study Record For participants continuing into Extension Phase, entering the sub-study and returning to Extension Phase: Before the sub-study: Date of Nominal Week 100 Visit <sup>[a]</sup> < Date < Date of First Sub-study Record After the sub-study: For participants continuing into LTFU Phase after return to extension phase: End of Sub-study Date <sup>[b]</sup> < Date ≤ LTFU ART Start Date <sup>[a]</sup> For participants transitioned to marketed product/alternative HAART and did not withdraw study due to safety related reason: End of Sub-study Date <sup>[b]</sup> < Date ≤ Date of end of study +35 days (Q4W) or +63 days (Q8W) |

| Sub-study | For participants entering the sub-study and not receiving any thigh |
|---|---|
| Screening | injection: |
| | If participants continued into LTFU Phase after the sub-study, then |
| | Date of First sub-study record ≤ Date < LTFU ART Start Date <sup>[b]</sup> |
| | If participants transitioned to marketed product/alternative HAART and did not withdraw study due to safety related reason, then |
| | Date of First sub-study record ≤ Date < Date of end of study +35 days (Q4W) |
| | or + 63 days (Q8W) |
| | If participants continued into Extension Phase after the sub-study, then |
| | Date of First sub-study record ≤ Date ≤ End of Sub-study Date[c] |
| | For participants entering the sub-study and receiving thigh injection(s): |
| T1:11:0 | Date of First sub-study record ≤ Date ≤ Date of First Thigh Injection <sup>[d]</sup> |
| Thigh Injection | For participants continuing into Return to Gluteal Injection Phase: |
| | Date of First Thigh Injection <sup>[d]</sup> < Date ≤ Date of Nominal Sub-study Week 16 |
| | Visit <sup>[e]</sup> |
| | For participants not continuing into Return to Gluteal Injection Phase: |
| | If participants continued into LTFU Phase after the sub-study, then |
| | Date of First Thigh Injection <sup>[d]</sup> < Date ≤ LTFU ART Start Date <sup>[b]</sup> |
| | If participants continued into Extension Phase after the sub-study, then |
| | Date of First Thigh Injection <sup>[d]</sup> < Date ≤ End of Sub-study Date <sup>[c]</sup> |
| | If participants transitioned to marketed product/alternative HAART and did not |
| | withdraw study due to safety related reason, then |
| | Date of First Thigh Injection ≤ Date ≤ Date of end of study +35 days (Q4W) or + 63 days (Q8W) |
| Return to | For participants continuing into Return to Extension Phase after the |
| Gluteal | sub-study: |
| Injection | Date of Nominal Sub-study Week 16 Visit <sup>[e]</sup> < Date ≤ End of Sub-study Date <sup>[c]</sup> |
| ,000.011 | For participants continuing into LTFU Phase after the sub-study: |
| | Date of Nominal Sub-study Week 16 Visit <sup>[e]</sup> < Date ≤ LTFU ART Start Date <sup>[b]</sup> |
| | For participants transitioned to marketed product/alternative HAART |
| | and did not withdraw study due to safety related reason: |
| | Date of Nominal Sub-study Week 16 Visit <sup>[c]</sup> < Date ≤ Date of end of study +35 |
| | days (Q4W) or + 63 days (Q8W) |
| | adjo (Q 111) or . oo dajo (Q011) |

- Date = start or assessment date
- [a] If the collected time of the assessment is available, the assessment taken on the same day as nominal Week 100 visit date but after the Week 100 injection will be assigned to Extension Phase.
- [b] If participants have missing LFTU ART start date (i.e. the participants have not started ART in LFTU yet), only the lower bound of the window will be considered in the derivation.
- [c] End of Sub-study Date is defined in Section 15.6.1.
- [d] The post-dose assessments (e.g. 2-hour post-dose ECG, 2-hour post-dose PK and NRS) taken on the date of first thigh injection will be assigned Thigh Injection Phase, instead of Sub-study Screening Phase.
- [e] The Date of Nominal Sub-study Week 16 is defined in Section 15.6.1. The post-dose assessment (e.g. NRS) taken on the date of Sub-study Week 16 injection will be assigned Return to Gluteal Injection Phase, instead of Thigh Injection Phase.

Table 19 Assignment to Long-term Follow-up Phase

| Study Phase | Definition |
|-------------|------------|
|-------------|------------|

| Long-term | Date > max (Last IM Injection Date, Last Oral Bridging End Date) |
|-----------|------------------------------------------------------------------|
| Follow-up | |

- Date = Assessment/Start Date
- For AEs leading to withdrawal and started on the same date as LTFU ART Start Date, appropriate study treatment associated phase, instead of long-term follow-up phase, will be assigned. Refer to Table 17 for details.

Only participants who received at least one CAB and/or RPV injection will enter the long-term follow-up. Participants transitioning to CAB+RPV LA marketed product or alternative HAART (except due to safety-related reasons) do not need to enter the LTFU Phase. Note that the long-term follow-up phase and maintenance/extension/sub-study screening/thigh injection/return to gluteal injection phases are not necessarily mutually exclusive and are to be defined with separate phase variables in the datasets. For example, an Q4W IM participant who has Week 44 injection and withdrawal at Week 48 without receiving Week 48 injection, the "Week 48 withdrawal visit" belongs to both the maintenance phase and long-term follow-up phase.

#### 15.4.2. Treatment State

Within each treatment study phase (i.e. Maintenance and Extension—based on assignment of study phase described in Section 15.4.1), only those assessments which occur within the ranges shown in Table 20 will be considered 'on-treatment' for the given phase. No treatment states will be assigned to medications.

Table 20 Treatment State within Study Phases<sup>b</sup>

| Study Phase <sup>a</sup> | Treatment State | Date Range |
|---|---|---|
| Screening | Pre-treatment | All assessments/events within the phase |
| Maintenance | On-treatment | Q8W arm: |
| | | Date ≤ max (Date of Last Injection + 63, Date of Last |
| | | Dose of Oral Study Treatment (CAB+RPV or SOC |
| | | Bridging) + 1) |
| | | Q4W arm: |
| | | Date ≤ max (Date of Last Injection + 35, Date of Last |
| | | Dose of Oral Study Treatment (CAB+RPV or SOC |
| | | Bridging) + 1) |
| | Post-treatment | Q8W arm: |
| | | Date > max (Date of Last Injection + 63, Date of Last |
| | | Dose of Oral Study Treatment (CAB+RPV or SOC |
| | | Bridging) + 1) |
| | | Q4W arm: |
| | | Date > max (Date of Last Injection + 35, Date of Last |
| | | Dose of Oral Study Treatment (CAB+RPV or SOC |
| Extension | On-treatment | Bridging) + 1) Q8W arm: |
| EXIGUSION | On-treatment | |
| | | Date ≤ max (Date of Last Injection + 63, Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC |
| | | Bridging) + 1) |
| | | Q4W arm: |

| | | Date ≤ max (Date of Last Injection + 35, Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1) |
|---|---|---|
| | Post-treatment | Q8W arm: Date > max (Date of Last Injection + 63, Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1) |
| | | Q4W arm: Date > max (Date of Last Injection + 35, Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1) |
| Long-term Follow-<br>up | On-treatment | Q8W arm: Date ≤ min (LTFU ART start date, max (Date of Last Injection + 63, Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)) |
| | | Q4W arm: Date ≤ min (LTFU ART start date, max (Date of Last Injection + 35, Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)) |
| | Post-treatment | Q8W arm: Date > min (LTFU ART start date, max (Date of Last Injection + 63, Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)) |
| | | Q4W: Date > min (LTFU ART start date, max (Date of Last Injection + 35, Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)) |

- Date = Assessment/Start Date.
- For Sub-study Screening, Thigh Injection and Return to Gluteal Injection phases, the same on-treatment and post-treatment algorithms as those in Extension Phase will be applied.
- a. Treatment State is determined after data has been assigned to the study phases as defined in Section 15.4.1.
- b. Last injection and/or last dose of oral study treatment (CAB+RPV or SOC bridging) are only applied to participants who permanently discontinued the study treatment. The assessments for participants who did not permanently discontinue the study treatment will be considered 'On-treatment'. For participants continuing into extension phase, all data assigned to maintenance phase per Section 15.4.1 will be considered 'On-treatment'.

#### 15.4.2.1. Treatment States for AE Data

For adverse events, partial AE start date will use imputation as described in Section 15.7.2.1. In the case of a completely missing start date, the event will be considered to have started On-treatment in the Maintenance phase unless an end date for the AE is provided which is before start of study treatment at Maintenance phase; in such a case the AE is assigned as Pre-treatment.

Additional variables will be derived as shown in Table 21.
Table 21 Days since First Dose of Each Study Phase, Days since Phase Start, AE Duration and Relation to Study Treatment

| | Definition |
|---|---|
| Days since<br>First Dose<br>(Days) <sup>a</sup> | AE Start Date – Maintenance Treatment Start Date + 1 |
| Days since<br>Last Dose<br>(Days) <sup>a</sup> | AE Start Date – Date of Last Dose of Study Treatment prior to/on the Start Date of AE + 1 |
| Days since | For AEs in Maintenance Phase: |
| Phase Start | AE Start Date - Maintenance Treatment Start Date + 1 |
| | For AEs in Extension Phase before Sub-study: |
| | AE Start Date – Date of Nominal Week 100 Visit + 1 |
| | For AEs in Extension Phase after Sub-study: |
| | AE Start Date – End of Sub-study Date <sup>c</sup> + 1 |
| | For AEs in Long-term Follow-up Phase: |
| | AE Start Date – Date of Last Dose of Study Treatment <sup>b</sup> |
| | For AEs in Sub-study Screening Phase: |
| | AE Start Date – Date of First Sub-study Record + 1 |
| | For AEs in Sub-study Thigh Injection Phase: |
| | AE Start Date - Date of First Thigh Injection + 1 |
| | For AEs in Return to Gluteal Injection Phase: |
| | AE Start Date - Date of Nominal Sub-study Week 16 Visit + 1 |
| Duration<br>(Days) | AE Resolution Date – AE Start Date + 1 |
| Drug-related | If relationship is marked 'YES' on Inform/eCRF or value is missing. |

#### NOTES:

- a. Days since First/Last Dose will only be derived for AEs assigned to maintenance phase, extension phase and long-term follow-up phase.
- b. Date of Last Dose of Study Treatment = max (Last IM Injection Date, Last Oral Bridging End Date), only applicable to participants who permanently discontinued study treatment.
- c. End of Sub-study Date is defined in Section 15.6.1.

## 15.4.3. Study Period

Certain displays will be produced for data collected during the oral lead-in. The study period variable is defined in Table 22 and Table 23. Study period is assigned after the study phase is assigned (screening, maintenance, extension, or long-term follow-up) based on the Tables in Section 15.4.1.

Table 22 Assignment of Study Period for AE Data

| Study Period | Date range |
|--------------|------------|

| Oral Lead-in | For participants receiving at least one Injection: Maintenance Treatment Start Date ≤ Date < Date of First IM Injection |
|---|---|
| | For participants withdrawing prior to first Injection: Date ≥ Maintenance Treatment Start Date |
| | Note that the oral lead-in period is only applicable to the participants who received at least one dose of study treatment during the oral lead-in period in the study. Oral lead-in period is within the maintenance phase. |

#### NOTES:

• Date = AE Start date.

 Table 23
 Assignment of Study Period for Lab Assessments:

| Period | Date range |
|---|---|
| Oral Lead-in | For participants receiving at least one Injection: Maintenance Treatment Start Date < Date ≤ Date of First IM Injection |
| | For participants withdrawing prior to first Injection: Date > Maintenance Treatment Start Date |
| | Note that the oral lead-in period is only applicable to the participants who received at least one dose of study treatment during the oral lead-in period in the study. Oral lead-in period is within the maintenance phase. |

### NOTES:

• Date = Date of assessment.

# 15.5. Appendix 5: Data Display Standards & Handling Conventions

## 15.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : us1salx00259 |
| HARP Compound | : \ARPROD\GSK1265744\mid207966 |
| Analysis Datasets | |

#### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for every reporting effort described in the RAP.

### 15.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### Planned and Actual Time

- Reporting for tables, figures and formal statistical analyses:
  - Actual time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - If space allows, planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).

- Unscheduled or unplanned readings will be presented within the participant's listings.
- When data falls within both maintenance / extension and long-term follow-up phases, it will be presented in maintenance / extension phase, unless otherwise specified.
- Unless otherwise specified, when data falls within both screening and baseline visits per analysis visit windows, it will be presented at baseline visit.

#### **Unscheduled Visits**

- Unscheduled visits will be assigned to a study visit using the all-inclusive windows defined in Section 15.2.3.
- However, data summaries will only report visits that are planned assessment time points for each parameter (according to the Time and Events table).
- Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1. First and third quartiles will also |
| | be included in the summary. |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 15.5.3. Reporting Standards for Pharmacokinetic

| Reporting of Pharmacokinetic Concentration Data | |
|---|---|
| Descriptive | Refer to IDSL PK Display Standards. |
| Summary Statistics, | Refer to IDSL Statistical Principle 6.06.1 |
| Graphical Displays | Assign the low limit of quantification (CAB 0.025 ug/mL, RPV 1 ng/mL) |
| and Listings | NQ values. |
| Reporting of Pharmacokinetic Parameters | |
| Descriptive | N, n, geometric mean, 95% CI of geometric mean, standard deviation |
| Summary Statistics | (SD) of loge transformed data and between participant coefficient of |
| (Log <sub>e</sub> Transformed) | variation (CV <sub>b</sub> (%)) will be reported. |
| | $\circ CV_b(\%) = \sqrt{\exp(SD^2) - 1} \times 100$ |
| | (SD = SD of log <sub>e</sub> transformed data) |

## 15.6. Appendix 6: Derived and Transformed Data

#### 15.6.1. General

#### **Multiple Measurements at One Time Point**

• If after window assignment there are multiple valid assessments of a parameter within the same window, refer to Section 15.3.5.1 for determination of the value to be used for summary statistics of observed values. Assessments not chosen for use in summary statistics will still appear in the associated listings. Assessments not chosen for use in summary statistics by this algorithm will still appear in the associated listings. Also, all applicable valid assessments, irrespective of proximity to the target study day, will be used when categorizing values across visits, such as 'maximum grade' or 'at any time', and for any algorithm that has specific rules for which observation to use (e.g. snapshot algorithm, LOCF or CVF identification).

#### **Nominal Week 100 Visit Date**

- For participants who received Week 100 injection, nominal Week 100 visit date is defined by the Week 100 injection date.
- Otherwise, nominal Week 100 visit date is defined by the date of latest Week 100 assessment.
- For participants who continued into Extension Phase however missed Week 100 visit, nominal Week 100 visit date is defined by the end of Maintenance Phase date (i.e. date for the Maintenance Phase conclusion record in the SDTM DS domain) for the analysis purpose.

## Nominal Sub-study Week 16 Visit Date

- For participants who received Sub-study Week 16 injection, nominal Sub-study Week 16 visit date is defined by the Sub-study Week 16 injection date.
- Otherwise, nominal Sub-study Week 16 visit date is defined by the date of latest Substudy Week 16 assessment.
- For participants who continued into Return to Gluteal Injection Phase however missed Sub-study Week 16 visit, nominal Sub-study Week 16 visit date is defined by the end of Thigh Injection Phase date (i.e. date for the Thigh Injection Phase conclusion record in the SDTM DS domain) for the analysis purpose.

#### **End of Sub-study Date**

- For sub-study screen failures, the end of sub-study date is defined by the date they failed to meet the inclusion/exclusion criteria in the sub-study.
- For other sub-study participants, the end of sub-study date is defined by the date of completion or withdrawal available in the sub-study conclusion eCRF form.

#### **Study Day**

The Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the start date of study treatment during the Maintenance Phase as follows:

if date of event ≥ start date of study treatment, then

Study Day=date of event - start date of Maintenance Phase treatment +1

if date of event < start date of study treatment, then

Study Day=date of event - start date of Maintenance Phase treatment

Note that the start date of study treatment during maintenance phase is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

#### **Extension Phase Study Day**

The Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the date of nominal Week 100 visit as follows:

if date of event ≥ date of nominal Week 100 visit, then

Study Day=date of event - date of nominal Week 100 visit + 1

if date of event < date of nominal Week 100 visit, then

Study Day=date of event - date of nominal Week 100 visit

Note that the date of nominal Week 100 visit is considered to be on Extension Phase Study Day 1 and the day before this is Extension Phase Study Day -1; i.e., there is no Extension Phase Study Day 0.

#### **Sub-study Phase Study Day**

Each phase Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the reference date for each phase of the sub-study as follows:

if date of event ≥ reference date, then

Study Day=date of event - reference date + 1

if date of event < reference date, then

Study Day=date of event - reference date

The reference date for the Screening Phase is the date of first screening visit in the sub-study, for the Thigh Injection Phase is the date of first thigh injection, and for the Return to Gluteal Injection Phase is the nominal sub-study Week 16 visit date as specified in this section.

### Long-term Follow-up Study Day

The Long-Term Follow Up (LTFU) Study Day of an event (e.g., lab assessment, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the end of study treatment [i.e. max(Last IM Injection Date, Last Oral Bridging End Date)]

as follows:

If the date of event falls in Long-term Follow up phase, then

LTFU Study Day = Date of Event - End Date of IP

#### **Change from Baseline**

- Post-Dose Visit Value Baseline
  - Unless otherwise specified, the baseline definitions specified in Section 5.2 will be used for derivations for endpoints / parameters.

### 15.6.2. Study Population

#### **Demographics and Baseline Characteristics**

#### Age

- Age, in whole years, will be calculated with respect to the participant's Screening visit. For substudy, age will be calculated with respect to the participant's first sub-study screening visit.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied.
   Consequently, the age of the participant will not be calculated and will remain missing.

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / Height (m)<sup>2</sup>

#### **Hepatitis Status**

- Hepatitis C status will be determined using antibody and/or hepatitis C virus (HCV) RNA assessments performed during screening or during the conduct of the study.
- If both antibody and virus RNA assessments are available, then the latter will take precedence
  and positive/negative status will be based on whether HCV RNA is detectable (i.e., ≥ limit of
  quantification) or not.
- A participant will be considered positive for hepatitis B virus (HBV) if they have a positive surface antigen or detectable HBV DNA result. "HBV DNA DETECTED" in the lab comment takes precedence over HBV DNA test result for positive hepatitis B status, for example, if a participant has HBV test result below level of detection, however, the lab comment shows that HBV DNA detected, this participant will be considered positive for hepatitis B. If HBV DNA result is available, it will be used to qualify hepatitis B status as positive or negative (positive if ≥ limit of quantification); otherwise Hepatitis B status will be determined using the surface antigen result.
- Hepatitis status at entry will be based on the assessments prior to/on the start of the study treatment.

#### Framingham Risk Equation

#### **Demographics and Baseline Characteristics**

• The predicted probability,  $\hat{p}$ , of having a cardiovascular disease (CVD) within the next 10-years according to the Framingham formula [D'Agostino, 2008] is

#### For females:

$$\widehat{p}_F = 1 - S_0(t)^{exp} \begin{cases} 2.32888 \times \log(age) + 1.20904 \times \log(TC) - 0.70833 \times \log(HDL) + 2.76157 \times \log(SBP_u) + 1.20904 \times \log(SBP_t) + 0.52873 \times I_s + 0.69154 \times I_d - 26.1931 \end{cases}$$

For males:

$$\widehat{p}_{M} = 1 - S_{0}(t)^{exp} \begin{cases} 3.06117 \times \log(age) + 1.12370 \times \log(TC) - 0.93263 \times \log(HDL) + 1.93303 \times \log(SBP_{u}) + 1.99881 \times \log(SBP_{t}) + 0.65451 \times I_{s} + 0.57367 \times I_{d} - 23.9802 \end{cases}$$

where

$$S_0(t) = \begin{cases} 0.95012, \text{ females} \\ 0.88936, \text{ males} \end{cases}$$

$$I_s = \begin{cases} 1, \text{ current smoker} \\ 0, & otherwise \end{cases}$$

$$I_d = \begin{cases} 1, & \text{diabetic} \\ 0, & otherwise \end{cases}$$

TC = total serum cholesterol (mg/dL),

HDL = serum HDL cholesterol (mg/dL).

SBPu = systolic blood pressure (mmHg) if participant is not treated for high blood pressure (note that if a participant is treated for high blood pressure then log(SBPu) = 0)
SBPt = systolic blood pressure (mmHg) if participant is treated for high blood pressure (note that if a participant is not treated for high blood pressure then log(SBPt) = 0)

- A participant will be considered as treated for high blood pressure if during screening it has specified that is suffering from hypertension.
- A participant is classified as diabetic if current or past is indicated in the medical conditions eCRF for Type 1 or Type 2 diabetes mellitus, or if baseline fasting glucose ≥7.00 mmol/L (126 mg/dL).
- Smoking status is collected in the eCRF at Day 1. A current smoker is defined as currently smoking/using tobacco or has smoked/used tobacco within the previous 6 months; a former smoker is defined as previously smoked/used tobacco products and has not smoked/used tobacco products within the previous 6 months.
- This calculation will not be performed for participants who have indicated current or past
  myocardial infarction conditions on the eCRF. These participants will not be included in
  summary statistics of risk, but they will be counted in the highest category of risk in the
  summary by category.

## **Prior Exposure to CAB+RPV**

 For participants transitioning from ATLAS study and having prior exposure to CAB+RPV in ATLAS study: Duration of Prior Exposure to CAB+RPV = Randomization Date – Prior Oral CAB Start Date in ATLAS Study + 1.

### **Demographics and Baseline Characteristics**

- For participants transitioning from ATLAS study and not having prior exposure to CAB+RPV in ATLAS study, or for participants randomized from current SOC, Duration of Prior Exposure to CAB+RPV = 0.
- Duration of Prior Exposure to CAB+RPV will be categorized to 0 weeks, 1-24 weeks and >24 weeks.

### **Lipid-modifying Agents**

- The following ATC codes correspond to lipid-modifying agents:
  - o ATC Level 2: C10
  - o ATC Level 3: C10A, C10B (if Level 2 is not available)
  - ATC Level 4: C10AA, C10AB, C10AC, C10AD, C10AX, C10BA, C10BX (if level 2, 3 are not available)
- Participants are considered to have used a lipid-modifying agent at baseline if they are taking the medication at the time of their baseline fasting lipid testing date.
- Participants are also considered to have used a lipid-modifying agent at baseline if they stopped their lipid modifying medication within 12 weeks prior to their baseline fasting lipid testing date.

## 15.6.3. **Efficacy**

#### Snapshot

- The Snapshot algorithm is intended to be primarily a virologic assessment of the endpoint, and as such follows a "virology first" hierarchy.
- 'HIV-1 RNA < 50 c/mL' or 'HIV-1 RNA ≥ 50 c/mL' within an analysis window (see Table 10 and Table 13) is typically determined by the last available HIV-1 RNA measurement in that window while the participant is On-treatment in the Maintenance Phase (as assigned based on Section 15.4).
- When no HIV-1 RNA data is available within a window, a participant cannot be assigned to the category of 'HIV-1 RNA < 50 c/mL'. Depending on the reason for lack of data, the participant will be classified as 'HIV-1 RNA < 50 c/mL' or reported as 'No Virologic Data at Week X'; in the latter case, the algorithm further classifies the nature of the missing data. Typically, a participant withdrawn (i) due to AE or, (ii) for another reason yet was suppressed at the time, will be counted as 'No Virologic Data at Week X'. Should a participant withdraw for reasons other than AE and was not suppressed at the time, they will be categorized as 'HIV-1 RNA ≥ 50 c/mL'.</p>
- Full details of the algorithm, including the handling of special cases, are included in Section 15.9

### Plasma HIV-1 RNA

- For summaries and analyses which use HIV-1 RNA level as a continuous measure, the logarithm to base 10 of the value will be used.
- HIV-1 RNA results may be provided as censored values, such as <40 or >9,999,999 c/mL. For
  the purposes of summary statistics, such values will be replaced by the next value beyond the
  limit of detection, e.g., 39 or 10,000,000 c/mL, respectively, for the given examples. Data
  listings will show the censored values as provided.

## Target Detected / Target Not Detected / Super Low Viral Load Testing

- When a measurement of plasma HIV-1 RNA is below the limit of quantification (i.e. 40 c/mL) and is qualitatively observable that will be denoted as a "Target Detected" measure, while HIV-1 RNA below the limit of quantification that is not qualitatively observable that will be denoted as "Target Not Detected". Any measurements <40 c/mL characterised as "Target Not Detected" or "Target Detected" will be captured in the database.</p>
- Super low viral load will also be tested by BioMONTR Labs for viral loads below the limit of quantification at some visits (e.g. Week 48).

## Confirmed Virologic Failure (CVF)

- The definition of CVF is provided in the Protocol, Section 5.5.4 Definition of Confirmed Virologic Failure.
- In case there are multiple plasma HIV-1 RNA results on the same day, the worst result (i.e. the largest value) will be used in determination of CVF.

## Treatment (TRDF) and Efficacy Related (ERDF) Discontinuation = Failure

• The analysis of time to confirmed virologic failure (CVF) or discontinuation due to treatment related reasons (i.e., drug-related AE, intolerability of injections, protocol defined safety stopping criteria, or lack of efficacy) will censor participants who have not met CVF criteria and are ongoing in the study, or who have discontinued for reasons other than those related to treatment. This will be the Treatment Related Discontinuation = Failure (TRDF) data.

- Participants who have not met CVF criteria and are ongoing in the study, or who have discontinued for reasons other than lack of efficacy, will be censored in the analysis of the Efficacy Related Discontinuation = Failure (ERDF) data.
- Proportion of Participants without virologic (ERDF) or tolerability (TRDF) failure will be
  estimated using the Kaplan-Meier nonparametric method based on the time to ERDF or TRDF.
  The estimated proportion at time point of interest will be presented by treatment group, along
  with estimated difference in proportions between treatment groups and its associated two-sided
  95% CI. The estimate of the standard error used to derive confidence intervals will be based on
  Greenwood's formula [Kalbfleisch,1980].
- See Appendix 10: Variables Defined for Time to Event Analysis for additional details.

## Summary for Participants per Viral Load Category by Visit

- Summary will be based on observed available data, with no imputation for missing values. The
  proportion of participants in each viral load category will be calculated using the denominator
  and numerator specified below:
  - Denominator: Number of participants with on-treatment viral load within the snapshot visit window.
  - Numerator: Number of participants with plasma HIV-1 RNA in the specified category based on the last on-treatment viral load assessment collected within the snapshot visit window.

#### **HIV-1 Disease progression Stage**

- Categories:
  - CDC Stage 1 at Baseline to CDC Stage II;
  - CDC Stage I at Baseline to CDC Stage III;
  - CDC Stage II at Baseline to CDC Stage III;
  - CDC Stage III at Baseline to new CDC Stage III event;
  - o CDC Stage I, II, III at Baseline to Death.

Please refer to Protocol (Appendix 4: CDC Classification for HIV-1 Infection) for defining Stage.

- For the purpose of analysis, the CDC at Baseline and at post-baseline during Maintenance Phase will be derived as below:
  - At Baseline, the 'Baseline CDC stage' for each participant was assessed by investigator and recorded in the eCRF. However, for the analysis, Baseline CDC stage will be rederived based Baseline CD4+ values as well as whether any HIV-associated/AIDS-defining conditions present at baseline per the Criteria's thresholds (Appendix 4 in Protocol).
  - To analyse disease progression, the most advanced post-baseline CDC stage within the period of interest (e.g. Maintenance Phase) will be derived based on the occurrences of new AIDs-defining conditions (please refer to Appendix 4 in Protocol for the list of AIDsdefining Conditions) as well as the nadir value of post-baseline CD4+.
    - ➤ For example, if a participant with CDC 'Stage I' at Baseline had the lowest Maintenance Phase CD4+ =120 cell/mm³ without new AIDs-defining conditions, then HIV disease progression for this participant during the Maintenance Phase would be considered as 'CDC stage I at Baseline to CDC stage III'.
    - ➤ If a participant with CDC 'Stage II' at Baseline had the lowest Maintenance Phase CD4+ =220 cell/mm3 AND had at least one new AIDs-defining condition, then HIV

disease progression for this participant during the Maintenance Phase would be considered as 'CDC stage II at Baseline to CDC stage III'.

### **Delay in IP Injection**

- For participants on the Q4W arm, IM dosing is expected to occur every 4 weeks from Week 4B onwards for those transitioning from SOC (i.e. those requiring oral lead-in) and from Day 1 onwards for those transitioning from CAB+RPV Q4W in ATLAS (i.e. those not requiring oral lead-in). The Delay in IP injection (days) will be calculated as:
  - Delay in IP Injection (days) = Injection date date of preceding injection 28 days
- For participants on the Q8W arm, IM dosing is expected to occur at Week 4B and then every 8 weeks from Week 8 onwards for those transitioning from SOC (i.e. those requiring oral lead-in) and every 8 weeks from Day 1 for those transitioning from CAB+RPV Q4W (i.e. those not requiring oral lead-in) in ATLAS. If participants receive reloading dose injection after oral bridging, the next IM dosing is expected to be 4 weeks from the reloading injection and then every 8 weeks onwards.
  - For participants transitioning from SOC on the Q8W arm, if the preceding injection occurs at Week 4B, the Delay in IP injection (days) will be calculated as:
     Delay in IP Injection (days) = Date of Week 8 injection - date of Week 4B injection - 28 days
  - For participants receiving oral bridging medication and then returning to LA injections, if the
    preceding injection occurs at a reloading dose visit, the Delay in IP injection (days) will be
    calculated as:
    - Delay in IP Injection (days) = Injection date date of preceding injection 28 days
  - For participants transitioning from SOC on the Q8W arm, if the preceding injection occurs at a visit later than Week 4B or at non-reloading visit, the Delay in IP injection (days) will be calculated as:
    - Delay in IP Injection (days) = Injection date date of preceding injection 56 days
  - For participants transitioning from CAB+RPV Q4W in ATLAS on the Q8W arm, if the preceding injection occurs at non-reloading visit, the Delay in IP injection (days) will be calculated as:
    - Delay in IP Injection (days) = Injection date date of preceding injection 56 days
- If the preceding study treatment is oral (e.g. CAB+RPV or SOC oral bridging), the Delay in IP injection (days) will be calculated as:
  - Delay in IP Injection (days) = Injection date date of last oral dose on/prior to the injection date
- Delay in IP injection will be grouped into: ≤1, 2-3, 4-7, >7 days.
- The proportion of participants with HIV-1 RNA ≥50 c/mL at Week 48 (Snapshot) will be summarized by last delay in IP Injection. The last delay in IP injection will be the delay in IP injection at Week 48, or the delay in last IP injection prior to Week 48 if a participant did not receive Week 48 injection (i.e. missing visit or withdrawal). The similar analysis will be done for Week 96 and Week 152 timepoints where the proportion of participants with HIV-1 RNA ≥50 c/mL at Weeks 96 and 152 (Snapshot) and the delay in IP injection at Weeks 96 and 152 are considered respectively.

### 15.6.4. Safety

#### **Adverse Events**

## **DAIDS Grading**

 Clinical adverse events will be graded based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.1, March 2017, as specified in the protocol Appendix 11.2.

## Potential QTc Interval Prolonging Events of Interest

Potential QTc Interval Prolonging Events of Interest will be identified based on Standardised MedDRA Query (SMQ) for Torsade de pointes/QT prolongation, broad (MedDRA). The terms per this reference are listed below.

| AE preferred term |
|----------------------------------------------|
| Electrocardiogram QT interval abnormal |
| Electrocardiogram QT prolonged |
| Long QT syndrome |
| Long QT syndrome congenital |
| Torsade de pointes |
| Ventricular tachycardia |
| Cardiac arrest |
| Cardiac death |
| Cardiac fibrillation |
| Cardio-respiratory arrest |
| Electrocardiogram repolarisation abnormality |
| Electrocardiogram U wave inversion |
| Electrocardiogram U wave present |
| Electrocardiogram U-wave abnormality |
| Loss of consciousness |
| Sudden cardiac death |
| Sudden death |
| Syncope |
| Ventricular arrhythmia |
| Ventricular fibrillation |
| Ventricular flutter |
| Ventricular tachyarrhythmia |

## **Laboratory Parameters**

• If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to

### **Laboratory Parameters**

determine how much to add or subtract in order to impute the corresponding numeric value. If a character value starting with "<=x", then the numeric value will be x.

- Example 1: 2 Significant Digits = '< x ' becomes x 0.01
- Example 2: 1 Significant Digit = '> x' or '>=x' becomes x + 0.1
- Example 3: 0 Significant Digits = '< x' becomes x 1</li>

#### Estimate of Glomerular Filtration Rate (GFR) (Levey, 2012)

• Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation [Levey, 2012] will be used by the central laboratory to provide an estimate of GFR, in mL/min per 1.73 m², as follows:

$$GFR = 141 \times min \left(\frac{CRT_{mg/dL}}{\kappa}, 1\right)^{\alpha} \times max \left(\frac{CRT_{mg/dL}}{\kappa}, 1\right)^{-1.209} \times 0.993^{Age} \times [1.018 \text{ if Female}] \times [1.159 \text{ if Black}]$$

where age (in years) is at time of assessment,  $\kappa$  = 0.7 if female or 0.9 if male,  $\alpha$  = -0.329 if female and -0.411 if male, min() indicates the minimum of CRT/ $\kappa$  or 1, max() indicates the maximum of CRT/ $\kappa$  or 1, and CRTmg/dL is serum creatinine concentration in mg/dL. The serum creatinine concentration in mg/dL is obtained from GSK standard units of  $\mu$ mol/L as CRTmg/dL =0.0113x CRT $\mu$ mol/L.

The CKD-EPI GFR will also be calculated using Cystatin C, as follows

133 X min(Scys/0.8, 1) -0.499 X max (Scys/0.8, 1)-1.328 X 0.996 Age X[0.932 if female]

Where Scys is serum cystatin C mg/Liter, min indicates the minimum of Scr/0.8 or 1, and max indicates the maximum of Scys/0.8 or 1.

**Lab Toxicities – DAIDS Grading based on** Version 2.1, March 2017, as specified in the protocol of Appendix 11.2.

- Toxicities will be based on the Division of AIDS (DAIDS) grading system, Version 2.1, March 2.17, as specified in the protocol of Appendix 11.2
- Toxicity grades provided by the central laboratory do not distinguish between abnormally high or low criteria, when both are relevant for a parameter.
- When summarising toxicity grades for such parameters, they will be categorised as to whether they are above or below the midpoint of normal range.

| Parameter | Below Midpoint for those ≥Grade 1 | Above Midpoint for those ≥Grade 1 |
|---|---|---|
| Fasted glucose | Hypoglycemia | Hyperglycemia |
| Sodium | Hyponatremia | Hypernatremia |
| Potassium | Hypokalemia | Hyperkalemia |

#### National Cholesterol Education Program (NCEP) Lipid Categories

 In addition to DAIDS toxicity grades (see protocol), lipid values will be categorized according to the 2001 NCEP Adult Lipid Guidelines [Grundy, 2001]

| boratory Parameters | | | |
|---|---|---|---|
| Parameter | Value Range (mmol/L) | Value Range (mg/dL) | Category |
| Triglycerides | <1.70 | <150 | Normal |
| | 1.70 to <2.26 | 150 to <200 | Borderline High |
| | 2.26 to <5.65 | 200 to <500 | High |
| | ≥5.65 | ≥500 | Very High |
| Total Cholesterol | <5.18 | <200 | Desirable |
| | 5.18 to <6.21 | 200 to <240 | Borderline High |
| | ≥6.21 | ≥240 | High |
| HDL Cholesterol | <1.04 | <40 | Low |
| | 1.04 to <1.56 | 40 to <60 | Normal |
| | ≥1.56 | ≥60 | High |
| LDL Cholesterol | <2.59 | <100 | Optimal |
| | 2.59 to <3.37 | 100 to <130 | Near/Above Optimal |
| | 3.37 to <4.14 | 130 to <160 | Borderline High |
| | 4.14 to <4.92 | 160 to <190 | High |
| | ≥4.92 | ≥190 | Very High |

## Percentage change for lipids

The percentage change from baseline is calculated as:

% change from baseline =  $\frac{\text{value at Week 48 or 96-baseline value}}{\text{baseline value}} \times 100\%$ 

#### **Total Cholesterol / HDL Cholesterol Ratio**

When both total cholesterol and HDL cholesterol results are available from the same date for a
participant, then the ratio will be calculated by dividing the total cholesterol result by the HDL
cholesterol result. The ratio can be classified as follows:

| Parameter | Value Range |
|-------------------|--------------|
| Total Cholesterol | < 3.5 |
| / HDL Ratio | 3.5 to < 4.4 |
| | 4.4 to < 5 |
| | ≥5 |

## **Other Safety Endpoints**

### Corrected QT (QTc)

When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.

If RR interval (in msec) is provided then missing QTcB and/or QTcF will be derived as

$$QTcB = \frac{QT}{\sqrt{RR/1000}} \qquad \qquad QTcF = \frac{QT}{\sqrt[3]{RR/1000}}$$

where uncorrected QT interval is also measured in msec.

### Other Safety Endpoints

If RR interval is not provided directly and one of QTcB or QTcF has been entered, then RR interval can be obtained from the above formulas and used to calculate the other correction method value; i.e.,

$$QTcB = \sqrt{\frac{QTcF^{3}}{QT}} \qquad \qquad QTcF = \sqrt[3]{QT \cdot QTcB^{2}}$$

#### **Extent of Exposure**

- Exposure to CAB+RPV (oral lead-in or oral bridging) and CAB LA+RPV LA will be calculated from the IP eCRF pages.
- For Maintenance Phase:
  - Exposure to oral CAB+RPV (oral lead-in) = IP (oral lead-in) stop date IP (oral lead-in) start date +1
  - Exposure to CAB LA + RPV LA = Number of IP injection visits received during maintenance phase (up to but not including injections administered at Week 100)
  - Exposure to SOC oral bridging: Duration of the SOC ART medication taken as oral bridging during the Maintenance Phase. If the SOC oral bridging is taken in different periods during the Maintenance Phase, the duration will be calculated by the sum of the non-overlapped periods.
  - Exposure to CAB+RPV oral bridging: Duration of the CAB+RPV taken as oral bridging during the Maintenance Phase. If the CAB+RPV oral bridging is taken in different periods during the Maintenance Phase, the duration will be calculated by the sum of the non-overlapped periods.
  - Overall exposure to study treatment:
     For participants on Q4W arm: min [Date of Latest Maintenance Phase Visit up to and including Week 100, max (Date of Last Injection + 35, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] min (Start Date for Oral lead-in CAB+RPV, Date of First Study Injection) + 1
     For participants on Q8W arm: min [Date of Latest Maintenance Phase Visit up to and including Week 100, max (Date of Last Injection + 63, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] min (Start Date for Oral lead-in CAB+RPV, Date of First Study Injection) + 1
  - Overall exposure to IP = Overall exposure to Study Treatment Exposure to SOC Oral Bridging
- For Maintenance + Extension Phase
  - Exposure to CAB LA + RPV LA = Number of IP injection visits received during Maintenance Phase and Extension Phase
  - Exposure to SOC or CAB+RPV oral bridging during the Maintenance and Extension Phase will be calculated similarly to that during the Maintenance Phase except that the exposure includes both Maintenance and Extension Phase.
  - Overall exposure to study treatment:

#### **Other Safety Endpoints**

For participants on Q4W arm: min [Date of Latest Maintenance/Extension Phase Visit, max (Date of Last Injection + 35, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] – min (Start Date for Oral lead-in CAB+RPV, Date of First Study Injection) + 1

For participants on Q8W arm: min [Date of Latest Maintenance/Extension Phase Visit, max (Date of Last Injection + 63, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] – min (Start Date for Oral lead-in CAB+RPV, Date of First Study Injection) + 1

- Overall exposure to IP = Overall exposure to Study Treatment Exposure to SOC Oral Bridging
- For Thigh Injection Phase
  - Exposure to CAB LA + RPV LA = Number of IP injection visits received during Thigh Injection Phase. Note that the planned Sub-study Week 16 injections belong to Return to Gluteal Injection Phase.
  - o The SOC or CAB+RPV oral bridging are not allowed in this phase.
  - Overall exposure to IP:

For participants on Q4W arm: min [Date of Latest Thigh Injection Phase Visit up to the Nominal Sub-study Week 16 Visit Date, max (Date of Last Injection + 35, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] – Date of First Thigh Injection) + 1

For participants on Q8W arm: min [Date of Latest Thigh Injection Phase Visit up to the Nominal Sub-study Week 16 Visit Date, max (Date of Last Injection + 63, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] – Date of First Thigh Injection + 1

Note that the Nominal Sub-study Week 16 visit date is defined in Section 15.6.1.

- Overall exposure to IP = Overall exposure to Study Treatment.
- For Thigh Injection + Return to Gluteal Injection Phase
  - Exposure to CAB LA + RPV LA = Number of IP injection visits received during Thigh Injection or Return to Gluteal Injection Phase. Note that the injections received on the date of Sub-study Week 24 visit belong to the Extension Phase in main study.
  - The SOC or CAB+RPV oral bridging are not allowed in these two phases.
  - Overall exposure to IP:
    - For participants on Q4W arm: min [End of Sub-study Date, max (Date of Last Injection + 35, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] Date of First Thigh Injection) + 1
    - For participants on Q8W arm: min [End of Sub-study Date, max (Date of Last Injection + 63, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] Date of First Thigh Injection + 1
    - Note that the End of Sub-study Date is defined in Section 15.6.1.
  - Overall exposure to IP = Overall exposure to Study Treatment.
- Last Injection and/or Last Dose of Oral CAB+RPV and/or Last Dose of SOC Oral Bridging are only applicable to those who permanently discontinued study treatment.

#### **Other Safety Endpoints**

- Duration of dosing in participant years will be calculated as the sum of participant duration of dosing in days (across all participants)/365.25
- Participants who were randomized but did not report an IP start date will be categorised as having zero days of exposure.

## Adherence to CAB/RPV Injection Schedule

Timeliness of Injections relative to Date of Projected Dosing Visits are assessed by using "actual injection visit date - projected visit date from first injection". The injections of interest in adherence analysis are those after first injection. For participants requiring the oral CAB+RPV lead-in, the first injection is planned to be taken at Week 4B. For participants not requiring the oral CAB+RPV lead-in, the first injection is planned to be taken at Baseline/Day 1. For participants receiving the oral bridging and then returning to injections, if the first injection upon return is a reloading dose injection, the immediate next injection visit is planned to be four weeks after the reloading injection visit. If a participant has multiple oral bridging episodes, he or she may have more than one reloading dose injection visits during the study. Each injection visit is counted only once. Individual CAB and RPV injections administered at the same visit are not counted twice. "Extra" unscheduled injections are excluded from all derivations. For example, if during a scheduled visit a participant receives 1 ml of injection instead of 2 ml due to a dosing error, but this participant returns one week later for the remaining 1 ml injection, then the additional visit is excluded. If a participant receives an extra injection at an unscheduled visit by mistake, this visit will also be excluded.

The categories of Timeliness of Injections relative to Date of Projected Dosing Visits for summary are listed below:

```
-14 to -8 days

-7 to -4 days

-3 to -2 days

-1 day

0 day

1 day

2 to 3 days
```

< -14 days

4 to 7 days

8 to 14 days

>14 days

Missed Reloading Injection (Non-COVID-19)

Missed Reloading Injection (COVID-19)

Missed Injection w/o OB (Non-COVID-19)

Missed Injection w/o OB (COVID-19)

Missed Injection with CAB+RPV OB (Non-COVID-19)

Missed Injection with CAB+RPV OB (COVID-19)

### **CONFIDENTIAL**

207966

## **Other Safety Endpoints**

Missed Injection with SOC OB (COVID-19)

## Columbia Suicide Severity Rating Scale (C-SSRS)

Missing data will not have any imputation performed (Nilsson, 2013).

#### 15.6.5. Pharmacokinetic

This document is intended for planning analysis of PK concentration data and PK parameters only. Population pharmacokinetics and identification of important determinants of variability will be described in a separate document.

#### **Pharmacokinetic Analyses**

#### Plasma CAB and RPV Concentration-time Data

Plasma samples for determination of CAB and RPV concentration will be collected throughout the Maintenance Phase, at Week 152 and at the withdrawal visit in the main study, and up to Week 17 in the sub-study. Additional samples will be collected for storage during the Long-Term Follow-Up Phase and for female participants who become pregnant during the study.

In rare occasions, PK samples are collected post-dose on the same day as the study treatment administration during the main study. The data from these PK samples will be excluded from the pre-dose and/or 1-week post-dose summaries in the main study. If time was not collected for the oral study treatment, the PK sample collected on the same day as the oral study treatment is assumed to be taken prior to the oral dose unless medical monitor or data querying informs otherwise.

PK data collected for liver event will be listed but will not be included in the summaries or figures.

#### Plasma CAB and RPV PK Parameters

The following PK parameters will be determined from the sub-study concentration-time data for each treatment, analyte and dosing interval, as data permit: maximum concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve through the end of the dosing interval (AUC(0-tau)). These PK parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin 8.3. All calculations of non-compartmental parameters will be based on actual sampling times. Derivation of PK parameters will be performed by, or under the direct auspices of, Clinical Pharmacology Modelling and Simulation (CPMS), GlaxoSmithKline.

In addition, the concentration at the end of a dosing interval (Ctau) will be obtained from the evaluable pre-dose (trough) concentration collected at start of the subsequent interval. For example, the Ctau for last thigh injection interval will be obtained from the evaluable pre-dose PK concentration collected at the Sub-study Week 16 visit.

| Treatment Arm | Dosing Interval in Sub-study | | |
|---|---|---|---|
| | Gluteal Injection | First Thigh Injection | Last Thigh Injection |
| Q8W | Week -8 to Day 1 | Day 1 to Week 8 | Week 8 to Week 16 |
| Q4W | Week -4 to Day 1 | Day 1 to Week 4 | Week 12 to Week 16 |

#### **Evaluable Concentration**

#### **Pharmacokinetic Analyses**

PK concentration will be summarized in two ways: 'all data' without regard to timing relative to scheduled time and 'evaluable data'.

The 'evaluable data' are from the samples that met sample collection window criteria. Sampling windows are set relative to the previous dose as follows:

- 20-28 hrs after last oral dose taken and properly administered last 3 oral doses for pre-dose sample at Week 4B for participants requiring oral lead-in
- ± 4 days for pre-dose sample at visits other than Week 4B, and for pre-dose samples at Week 4B for participants not requiring oral lead-in (e.g. participants transitioning from ATLAS Q4W and remain on Q4W arm in this study)
- 3-10 days post last injection for 1-week post injection visits
- 21-35 days post last injection for 4-week post-dose samples (e.g. collected at substudy Week -4, Week 4 and Week 12 visits). Note that 4-week post-dose samples will be collected from subjects on Q8W arm only.
- 1-3 hours post last injection for 2-hour post-dose samples
- Samples impacted by dosing errors (wrong dose) or oral bridging will also be excluded

| Timepoint | Evaluable<br>Window | For Programming: |
|---|---|---|
| Pre-dose: WK4B<br>for participants<br>requiring oral<br>lead-in | 20-28 hrs after last oral dose taken and the last 3 oral doses administered properly | 20 hrs ≤ Time since Last Oral Dose ≤ 28 hrs and the last 3 oral doses administered on the three consecutive days prior to WK4B. |
| Pre-dose at other visits, Pre-dose WK4B for participants not requiring oral lead-in | ± 4 days | For Q4W arm, Day 1 pre-dose, Week 8 for those transitioning from SOC (i.e. requiring oral lead-in), and the immediate next visit after reloading on Q8W arm: 24 days ≤ Days Since Last Injection ≤ 32 days For visits other than above on Q8W arm: 52 days ≤ Days Since Last Injection ≤ 60 days |
| 1-WK-Post: | 3-10 days post last injection | 3 days ≤ Days Since Last Injection ≤ 10 days |
| 4-WK-Post: | 21-35 days<br>post last<br>injection | 21 days ≤ Days Since Last Injection ≤ 35 days |
| 2-HR-Post: | 1-3 hours post last injection | 1 hr ≤ Time since Last Oral Dose ≤ 3 hrs |

Relative Time is calculated relative to the date and time of last dose. For example, if the time of the last dose (e.g. oral lead-in/oral bridging) is missing, then the relative time for PK sample will be set to missing and the sample will not be considered 'evaluable'.

#### **Pharmacokinetic Analyses**

If a pre-dose sample is collected on the same day as the first dose of oral bridging, the time of the first dose (not recorded in eCRF) is assumed to be 'after' the collection of pre-dose sample, unless medical monitor or Data querying informs otherwise.

The time-deviation (hours) from the targeted timepoint will be calculated for the post-dose samples using the following formula:

Time\_deviation (hrs) for '2-Hour POST' = Sample date.time - last injection date.time - 2 hours

Time\_deviation (hrs) for '1-Week POST' = Sample date.time - last injection date.time - 7\*24 hours

Time\_deviation (hrs) for '4-Week POST' = Sample date.time - last injection date.time - 28\*24 hours

The following windows are for defining 'evaluable' Long-term Follow-up phase PK concentrations.

| Timepoint | Evaluable Window | For Programming: |
|---|---|---|
| LTFU MONTH<br>1/WD | ± 4 days | 24 days ≤ Days Since Last Injection ≤ 32 days |
| LTFU MONTH 3 | ± 1 Weeks | 77 days ≤ Days Since Last Injection ≤ 91 days |
| LTFU MONTH 6 | ± 2 Weeks | 154 days ≤ Days Since Last Injection ≤ 182 days |
| LTFU MONTH 9 | ± 2 Weeks | 238 days ≤ Days Since Last Injection ≤ 266 days |
| LTFU MONTH 12 | ± 2 Weeks | 322 days ≤ Days Since Last Injection ≤ 350 days |

#### 15.6.6. Health Outcomes





## **Total Treatment Satisfaction Score (change)**

- Total Treatment Satisfaction Score is computed with items 1-11. Items 1-11 are summed to produce a score with a possible range of -33 to 33
- Item 12 will be computed as an individual item only.
- The higher the score, the greater the improvement in satisfaction with treatment; the lower the score, the greater the deterioration in satisfaction with treatment. A score of columns are stated in the score of columns are stated in the score of columns.
- A maximum of 5 items can be missing, the missing scores will be imputed with the mean of the
  completed item scores. If 6 or more items are missing, then the overall treatment satisfaction
  scale score should not be computed and will remain missing.

## **Individual Treatment Satisfaction Change Item Scores**

- Items are rated as +3 CCI
- The higher the score, the greater the improvement in satisfaction with each aspect of treatment and the lower the score, the greater the deterioration in satisfaction with each aspect of treatment.

#### **Questionnaire Version**

to -3 CCI

- In main study, three versions of the HIVTSQc questionnaire are available with the questions the same and only the overhead text is different.
  - Q4W ATLAS to Q4W ATLAS-2M: for participants who randomized to Q4W arm in ATLAS and then randomized to Q4W arm in ATLAS-2M
  - Q4W ATLAS to Q8W ATLAS-2M: for participants who randomized to Q4W arm in ATLAS and then randomized to Q8W arm in ATLAS-2M
  - SOC to Q4W or Q8W ATLAS-2M: for participants who either were randomized to SOC arm in ATLAS or did not participate in ATLAS
- If a participant takes a wrong version of the questionnaire in main study, the data collected from the wrong version will be considered invalid and will not be included in the summary.
- In sub-study, all participants will take the same version of the questionnaire.

#### PIN

Questionnaire (Each question is scored 1-5)

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by this |
|---|
| arty copyright laws and therefore have been excluded. |
| Dimension Score (Chevat, 2008) |
| Domains and Clusters |
| O CCI |
| O CCI |
| 5 items not included in any of these domains and maintained as individual items (items |
| No everall ecore is calculated per the guidence |
| No overall score is calculated per the guidance The course of a developing is calculated as the group of all items with the develop. High an accusa- |
| The score of a domain is calculated as the mean of all items with the domain. Higher scores |
| represent worse perception of injection. |
| A maximum of <50% items can be missing within a domain, which can be imputed to reflect the |
| mean of the completed item scores within the domain. Thus, if the number of missing items is |
| ≥3 <mark>cci ), ≥2 cci ), ≥1 cci , then the</mark> |
| total score for the domain should not be computed and instead be imputed using LOCF |
| (Section 15.7.2.2) |
| Individual Item Scores |
| Items are rated on a 5-point scale, ranging from 1(CC) to 5 (CC) |

etc.).

- Lower scores represent worse perception of injection
- For individual item scores outputs, missing scores will not be computed and instead be imputed using LOCF (Section 15.7.2.2).

HAT-QoL (Holmes, 1999)

Questionnaire (Questions 1-14 are scored 1 to 5)



## Life satisfaction, HIV medications, disclosure worries

The ratings for Items (a, b, c, d, e) will be recoded as below for analysis:
 Response option
 Life Satisfaction
 Medication/disclosure worries

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

A maximum of 50% question items can be missing within a domain, which can be computed and replaced with the mean of the completed item scores within the domain. Thus, if there are more than 1 item missing for Life Satisfaction, and more than 2 items missing for

Medication/disclosure worries, then the total score for the domain should not be computed and instead be imputed using LOCF (Section 15.7.2.2). A computed score for missing value will be added to calculate a total score for the domain. Total score for each of the three domains will be calculated and will be denoted as 'LISAT' for life satisfaction, 'MEDWO' for medication worries, and 'DISWO' for disclosure worries.

 Transform each dimension's total imputed value score to the 0-100 scale using the following formulae:

Life satisfaction: LISAT100=(100/(20-4))\*(LISAT-4)

Medication worries: MEDWO100=(100/(25-5))\*(MEDWO-5) Disclosure worries: DISWO100=(100/(25-5))\*(DISWO-5)

The higher the score, the greater satisfaction to life and the less worry. The transformed dimension score for each domain will be summarized and analysed.

#### Individual Item Scores

 For individual item scores outputs, missing scores will not be computed and instead be imputed using LOCF (Section 15.7.2.2).

## ACCEPT (Acceptance/General Dimension) (Gilet, 2014)

Questionnaire (Questions 1-3 constitute to Acceptance/General Dimension)

third party copyright laws and therefore have been excluded.

Proportion of participants with individual item scores will be calculated.

#### Individual Item Scores

• Items are rated as 1 ccl . and '5' with ccl

- Acceptance/General dimension score is calculated only if at least 2 items in the dimension are completed
- Items will be recoded to score as follows:

| Rating | Recode |
|-----------------------------------------------------------------|--------|
| Totally disagree/Not at all acceptable/ Not at all convinced: | 1 |
| 2. Somewhat disagree/Not very acceptable/ Not really convinced: | 1 |
| 3. Somewhat agree/ Somewhat acceptable/ Somewhat convinced: | 2 |
| 4. Totally agree/ Totally acceptable/ Totally convinced: | 3 |
| 5. I don't know: | 1 |

 The total score of the dimension is calculated as the mean of the recoded items of the dimension and then linearly transformed to be on a scale from 0 to 100: score, as below:

Total Score = (mean of the recoded items in the dimension - 1)/2 \*100

For individual item scores outputs, missing scores will not be computed and instead be imputed

using LOCF (Section 15.7.2.2). **Preference** Questionnaire 1. Based on your experience which HIV treatment do you prefer?

□ Injectable Long-Acting HIV Treatment every 4 weeks

□ Injectable Long-Acting HIV Treatment every 8 weeks (only select this answer if you received the 8-week injectable regimen of CAB LA + RPV LA during study)

□ Oral daily HIV Treatment

□ No preference

If you selected no preference, skip questions 2 and 3.

If you selected any other response, please continue and complete all questions.

What is the main practical attribute of this HIV therapy supporting your preference?

Mode of administration

□ Frequency of administration

Time required for administration

Scheduling visits

Storing medications

□ Impact of side effects

□ Other, please specify

3. What is the main benefit related to this HIV therapy supporting your preference?

□ More convenient, easier to integrate into one's daily life

□ Less stressful

□ Less stigma

Easier to take the drug exactly as prescribed

More efficacious

□ Other, please specify

#### **Questionnaire Version**

- Two versions of questionnaire are available. The questions in each version of the questionnaire are the same and only the overhead text is different.
  - ATLAS (from Q4W ATLAS): for participants randomized to Q4W arm in ATLAS.
  - ATLAS-2M (from SOC ATLAS or out): for participants who either were randomized to SOC arm in ATLAS or did not participate in ATLAS.

#### Data Handling

Any missing values will remain missing (i.e. no imputation).

### Reasons for Oral Bridging and Preference

#### Questionnaire

This questionnaire will be administered to participants receiving oral bridging during the Maintenance and/or Extension phase. It includes three questions regarding contact mode, main reasons for switch back to daily oral HIV medication and the HIV treatment preference. For the preference question, it asks participants to provide the statements supporting their preference. The details can be found in the eCRF.

#### **Data Handling**

Any missing values will remain missing (i.e. no imputation).

#### **Preference Thigh Injection vs Gluteal Injection**

#### Questionnaire

This questionnaire will be administered to sub-study participants. It includes two questions regarding injection site preference and contact mode. For the preference question, it asks participants to provide the statements supporting their preference. The details can be found in the eCRF.

## **Data Handling**

• Any missing values will remain missing (i.e. no imputation).

#### **Tolerability of Injection (NRS)**

#### Questionnaire

• This questionnaire will be administered to sub-study participants. It includes two questions regarding the maximum level of pain experienced with the most recent injections and contact mode. The score for the maximum level of pain ranges from no pain (0) to extreme pain (10).

## **Data Handling**

Any missing values will remain missing (i.e. no imputation).

#### Reasons for Continuation/Switch

#### Questionnaires

- Reasons for Continuation questionnaire is collected for participants who were randomized to Q4W arm in ATLAS.
- Reason for Switch questionnaire is collected for participants who either were randomized to SOC arm in ATLAS or did not participate in ATLAS.

## **Data Handling**

- If a participant takes a wrong questionnaire, for example, the participant randomized to SOC arm in ATLAS took Reasons for Continuation questionnaire, the data collected from this wrong version will be considered invalid and will not be included in the summary.
- If the questionnaire is taken beyond ± 2 weeks window from maintenance phase treatment start date (i.e. Study Day < -14 or Study Day > 14) will be consider not evaluable and will not be included in the summary.
- Any missing values will remain missing (i.e. no imputation).

#### 15.6.7. Virology

#### Genotype

#### **Amino Acid Changes**

- A mutation is considered present whenever the encoded amino acid residue differs from the amino acid that would have been encoded by the wild-type (e.g., HXB2, NL43) comparator gene; e.g., Q148K.
- If the encoded amino acid is seen as a mixture of wild-type and mutant amino acid, e.g., Q148Q/K, the mutated amino acid is considered present at the codon of interest.
- If the encoded amino acid is seen as a mixture of two or more amino acids, which may or may not include wild type, e.g., Q184K/H or Q184K/H/Q, etc., for the purposes of calculating the number of mutated amino acids, only one mutation is considered to be present at the codon of

interest.

### **Representation of Amino Acid Changes**

| Mutations | Amino acid change |
|---|---|
| T69S | Single mutation from amino acid 'T' (vendor reference) to 'S' (sample) at codon '69' |
| Q148H/K/R | Mixture of amino acid mutations 'H', 'K' and 'R' (sample) from amino acid 'Q' |
| | (vendor reference) at codon '148' |
| _69_1T | First insertion of amino acid 'T' (sample) at codon '69' |
| _69_2S | Second insertion of amino acid 'S' (sample) at codon '69' |
| _69_3S/A | Third insertion of a mixture of amino acids 'S' and 'A' (sample) at codon '69' |
| L74L/- | Mixture of amino acid 'L' (sample) and a deletion at codon '74' |
| V75- | Single deletion of amino acid (sample) at codon '75' |

#### **Resistance Associated Mutations**

 Known INI mutations associated with the development of resistance to CAB, BIC, RAL, EVG or DTG:

| Amino Acids in<br>HIV Integrase for<br>Analysis | H51Y, <b>T66A/I/K</b> , <b>E92Q/V</b> /G, Q95K, T97A, <b>G118R</b> , <b>F121C/Y</b> , E138A/K/T, G140A/C/ <b>R</b> /S**, <b>Y143C/H/R/K/S/G/A</b> , <b>P145S</b> , <b>Q146P</b> , <b>S147G</b> , <b>Q148H/K/R/</b> N, <b>V151</b> A/L, S153F/Y, <b>N155H</b> /S/T, E157Q, G163R/K, S230R, R263K, |
|---|---|
| , | L68V/I*, L74I/M*, E138D*, V151I*, G193E* |

#### NOTES:

- Draft listing; may be modified in case of additional substantive data availability.
- INI mutations listed taken from Stanford HIV Resistance Database (<a href="http://hivdb.stanford.edu/DR/cgi-bin/rules\_scores\_hivdb.cgi?class=INI">http://hivdb.stanford.edu/DR/cgi-bin/rules\_scores\_hivdb.cgi?class=INI</a> cited 22Feb2021) and accessed on 28Mar2022.
- INI substitutions listed above in bold had a score of =60.
- \* Denotes additional INI mutations added as they were identified during in vitro passage of DTG or seen in a previous DTG study in INI-experienced participants (ING112574).
- \*\*G140R is potentially associated with CAB based on in-stream data monitoring of CVF participants.
- Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA). The most up to date IAS-USA guidelines available at the time of DBL will be used in the analysis [Wensing, 2019].

| Class | Major Mutations |
|---|---|
| NRTIs | M41L, A62V, K65R/E/N, D67N, 69 insert, K70E/R, L74V, V75I, F77L, Y115F, F116Y, |
| | Q151M, M184V/I, L210W, T215Y/F, K219Q/E |
| NNRTIs | L100I, K101E/P, K103N/S, V106A/M, V108I, E138/A/G/K/Q/R, V179L, |
| | Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L |
| Pls | D30N, V32I, M46I/L, I47A/V, G48V, I50V/L, I54M/L/V, Q58E, T74P, L76V, |
| | V82A/T/F/L/S, N83D, I84V, N88S, L90M |

Note: List generated from IAS USA Guideline, [Wensing, 2019]

- The pre-specified INSTI Mutations are identified as below:
  - Per the IAS-USA list of mutations associated with resistance to Bictegravir, Cabotegravir, Dolutegravir, Elvitegravir, or Raltegravir (IAS-USA 2019 resistance mutations update volume 27 issue 3, 2019): T66A/I/K, L74M, E92Q/G, T97A, G118R, F121Y, E138A/K/T, G140A/C/R/S, Y143C/H/R, S147G, Q148H/K/R, S153F/Y, N155H, R263K

- Observed mutations during in vitro passage of DTG or seen in a previous DTG study in INI-experienced subjects (study ING112574): H51Y, L74I, L68V/I, E92V, Q95K, E138D, Y143K/S/G/A, P145S, Q146P, V151I/L/A, N155S/T, E157Q, G163R/K, G193E, S230R
- Mutations per FDA request for Study 201584: Q146L, T124A
- The NNRTI resistance associated mutations (RAMs) are identified per IAS-USA NNRTI mutations (IAS-USA 2019 resistance mutations update volume 27 issue 3, 2019):
  - V90I, A98G, L100I, K101E/H/P, K103N/S, V106A/I/M/T, V108I, E138A/G/K/Q/R, V179D/F/L/T, Y181C/I/V, Y188C/H/L, G190A/E/S, H221Y, P225H, F227C/L/R, M230I/L, L234I
- The RPV RAMs are identified per IAS-USA NNRTI mutations (IAS-USA 2019 resistance mutations update volume 27 issue 3, 2019):
  - L100I, K101E/P, E138A/G/K/Q/R, V179L, Y181C/I/V, Y188L, H221Y, F227C, M230I/L

#### Phenotype

#### Phenotypic Susceptibility

Phenotypic susceptibility to all licensed antiretroviral drugs and CAB will be determined using PhenoSense HIV assays from Monogram Inc. and will be reported as fold change (FC) in IC50 relative to wild-type control virus NL4-3, i.e., FC of sample virus = IC50 of sample virus/IC50 of control virus.

Phenotypic susceptibilities will be categorised according to FC as shown in tables below (based on Monogram PhenoSense assay). Clinical cutoffs (where available) or biological cutoffs by PhenoSense will be used to define the phenotypic susceptibility of background treatment by Monogram.

Replication capacity is generated as part of standard phenotypic assays.

## PhenoSense Algorithm

| Drug | Abbreviation | Class | PhenoSense cutoff |
|-----------------|--------------|-------|--------------------------|
| Abacavir | ABC | NRTI | (4.5 – 6.5) <sup>a</sup> |
| Lamivudine | 3TC | NRTI | 3.5 a |
| Didanosine | ddl | NRTI | (1.3 – 2.2) a |
| Stavudine | d4T | NRTI | 1.7 a |
| Zidovudine | AZT (ZDV) | NRTI | 1.9 |
| Emtricitabine | FTC | NRTI | 3.5 |
| Tenofovir | TDF (TAF) | NRTI | (1.4 – 4) <sup>a</sup> |
| Delavirdine | DLV | NNRTI | 6.2 |
| Efavirenz | EFV | NNRTI | 3 |
| Nevirapine | NVP | NNRTI | 4.5 |
| Etravirine | ETR | NNRTI | (2.9-10) a |
| Rilpivirine | RPV | NNRTI | 2.0 |
| Doravirine | DOR | NNRTI | 3 |
| Fosamprenavir/r | FPV/r | PI | (4-11) a |
| Atazanavir | ATV | PI | 2.2ª |
| Atazanavir/r | ATV/r | PI | 5.2 a |
| Indinavir/r | IDV/r | PI | 10 a |
| Lopinavir/r | LPV/r | PI | (9 – 55) <sup>a</sup> |
| Nelfinavir | NFV | PI | 3.6 |

| Saquinavir/r | SQV/r | PI | (2.3 – 12) a |
|--------------|-------|-----|--------------|
| Tipranavir/r | TPV/r | PI | (2 – 8) a |
| Darunavir/r | DRV/r | PI | (10 – 90) a |
| Ritonavir | RTV | PI | 2.5 |
| Enfuvirtide | T20 | FI | 6.48 |
| Cabotegravir | CAB | INI | 2.5 |
| Raltegravir | RAL | INI | 1.5 |
| Elvitegravir | EVG | INI | 2.5 |
| Dolutegravir | DTG | INI | (4-13) a |
| Bictegravir | BIC | INI | (2.5- 10) |

a. clinical cutoff (lower cutoff – higher cutoff).

#### Phenotypic Susceptibility

Phenotypic susceptibility to each drug in a participant's background regimen is determined by applying drug-associated cutoffs as defined by the PhenoSense algorithm to the phenotypic fold resistance as below:

#### **Full Sensitivity**

| Fold Change | Interpretation |
|----------------------------------------------|----------------|
| > clinical lower cutoff or biological cutoff | resistant |
| ≤ clinical lower cutoff or biological cutoff | sensitive |

#### **Partial Sensitivity**

| Fold Change | Interpretation |
|------------------------------------------------------|---------------------|
| > clinical higher cutoff | resistant |
| ≤ clinical higher cutoff and > clinical lower cutoff | partially sensitive |
| ≤ clinical lower cutoff | sensitive |

PHENOTYP dataset from Monogram contains the phenotypic susceptibility for each drug derived from the cutoff listed above. Thus, phenotypic susceptibility (i.e. full sensitivity and partial sensitivity) will not be re-derived for our analysis.

#### **Genotypic and Net Assessment Susceptibility**

Genotypic and Net assessment susceptibility to all licensed antiretroviral drugs and CAB will be determined from Monogram Inc. Net assessment susceptibility will be reported with the categories of 'resistant', 'partially sensitive', and 'sensitive' as what will be performed for phenotypic susceptibility. Genotypic susceptibility will be reported with the categories of 'resistant', 'resistance possible' and 'sensitive'. Genotypic and Net assessment susceptibility will be assessed at time of CVF using plasma sample, Genotypic susceptibility may be assessed at baseline using PBMC.

## 15.7. Appendix 7: Reporting Standards for Missing Data

## 15.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as <ul> <li>Randomly assigned to either treatment group, completed the randomized Maintenance Phase including Week 100 and did not enter the Extension Phase;</li> <li>Randomly assigned to either treatment group, completed the randomized Maintenance Phase including Week 100, and entered and completed the Extension Phase (defined as remaining on study until commercial supplies of CAB LA + RPV LA Q4W or Q8W regimen become locally available or development of CAB LA + RPV LA is terminated).</li> </ul> </li> </ul> |
| | Participants who withdraw from CAB LA + RPV LA and go into the LTFU Phase, and participants who withdraw from oral lead-in will be considered to have prematurely withdrawn from the study treatment. |
| | In addition to the 52-week Follow-Up phase required for participants who receive one or more injections with CAB LA or RPV LA, an in-clinic Follow-Up visit will be conducted approximately 4 weeks after the last dose of study medication for participants who withdraw during the oral lead-in period with ongoing AEs, and serious adverse events (SAEs) and also any laboratory abnormalities that are considered to be AEs or potentially harmful to the participant, at the last on-study visit. Assessments at the Follow-up visit should reflect any ongoing complaints (e.g., blood draws to follow a laboratory abnormality). Follow-Up visits are not required for successful completion of the study. |
| | Withdrawn participants were not replaced in the study. |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures, unless<br/>otherwise specified.</li> </ul> |
| | <ul> <li>Withdrawal visits will be slotted as per Error! Not a valid result for table.: Assessment<br/>Windows or will be summarised as withdrawal visits.</li> </ul> |

## 15.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 15.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment State.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the last contact date; in this case the last contact date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| ART/Non-<br>ART<br>Medications<br>or Medical<br>History | <ul> <li>Partial dates recorded in the eCRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month. If medications recorded in the eCRF as prior (e.g. recorded in prior ART or prior ATLAS ART forms), the earlier date of the imputed and the day prior to the maintenance phase treatment start date will be used, i.e. min (imputed stop date, maintenance phase treatment start date - 1).</li> </ul> </li> <li>For medications with completely missing start date, they will be considered started prior to the maintenance phase treatment start date.</li> <li>For medications with completely missing stop date, they will be considered ongoing unless recorded in eCRF as prior (e.g. recorded in prior ART or prior ATLAS ART forms).</li> <li>For ART booster medications, the start and stop dates are not recorded in the database (i.e. missing), the dates will be imputed to be the same as the dates of their parent medications.</li> <li>The recorded partial or missing date will be displayed in listings.</li> </ul> |
| Health | For the health outcomes questionnaire data, please refer to Section 12. |
| outcomes | <ul> <li>For the summary of individual item scores outputs, missing scores will not be<br/>computed.</li> </ul> |

## 15.7.2.2. Handling of Missing data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Snapshot | <ul> <li>In the Snapshot dataset, participants without HIV-1 RNA data in the assessment<br/>window for the visit of interest (due to missing data or discontinuation of IP prior<br/>to the visit window) do not belong to 'HIV-1 RNA &lt; 50 c/mL (or &lt;200 c/mL)'.</li> </ul> |
| | The nature of this missing data will be further classified in Snapshot summaries as either 'HIV-1 RNA ≥ 50 c/mL' (or "HIV-1 RNA ≥ 200 c/mL') or 'No Virologic |
| | Data at Week X'; Appendix 9: Snapshot Algorithm Details for full details |
| LOCF | <ul> <li>In the LOCF dataset, missing values will be carried forward from the previous,<br/>non-missing available on-treatment assessment. If the baseline value is missing<br/>any missing values until the first non-missing value will remain missing.</li> </ul> |
| Lipid LOCF | Baseline for Lipids LOCF Analyses in main study: |
| | Last evaluable lipids assessment up to and including the start of IP, where<br>'evaluable' is defined as: Lipid-modifying agents not taken within 12 weeks of the date of assessment and Lipids are collected in a fasting state. |
| | During the Maintenance or Extension Phase: |
| | If participants initiate serum lipid-modifying agents during the Maintenance or Extension Phase, then the last available fasted on-treatment lipid values prior to the initiation will be used in place of future, observed on-treatment values. |
| | <ul> <li>Imputation at planned visits will continue even if the participant discontinues the<br/>lipid-modifying agent. Missing assessments will not be imputed if there is no<br/>last available fasting on-treatment lipid value prior to the initiation of serum lipid-<br/>modifying agent.</li> </ul> |
| | If participants take lipid modifying agents within 12 weeks prior to the start of the study treatment, all the post-baseline values will be missing. |
| | Baseline for Lipids LOCF Analyses in sub-study: |
| | Last evaluable lipids assessment up to and including the start of thigh injection, where 'evaluable' is defined as: Lipid-modifying agents not taken within 12 weeks of the date of assessment and Lipids are collected in a fasting state. |
| | During the Thigh Injection or Return to Gluteal Injection Phase: |
| | If participants initiate serum lipid-modifying agents during the Thigh injection or<br>Return to Gluteal Injection Phase, then the last available fasted on-treatment<br>lipid values prior to the initiation will be used in place of future, observed on-treatment values in sub-study. |
| | <ul> <li>Imputation at planned visits will continue even if the participant discontinues the<br/>lipid-modifying agent. Missing assessments will not be imputed if there is no<br/>last available fasting on-treatment lipid value prior to the initiation of serum lipid-<br/>modifying agent.</li> </ul> |
| | If participants take lipid modifying agents within 12 weeks prior to the start of the thigh injection, all the post-baseline values in sub-study will be missing. |
| | Analyses Evaluated with Lipid LOCF Dataset: |

| Element | Reporting Detail |
|---|---|
| | Week 48 analysis: |
| | This dataset will be used to summarize fasting lipids parameters in the following displays: |
| | Summary of Fasting TC/HDL ratio Change from Baseline |
| | Summary of Fasting Lipids Percentage Changes from Baseline |
| | Summary of Chemistry Changes from Baseline |
| | Summary of Chemistry Values |
| | All other displays of lipids (e.g. toxicity tables and NCEP tables) will use observed fasting data, without LOCF imputation. |
| | Post-Week 48 analysis: |
| | Lipid LOCF dataset will be used for all lipid analysis except for the Summary of Maximum Post-Baseline Emergent Chemistry Toxicities. |
# 15.8. Appendix 8: Values of Potential Clinical Importance

ECG values of potential clinical importance are defined as QTc > 500 msec or increase from baseline in QTc  $\geq$  60 msec.

#### 15.9. Appendix 9: Snapshot Algorithm Details

o HIV-1 RNA < 50 c/mL

#### **Detailed Algorithm Steps**

- Consider an analysis visit window for Week X as defined in Table 10 and Table 13.
- The HIV-1 RNA threshold of 50, 200 c/mL will be analysed, respectively, in this study
- The COVID-19 pandemic presents significant logistical challenges for many clinical sites around the world, with variable restrictions being placed on site resources and operations, and on an individual participants ability to attend clinic visits. The snapshot algorithm is modified to allow for the presentation of full scope of COVID-19 relatedness. The analysis window 'Week 48' and HIV-1 RNA threshold of '50 c/mL' are used for the purpose of illustration. A participant's Snapshot response and reason at Week 48 are categorized as below.

```
o HIV-1 RNA \geq 50 c/mL
  Data in window not below 50
    Non-COVID-19 related
         Discontinued for lack of efficacy
         Discontinued for other reason while not below 50
         Change in background therapy*
     COVID-19 related
         Discontinued for lack of efficacy
         Discontinued for other reason while not below 50
         Change in background therapy*
 No Virologic Data at Week 48 Window
     Non-COVID-19 related
         Discontinued study due to AE or death
         Discontinued study for other reasons
         On study but missing data in window
     COVID-19 related
         Discontinued study due to AE or death
         Discontinued study for other reasons
         On study but missing data in window
```

<sup>\*</sup> Note: since permanent change in ART are not permitted in this protocol, all such participants who permanently change ART will be considered 'HIV-1 RNA ≥ 50 c/mL' if the permanent change in ART is made prior to an analysis timepoint. Participants with protocol permitted temporary oral bridging treatment (CAB+RPV or SOC, the SOC oral bridging medication is permitted during COVID-19 pandemic due to the unavailability of the CAB/RPV IM injections and oral CAB+RPV) or a temporary change in ART by mistake prior to an analysis timepoint (e.g. participant took the ART different from study treatment during oral lead-in by mistake for a short period and then went back to the study treatment) will not be considered 'HIV-1 RNA ≥ 50 c/mL' due to 'change in ART'.

- The steps in determining response and reasons are indicated in the table below, in the order stated.
- Background therapy is not given to participants while on study. The "change in background therapy" in detailed steps below refers to the "change in ART" in this study.

#### **Detailed steps**

Please note that the following scenarios will NOT be penalized Per Snapshot algorithm (i.e. please exclude these scenarios from **Condition** 1-4).

- Dose reduction, dropping a component, or change in formulation (e.g. 'Tivicay + Kivexa' to 'Triumeq' with the identical ingredients)
- Protocol permitted temporary oral bridging, or temporary change in ART by mistake

| Protocol permitted temporary oral bridging, or temporary change in ART by mistake | | |
|---|---|---|
| Condition ('Week 48' indicates Week 48 window) | Response | Reasons |
| If non-permitted change in background therapy prior to Week 48 | | |
| 1.1. If the change in background therapy is not due to COVID-19 | HIV-1 RNA ≥ 50 | Change in background therapy (non-COVID-19 related) |
| 1.2. If the change in background therapy is due to COVID-19 | HIV-1 RNA ≥ 50 | Change in background therapy (COVID-19 related) |
| <ol> <li>If permitted change<sup>[a]</sup> in background therapy<br/>prior to Week 48 AND the latest on-treatment<br/>VL prior to/on the date of change is ≥ 50 c/mL<br/>(NA to this study)</li> </ol> | | |
| 2.1 If the change in background therapy is not due to COVID-19 | HIV-1 RNA ≥ 50 | Change in background therapy (Non-COVID-19 related) |
| 2.2 If the change in background therapy is due to COVID-19 | HIV-1 RNA ≥ 50 | Change in background therapy (COVID-19 related) |
| If non-permitted change in background therapy during Week 48 | | |
| <ul> <li>Last on-treatment VL during Week 48 prior<br/>to/on the date of change ≥ 50 c/mL</li> </ul> | HIV-1 RNA ≥ 50 | Data in window not below 50 |
| Last on-treatment VL during Week 48 prior<br>to/on the date of change < 50 c/mL | HIV-1 RNA < 50 | |
| <ul> <li>No VL during Week 48 prior to/on the date<br/>of change and the change in background<br/>therapy is not due to COVID-19</li> </ul> | HIV-1 RNA ≥<br>50 | Change in background therapy (Non-COVID-19 related) |

| <ul> <li>No VL during Week 48 prior to/on the date<br/>of change and the change in background<br/>therapy is due to COVID-19</li> </ul> | HIV-1 RNA ≥<br>50 | Change in background therapy (COVID-19 related) |
|---|---|---|
| <ol> <li>If permitted change<sup>[a]</sup> in background therapy<br/>during Week 48 AND the last on-treatment VL<br/>prior to/on the date of change is ≥ 50 c/mL (NA<br/>to this study)</li> </ol> | | |
| 4.1 This last on-treatment VL occurs prior to Week 48 | | |
| 4.1.1 The change in background therapy is not due to COVID-19 | HIV-1 RNA ≥<br>50 | Change in background therapy (Non-COVID-19 related) |
| 4.1.2 The change in background therapy is due to COVID-19 | HIV-1 RNA ≥<br>50 | Change in background therapy (COVID-19 related) |
| 4. 2 This last on-treatment VL occurs during Week 48 but prior to/on the date of change | HIV-1 RNA ≥<br>50 | Data in window not below 50 |
| 5. If none of the above conditions met | | |
| 5.1 On-treatment VL available during Week 48 | | |
| <ul> <li>Last on-treatment VL during Week 48</li> <li>≥ 50 c/mL</li> </ul> | HIV-1 RNA ≥<br>50 | Data in window not below 50 |
| <ul> <li>Last on-treatment VL during Week 48</li> <li>&lt; 50 c/mL</li> </ul> | HIV-1 RNA <<br>50 | |
| 5.2 No on-treatment VL during Week 48 | | |
| 5.2.1 If participants are still on study, i.e. a participant has not permanently discontinued the study treatment yet, or if a participant permanently discontinued the study treatment and the upper bound of analysis snapshot window is prior to the following date: Q8W arm: Min[max(Date of last injection + 63, Date of Last Dose of Oral Study Treatment (CAB+RPV, SOC Bridging + 1), Withdrawal | | |
| Date, LTFU ART Start Date] Q4W arm: Min[max(Date of last injection + 35, Date of Last Dose of Oral Study Treatment (CAB+RPV, SOC Bridging) + 1), Withdrawal Date, LTFU ART Start Date] , where 'Withdrawal Date' refers to the date the participant failed to complete or completed per study conclusion form. | | |

| 5.2.1.1 If no on-treatment VL during Week 48 is not due to COVID-19 | No virologic<br>data at Week | On study but missing data in |
|---|---|---|
| | 48 Window | window (Non-<br>COVID-19 related) |
| 5.2.1.2 If no on-treatment VL during Week 48 is due to COVID-19 | No virologic<br>data at Week<br>48 Window | On study but<br>missing data in<br>window (COVID-19<br>related) |
| 5.2.2 If participants withdraw <sup>[b]</sup> before/during Week 48 due to | | |
| 5.2.2.1 Non-COVID-19 related safety reasons (e.g AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria etc, as recorded in eCRF Conclusion form) | _ | Disc due to<br>AE/death (Non-<br>COVID-19 related) |
| 5.2.2.2 COVID-19 related safety reasons (e.g. AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria etc, as recorded in eCRF Conclusion form) | No virologic<br>data at Week<br>48 Window | Disc due to<br>AE/death (COVID-<br>19 related) |
| 5.2.2.3 Non-safety and Non-COVID-19 related reasons (e.g. Lack of efficacy, protocol deviation, withdrew consent, loss to follow-up, study closed/terminated, investigator discretion etc, as recorded in eCRF Conclusion Form) | | |
| <ul> <li>Last on-treatment VL &lt;50 c/mL OR no<br/>on-treatment VL available during study</li> </ul> | No virologic<br>Data at Week<br>48 Window | Disc for other reasons (Non-COVID-19 related) |
| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND<br/>withdrawal due to Lack of efficacy</li> </ul> | HIV-1 RNA ≥<br>50 | Disc. for lack of<br>efficacy (Non-<br>COVID-19 related) |
| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND<br/>withdrawal due to all other non-safety<br/>related reasons</li> </ul> | HIV-1 RNA ≥<br>50 | Disc. for other reason while not below 50 (Non-COVID-19 related) |
| 5.2.2.4 Non-safety and COVID-19 related reasons (e.g. protocol deviation, withdrew consent, loss to follow-up, study closed/terminated, investigator discretion etc, as recorded in eCRF Conclusion Form) | | |
| <ul> <li>Last on-treatment VL &lt;50 c/mL OR no<br/>on-treatment VL available during study</li> </ul> | No virologic<br>Data at Week<br>48 Window | Disc for other reasons (COVID-19 related) |

| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND<br/>withdrawal due to Lack of efficacy</li> </ul> | HIV-1 RNA ≥ 50 | Disc. for lack of<br>efficacy (COVID-19<br>related) |
|---|---|---|
| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND<br/>withdrawal due to all other non-safety<br/>related reasons</li> </ul> | HIV-1 RNA ≥ 50 | Disc. for other<br>reason while not<br>below 50 (COVID-19<br>related) |

- a. Excluding permitted change in background therapy where change or decision to change is made prior to/on the first on-treatment viral result
- b. Including participants who either prematurely withdraw or complete the study per study conclusion form. In this study, participants who completed the Maintenance phase and decided not to enter the Extension phase without the reason beyond the completion of the study commitment are considered completers per study conclusion form.

#### **Examples from FDA guidance**

#### Data in Window

Virologic outcome should be determined by the last available measurement while the patient is on treatment and continued on trial within the time window:

 HIV-1 RNA = 580 c/mL at Day 336, HIV-1 RNA below 50 c/mL on Day 350. This should be categorized as HIV-1 RNA below 50 c/mL.

#### No Data in Window

Discontinued study due to Adverse Event or Death:

- Any patient who discontinues because of an AE or death before the window should be classified as *Discontinued due to AE or Death* (as appropriate), regardless of the HIV-1 RNA result, even if the HIV-1 RNA is below 50 c/mL at the time of discontinuation.
- However, if a patient has an HIV-1 RNA value in the time window and also discontinues in the time window, the viral load data should be used to classify the patient's response. This is the Virology First hierarchy:
  - a. HIV-1 RNA below 50 c/mL at Day 336 and discontinues because of AE or even dies on Day 360 — this person is categorized as having HIV-1 RNA below 50 c/mL.
  - b. HIV-1 RNA is 552 c/mL on Day 336 and the patient discontinues on Day 360, the patient is categorized as having HIV-1 RNA ≥ 50 c/mL.

#### Discontinued for Other Reasons:

- Only patients who have achieved virologic suppression can be counted as Discontinued for Other Reasons.
- If a patient discontinues the study before the time window because of *lack of efficacy* then the patient should be included in the HIV-1 RNA ≥ 50 row and not in the Discontinued for Other Reasons row.
- If a patient discontinues because participant withdrew consent and his or her HIV-1 RNA
  result at the time of discontinuation was equal to or above 50 c/mL, then he or she
  should be categorized as HIV-1 RNA ≥ 50 and NOT as Discontinued for Other
  Reasons.

- If a patient discontinued because of *Lost to Follow-Up* and the last HIV-1 RNA result was 49 c/mL, then the patient can be categorized as Discontinued for Other Reasons.
- If patients changed background treatment not permitted by protocol— they should be considered an efficacy failure and captured in the HIV-1 RNA ≥ 50 c/mL row.

On study but missing data in window:

- If there are no data during Days 294 to 377, but there is an HIV-1 RNA below 50 c/mL on Day 380, this patient should be considered On Study but Missing Data in Window.
- If there are no data during Days 294 to 377, but there is an HIV-1 RNA equal to or above 50 c/mL on Day 280, this patient also should be classified as On Study but Missing Data in Window.

# 15.10. Appendix 10: Variables Defined for Time to Event Analysis

Programming Instructions for the Kaplan-Meier analysis of treatment-related discontinuation equals failure (TRDF) for Week 24 IDMC / Week 24 / Week 48 / Week 96 Analyses

| discontinuation equals failure (TRDF) for Week 24 IDMC / Week 24 / Week 48 / Week 96 Analyses | | |
|---|---|---|
| Condition | Censor<br>Status | Event Description/AVAL |
| 1. Participant met CVF event criteria during the Maintenance Phase (based on derived CVF) 2. Participant with Maintenance Phase withdrawal due to 'Lack of Efficacy', 'Treatment Related AE', 'Intolerability due to Injection', or 'Protocol Defined Safety Stopping Criteria' during Maintenance Phase Note: primary reason and/or | Status<br>CNSR=0 | EVNTDESC=CVF AVAL=Study Day of SVF* *immediately preceding CVF EVNTDESC= terms in italic, respectively. For Q4W arm: AVAL= min [Study Day of Maintenance Phase Discontinuation, max (Study Day of Last Injection + 35, Study Day of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)] For Q8W arm: AVAL= min [Study Day of Maintenance Phase Discontinuation, max (Study Day of Last Injection + |
| standardized subreason for discontinuation based on Maintenance Conclusion form in the eCRF. 'Protocol Defined Safety Stopping Criteria' includes GSK defined liver chemistry stopping criteria, renal toxicity criteria and QTc withdrawal criteria. Treatment Related AE' is defined as participants who have primary reason for withdrawal =AE and who have at least one AE considered drug related and leading to withdrawal/permanent discontinuation of investigational product. | | 63, Study Day of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)] Note: Date of Maintenance Phase discontinuation is from the Maintenance Phase Conclusion form in the eCRF. |
| conditions met | CNCD-4 | EVAITABLE CONSERVED AND TO CANADA |
| Participant with Maintenance Phase withdrawal due to other | CNSR=1 | EVNTDESC='Censored due to Study Discontinuation for Other Reasons' |
| reasons | | AVAL will be defined as the same as above 2 |

| Programming Instructions for the Kaplan-Meier analysis of treatment-related |
|---|
| discontinuation equals failure (TRDF) for Week 24 IDMC / Week 24 / Week 48 / Week 96 |
| Analyses |

| Condition | Censor<br>Status | Event Description/AVAL |
|---|---|---|
| Participant who did not have premature withdrawal from the Maintenance | CNSR=1 | EVNTDESC='Censored due to data cutoff for analysis' |
| Phase | | AVAL = Study Day of last on-treatment date during the maintenance phase, which is defined as follows: |
| | | For Q4W arm: min [Study Day of Nominal Week 100 Visit, Study Day of LTFU ART Start Date, Study Day of Last Contact Date at time of analysis, max (Study Day of Last Injection + 35, Study Day of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)] |
| | | For Q8W arm min [Study Day of Nominal Week 100 Visit, Study Day of LTFU ART Start Date, Study Day of Last Contact Date at time of analysis, max (Study Day of Last Q8W IM Dose + 63, Study Day of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)] |

| Programming Instructions for the Kaplan-Meier analysis of treatment-related discontinuation equals failure (TRDF) for Week 152 Analysis | | |
|---|---|---|
| Condition | Censor<br>Status | Event Description/AVAL |
| Participant met CVF event criteria during the Maintenance and Extension Phase (based on derived CVF) | CNSR=0 | EVNTDESC=CVF AVAL=Study Day of SVF* *immediately preceding CVF |
| 2. Participant with study withdrawal due to 'Lack of Efficacy', 'Treatment Related AE', 'Intolerability due to Injection', or 'Protocol Defined Safety Stopping Criteria' | CNSR=0 | EVNTDESC= terms in italic, respectively. For Q4W arm: AVAL= min [Study Day of Study Discontinuation, max (Study Day of Last Injection + 35, Study Day of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)] |
| Note: primary reason and/or standardized subreason for discontinuation based on | | For Q8W arm: AVAL= min [Study Day of Study Discontinuation, max (Study Day of Last Injection + 63, Study Day of |

| Programming Instructions for the Kaplan-Meier analysis of treatment-related discontinuation equals failure (TRDF) for Week 152 Analysis | | |
|---|---|---|
| Condition | Censor<br>Status | Event Description/AVAL |
| Study Conclusion form in the eCRF. 'Protocol Defined Safety Stopping Criteria' includes GSK defined liver chemistry stopping criteria, renal toxicity criteria and QTc withdrawal criteria. Treatment Related AE' is defined as participants who have primary reason for withdrawal =AE and who have at least one AE considered drug related and leading to withdrawal/permanent discontinuation of investigational product. | | Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)] Note: Date of Study discontinuation is from the Study Conclusion form in the eCRF. |
| If none of the above conditions met | | |
| Participant with study withdrawal due to other reasons | CNSR=1 | EVNTDESC='Censored due to Study Discontinuation for Other Reasons' AVAL will be defined as the same as above 2 |
| Participant who did not have premature withdrawal | CNSR=1 | EVNTDESC='Censored due to data cutoff for analysis' AVAL = Study Day of last on-treatment date, which is defined as follows: For Q4W arm: min [Study Day of LTFU ART Start Date, Study Day of Last Contact Date at time of analysis, max (Study Day of Last Injection + 35, Study Day of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)] For Q8W arm min [Study Day of LTFU ART Start Date, Study Day of Last Contact Date at time of analysis, max (Study Day of Last Q8W IM Dose + 63, Study Day of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1)] |


207966

Note that last injection and last dose of oral study treatment (CAB+RPV or SOC bridging) mentioned in table above are only applied to participants who permanently discontinued from the study treatment. The similar approach will be used to derive for Kaplan-Meier analysis of efficacy-related discontinuation equals failure (ERDF), except that the reason of withdrawal in Condition 2 will be restricted to 'Lack of Efficacy'.

# 15.11. Appendix 11: Identification of Adverse Events of Special Interest

The adverse events of special interest are identified based on MedDRA coded values and/or AE data available in the study database. The system organ classes (SOCs), preferred terms (PTs) or codes, Standardised MedDRA Queries (SMQs), High Level Group Terms (HLGTs), and High Level Terms (HLTs) below are from MedDRA 21.1. SMQs use narrow terms unless otherwise specified. In case there is a change to the version of MedDRA at time of reporting, the coded values based on the MedDRA version at the time of reporting will be used. The additional events may also be added based on the blinded review of AE data collected on study prior to the database freeze.

#### 1. Hepatic Safety Profile: Assessment of risk of hepatoxicity

#### Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions (SMQ)

| PT | PT Code |
|--------------------------------------|----------|
| Acquired hepatocerebral degeneration | 10080860 |
| Acute hepatic failure | 10000804 |
| Acute on chronic liver failure | 10077305 |
| Acute yellow liver atrophy | 10070815 |
| Ascites | 10003445 |
| Asterixis | 10003547 |
| Bacterascites | 10068547 |
| Biliary cirrhosis | 10004659 |
| Biliary fibrosis | 10004664 |
| Cholestatic liver injury | 10067969 |
| Chronic hepatic failure | 10057573 |
| Coma hepatic | 10010075 |
| Cryptogenic cirrhosis | 10063075 |
| Diabetic hepatopathy | 10071265 |
| Drug-induced liver injury | 10072268 |
| Duodenal varices | 10051010 |
| Gallbladder varices | 10072319 |
| Gastric variceal injection | 10076237 |
| Gastric variceal ligation | 10076238 |
| Gastric varices | 10051012 |
| Gastric varices haemorrhage | 10057572 |
| Hepatectomy | 10061997 |
| Hepatic atrophy | 10019637 |
| Hepatic calcification | 10065274 |
| Hepatic cirrhosis | 10019641 |
| Hepatic encephalopathy | 10019660 |
| Hepatic encephalopathy prophylaxis | 10066599 |

| PT | PT Code |
|--------------------------------------|----------|
| Hepatic failure | 10019663 |
| Hepatic fibrosis | 10019668 |
| Hepatic hydrothorax | 10067365 |
| Hepatic infiltration eosinophilic | 10064668 |
| Hepatic lesion | 10061998 |
| Hepatic necrosis | 10019692 |
| Hepatic steato-fibrosis | 10077215 |
| Hepatic steatosis | 10019708 |
| Hepatitis fulminant | 10019772 |
| Hepatobiliary disease | 10062000 |
| Hepatocellular foamy cell syndrome | 10053244 |
| Hepatocellular injury | 10019837 |
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Hepatotoxicity | 10019851 |
| Intestinal varices | 10071502 |
| Intestinal varices haemorrhage | 10078058 |
| Liver and small intestine transplant | 10052280 |
| Liver dialysis | 10076640 |
| Liver disorder | 10024670 |
| Liver injury | 10067125 |
| Liver operation | 10062040 |
| Liver transplant | 10024714 |
| Lupoid hepatic cirrhosis | 10025129 |
| Minimal hepatic encephalopathy | 10076204 |
| Mixed liver injury | 10066758 |
| Nodular regenerative hyperplasia | 10051081 |
| Non-alcoholic fatty liver | 10029530 |
| Non-alcoholic steatohepatitis | 10053219 |
| Non-cirrhotic portal hypertension | 10077259 |
| Oedema due to hepatic disease | 10049631 |
| Oesophageal varices haemorrhage | 10030210 |
| Peripancreatic varices | 10073215 |
| Portal fibrosis | 10074726 |
| Portal hypertension | 10036200 |
| Portal hypertensive colopathy | 10079446 |
| Portal hypertensive enteropathy | 10068923 |
| Portal hypertensive gastropathy | 10050897 |

| PT | PT Code |
|---------------------------------------|----------|
| Portal vein cavernous transformation | 10073979 |
| Portal vein dilatation | 10073209 |
| Portopulmonary hypertension | 10067281 |
| Primary biliary cholangitis | 10080429 |
| Regenerative siderotic hepatic nodule | 10080679 |
| Renal and liver transplant | 10052279 |
| Retrograde portal vein flow | 10067338 |
| Reye's syndrome | 10039012 |
| Reynold's syndrome | 10070953 |
| Splenic varices | 10067823 |
| Splenic varices haemorrhage | 10068662 |
| Steatohepatitis | 10076331 |
| Subacute hepatic failure | 10056956 |
| Varices oesophageal | 10056091 |
| Varicose veins of abdominal wall | 10072284 |
| White nipple sign | 10078438 |

# Hepatitis, non-infectious (SMQ)

| PT | PT Code |
|--------------------------------------------|----------|
| Acute graft versus host disease in liver | 10066263 |
| Allergic hepatitis | 10071198 |
| Alloimmune hepatitis | 10080576 |
| Autoimmune hepatitis | 10003827 |
| Chronic graft versus host disease in liver | 10072160 |
| Chronic hepatitis | 10008909 |
| Graft versus host disease in liver | 10064676 |
| Hepatitis | 10019717 |
| Hepatitis acute | 10019727 |
| Hepatitis cholestatic | 10019754 |
| Hepatitis chronic active | 10019755 |
| Hepatitis chronic persistent | 10019759 |
| Hepatitis fulminant | 10019772 |
| Hepatitis toxic | 10019795 |
| Immune-mediated hepatitis | 10078962 |
| Ischaemic hepatitis | 10023025 |
| Lupus hepatitis | 10067737 |
| Non-alcoholic steatohepatitis | 10053219 |
| Radiation hepatitis | 10051015 |
| Steatohepatitis | 10076331 |

#### 2. Hypersensitivity Reactions (HSR)

# Drug reaction with eosinophilia and systemic symptoms syndrome (SMQ)

| PT | PT Code |
|-------------------------------------------------------|----------|
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Pseudolymphoma | 10037127 |

# PTs (Selective)

| PT | PT Code |
|-----------------------------------|----------|
| Drug hypersensitivity | 10013700 |
| Hypersensitivity | 10020751 |
| Type IV Hypersensitivity reaction | 10053613 |
| Eosinophillia | 10014950 |
| Eye swelling | 10015967 |
| Eyelid oedema | 10015993 |
| Lip swelling | 10024570 |
| Angioedema | 10002424 |
| Circumoral oedema | 10052250 |
| Face oedema | 10016029 |
| Idiopathic angioedema | 10073257 |
| Lip oedema | 10024558 |
| Mouth swelling | 10075203 |
| Oedema mouth | 10030110 |
| Periorbital oedema | 10034545 |
| Swelling face | 10042682 |
| Periorbital swelling | 10056647 |
| Swelling of eyelid | 10042690 |

#### 3. Rash

#### Severe cutaneous adverse reactions (SMQ)

| PT | PT Code |
|-------------------------------------------------------|----------|
| Acute generalised exanthematous pustulosis | 10048799 |
| Cutaneous vasculitis | 10011686 |
| Dermatitis bullous | 10012441 |
| Dermatitis exfoliative | 10012455 |
| Dermatitis exfoliative generalised | 10012456 |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |

| PT | PT Code |
|-----------------------------|----------|
| Epidermal necrosis | 10059284 |
| Erythema multiforme | 10015218 |
| Exfoliative rash | 10064579 |
| Oculomucocutaneous syndrome | 10030081 |
| Skin necrosis | 10040893 |
| Stevens-Johnson syndrome | 10042033 |
| Toxic epidermal necrolysis | 10044223 |
| Toxic skin eruption | 10057970 |

# PTs (Selective)

| PT | PT Code |
|----------------------|----------|
| Eyelid rash | 10074620 |
| Genital rash | 10018175 |
| Mucocutaneous rash | 10056671 |
| Nodular rash | 10075807 |
| Perineal rash | 10075364 |
| Rash | 10037844 |
| Rash erythematous | 10037855 |
| Rash generalised | 10037858 |
| Rash macular | 10037867 |
| Rash maculo-papular | 10037868 |
| Rash maculovesicular | 10050004 |
| Rash morbilliform | 10037870 |
| Rash papular | 10037876 |
| Rash rubelliform | 10057984 |
| Rash scarlatiniform | 10037890 |
| Rash vesicular | 10037898 |
| Rash pruritic | 10037884 |
| Rash follicular | 10037857 |
| Rash pustular | 10037888 |
| Drug eruption | 10013687 |

# 4. Prolongation of the Corrected QT Interval of the ECG in Supratherapeutic Doses Torsade de pointes/QT prolongation (SMQ)

| PT | PT Code |
|----------------------------------------|----------|
| Electrocardiogram QT interval abnormal | 10063748 |

| PT | PT Code |
|--------------------------------|----------|
| Electrocardiogram QT prolonged | 10014387 |
| Long QT syndrome | 10024803 |
| Long QT syndrome congenital | 10057926 |
| Torsade de pointes | 10044066 |
| Ventricular tachycardia | 10047302 |

# PTs (Selective)

| PT | PT Code |
|----------------------------------------------|----------|
| Electrocardiogram repolarisation abnormality | 10052464 |

#### 5. Suicidal Ideation/Behaviour

# Suicide/self-injury (SMQ)

| PT | PT Code |
|-------------------------------------------------|----------|
| Assisted suicide | 10079105 |
| Columbia suicide severity rating scale abnormal | 10075616 |
| Completed suicide | 10010144 |
| Depression suicidal | 10012397 |
| Intentional overdose | 10022523 |
| Intentional self-injury | 10022524 |
| Poisoning deliberate | 10036000 |
| Self-injurious ideation | 10051154 |
| Suicidal behaviour | 10065604 |
| Suicidal ideation | 10042458 |
| Suicide attempt | 10042464 |
| Suicide threat | 10077417 |
| Suspected suicide attempt | 10081704 |

# 6. Depression

# Depression (excl suicide and self injury) (SMQ)

| PT | PT Code |
|-----------------------------------------------------------|----------|
| Activation syndrome | 10066817 |
| Adjustment disorder with depressed mood | 10001297 |
| Adjustment disorder with mixed anxiety and depressed mood | 10001299 |
| Agitated depression | 10001496 |
| Anhedonia | 10002511 |

| PT | PT Code |
|---------------------------------------|----------|
| Antidepressant therapy | 10054976 |
| Childhood depression | 10068631 |
| Decreased interest | 10011971 |
| Depressed mood | 10012374 |
| Depression | 10012378 |
| Depression postoperative | 10012390 |
| Depressive symptom | 10054089 |
| Dysphoria | 10013954 |
| Electroconvulsive therapy | 10014404 |
| Feeling guilty | 10049708 |
| Feeling of despair | 10016344 |
| Feelings of worthlessness | 10016374 |
| Helplessness | 10077169 |
| Major depression | 10057840 |
| Menopausal depression | 10067371 |
| Mixed anxiety and depressive disorder | 10080836 |
| Perinatal depression | 10078366 |
| Persistent depressive disorder | 10077804 |
| Post stroke depression | 10070606 |
| Postictal depression | 10071324 |

# 7. Bipolar Disorder

# **HLGT Manic and Bipolar mood disorders and disturbances**

| PT | PT Code |
|----------------------|----------|
| Bipolar I disorder | 10004939 |
| Bipolar II disorder | 10004940 |
| Bipolar disorder | 10057667 |
| Cyclothymic disorder | 10011724 |
| Hypomania | 10021030 |
| Mania | 10026749 |

# 8. Psychosis

# Psychosis and psychotic disorders (SMQ)

| PT | PT Code |
|---------------------|----------|
| Acute psychosis | 10001022 |
| Alcoholic psychosis | 10001632 |

| PT | PT Code |
|---------------------------------------------------|----------|
| Alice in wonderland syndrome | 10001666 |
| Brief psychotic disorder with marked stressors | 10048549 |
| Brief psychotic disorder without marked stressors | 10056395 |
| Brief psychotic disorder, with postpartum onset | 10006362 |
| Charles Bonnet syndrome | 10063354 |
| Childhood psychosis | 10061040 |
| Clang associations | 10009232 |
| Cotard's syndrome | 10059591 |
| Delusion | 10012239 |
| Delusion of grandeur | 10012241 |
| Delusion of reference | 10012244 |
| Delusion of replacement | 10012245 |
| Delusional disorder, erotomanic type | 10012249 |
| Delusional disorder, grandiose type | 10012250 |
| Delusional disorder, jealous type | 10012251 |
| Delusional disorder, mixed type | 10012252 |
| Delusional disorder, persecutory type | 10053195 |
| Delusional disorder, somatic type | 10012254 |
| Delusional disorder, unspecified type | 10012255 |
| Delusional perception | 10012258 |
| Dementia of the Alzheimer's type, with delusions | 10012295 |
| Depressive delusion | 10063033 |
| Derailment | 10012411 |
| Epileptic psychosis | 10059232 |
| Erotomanic delusion | 10015134 |
| Flight of ideas | 10016777 |
| Hallucination | 10019063 |
| Hallucination, auditory | 10019070 |
| Hallucination, gustatory | 10019071 |
| Hallucination, olfactory | 10019072 |
| Hallucination, synaesthetic | 10062824 |
| Hallucination, tactile | 10019074 |
| Hallucination, visual | 10019075 |
| Hallucinations, mixed | 10019079 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Hysterical psychosis | 10062645 |
| Ideas of reference | 10021212 |
| Illusion | 10021403 |

| PT | PT Code |
|-------------------------------------------------------|----------|
| Jealous delusion | 10023164 |
| Loose associations | 10024825 |
| Mixed delusion | 10076429 |
| Neologism | 10028916 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Paranoia | 10033864 |
| Paranoid personality disorder | 10033869 |
| Parkinson's disease psychosis | 10074835 |
| Paroxysmal perceptual alteration | 10063117 |
| Persecutory delusion | 10034702 |
| Postictal psychosis | 10070669 |
| Post-injection delirium sedation syndrome | 10072851 |
| Posturing | 10036437 |
| Psychosis postoperative | 10065617 |
| Psychotic behaviour | 10037249 |
| Psychotic disorder | 10061920 |
| Psychotic disorder due to a general medical condition | 10061921 |
| Reactive psychosis | 10053632 |
| Rebound psychosis | 10074833 |
| Schizoaffective disorder | 10039621 |
| Schizoaffective disorder bipolar type | 10068889 |
| Schizoaffective disorder depressive type | 10068890 |
| Schizophrenia | 10039626 |
| Schizophreniform disorder | 10039647 |
| Schizotypal personality disorder | 10039651 |
| Senile psychosis | 10039987 |
| Shared psychotic disorder | 10040535 |
| Somatic delusion | 10041317 |
| Somatic hallucination | 10062684 |
| Substance-induced psychotic disorder | 10072388 |
| Tangentiality | 10043114 |
| Thought blocking | 10043495 |
| Thought broadcasting | 10052214 |
| Thought insertion | 10043496 |
| Thought withdrawal | 10043497 |
| Transient psychosis | 10056326 |
| Waxy flexibility | 10047853 |

#### 9. Mood Disorders

# **HLGT Mood disorders and disturbances NEC, Psychiatric disorders SOC**

| PT | PT Code |
|----------------------------------------|----------|
| Crying | 10011469 |
| Mood swings | 10027951 |
| Boredom | 10048909 |
| Mood altered | 10027940 |
| Apathy | 10002942 |
| Affective ambivalence | 10077173 |
| Emotional poverty | 10014557 |
| Euphoric mood | 10015535 |
| Premenstrual dysphoric disorder | 10051537 |
| Alexithymia | 10077719 |
| Laziness | 10051602 |
| Blunted affect | 10005885 |
| Constricted affect | 10010778 |
| Affect lability | 10054196 |
| Anger | 10002368 |
| Affective disorder | 10001443 |
| Lethargy | 10024264 |
| Listless | 10024642 |
| Inappropriate affect | 10021588 |
| Dysphoria | 10013954 |
| Mood disorder due to a general medical | |
| condition | 10027944 |
| Morose | 10027977 |
| Screaming | 10039740 |
| Steroid withdrawal syndrome | 10042028 |
| Emotional disorder | 10014551 |
| Irritability | 10022998 |
| Moaning | 10027783 |
| Premenstrual syndrome | 10036618 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Substance-induced mood disorder | 10072387 |
| Flat affect | 10016759 |
| Diencephalic syndrome of infancy | 10012774 |
| Emotional distress | 10049119 |
| Frustration tolerance decreased | 10077753 |
| Seasonal affective disorder | 10039775 |

# 10. Anxiety

# **HLGT Anxiety disorders and symptoms**

| PT | PT Code |
|-----------------------------------------------------|----------|
| Acrophobia | 10000605 |
| Activation syndrome | 10066817 |
| Acute stress disorder | 10001084 |
| Aerophobia | 10080300 |
| Agitation | 10001497 |
| Agitation neonatal | 10001500 |
| Agitation postoperative | 10049989 |
| Agoraphobia | 10001502 |
| Akathisia | 10001540 |
| Algophobia | 10078056 |
| Animal phobia | 10002518 |
| Anniversary reaction | 10074066 |
| Anticipatory anxiety | 10002758 |
| Anxiety | 10002855 |
| Anxiety disorder | 10057666 |
| Anxiety disorder due to a general medical condition | 10002859 |
| Arachnophobia | 10051408 |
| Astraphobia | 10078372 |
| Autophobia | 10071070 |
| Body dysmorphic disorder | 10052793 |
| Burnout syndrome | 10065369 |
| Claustrophobia | 10009244 |
| Compulsions | 10010219 |
| Compulsive cheek biting | 10076510 |
| Compulsive handwashing | 10071263 |
| Compulsive hoarding | 10068007 |
| Compulsive lip biting | 10066241 |
| Compulsive shopping | 10067948 |
| Dermatillomania | 10065701 |
| Dysmorphophobia | 10049096 |
| Emetophobia | 10070637 |
| Fear | 10016275 |
| Fear of animals | 10016276 |
| Fear of closed spaces | 10016277 |
| Fear of crowded places | 10050365 |
| Fear of death | 10066392 |

| PT | PT Code |
|-------------------------------------------------------------|----------|
| Fear of disease | 10016278 |
| Fear of eating | 10050366 |
| Fear of falling | 10048744 |
| Fear of injection | 10073753 |
| Fear of open spaces | 10016279 |
| Fear of pregnancy | 10067035 |
| Fear of weight gain | 10016280 |
| Fear-related avoidance of activities | 10080136 |
| Generalised anxiety disorder | 10018075 |
| Glossophobia | 10080077 |
| Haemophobia | 10073458 |
| Haphephobia | 10067580 |
| Hydrophobia | 10053317 |
| Hyperarousal | 10080831 |
| Immunisation anxiety related reaction | 10075205 |
| Kinesiophobia | 10078430 |
| Limited symptom panic attack | 10024511 |
| Mysophobia | 10078769 |
| Nail picking | 10066779 |
| Nervousness | 10029216 |
| Neurosis | 10029333 |
| Noctiphobia | 10057946 |
| Nocturnal fear | 10057948 |
| Nosophobia | 10063546 |
| Obsessive need for symmetry | 10077179 |
| Obsessive rumination | 10056264 |
| Obsessive thoughts | 10029897 |
| Obsessive-compulsive disorder | 10029898 |
| Obsessive-compulsive symptom | 10077894 |
| Ochlophobia | 10050095 |
| Osmophobia | 10060765 |
| Paediatric autoimmune neuropsychiatric disorders associated | |
| with streptococcal infection | 10072147 |
| Panic attack | 10033664 |
| Panic disorder | 10033666 |
| Panic reaction | 10033670 |
| Paruresis | 10069024 |
| Performance fear | 10034432 |
| Phagophobia | 10050096 |
| Pharmacophobia | 10069423 |

| PT | PT Code |
|--------------------------------|----------|
| Phobia | 10034912 |
| Phobia of driving | 10056676 |
| Phobia of exams | 10034913 |
| Phobic avoidance | 10034918 |
| Phonophobia | 10054956 |
| Photaugiaphobia | 10064420 |
| Post-traumatic stress disorder | 10036316 |
| Postpartum neurosis | 10036419 |
| Postpartum stress disorder | 10056394 |
| Procedural anxiety | 10075204 |
| Pseudoangina | 10056610 |
| Selective mutism | 10039917 |
| Separation anxiety disorder | 10040045 |
| Sitophobia | 10080170 |
| Social anxiety disorder | 10041242 |
| Social fear | 10041247 |
| Stress | 10042209 |
| Tension | 10043268 |
| Terminal agitation | 10077416 |
| Thanatophobia | 10064723 |
| Thermophobia | 10075147 |
| Trichotemnomania | 10072752 |
| Trichotillomania | 10044629 |

# 11. Sleep Disorders

# **HLGT Sleep Disorders and Disturbances**

| PT | PT Code |
|-----------------------------------|----------|
| Behavioural insomnia of childhood | 10072072 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Middle insomnia | 10027590 |
| Terminal insomnia | 10068932 |
| Breathing-related sleep disorder | 10006344 |
| Dyssomnia | 10061827 |
| Hypersomnia | 10020765 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |

| РТ | PT Code |
|-------------------------------------------------------------|----------|
| Poor quality sleep | 10062519 |
| Sleep apnoea syndrome | 10040979 |
| Somnolence | 10041349 |
| Somnolence neonatal | 10041350 |
| Stupor | 10042264 |
| Upper airway resistance syndrome | 10063968 |
| Cataplexy | 10007737 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Narcolepsy | 10028713 |
| Sleep attacks | 10040981 |
| Sleep paralysis | 10041002 |
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Confusional arousal | 10067494 |
| Exploding head syndrome | 10080684 |
| Loss of dreaming | 10065085 |
| Nightmare | 10029412 |
| Parasomnia | 10061910 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Sleep inertia | 10067493 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Hypersomnia related to another mental condition | 10020767 |
| Hypersomnia-bulimia syndrome | 10053712 |
| Insomnia related to another mental condition | 10022443 |
| Sleep disorder | 10040984 |
| Sleep disorder due to a general medical condition | 10063910 |
| Sleep disorder due to general medical condition, | |
| hypersomnia type | 10040985 |
| Sleep disorder due to general medical condition, | 40040000 |
| insomnia type | 10040986 |
| Sleep disorder due to general medical condition, mixed type | 10040987 |
| Sleep disorder due to general medical condition, | 10070301 |
| parasomnia type | 10040988 |
| Sopor | 10058709 |

| PT | PT Code |
|--------------------------------------|----------|
| Advanced sleep phase | 10001423 |
| Circadian rhythm sleep disorder | 10009191 |
| Delayed sleep phase | 10012209 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Shift work disorder | 10078088 |

# **HLGT Sleep disturbances (incl subtypes)**

| PT | PT Code |
|--------------------------------------|----------|
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Confusional arousal | 10067494 |
| Loss of dreaming | 10065085 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Behavioural insomnia of childhood | 10072072 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Middle insomnia | 10027590 |
| Terminal insomnia | 10068932 |
| Advanced sleep phase | 10001423 |
| Circadian rhythm sleep disorder | 10009191 |
| Delayed sleep phase | 10012209 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Shift work disorder | 10078088 |
| Cataplexy | 10007737 |
| Hypersomnia | 10020765 |
| Narcolepsy | 10028713 |
| Central-alveolar hypoventilation | 10007982 |
| Sleep apnoea syndrome | 10040979 |

| PT | PT Code |
|---------------------------------------------|----------|
| Breathing-related sleep disorder | 10006344 |
| Dyssomnia | 10061827 |
| Fatal familial insomnia | 10072077 |
| Microsleep | 10076954 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Sleep deficit | 10080881 |
| Sudden onset of sleep | 10050014 |
| Upper airway resistance syndrome | 10063968 |

#### 12. Injection Site Reactions (ISR) from Study Drug Injections

Study drug ISR data available in the database, i.e. data collected from non-serious ISR AE eCRF form and collected serious adverse events with 'STUDY DRUG INJECTION SITE' included in the AE term.

#### 13. Seizures and Seizure-like Events

# Convulsions (SMQ)

| PT | PT Code |
|-----------------------------------------------------------------|----------|
| 2-Hydroxyglutaric aciduria | 10078971 |
| Acquired epileptic aphasia | 10052075 |
| Acute encephalitis with refractory, repetitive partial seizures | 10076948 |
| Alcoholic seizure | 10056347 |
| Aspartate-glutamate-transporter deficiency | 10079140 |
| Atonic seizures | 10003628 |
| Atypical benign partial epilepsy | 10056699 |
| Automatism epileptic | 10003831 |
| Autonomic seizure | 10049612 |
| Baltic myoclonic epilepsy | 10054895 |
| Benign familial neonatal convulsions | 10067866 |
| Benign rolandic epilepsy | 10070530 |
| Biotinidase deficiency | 10071434 |
| Change in seizure presentation | 10075606 |
| Clonic convulsion | 10053398 |
| Convulsion in childhood | 10052391 |

| PT | PT Code |
|---|---|
| Convulsion neonatal | 10010911 |
| Convulsions local | 10010920 |
| Convulsive threshold lowered | 10010927 |
| CSWS syndrome | 10078827 |
| Deja vu | 10012177 |
| Double cortex syndrome | 10073490 |
| Dreamy state | 10013634 |
| Drug withdrawal convulsions | 10013752 |
| Early infantile epileptic encephalopathy with burst-<br>suppression | 10071545 |
| Eclampsia | 10014129 |
| Epilepsy | 10015037 |
| Epilepsy surgery | 10079824 |
| Epilepsy with myoclonic-atonic seizures | 10081179 |
| Epileptic aura | 10015049 |
| Epileptic psychosis | 10059232 |
| Febrile convulsion | 10016284 |
| Febrile infection-related epilepsy syndrome | 10079438 |
| Focal dyscognitive seizures | 10079424 |
| Frontal lobe epilepsy | 10049424 |
| Generalised non-convulsive epilepsy | 10018090 |
| Generalised tonic-clonic seizure | 10018100 |
| Glucose transporter type 1 deficiency syndrome | 10078727 |
| Gray matter heterotopia | 10080533 |
| Hemimegalencephaly | 10078100 |
| Hyperglycaemic seizure | 10071394 |
| Hypocalcaemic seizure | 10072456 |
| Hypoglycaemic seizure | 10048803 |
| Hyponatraemic seizure | 10073183 |
| Idiopathic generalised epilepsy | 10071081 |
| Infantile spasms | 10021750 |
| Juvenile myoclonic epilepsy | 10071082 |
| Lafora's myoclonic epilepsy | 10054030 |
| Lennox-Gastaut syndrome | 10048816 |
| Migraine-triggered seizure | 10076676 |
| Molybdenum cofactor deficiency | 10069687 |
| Multiple subpial transection | 10079825 |
| Myoclonic epilepsy | 10054859 |
| Myoclonic epilepsy and ragged-red fibres | 10069825 |
| Partial seizures | 10061334 |

| PT | PT Code |
|------------------------------------------------|----------|
| Partial seizures with secondary generalisation | 10056209 |
| Petit mal epilepsy | 10034759 |
| Polymicrogyria | 10073489 |
| Post stroke epilepsy | 10076982 |
| Post stroke seizure | 10076981 |
| Postictal headache | 10052470 |
| Postictal paralysis | 10052469 |
| Postictal psychosis | 10070669 |
| Postictal state | 10048727 |
| Post-traumatic epilepsy | 10036312 |
| Schizencephaly | 10073487 |
| Seizure | 10039906 |
| Seizure anoxic | 10039907 |
| Seizure cluster | 10071350 |
| Seizure like phenomena | 10071048 |
| Severe myoclonic epilepsy of infancy | 10073677 |
| Simple partial seizures | 10040703 |
| Status epilepticus | 10041962 |
| Sudden unexplained death in epilepsy | 10063894 |
| Temporal lobe epilepsy | 10043209 |
| Tonic clonic movements | 10051171 |
| Tonic convulsion | 10043994 |
| Tonic posturing | 10075125 |
| Topectomy | 10073488 |
| Transient epileptic amnesia | 10081728 |
| Tuberous sclerosis complex | 10080584 |
| Uncinate fits | 10045476 |

# PTs (Selective)

| PT | PT Code |
|----------------------------------|----------|
| Confusional state | 10010305 |
| Loss of consciousness | 10024855 |
| Syncope | 10042772 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Altered state of consciousness | 10050093 |
| Depressed level of consciousness | 10012373 |
| Consciousness fluctuating | 10050093 |

#### 14. Weight Gain

#### **HLT General nutritional disorders NEC (Selective)**

| PT | PT Code |
|----------------------|----------|
| Abdominal fat apron | 10077983 |
| Overweight | 10033307 |
| Abnormal weight gain | 10000188 |
| Central obesity | 10065941 |
| Obesity | 10029883 |

#### HLT Physical examination procedures and organ system status (Selective)

| PT | PT Code |
|-------------------------------|----------|
| Weight abnormal | 10056814 |
| Weight increased | 10047899 |
| Waist circumference increased | 10064863 |
| Body mass index abnormal | 10074506 |
| Body mass index increased | 10005897 |

#### General signs and symptoms NEC (Selective)

| PT | PT Code |
|----------------------|----------|
| Fat tissue increased | 10016251 |

#### 15. Rhabdomyolysis

#### Rhabdomyolysis/myopathy (SMQ)

| PT | PT Code |
|---------------------------|----------|
| Muscle necrosis | 10028320 |
| Myoglobin blood increased | 10028625 |
| Myoglobin blood present | 10059888 |
| Myoglobin urine present | 10028631 |
| Myoglobinaemia | 10058735 |
| Myoglobinuria | 10028629 |
| Myopathy | 10028641 |
| Myopathy toxic | 10028648 |
| Necrotising myositis | 10074769 |

| PT | PT Code |
|---------------------|----------|
| Rhabdomyolysis | 10039020 |
| Thyrotoxic myopathy | 10081524 |

# PTs (Selective)

| PT | PT Code |
|----------|----------|
| Myalgia | 10028411 |
| Myositis | 10028653 |

#### 16. Pancreatitis

# Acute pancreatitis (SMQ)

| PT | PT Code |
|------------------------------------|----------|
| Cullen's sign | 10059029 |
| Grey Turner's sign | 10075426 |
| Haemorrhagic necrotic pancreatitis | 10076058 |
| Hereditary pancreatitis | 10056976 |
| Ischaemic pancreatitis | 10066127 |
| Oedematous pancreatitis | 10052400 |
| Pancreatic abscess | 10048984 |
| Pancreatic haemorrhage | 10033625 |
| Pancreatic necrosis | 10058096 |
| Pancreatic phlegmon | 10056975 |
| Pancreatic pseudoaneurysm | 10081762 |
| Pancreatic pseudocyst | 10033635 |
| Pancreatic pseudocyst drainage | 10033636 |
| Pancreatitis | 10033645 |
| Pancreatitis acute | 10033647 |
| Pancreatitis haemorrhagic | 10033650 |
| Pancreatitis necrotising | 10033654 |
| Pancreatitis relapsing | 10033657 |
| Pancreatorenal syndrome | 10056277 |

# 17. Impact on Creatinine

# Acute renal failure (SMQ)

| PT | PT Code |
|-----------------------------|----------|
| Acute kidney injury | 10069339 |
| Acute phosphate nephropathy | 10069688 |

| PT | PT Code |
|----------------------------------|----------|
| Anuria | 10002847 |
| Azotaemia | 10003885 |
| Continuous haemodiafiltration | 10066338 |
| Dialysis | 10061105 |
| Foetal renal impairment 10078987 | |
| Haemodialysis | 10018875 |
| Haemofiltration | 10053090 |
| Hyponatriuria | 10077515 |
| Neonatal anuria | 10049778 |
| Nephropathy toxic | 10029155 |
| Oliguria | 10030302 |
| Peritoneal dialysis | 10034660 |
| Prerenal failure | 10072370 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |
| Renal impairment | 10062237 |
| Renal impairment neonatal | 10049776 |

# Renal Failure and Impairment HLT

| PT | PT Code |
|--------------------------------------|----------|
| Acute Kidney injury | 10069339 |
| Anuria | 10002847 |
| Atypical haemolytic uraemic syndrome | 10079840 |
| Cardiorenal syndrome | 10068230 |
| Chronic kidney disease | 10064848 |
| Crush syndrome | 10050702 |
| Diabetic end stage renal disease | 10012660 |
| End stage renal disease | 10077512 |
| Foetal renal impairment | 10078987 |
| Haemolytic uraemic syndrome | 10018932 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Nail-patella syndrome | 10063431 |
| Neonatal anuria | 10049778 |
| Oliguria | 10030302 |
| Pancreatorenal syndrome | 10056277 |
| Postoperative renal failure | 10056675 |
| Postrenal failure | 10059345 |
| Prerenal failure | 10072370 |

| PT | PT Code |
|----------------------------|----------|
| Propofol infusion syndrome | 10063181 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |
| Renal impairment | 10062237 |
| Renal impairment neonatal | 10049776 |
| Renal injury | 10061481 |
| Scleroderma renal crisis | 10062553 |
| Traumatic anuria | 10044501 |

#### 18. Safety in Pregnancy

Use AE terms co-reported in pregnancy exposures to CAB and/or RPV.

#### 19. Hyperglycaemia

Medical concept of Hyperglycaemia/new onset diabetes mellitus - SMQs (1) 'Hyperglycaemia/new onset diabetes mellitus (SMQ) Narrow SMQ code 20000041

| PT | PT Code |
|-------------------------------------------|----------|
| Blood 1,5-anhydroglucitol decreased | 10065367 |
| Blood glucose increased | 10005557 |
| Diabetes complicating pregnancy | 10012596 |
| Diabetes mellitus | 10012601 |
| Diabetes mellitus inadequate control | 10012607 |
| Diabetes with hyperosmolarity | 10012631 |
| Diabetic arteritis | 10077357 |
| Diabetic coma | 10012650 |
| Diabetic coronary microangiopathy | 10080788 |
| Diabetic hepatopathy | 10071265 |
| Diabetic hyperglycaemic coma | 10012668 |
| Diabetic hyperosmolar coma | 10012669 |
| Diabetic ketoacidosis | 10012671 |
| Diabetic ketoacidotic hyperglycaemic coma | 10012672 |
| Diabetic ketosis | 10012673 |
| Diabetic metabolic decompensation | 10074309 |
| Diabetic wound | 10081558 |
| Euglycaemic diabetic ketoacidosis | 10080061 |
| Fructosamine increased | 10017395 |
| Fulminant type 1 diabetes mellitus | 10072628 |
| Gestational diabetes | 10018209 |
| Glucose tolerance impaired | 10018429 |
| Glucose tolerance impaired in pregnancy | 10018430 |

| PT | PT Code |
|-------------------------------------------------|----------|
| Glucose urine present | 10018478 |
| Glycated albumin increased | 10082836 |
| Glycosuria | 10018473 |
| Glycosuria during pregnancy | 10018475 |
| Glycosylated haemoglobin abnormal | 10018481 |
| Glycosylated haemoglobin increased | 10018484 |
| Hyperglycaemia | 10020635 |
| Hyperglycaemic hyperosmolar nonketotic syndrome | 10063554 |
| Hyperglycaemic seizure | 10071394 |
| Hyperglycaemic unconsciousness | 10071286 |
| Impaired fasting glucose | 10056997 |
| Insulin resistance | 10022489 |
| Insulin resistant diabetes | 10022491 |
| Insulin-requiring type 2 diabetes mellitus | 10053247 |
| Ketoacidosis | 10023379 |
| Ketonuria | 10023388 |
| Ketosis | 10023391 |
| Ketosis-prone diabetes mellitus | 10023392 |
| Latent autoimmune diabetes in adults | 10066389 |
| Monogenic diabetes | 10075980 |
| Neonatal diabetes mellitus | 10028933 |
| New onset diabetes after transplantation | 10082630 |
| Pancreatogenous diabetes | 10033660 |
| Steroid diabetes | 10081755 |
| Type 1 diabetes mellitus | 10067584 |
| Type 2 diabetes mellitus | 10067585 |
| Type 3 diabetes mellitus | 10072659 |
| Urine ketone body present | 10057597 |
| Hepatogenous diabetes | 10085610 |
| Maternally inherited diabetes and deafness | 10086189 |
| Neonatal hyperglycaemia | 10086425 |
| Acquired generalised lipodystrophy | 10087376 |
| Glycated serum protein increased | 10087214 |
| Hyperglycaemic crisis | 10087319 |

#### 15.12. Appendix 12: Identification of COVID-19 Adverse Events

COVID-19 adverse events are identified based on MedDRA coded values and/or AE referenced in the COVID-19 Coronavirus Infection assessment. The Lowest Level Terms (LLTs) and codes, Preferred Terms (PTs), High Level Terms (HLTs), High Level Group Terms (HLGTs), and System Organ Classes (SOCs), below are from MedDRA 23.0. In case there is a change to the version of MedDRA at time of reporting, the coded values based on the MedDRA version at the time of reporting will be used. The additional events may also be added based on the blinded review of AE data collected on study prior to the database freeze.

SOC: Infections and infestations

| LLT code | LLT | PT | HLT | HLGT |
|---|---|---|---|---|
| | | Asymptomatic | Coronavirus | Viral infectious |
| 10084459 | Asymptomatic COVID-19 | COVID-19 | infections | disorders |
| | Asymptomatic SARS- | Asymptomatic | Coronavirus | Viral infectious |
| 10084467 | CoV-2 infection | COVID-19 | infections | disorders |
| | | Coronavirus | Coronavirus | Viral infectious |
| 10053983 | Corona virus infection | infection | infections | disorders |
| | | Coronavirus | Coronavirus | Viral infectious |
| 10051905 | Coronavirus infection | infection | infections | disorders |
| | Coronavirus disease | | Coronavirus | Viral infectious |
| 10084382 | 2019 | COVID-19 | infections | disorders |
| | | | Coronavirus | Viral infectious |
| 10084268 | COVID-19 | COVID-19 | infections | disorders |
| | COVID-19 respiratory | | Coronavirus | Viral infectious |
| 10084401 | infection | COVID-19 | infections | disorders |
| | SARS-CoV-2 acute | | Coronavirus | Viral infectious |
| 10084270 | respiratory disease | COVID-19 | infections | disorders |
| | | | Coronavirus | Viral infectious |
| 10084272 | SARS-CoV-2 infection | COVID-19 | infections | disorders |
| | | COVID-19 | Coronavirus | Viral infectious |
| 10084381 | Coronavirus pneumonia | pneumonia | infections | disorders |
| | | COVID-19 | Coronavirus | Viral infectious |
| 10084380 | COVID-19 pneumonia | pneumonia | infections | disorders |
| | Novel COVID-19- | COVID-19 | Coronavirus | Viral infectious |
| 10084383 | infected pneumonia | pneumonia | infections | disorders |
| | | Suspected | Coronavirus | Viral infectious |
| 10084451 | Suspected COVID-19 | COVID-19 | infections | disorders |
| | Suspected SARS-CoV-2 | Suspected | Coronavirus | Viral infectious |
| 10084452 | infection | COVID-19 | infections | disorders |
| | | SARS-CoV-2 | Infectious | Ancillary infectious |
| 10084461 | SARS-CoV-2 carrier | carrier | disorders carrier | topics |

#### 15.13. Appendix 13: IDMC

Independent review will be provided by an IDMC to ensure external objective medical and/or statistical review of efficacy and safety in order to protect the ethical interests and well-being of participants and to protect the scientific validity of this study. An ad-hoc review of data by the IDMC will be triggered whenever the number of confirmed virologic failures in the Q8W arm exceeds thresholds pre-specified in the IDMC charter. Further, analyses including futility checking will be performed for the IDMC to evaluate the efficacy and safety when approximately 50% of participants have completed their visit at Week 24.

The list of required outputs is provided in the IDMC Charter, Section 12.3, Appendix C.

Data handing methods and derived data definitions will be the same as detailed in this RAP, unless otherwise stated.

#### 15.13.1. Adhoc CVF IDMC Analyses

The number of participants meeting Confirmed Virologic Failure (CVF) Criterion per the protocol will be monitored and may result in ad-hoc IDMC data reviews.

The Statistics Data Analysis Centre (SDAC) will be notified by the study virologist in writing every time a CVF occurs in the study. The SDAC will track the number of participants on Q8W arm past Week 4. The rate of CVF will be monitored against the thresholds specified in IDMC Charter Table 1 (See IDMC Charter, Section 3.5.2).

#### 15.13.2. Week 24 IDMC Analyses

Analyses including futility checking will be performed when approximately 50% of participants have completed their Week 24 visit.

A futility rule will assess the evidence that the CAB LA + RPV LA Q8W arm is non-inferior to the Q4W control arm. This rule will use the interim data (~ 50% participants completing Week 24) to calculate the Bayesian predictive probabilities that the CAB LA + RPV LA Q8W arm is non-inferior to the Q4W arm at Week 24. A 4% non-inferiority margin will be used. The details of statistical methods can be found in IDMC Charter, Section 12.6.1. The list of outputs is also provided in Section 15.15.4.
## 15.14. Appendix 14: Abbreviations & Trademarks

## 15.14.1. Abbreviations

| Abbreviation | Description |
|--------------|------------------------------------------------------------|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Events of Special Interest |
| BMI | Body Mass Index |
| CAB | Cabotegravir |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| СМН | Cochran-Mantel-Haenszel |
| COVID | Coronavirus Disease |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| eC-SSRS | Electronic Columbia Suicide Severity Rating Scale |
| CVb | Coefficient of Variation (Between) |
| CVD | Cardiovascular Disease |
| CVF | Confirmed Virologic Failure |
| DAIDS | Division of AIDS |
| DBF | Database Freeze |
| DBL | Database Lock |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Place |
| DTG | Dolutegravir |
| eCRF | Electronic Case Record Form |
| eGFR | Estimated Glomerular Filtration Rate |
| EMA | European Medicines Agency |
| ERDF | Efficacy Related Discontinuation Failure |
| FDA | Food and Drug Administration |
| FSFV | First Subject First Visit |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| HAT-QoL | Health-related Quality of Life |
| HBV | Hepatitis B Virus |
| HCV | Hepatitis C Virus |
| HIV | Human Immunodeficiency Virus |
| HIVTSQc | Change Version of HIV Treatment Satisfaction Questionnaire |
| HIVTSQs | Status Version of HIV Treatment Satisfaction Questionnaire |
| HLGT | High Level Group Term |
| HLT | High Level Term |
| HSR | Hypersensitivity Reaction |
| ICH | International Conference on Harmonisation |

| IDMC Independent Data Monitoring Committee |
|-------------------------------------------------------|
| IDSL Integrated Data Standards Library |
| IMMS International Modules Management System |
| INI Integrase Inhibitors |
| IP Investigational Product |
| ITT Intent-To-Treat |
| ITT-E Intent-To-Treat Exposed |
| LA Long Acting |
| LOCF Last Observation Carries Forward |
| MMRM Mixed Model Repeated Measures |
| NA Not Applicable |
| NCEP National Cholesterol Education Program |
| NNRTI Non-Nucleoside Reverse Transcriptase Inhibitors |
| NQ Non Quantifiable |
| NRTI Nucleoside Reverse Transcriptase Inhibitors |
| OC Observed Case |
| PBMC Peripheral Blood Mononuclear Cell |
| PCI Potential Clinical Importance |
| PD Pharmacodynamic |
| PDMP Protocol Deviation Management Plan |
| PI Protease Inhibitors |
| PIN Perception of Injection |
| PK Pharmacokinetic |
| PP Per Protocol |
| PT Preferred Term |
| QTcF Frederica's QT Interval Corrected for Heart Rate |
| QTcB Bazett's QT Interval Corrected for Heart Rate |
| RAM Resistance Associated Mutation |
| RAMOS Randomization & Medication Ordering System |
| RAP Reporting & Analysis Plan |
| RPV Rilpivirine |
| SAE Serious Adverse Event |
| SAC Statistical Analysis Complete |
| SD Standard Deviation |
| SDAC Statistics Data Analysis Centre |
| SDTM Study Data Tabulation Model |
| SMQ Standardised MedDRA Query |
| SOC System Organ Class |
| SOP Standard Operation Procedure |
| TFL Tables, Figures & Listings |
| TRDF Treatment Related Discontinuation Failure |

#### 15.14.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| Tivicay |
| Triumeq |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Edurant |
| NONMEM |
| SAS |
| WinNonlin |

#### 15.15. Appendix 15: List of Data Displays

#### 15.15.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|-----------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacokinetic / Pharmacodynamic | 5.1 to 5.n | 5.1 to 5.n |
| Health Outcomes | 6.1 to 6.n | 6.1 to 6.n |
| Virology | 7.1 to 7.n | 7.1 to 7.n |
| Section | List | ings |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

#### 15.15.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays will be provided in a separate document.

The example mock-up displays from other reporting efforts will be named in the format: Study Number/HARP Reporting Effort/Output Type (T/ F/L)/Display Number, where T stands for Table, F stands for Figure and L stands for Listing. For example, the Table 1.1 from primary\_02 reporting effort for Study 201585 will be named by 201585/primary\_02/T1.1.

Other example mock-up displays will be named using the following format.

| Section | Figure | Table | Listing |
|-----------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |
| Health Outcomes | HO_Fn | HO_Tn | HO_Ln |
| Virology | VIR_Fn | VIR_Tn | VIR_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column.

#### 15.15.3. Deliverables

| Delivery [1] | Description |
|---|---|
| IW24 | IDMC analyses when approximately 50% participants have completed their Week 24 visits |
| W24 | Week 24 when 100% participants have completed their Week 24 visits |
| HL | Headline at Week 48 or Week 96 |
| W48 | Week 48 |
| W96 | Week 96 |
| W152 | Week 152 |
| Sub-study | Sub-study |
| EOS | End of study |

#### NOTES:

# 15.15.4. List of Data Displays for Week 24 IDMC and Week 24 Planned Analyses

For Week 24 planned analyses, the Week 24 Futility population will be replaced by the Intent-to-Treat Exposed population. In addition, unless otherwise specified, present the listings by prior exposure to CAB+RPV (i.e. rederived randomization strata, 0, 1-24, >24 weeks, refer to Section 15.6.2 for calculation details) except for study population listings.

<sup>1.</sup> Indicates order in which displays will be generated for the reporting effort

## 15.15.4.1. Study Population Tables

| Study P | Study Population Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Subject | Disposition | on | | | , | |
| 1.1 | NA | Week 24<br>Futility | ES1 | Summary of Subject Accountability: Maintenance Phase Conclusion Record - Week 24 Futility | ICH E3, GSKCTR, FDAAA,<br>EudraCT, see also in<br>201585/primary_02/T1.7. | IW24 |
| 1.2 | 1.1 | Intent-to-<br>Treat<br>Exposed | ES1 | Summary of Subject Accountability:<br>Maintenance Phase Conclusion Record - ITT-E | ICH E3, GSKCTR, FDAAA,<br>EudraCT, see also in<br>201585/primary_02/T1.7. | IW24, W24 |
| Demog | raphic and | Baseline Cha | aracteristics | | | |
| 1.3 | NA | Week 24<br>Futility | 201585/primary_02/T1.16 | Summary of Demographic Characteristics - Week 24 Futility | ICH E3, FDAAA, EudraCT | IW24 |
| 1.4 | 1.2 | Intent-to-<br>Treat<br>Exposed | 201585/primary_02/T1.16 | Summary of Demographic Characteristics - ITT-E | ICH E3, FDAAA, EudraCT | IW24, W24 |
| 1.5 | NA | Week 24<br>Futility | 201584/idmc_03/T1.3 | Summary of Prior Exposure to CAB+RPV -<br>Week 24 Futility | Adjust footnote and row labels as appropriate. | IW24 |
| 1.6 | 1.3 | Intent-to-<br>Treat<br>Exposed | 201584/idmc_03/T1.3 | Summary of Prior Exposure to CAB+RPV - ITT-E | Adjust footnote and row labels as appropriate. | IW24, W24 |
| 1.7 | 1.4 | Intent-to-<br>Treat<br>Exposed | 201584/idmc_03/T1.7 | Summary of Prior Exposure to CAB+RPV by Country | Adjust footnote and row labels as appropriate. | IW24, W24 |
| 1.8 | 1.5 | Intent-to-<br>Treat<br>Exposed | 201585/primary_02/T1.19 | Summary of Hepatitis Status at Entry | Add footnote as appropriate for subjects classified as Hepatitis B positive in analysis. | IW24, W24 |

# 15.15.4.2. Efficacy Tables

| Efficac | Efficacy Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.1 | 2.1 | Week 24<br>Futility | 201585/primary_02/T2.1 | Summary of Analysis for<br>Proportion of Subjects with<br>Plasma HIV-1 RNA ≥50 c/mL at<br>Week 24 and Posterior<br>Predictive Probability of Success<br>for the Q8W Arm - Snapshot<br>Analysis | For Week 24 IDMC, add a column on right with 'Posterior Predictive Probability of Success" and adjust the footnotes as appropriate, also add a footnote "Target threshold for posterior predictive probability is 15%.". For planned Week 24, remove 'and Posterior Predictive Probability of Success for the Q8W Arm' from the title, adjust the footnote as appropriate. For proportions, keep one decimal place. The adjustment is based on rederived randomization strata. | IW24, W24 |
| 2.2 | 2.2 | Week 24<br>Futility | 201585/primary_02/T2.4 | Summary of Study Outcomes<br>(50 c/mL Threshold) at Week 24<br>(Maintenance Phase) - Snapshot<br>Analysis | For proportions, keep one decimal place. | IW24, W24 |
| 2.3 | 2.3 | Week 24<br>Futility | 201585/primary_02/T2.6 | Note that only by randomization strata summary is provided. Change the footnote to "[1] Difference: Proportion on Q8W - Proportion on Q4W. 95% Cls were calculated using an unconditional exact method with two inverted one-sided tests based on the score statistic." Add Footnote "Note: Randomization strata are rederived using the prior exposure to CAB+RPV in Study 201585, collected from eCRF." For proportions, keep one decimal place. | | IW24, W24 |

| Efficac | Efficacy Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.4 | 2.4 | Week 24<br>Futility | 201585/primary_02/T2.21 | Cumulative Proportion of<br>Subjects Meeting Confirmed<br>Virologic Failure by Visit (Up to<br>Week 24) | For proportions, keep one decimal place. Non-snapshot visit window will be used. | IW24, W24 |
| 2.5 | 2.5 | Week 24<br>Futility | 201585/primary_02/T2.21 | Cumulative Proportion of<br>Subjects Meeting Confirmed<br>Virologic Failure by Visit and<br>Randomization Strata (Up to<br>Week 24) | Add column for 'Analysis Strata', add footnote for randomization strata similar to T2.3. For proportions, keep one decimal place. Non-snapshot visit window will be used. | IW24, W24 |
| 2.6 | 2.6 | Intent-to-<br>Treat<br>Exposed | 201585/primary_02/T2.21 | Cumulative Proportion of<br>Subjects Meeting Confirmed<br>Virologic Failure during the<br>Maintenance Phase | Note that this is overall summary, not by visit. Replace the column 'Timepoint' with 'CVF Category'. For proportions, keep one decimal place. | IW24, W24 |
| 2.7 | 2.7 | Intent-to-<br>Treat<br>Exposed | 201584/idmc_03/T2.7 | Cumulative Proportion of<br>Subjects Meeting Confirmed<br>Virologic Failure by<br>Randomization Strata during the<br>Maintenance Phase | Adjust footnote and row labels as appropriate. For proportions, keep one decimal place. Use rederived Randomization strata. | IW24, W24 |
| 2.8 | 2.8 | Week 24<br>Futility | EFF_T1 | Summary of Kaplan-Meier<br>Estimates of Proportion of<br>Subjects without CVF at Week<br>24 - Treatment Related<br>Discontinuation = Failure | The non-snapshot visit window for Week 24 will be used. | IW24, W24 |

| Efficac | Efficacy Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.9 | 2.9 | Week 24<br>Futility | EFF_T2 | Summary of Kaplan-Meier Estimates of Proportion of Subjects without CVF at Week 24 - Efficacy Related Discontinuation=Failure | The non-snapshot visit window for Week 24 will be used. | IW24, W24 |
| 2.10 | 2.10 | Intent-to-<br>Treat<br>Exposed | 201584/idmc_03/T2.10 | Proportion of Subjects with<br>Plasma HIV-1 RNA < 50 c/mL by<br>Visit - Observed Case Analysis | Adjust the footnote as appropriate. The non-<br>snapshot visit window will be used. For W24, add<br>'(Up to Week 24)' to the title, only display visits up<br>to Week 24. | IW24, W24 |
| 2.11 | 2.11 | Intent-to-<br>Treat<br>Exposed | 201584/idmc_03/T2.11 | Proportion of Subjects with<br>Plasma HIV-1 RNA <50 c/mL by<br>Visit and Randomization Strata -<br>Observed Case Analysis | Adjust footnote and row labels as appropriate. The non-snapshot visit window and rederived randomization strata will be used. For W24, add '(Up to Week 24)' to the title, only display visits up to Week 24. | IW24, W24 |

## 15.15.4.3. Efficacy Figures

| Efficacy | Efficacy Figures | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 2.1 | 2.1 | Week 24<br>Futility | 201584/idmc_03/F2.1 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit for Subjects Who are in the Category of 'Viral Load ≥50 c/mL' at Week 24 per Snapshot Algorithm | Adjust the x-axis label and footnote as appropriate. The x-values are based on study day of the assessment. | IW24, W24 |
| 2.2 | 2.2 | Intent-to-Treat<br>Exposed | 201584/idmc_03/F2.2 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit for Subjects with a Viral Load ≥50 c/mL during the Maintenance Phase | Adjust the x-axis label and footnote as appropriate. The x-values are based on study day of the assessment. | IW24, W24 |

## 15.15.4.4. Safety Tables

| Safety T | ables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverabl<br>e |
| Adverse | Events | | | | | |
| 3.1 | 3.1 | Safety | AE3 | Summary of All Adverse Events by Overall Frequency - Maintenance Phase | See also in 201585/primary_02/T3.20. | IW24, W24 |
| 3.2 | 3.2 | Safety | AE1 | Summary of All Drug-Related Adverse Events by<br>System Organ Class - Maintenance Phase | See also in 201585/primary_02/T3.16. | IW24, W24 |
| 3.3 | 3.3 | Safety | AE3 | Summary of Grade 3-5 Adverse Events by Overall Frequency - Maintenance Phase | See also in 201585/primary_02/T3.20. | IW24, W24 |
| Serious | and Oth | er Significant | Adverse Events | | | |
| 3.4 | 3.4 | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class - Maintenance Phase | See also in 201585/primary_02/T3.21. | IW24, W24 |
| 3.5 | 3.5 | Safety | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class - Maintenance Phase | See also in 201585/primary_02/T3.31. | IW24, W24 |
| Injection | n Site Re | action Advers | e Events | | | |
| 3.6 | 3.6 | Safety | 201585/primary_02/T3.<br>40 | Summary of Injection Site Reaction Adverse Events (Event-Level Summary) - Maintenance Phase | For W24, add 'Study Drug' before 'Injection' in the title and only summarize ISR from study drug injections. | IW24, W24 |

| Safety T | ables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverabl<br>e |
| 3.7 | 3.7 | Safety | 201585/primary_02/T3.<br>43 | Summary of Subject-Level Characteristics of Injection<br>Site Reaction Adverse Events - Overall and Common<br>(Maintenance Phase) | Common ISR adverse events includes injection site pain, injection site induration, injection site nodules and any other ISR with ≥5% subjects in either treatment arm. For W24, add 'Study Drug' before 'Injection' in the title and only summarize ISR from study drug injections. | IW24, W24 |
| Laborat | ory: Che | mistry and He | matology | | | |
| 3.8 | 3.8 | Safety | 201584/idmc_03/T3.8 | Summary of Maximum Post-Baseline Emergent<br>Clinical Chemistry Toxicities Parameters of Special<br>Interest - Maintenance Phase | Replace "Day 1" with "Study Day 1" in the first footnote. Use the same parameter list as the one in 201584/idmc_03/T3.8. | IW24, W24 |
| 3.9 | 3.9 | Safety | 201584/idmc_03/T3.9 | Summary of Maximum Post-Baseline Emergent<br>Hematology Toxicities Parameters of Special Interest<br>- Maintenance Phase | Replace "Day 1" with "Study Day 1" in the first footnote. Adjust the second footnote to be: "Note: Parameters of Special Interest include Hemogoblin, Leukocytes, Neutrophils, and Platelets." In output, change the parameter label 'White Blood Cell count' to 'Leukocytes'. | IW24, W24 |

## 15.15.4.5. Safety Figures

| Safety | Safety Figures | | | | | |
|---|---|---|---|---|---|---|
| No.<br>in<br>IW24 | No.<br>in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Labora | atory: H | epatobiliary (Liver | ) | | | |
| 3.1 | 3.1 | Safety | 201584/idmc_03/F3.2 | Scatter Plot of Maximum Maintenance Phase vs.<br>Baseline for ALT | Adjust the legend as needed. Change the first footnote to "Axes are on a log10 scale". Remove the second footnote. Adjust the treatment label from empty triangle to solid triangle. | IW24, W24 |
| 3.2 | 3.2 | Safety | 201584/idmc_03/F3.1 | Matrix Plot of Maximum Liver Chemistries -<br>Maintenance Phase | Replace ">5.1" with ">5.0" in the second footnote. Make treatment labels in the plot consistent across figures. | IW24, W24 |

#### 15.15.4.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.1 | 4.1 | Pharmacokinetic | 201585/primary_02/T4.1 | Summary of Plasma CAB PK Concentrations (ug/mL) - Time Data by Treatment and Visit - Including Log-Transformed Statistics | Remove the first footnote "Note:". | IW24, W24 |
| 4.2 | 4.2 | Pharmacokinetic | 201585/primary_02/T4.2 | Summary of Plasma RPV PK Concentrations (ng/mL) - Time Data by Treatment and Visit - Including Log-Transformed Statistics | Remove the first footnote "Note:" | IW24, W24 |
| 4.3 | NA | Pharmacokinetic | 201584/idmc_03/T4.3 | Proportion of Subjects with Evaluable PK Concentration below Expected Values | | IW24 |

## 15.15.4.7. Pharmacokinetic Figures

| Pharma | Pharmacokinetic Figures | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.1 | NA | Pharmacokinetic | 201584/idmc_03/<br>F4.1 | Scatter Plot of Evaluable PK Concentrations in<br>Relation to Occurrence of CVF up to Week 16 for<br>Subjects on Q8W Arm by Visit and Randomization<br>Strata | Note that this plot is by visit and rederived randomization strata. Add footnote for strata as appropriate. | IW24 |

# 15.15.4.8. Virology Tables

| Virology | y Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverabl<br>e |
| 7.1 | 7.1 | Confirmed<br>Virologic Failure | 201585/primary<br>_02/T8.1 | Summary of the Prevalence of Known INI Resistance<br>Mutations at Time of CVF (Maintenance Phase) -<br>Plasma Sample | | IW24, W24 |
| 7.2 | 7.2 | Confirmed<br>Virologic Failure | 201585/primary<br>_02/T8.2 | Summary of the Prevalence of Major Resistance<br>Mutations of NNRTI, NRTI, and PI Class at Time of<br>CVF (Maintenance Phase) - Plasma Sample | | IW24, W24 |
| 7.3 | 7.3 | Confirmed<br>Virologic Failure | 201585/primary<br>_02/T8.3 | Summary of Phenotypic Susceptibility at Time of CVF (Maintenance Phase) - Plasma Sample | | IW24, W24 |
| 7.4 | 7.4 | Confirmed<br>Virologic Failure | 201585/primary<br>_02/T8.7 | Summary of Fold Change to CAB and RPV at Time of CVF (Maintenance Phase) - Plasma Sample | | IW24, W24 |
| 7.5 | 7.5 | Confirmed<br>Virologic Failure | 201585/primary<br>_02/T8.8 | Summary of Viral Load, Genotypic and Phenotypic Data for Subjects Who Met Confirmed Virologic Failure Criteria during the Maintenance Phase | Remove the Columns 'ARTs' and 'FC for ARTs'. Remove the footnotes [1] and [2]. Adjust the footnote as appropriate. | IW24, W24 |

# 15.15.4.9. ICH Listings

Note: Both unique subject ID and latest subject ID for a subject will be included in the listings, unless otherwise specified.

| ICH List | ICH Listings | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Study P | Study Population | | | | | |
| 1 | 1 | Randomized | 201584/idmc_03/L1.<br>3 | Listing of Randomized and Actual Strata and Treatment Assignment | Randomized and Actual Treatments will include oral lead-in information (e.g. Oral followed by Q4W). For W24 analyses, remove column for Futility Population. | IW24, W24 |
| Efficacy | 1 | | | | | |
| 2 | 2 | Week 24 Futility | 201585/primary_02/<br>L11 | Listing of Study Outcomes (50 c/mL<br>Threshold) at Week 24 - Snapshot Analysis | | IW24, W24 |
| Adverse | Events | | | | | |
| 3 | 3 | Safety | 201585/primary_02/<br>L17 | Listing of Adverse Events Leading to<br>Withdrawal/Permanent Discontinuation of<br>Investigational Product - Maintenance<br>Phase | Remove "Time Since Last Dose" from the column header. | IW24, W24 |
| 4 | 4 | Safety | 201585/primary_02/<br>L17 | Listing of All Serious Adverse Events -<br>Maintenance Phase | Remove "Time Since Last Dose" from the column header. | IW24, W24 |
| Laborat | ory | | | | | |
| 5 | NA | Safety | 201584/idmc_03/L3.<br>5 | Listing of All Parameters of Special Interest<br>Laboratory Data for Subjects with Grade 3<br>or 4 Maintenance Phase Emergent<br>Toxicities for Parameters of Special Interest | Replace 'Day 1' with 'Study Day 1' in the second footnote. | IW24 |

| ICH List | tings | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| PK | | | | | | |
| 6 | 5 | Pharmacokinetic | 201584/idmc_03/L4.<br>1 | Listing of Plasma CAB PK Concentration-<br>Time Data | Change the first footnote to "Relative Time is calculated relative to the date and time of last previous dose. If the time of the last previous dose (e.g. oral lead-in/oral bridging) is missing, then the relative time will be set to missing and the sample will not be considered 'evaluable'." Remove the second footnote. Change column header 'Visit' to 'Analysis Visit/Nominal Visit' to include both visits. | IW24, W24 |
| 7 | 6 | Pharmacokinetic | 201584/idmc_03/L4.<br>2 | Listing of Plasma RPV PK Concentration-<br>Time Data | Change the first footnote to "Relative Time is calculated relative to the date and time of last previous dose. If the time of the last previous dose (e.g. oral lead-in/oral bridging) is missing, then the relative time will be set to missing and the sample will not be considered 'evaluable'." Remove the second footnote. Change column header 'Visit' to 'Analysis Visit/Nominal Visit' to include both visits. | IW24, W24 |

## 15.15.4.10. Non-ICH Listings

Note: Both unique subject ID and latest subject ID for a subject will be included in the listings, unless otherwise specified.

| Non-ICH | l Listings | ; | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Study P | opulation | 1 | | | | |
| 8 | 7 | Intent-to-Treat<br>Exposed | ES2 | Listing of Reasons for Maintenance Phase Withdrawal | See also in 201585/primary_02/L30. | IW24, W24 |
| 9 | 8 | Screened | Shell POP_L2 | Listing of Subjects Who Were Rescreened | | IW24, W24 |
| 10 | 9 | Intent-to-Treat<br>Exposed | 201584/idmc_0<br>3/L1.1 | Listing of Prior Antiretroviral Therapy | Remove the column 'Treatment Phase/Treatment State'. Add a column for Route. | IW24, W24 |
| 11 | 10 | Intent-to-Treat<br>Exposed | 201584/idmc_0<br>3/L1.2 | Listing of Concomitant Antiretroviral Therapy | Change column 'Treatment<br>Phase/Actual Treatment State' to<br>'Phase during Which Concomitant',<br>remove 'Induction Study Day' from<br>column headers, and remove<br>'Maintenance' from 'Maintenance<br>Study Day' in column headers. | IW24, W24 |
| Efficacy | 1 | | | | | |
| 12 | 11 | Confirmed Virologic<br>Failure | 201585/primary<br>_02/L40 | Listing of All Plasma HIV-1 RNA Viral Load<br>Data for Subjects with Confirmed Virologic<br>Failure during the Maintenance Phase | Non-snapshot visit window will be used for deriving the visits in Column 'Actual Relative Time'. Replace 'Period' in column header with 'Phase'. | IW24, W24 |

| Non-ICH | l Listings | 3 | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 13 | 12 | Week 24 Futility | 201585/primary<br>_02/L40 | Listing of All Plasma HIV-1 RNA Viral Load Data for Subjects Who are in the Category of 'Viral load ≥50 c/mL' at Week 24 per Snapshot Algorithm | Non-snapshot visit window will be used for deriving the visits in Column 'Actual Relative Time'. Replace 'Period' in column header with 'Phase'. | IW24, W24 |
| Adverse | Events | | | | | |
| 14 | 13 | Safety | 201585/primary<br>_02/L17 | Listing of All Drug-Related Adverse Events - Maintenance Phase | Remove "Time Since Last Dose" from the column header. | IW24, W24 |
| 15 | 14 | Safety | 201585/primary<br>_02/L17 | Listing of All Grade 3-5 Adverse Events -<br>Maintenance Phase | Remove "Time Since Last Dose" from the column header. | IW24, W24 |
| 16 | 15 | Safety | 201585/primary<br>_02/L17 | Listing of All Adverse Events - Long-term Follow-up Phase | Remove "Time Since Last Dose" from the column header. | IW24, W24 |
| PK | | | | | | |
| 17 | NA | Pharmacokinetic | 201584/idmc_0<br>3/L4.3 | Listing of Plasma CAB PK Concentration-Time Data for Subjects with CAB Concentration <1.35 ug/mL (~8 X PAIC90) at Visits up to Week 16 | Change the first footnote to "Relative Time is calculated relative to the date and time of last previous dose. If the time of the last previous dose (e.g. oral lead-in/oral bridging) is missing, then the relative time will be set to missing and the sample will not be considered 'evaluable'." Remove the second footnote. Change column header 'Visit' to 'Analysis Visit/Nominal Visit' to include both visits. | IW24 |

| Non-ICH | Non-ICH Listings | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 18 | NA Pharmacekinetic 201584/idmc_0 Data for Subjects | | Listing of Plasma CAB PK Concentration-Time Data for Subjects with CAB Concentration <0.166 ug/mL (PAIC90) at Visits up to Week 16 | The same note as in Listing 17. | IW24 | |
| 19 | NA | Pharmacokinetic | 201584/idmc_0<br>3/L4.5 | Listing of Plasma RPV PK Concentration-Time Data for Subjects with RPV Concentration <12 ng/mL (PAIC90) at Visits up to Week 16 | The same note as in Listing 17. | IW24 |
| Virology | / | | | | | |
| 20 | 16 | Confirmed Virologic Failure | 201584/idmc_0<br>3/L7.1 | Listing of Genotypic Mutation Data at All Timepoints | | IW24, W24 |
| 21 | 17 | Confirmed Virologic Failure | 201584/idmc_0<br>3/L7.2 | Listing of Phenotypic Data at All Timepoints | | IW24, W24 |

## 15.15.5. List of Data Displays for Week 48/96/End-of-Study Planned Analyses

## 15.15.5.1. Study Population Tables

| Study F | opulation | n Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subject | Subject Disposition | | | | | | |
| 1.1 | 1.1 | 1.1 | Randomized | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | 'No Treatment' column is not needed. | W48, W96, EOS |
| 1.2 | 1.2 | 1.2 | Screened | ES6 | Summary of Screening Status and Reasons for Screening Failures | | W48, W96 |
| 1.3 | 1.3 | 1.3 | Intent-to-<br>Treat<br>Exposed | ES1 | Summary of Subject Accountability: Study<br>Conclusion Record | For WK 96 and EOS: Add a footnote [1] for Subject Status: "[1] Subject Status is derived based on the data collected from the Study Conclusion eCRF form. "COMPLETED" subjects are those completing the study without reasons beyond the completion of the study commitment. "WITHDRAWN" subjects are those either withdrawn from Maintenance / Extension phase, or those who completed Maintenance phase and decided not to enter Extension phase due to reasons beyond the completion of the study commitment (Subjects xxx, xxx, and xxx are in this group and | W48, W96, EOS |

| Study F | Study Population Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | | | their primary reasons for withdrawal are xxx, xxx and xxx respectively.)." Update the numbering of other footnotes accordingly. Footnotes may be adjusted as appropriate. Add a section "Type of Adverse Events Which Led to Study Withdrawal" with categories "COVID-19" and "Non-COVID-19". | |
| 1.4 | 1.4 | NA | Intent-to-<br>Treat<br>Exposed | ES1 | Summary of Subject Accountability:<br>Maintenance Phase Conclusion Record | For W96: Add a section "Type of Adverse Events Which Led to Study Withdrawal" with categories "COVID-19" and "Non-COVID-19". | HL, W48, W96 |
| NA | 1.5 | 1.4 | Intent-to-<br>Treat<br>Exposed | ES1 | Summary of Subject Accountability: Maintenance + Extension Phase Conclusion Record | For subject status, refer to 201584/primary_07/T1.10 for the layout. For W96 and EOS: Add a section "Type of Adverse Events Which Led to Study Withdrawal" with categories "COVID-19" and "Non-COVID-19". | W96, EOS |
| 1.5 | 1.6 | 1.5 | Long-term<br>Follow-up | ES1 | Summary of Subject Accountability: Long-term Follow-up Phase Conclusion Record | For W96 and EOS: Add a section "Type of Adverse Events Which Led to Study Withdrawal" with categories | W48, W96, EOS |

| Study F | Study Population Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | | | "COVID-19" and "Non-COVID-<br>19". | |
| 1.6 | 1.7 | 1.6 | Intent-to-<br>Treat<br>Exposed | ES4 | Summary of Subject Disposition at Each Study Phase | Replace 'Epoch' with 'Phase' in column header. Screening Phase will not be included. Add a footnote "Note: Entry into Long-Term Follow-up is based on presence of a long-term follow-up visit in the eCRF (i.e. LTFU Month 1, LTFU Month 3, etc.) or evidence of filling out the long-term follow-up phase conclusion form." For WK96 and EOS, update the last part of the footnote to be "or evidence of filling out the long-term follow-up phase conclusion form or indication of continuing into the long-term follow-up phase in the subject continuation form." | W48, W96, EOS |
| 1.7 | 1.8 | 1.7 | Intent-to-<br>Treat<br>Exposed | ES5 | Summary of Reasons for Withdrawal at Each Study Phase | The same comment as above. | W48, W96, EOS |
| 1.8 | 1.9 | 1.8 | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T1.9 | Summary of Subject Accountability: Withdrawals by Visit (Maintenance + Extension Phase) | | W48, W96, EOS |

| Study F | opulation | n Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.9 | 1.10 | 1.9 | Intent-to-<br>Treat<br>Exposed | ES1 | Summary of Study Drug Discontinuation | Update the row label to 'Primary Reason[1]/Subreason[2] for Study Drug Discontinuation'. For W96 and EOS: Add a section "Type of Adverse Events Which Led to Study Drug Discontinuation" with categories "COVID-19" and "Non-COVID-19". | W48, W96, EOS |
| 1.10 | 1.11 | NA | Intent-to-<br>Treat<br>Exposed | DV1a | Summary of Important Protocol Deviations | | W48, W96, EOS |
| NA | 1.12 | 1.10 | Intent-to-<br>Treat<br>Exposed | DV1a | Summary of Important Protocol Deviations (Maintenance + Extension Phase) | | W96, EOS |
| 1.11 | 1.13 | 1.11 | Intent-to-<br>Treat<br>Exposed | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | W48, W96 |
| 1.12 | 1.14 | 1.12 | Screened | 201585/primar<br>y_02/T1.1 | Summary of Study Populations | Adjust the footnote as appropriate. | HL, W48, W96,<br>EOS |
| 1.13 | 1.15 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.14 | Summary of Protocol Deviations Leading to Exclusion from the Per-Protocol Population | | W48, W96 |
| NA | 1.36 | 1.32 | Intent-to-<br>Treat<br>Exposed | DV1a | Summary of Important COVID-19 Related Protocol Deviations | Update the label for the first row to be "ANY IMPORTANT COVID-19 RELATED PROTOCOL DEVIATIONS". | W96, EOS |

| Study F | opulation | n Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| NA | 1.37 | 1.33 | Intent-to-<br>Treat<br>Exposed | DV1a | Summary of Important Non-COVID-19 Related Protocol Deviations | Update the label for the first row to be "ANY IMPORTANT NON-COVID-19 RELATED PROTOCOL DEVIATIONS". | W96, EOS |
| Demog | raphic an | d Baseli | ne Characteris | tics | | | |
| 1.14 | 1.16 | 1.13 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.16 | Summary of Demographic Characteristics | | HL, W48, W96,<br>EOS |
| 1.15 | 1.17 | 1.14 | Randomized | DM11 | Summary of Age Ranges | Also refer to 201585/primary_02/T1.4. Follow the footnote in 201585/primary_02/T1.4. | W48, W96 |
| 1.16 | 1.18 | 1.15 | Intent-to-<br>Treat<br>Exposed | DM5 | Summary of Race and Racial Combinations | | W48, W96, EOS |
| 1.17 | 1.19 | 1.16 | Intent-to-<br>Treat<br>Exposed | DM6 | Summary of Race and Racial Combinations<br>Details | | W48, W96, EOS |
| 1.18 | 1.20 | 1.17 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.19 | Summary of Hepatitis Status at Entry | Add footnote as appropriate for subjects classified as Hepatitis B positive in analysis. | W48, W96 |
| 1.19 | 1.21 | 1.18 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.20 | Summary of Derived Baseline CDC Stages of HIV Infection | | W48, W96 |
| 1.20 | 1.22 | 1.19 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.21 | Summary of Baseline Cardiovascular Risk<br>Assessments | | W48, W96 |

| Study F | opulation | n Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.21 | 1.23 | 1.20 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.22 | Distribution of CD4+ Cell Count Results at Screening and Baseline | | W48, W96 |
| 1.22 | 1.24 | 1.21 | Intent-to-<br>Treat<br>Exposed | Shell POP_T1 | Summary of Prior Exposure to CAB+RPV | | W48, W96 |
| 1.23 | 1.25 | 1.22 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.36 | Summary of HIV Risk Factors | | W48, W96 |
| Medica | Condition | ns and N | Medications | | | | |
| 1.24 | 1.26 | 1.23 | Intent-to-<br>Treat<br>Exposed | MH1 | Summary of Current Medical Conditions | | W48, W96, EOS |
| 1.25 | 1.27 | 1.24 | Intent-to-<br>Treat<br>Exposed | MH1 | Summary of Past Medical Conditions | | W48, W96, EOS |
| 1.26 | 1.28 | 1.25 | Intent-to-<br>Treat<br>Exposed | MH4 | Summary of Current Cardiac, Gastrointestinal,<br>Metabolism and Nutrition, Psychiatric, Renal<br>and Urinary, Nervous System Conditions, and<br>Hepatobiliary Disorders | | W48, W96, EOS |
| 1.27 | 1.29 | 1.26 | Intent-to-<br>Treat<br>Exposed | MH4 | Summary of Past Cardiac, Gastrointestinal,<br>Metabolism and Nutrition, Psychiatric, Renal<br>and Urinary, Nervous System Conditions, and<br>Hepatobiliary Disorders | | W48, W96, EOS |
| 1.28 | 1.30 | 1.27 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.28 | Summary of Prior ART Medications | Remove the footnote. Follow definitions in Section 6.2 to | W48, W96 |

| Study F | Study Population Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | | | determine the prior ART medications. | |
| 1.29 | 1.31 | NA | Intent-to-<br>Treat<br>Exposed | CM8 | Summary of Concomitant Non-ART Medication Ingredient Combinations (Maintenance Phase) | | W48, W96 |
| NA | 1.32 | 1.28 | Intent-to-<br>Treat<br>Exposed | CM8 | Summary of Concomitant Non-ART<br>Medication Ingredient Combinations<br>(Maintenance + Extension Phase) | | W96, EOS |
| 1.30 | 1.33 | 1.29 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.33 | Summary of Lipid Modifying Agent Use at Baseline | | W48, W96 |
| 1.31 | 1.34 | 1.30 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.34 | Summary of Lipid Modifying Agent Use<br>Started during the Maintenance Phase | | W48, W96 |
| 1.32 | 1.35 | 1.31 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.35 | Summary of Substance Use at Entry | | W48, W96 |

#### 15.15.5.2. Efficacy Tables

**Note:** For subgroup analyses, include rederived randomization strata (i.e. prior exposure to CAB+RPV: 0, 1-24, >24 weeks), all demographic and baseline characteristic subgroups as mentioned in EMA Subgroup Category 2 in Section 5.4.2, unless otherwise specified. Not all subjects on Q8W arm are planned to have viral load data collected at Week 4 (Week 4A or 4B), so leave Week 4 data blank for Q8W arm in by-visit snapshot analysis.

| Efficacy | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Primary | Efficacy | Analyse | s | | | | |
| 2.1 | 2.1 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis – ITT-E | Adjust the footnotes as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. | HL, W48, W96 |
| 2.2 | 2.2 | NA | Per-<br>Protocol | 201584/primar<br>y_01/T2.2 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis – Per-Protocol | Adjust the footnotes as appropriate. For WK96: replace 'Week 48' with 'Week 96' in title. | HL, W48, W96 |
| 2.3 | 2.3 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.3 | Summary of Study Outcomes (50 c/mL Threshold) at Week 48 (Maintenance Phase) – Snapshot Analysis | For WK96: replace 'Week 48' with 'Week 96' in title. Use shell EFF_T5 for mock-up. | HL, W48, W96 |
| 2.4 | 2.4 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T3 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 48 (Maintenance Phase) - Snapshot Analysis | For WK96, replace 'Week 48' with 'Week 96' in title. | HL, W48, W96 |

| Efficacy | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.5 | 2.5 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.5 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 48 by Subgroup (Maintenance Phase) - Snapshot Analysis | Adjust the footnote/column header label as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. Do not include rederived randomization strata in the table. | W48, W96 |
| 2.6 | 2.6 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T4 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 48 among Subjects with >=1 Weeks Prior Exposure to CAB+RPV (Maintenance Phase) - Snapshot Analysis | For WK96, replace 'Week 48' with 'Week 96' in title. | W48, W96 |
| 2.7 | 2.7 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.6 | Summary of Study Outcomes (50 c/mL Threshold) at Week 48 by Subgroup (Maintenance Phase) – Snapshot Analysis | For WK96: replace 'Week 48' with 'Week 96' in title. Use shell EFF_T5 for mock-up of each subgroup's study outcomes. | W48, W96 |
| Seconda | ary and E | Explorato | ory Efficacy A | nalyses | | | |
| 2.8 | 2.8 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.7 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis – ITT-E | Adjust the footnotes as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. | HL, W48, W96 |
| 2.9 | 2.9 | NA | Per-<br>Protocol | 201584/primar<br>y_01/T2.8 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis – Per-Protocol | Adjust the footnotes as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. | HL, W48, W96 |

| Efficacy | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.10 | 2.10 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T3 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 (Maintenance Phase) - Snapshot Analysis | Replace 'Number of HIV-1<br>RNA >=50 c/mL' with<br>'Number of HIV-1 RNA <50<br>c/mL' in column header. For<br>WK96, replace 'Week 48'<br>with 'Week 96' in title. | HL, W48, W96 |
| 2.11 | 2.11 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.10 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 by Subgroup (Maintenance Phase) - Snapshot Analysis | Adjust the footnote/column header label as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. Do not include rederived randomization strata in the table. | W48, W96 |
| 2.12 | 2.12 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T4 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 among Subjects with >=1 Weeks Prior Exposure to CAB+RPV (Maintenance Phase) - Snapshot Analysis | Replace 'Number of HIV-1<br>RNA >=50 c/mL' with<br>'Number of HIV-1 RNA <50<br>c/mL' in column header. For<br>WK96, replace 'Week 48'<br>with 'Week 96' in title. | W48, W96 |
| 2.13 | 2.13 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.11 | Proportion of Subjects with Plasma HIV-1 RNA<br>>=50 c/mL by Visit (Maintenance Phase) –<br>Snapshot Analysis | | W48, W96 |
| 2.14 | 2.14 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.12 | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Subgroup and Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.15 | 2.15 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.15 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |

| Efficacy | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.16 | 2.16 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.16 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Subgroup and Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.17 | 2.17 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.17 | Proportion of Subjects with Plasma HIV-1 RNA <200 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.18 | 2.18 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.17 | Proportion of Subjects with Plasma HIV-1 RNA >=200 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | Adjust column headers as appropriate. Keep one decimal place for proportion. | W48, W96 |
| 2.19 | 2.19 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T1 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Failure at Week 48 - Treatment Related Discontinuation = Failure | Adjust the row labels and footnotes as appropriate. For WK96, replace 'Week 48' with 'Week96' in title. | W48, W96 |
| 2.20 | 2.20 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T2 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Failure at Week 48 - Efficacy Related Discontinuation = Failure | Adjust the row labels and footnotes as appropriate. For WK96, replace 'Week 48' with 'Week96' in title. | W48, W96 |

| Efficacy | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.21 | 2.21 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.19 | Proportion of Subjects with HIV-1 RNA >=50 c/mL at Week 48 (Snapshot) by Last Delay in IP Injection (Maintenance Phase) | Display both arms. Change the footnote to 'The last delay in IP injection will be the delay in IP injection at Week 48, or the delay in last IP injection prior to Week 48 if a participant did not receive Week 48 injection (i.e. missing visit or withdrawal).'. For WK96, replace 'Week 48' with 'Week 96' in the title and footnote accordingly. | W48, W96 |
| 2.22 | 2.22 | 2.1 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.20 | Summary of Plasma HIV-1 RNA (log10 c/mL) by<br>Visit (Maintenance + Extension Phase) | | W48, W96,<br>EOS |
| 2.23 | 2.23 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.21 | Cumulative Proportion of Subjects Meeting<br>Confirmed Virology Failure Criteria by Visit during<br>the Maintenance Phase (Up to Week 48) | For WK96, remove 'Up to Week 48' in title. | HL, W48, W96 |
| 2.24 | 2.24 | 2.2 | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.21 | Cumulative Proportion of Subjects Meeting Confirmed Virology Failure Criteria (Maintenance + Extension Phase) | | HL, W48,<br>W96, EOS |
| 2.25 | 2.25 | NA | Confirmed<br>Virologic<br>Failure | 201584/primar<br>y_01/T2.24 | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmation of Confirmed Virologic Failure (Maintenance Phase) | | W48, W96 |

| Efficacy | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.26 | 2.26 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.34 | Proportion of Subjects with Plasma HIV-1 RNA <2 c/mL by Visit (Maintenance Phase) | Change footnote to 'Note: Data come from BioMontr low-level assay. Only visits with available data from this assay are included.' | W48, W96 |
| 2.27 | 2.27 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.51 | Summary of Study Outcomes (200 c/mL Threshold) at Week 48 (Maintenance Phase) – Snapshot Analysis | For WK96: replace 'Week 48' with 'Week 96' in title. Use shell EFF_T5 for mock-up. | W48, W96 |
| 2.28 | 2.28 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.37 | Summary of Subjects per Viral Load Category by Visit (Maintenance Phase) | Refer to 'Summary for Participants per Viral Load Category by Visit' in Section 15.6.3. Remove footnote [2]. Add a footnote "Note: The visit windows are based on snapshot analysis windows'. | W48, W96 |
| 2.29 | 2.29 | 2.3 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.25 | Summary of Change from Baseline in CD4+ Cell<br>Count (cells/mm^3) by Visit (Maintenance +<br>Extension Phase) | | W48, W96,<br>EOS |
| 2.30 | 2.30 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.38 | Summary of Change from Baseline in CD4+ Cell<br>Count (cells/mm^3) at Week 48 by Subgroup<br>(Maintenance Phase) | For WK96, replace 'Week 48' with 'Week 96' in title. | W48, W96 |
| 2.31 | 2.31 | 2.4 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.26 | Summary of CD4+ Cell Count (cells/mm^3) by Visit (Maintenance + Extension Phase) | | W48, W96,<br>EOS |
| 2.32 | 2.32 | 2.5 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.28 | Summary of Change from Baseline in CD8+ Cell Count (cells/mm^3) by Visit (Maintenance Phase) | | W48, W96,<br>EOS |

| Efficacy Tables | | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.33 | 2.33 | 2.6 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.27 | Summary of CD8+ Cell Count (cells/mm^3) by Visit (Maintenance Phase) | | W48, W96,<br>EOS |
| 2.34 | 2.34 | 2.7 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.29 | Summary of CD4+/CD8+ Ratio Cell Count (cells/mm^3) by Visit (Maintenance Phase) | Ratio will be taken when both CD4+ and CD8+ are available on the same date. | W48, W96,<br>EOS |
| 2.35 | 2.35 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.30 | Summary of HIV-1 Associated Conditions Including Recurrences (Maintenance Phase) | | W48, W96 |
| NA | NA | 2.8 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.30 | Summary of HIV-1 Associated Conditions Including Recurrences (Maintenance +Extension Phase) | | EOS |
| 2.36 | 2.36 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.31 | Summary of HIV-1 Associated Conditions Excluding Recurrences (Maintenance Phase) | | W48, W96 |
| NA | NA | 2.9 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.31 | Summary of HIV-1 Associated Conditions Excluding Recurrences (Maintenance +Extension Phase) | | EOS |
| 2.37 | 2.37 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.47 | Summary of HIV-1 Disease Progression and/or Deaths (Maintenance Phase) | For WK96: add a superscript [1] to the first n and add a footnote: "Note: It is the denominator for all percentages." | W48, W96 |

| Efficacy Tables | | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| NA | NA | 2.10 | Intent-to-<br>Treat<br>Exposed | 207966/primar<br>y_02/T2.37 | Summary of HIV-1 Disease Progression and/or Deaths (Maintenance + Extension Phase) | Replace "maintenance" with "maintenance and extension" in the footnote; add a superscript [1] to the first n and add a footnote: "Note: It is the denominator for all percentages." | EOS |
| 2.38 | 2.38 | 2.11 | Intent-to-<br>Treat<br>Exposed | 207966/primar<br>y_02/T2.38 | Summary of Change from Baseline in Plasma HIV-1<br>RNA (log10 c/mL) by Visit (Maintenance +<br>Extension Phase) | | W48, W96,<br>EOS |
#### 15.15.5.3. Efficacy Figures

**Note:** For subgroup analyses, include rederived randomization strata (i.e. prior exposure to CAB+RPV: 0, 1-24, >24 weeks), all demographic and baseline characteristic subgroups as mentioned in EMA Subgroup Category 2 in Section 5.4.2, unless otherwise specified. Not all subjects on Q8W arm are planned to have viral load data collected at Week 4 (Week 4A or 4B), so leave Week 4 data blank for Q8W arm in by-visit snapshot analysis.

| Efficacy | / Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Primary | Efficacy | Analyses | | | | | |
| 2.1 | 2.1 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F2.1 | Proportion (95% CI) of Subjects with HIV-1 RNA<br>≥50 c/mL by Visit (Maintenance Phase) –<br>Snapshot Analysis | | HL, W48, W96 |
| 2.2 | 2.2 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primary<br>_01/F2.2 | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA ≥50 c/mL at Week 48 by Subgroup – Snapshot Analysis | Non-inferiority margin is 4%.<br>Adjust the footnotes,<br>reference line and labels as<br>appropriate. For WK96,<br>replace 'Week 48' with<br>'Week 96' in title. | W48, W96 |
| Second | ary and E | xploratory | / Efficacy Ana | llyses | | | |
| 2.3 | 2.3 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F2.3 | Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | HL, W48, W96 |
| 2.4 | 2.4 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primary<br>_01/F2.4 | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL at Week 48 by Subgroup – Snapshot Analysis | Adjust the footnotes, reference line and labels as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. | W48, W96 |

| Efficacy | / Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.5 | 2.5 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F2.10 | Proportion (95% CI) of Subjects with HIV-1 RNA >=200 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.6 | 2.6 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F2.5 | Proportion (95% CI) of Subjects with HIV-1 RNA <200 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.7 | 2.7 | 2.1 | Intent-to-<br>Treat<br>Exposed | 207966/idmc_0<br>3/F2.1 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit – for CVF Subjects | | HL, W48,<br>W96, EOS |
| 2.8 | 2.8 | NA | Intent-to-<br>Treat<br>Exposed | 207966/idmc_0<br>3/F2.1 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit for subjects Who are in the Category of 'HIV-1 RNA >=50 c/mL' at Week 48 per Snapshot Algorithm | For WK96, replace 'Week 48' with 'Week 96' in the title. | HL, W48, W96 |

## 15.15.5.4. Safety Tables

| Safety 7 | Safety Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Exposu | re | | | | | | |
| 3.1 | 3.1 | 3.1 | Safety | 201585/primar<br>y_02/T3.1 | Summary of Extent of Exposure to Investigational Product (Maintenance Phase) | No need for the first two footnotes. Update the last footnote to be below: Note: The injection at nominal visit of Week 100 was not included in the summary of Exposure (No. of IP injections). For W96 and EOS: Replace "Investigational Product" with "Study Treatment including SOC Oral Bridging" in the title; Add sections after Section "Exposure (No. of IP injection visits)" for exposure to CAB+RPV oral bridging and exposure to SOC oral bridging similarly to exposure to oral lead-in; Add sections for overall exposure to IP similarly to overall exposure; the levels for categorical summaries will be selected as appropriate. | W48, W96 |
| NA | 3.2 | 3.2 | Safety | 201585/primar<br>y_02/T3.1 | Summary of Extent of Exposure to Investigational Product (Maintenance + Extension Phase) | Remove the footnotes. For W96 and EOS: update similarly to the table above. | W96, EOS |
| 3.2 | 3.3 | NA | Safety | 201585/primar<br>y_03/T3.102 | Summary of Needle Length and Gauge for CAB Injection (Maintenance Phase) | Display both arms. | W48, W96 |
| 3.3 | 3.4 | NA | Safety | 201585/primar<br>y_03/T3.103 | Summary of Needle Length and Gauge for RPV Injection (Maintenance Phase) | Display both arms. | W48, W96 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.4 | 3.5 | NA | Safety | 201585/primar<br>y_02/T3.6 | Summary of Adherence to CAB/RPV Injection Dosing Schedule (Maintenance Phase) | Display both arms. Adjust the footnotes as appropriate. For W96, present "Missed Injection with CAB+RPV Oral Bridging" and "Missed Injection with SOC Oral Bridging" separately. | W48, W96 |
| Adverse | Events | | | | | | |
| 3.5 | 3.6 | NA | Safety | 201585/primar<br>y_02/T3.7 | Summary of All Adverse Events by System Organ Class (Maintenance Phase) | | W48, W96 |
| 3.6 | 3.7 | NA | Safety | 201585/primar<br>y_02/T3.8 | Summary of All Adverse Events by System Organ Class and Maximum Toxicity (Maintenance Phase) | | HL, W48,<br>W96 |
| NA | 3.8 | 3.3 | Safety | 201585/primar<br>y_02/T3.8 | Summary of All Adverse Events by System Organ Class and Maximum Toxicity (Maintenance + Extension Phase) | | W96, EOS |
| 3.7 | 3.9 | NA | Safety | 201585/primar<br>y_02/T3.8 | Summary of All Adverse Events Excluding<br>Study Drug Injection Site Reactions by<br>System Organ Class and Maximum<br>Toxicity (Maintenance Phase) | | HL, W48,<br>W96 |
| NA | NA | 3.4 | Safety | 201585/primar<br>y_02/T3.8 | Summary of All Adverse Events Excluding<br>Study Drug Injection Site Reactions by<br>System Organ Class and Maximum<br>Toxicity (Maintenance + Extension Phase) | | EOS |
| NA | NA | 3.5 | Long-term<br>Follow-up | 201585/primar<br>y_02/T3.8 | Summary of All Adverse Events by System Organ Class and Maximum Toxicity (Longterm Follow-up Phase) | | EOS |
| 3.8 | 3.10 | NA | Safety | 201585/primar | Summary of All On-treatment Adverse | | W48, W96 |

| Safety 1 | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | y_02/T3.11 | Events by System Organ Class and Maximum Toxicity (Maintenance Phase) | | |
| 3.9 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.13 | Summary of All Adverse Events by System<br>Organ Class and Maximum Toxicity (Oral<br>Lead-in Period during the Maintenance<br>Phase) | Remove the footnote. Display both arms. | W48 |
| 3.10 | 3.11 | NA | Safety | 201585/primar<br>y_02/T3.14 | Summary of Common Adverse Events (>=5%) by Overall Frequency (Maintenance Phase) | | W48, W96 |
| 3.11 | 3.12 | NA | Safety | 201585/primar<br>y_02/T3.15 | Summary of Common Grade 2-5 Adverse<br>Events (>=1%) by Overall Frequency<br>(Maintenance Phase) | | W48, W96 |
| 3.12 | 3.13 | NA | Safety | 201585/primar<br>y_02/T3.16 | Summary of All Drug-related Adverse<br>Events by System Organ Class<br>(Maintenance Phase) | | W48, W96 |
| 3.13 | 3.14 | NA | Safety | 201585/primar<br>y_02/T3.17 | Summary of All Drug-related Adverse<br>Events by System Organ Class and<br>Maximum Toxicity (Maintenance Phase) | | HL, W48,<br>W96 |
| NA | 3.15 | 3.6 | Safety | 201585/primar<br>y_02/T3.17 | Summary of All Drug-related Adverse<br>Events by System Organ Class and<br>Maximum Toxicity (Maintenance +<br>Extension Phase) | | W96, EOS |
| 3.14 | 3.16 | NA | Safety | 201585/primar<br>y_02/T3.101 | Summary of All Drug-related Adverse<br>Events Excluding Study Drug Injection Site<br>Reactions by System Organ Class and<br>Maximum Toxicity (Maintenance Phase) | | HL, W48,<br>W96 |
| NA | NA | 3.7 | Safety | 201585/primar | Summary of All Drug-related Adverse | | EOS |

| Safety 1 | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | y_02/T3.101 | Events Excluding Study Drug Injection Site<br>Reactions by System Organ Class and<br>Maximum Toxicity (Maintenance +<br>Extension Phase) | | |
| 3.15 | 3.17 | NA | Safety | 201585/primar<br>y_02/T3.20 | Summary of All Drug-Related Grade 2-5<br>Adverse Events by Overall Frequency<br>(Maintenance Phase) | | W48, W96 |
| Serious | and Othe | r Signific | ant Adverse E | vents | | | |
| 3.16 | 3.18 | NA | Safety | 201585/primar<br>y_02/T3.21 | Summary of Serious Adverse Events by<br>System Organ Class (Maintenance Phase) | | HL, W48,<br>W96 |
| NA | 3.19 | 3.8 | Safety | 201585/primar<br>y_02/T3.21 | Summary of Serious Adverse Events by<br>System Organ Class (Maintenance +<br>Extension Phase) | | W96, EOS |
| 3.17 | 3.20 | 3.9 | Long-term<br>Follow-up | 201585/primar<br>y_02/T3.24 | Summary of Serious Adverse Events by<br>System Organ Class (Long-term Follow-up<br>Phase) | | W48, W96,<br>EOS |
| 3.18 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.25 | Summary of Serious Adverse Events by<br>System Organ Class (Oral Lead-in Period<br>during the Maintenance Phase) | Display both arms. | W48 |
| 3.19 | 3.21 | NA | Safety | 201585/primar<br>y_02/T3.26 | Summary of Drug-related Serious Adverse<br>Events by System Organ Class<br>(Maintenance Phase) | | W48, W96 |
| NA | 3.22 | 3.10 | Safety | 201585/primar<br>y_02/T3.26 | Summary of Drug-related Serious Adverse<br>Events by System Organ Class<br>(Maintenance + Extension Phase) | | W96, EOS |
| 3.20 | 3.23 | NA | Safety | 201585/primar<br>y_02/T3.29 | Summary of Non-Fatal Serious Adverse<br>Events by Overall Frequency (Maintenance | | W48, W96 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | | Phase) | | |
| 3.21 | 3.24 | NA | Safety | 201585/primar<br>y_02/T3.30 | Summary of Drug-related Non-Fatal<br>Serious Adverse Events by Overall<br>Frequency (Maintenance Phase) | | W48, W96 |
| 3.22 | 3.25 | NA | Safety | 201585/primar<br>y_02/T3.31 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class (Maintenance Phase) | | HL, W48,<br>W96 |
| NA | 3.26 | 3.11 | Safety | 201585/primar<br>y_02/T3.31 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class (Maintenance + Extension Phase) | | W96, EOS |
| 3.23 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.34 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class (Oral Lead-in Period during the Maintenance Phase) | Remove the footnote. Display both arms. | W48 |
| 3.24 | 3.27 | NA | Safety | 201585/primar<br>y_02/T3.35 | Summary of Common (>=5%) Non-Serious<br>Adverse Events (Maintenance Phase) | | W48, W96 |
| 3.25 | 3.28 | NA | Safety | 201585/primar<br>y_02/T3.36 | Summary of Subjects and Number of<br>Occurrences of Common (>=5%) Non-<br>Serious Adverse Events by System Organ<br>Class (Maintenance Phase) | | W48, W96 |
| 3.26 | 3.29 | NA | Safety | 201585/primar<br>y_02/T3.37 | Summary of Subjects and Number of occurrences of SAEs, Fatal SAEs, and Drug-related SAEs (Maintenance Phase) | | W48, W96 |
| 3.27 | 3.30 | NA | Safety | 201585/primar | Summary of Cumulative Adverse Events | Note that this table only display AEs | W48, W96 |

| Safety 1 | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | y_02/T3.38 | by Visit (Maintenance Phase) | occurring >=5% subjects during Maintenance Phase. | |
| Study D | rug Inject | ion Site R | Reaction Adve | rse Events (displ | ay for both arms) | | |
| 3.28 | 3.31 | NA | Safety | 201585/primar<br>y_02/T3.40 | Summary of Study Drug Injection Site<br>Reaction Adverse Events (Event-level<br>Summary) - Maintenance Phase | | HL, W48,<br>W96 |
| NA | 3.32 | 3.12 | Safety | 201585/primar<br>y_02/T3.40 | Summary of Study Drug Injection Site<br>Reaction Adverse Events (Event-level<br>Summary) - Maintenance + Extension<br>Phase | | W96, EOS |
| 3.29 | 3.33 | NA | Safety | 201585/primar<br>y_02/T3.43 | Summary of Subject-level Characteristics of Study Drug Injection Site Reaction Adverse Events – Overall and Common (Maintenance Phase) | | W48, W96 |
| NA | 3.34 | 3.13 | Safety | 201585/primar<br>y_02/T3.43 | Summary of Subject-level Characteristics of Study Drug Injection Site Reaction Adverse Events – Overall and Common (Maintenance + Extension Phase) | | W96, EOS |
| 3.30 | 3.35 | NA | Safety | 201585/primar<br>y_02/T3.46 | Summary of Study Drug Injection Site<br>Reaction Adverse Events by Visit and<br>Maximum Severity – Overall and Common<br>(Maintenance Phase) | Change the second footnote to 'Note:<br>Common ISR includes pain,<br>induration, nodules and any other<br>ISR with >=5% subjects in either<br>treatment arm.' Footnote may be<br>adjusted for clarifications. | W48, W96 |
| 3.31 | 3.36 | NA | Safety | 201585/primar<br>y_02/T3.47 | Summary of Drug-related Study Drug<br>Injection Site Reaction Adverse Events<br>(Event-level Summary) - CAB | | W48, W96 |

| Safety 1 | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | | (Maintenance Phase) | | |
| 3.32 | 3.37 | NA | Safety | 201585/primar<br>y_02/T3.48 | Summary of Drug-related Subject-level<br>Characteristics of Study Drug Injection Site<br>Reaction Adverse Events (Maintenance<br>Phase) - Overall and Common (CAB) | | W48, W96 |
| 3.33 | 3.38 | NA | Safety | 201585/primar<br>y_02/T3.49 | Summary of Overall and Common Drug-<br>related Study Drug Injection Site Reaction<br>Adverse Events by Visit and Maximum<br>Severity (Maintenance Phase) - CAB | Footnote may be adjusted for clarifications. | W48, W96 |
| 3.34 | 3.39 | NA | Safety | 201585/primar<br>y_02/T3.50 | Summary of Maximum Drug-related Study<br>Drug Injection Site Reaction Adverse Event<br>Grade by Needle Length (Maintenance<br>Phase) – Common (CAB) | Update the needle length in column header to be "<=1.5 inches', '>1.5 to <2 inches' and '>=2 inches' respectively. Change the first footnote to 'Note: Common ISR includes pain, induration, nodules and any other ISR with >=5% subjects in either treatment arm.'. Remove the second footnote. | W48, W96 |
| 3.35 | 3.40 | NA | Safety | 201585/primar<br>y_02/T3.51 | Summary of Drug-related Study Drug<br>Injection Site Reaction Adverse Events<br>(Event-level Summary) - RPV<br>(Maintenance Phase) | | W48, W96 |
| 3.36 | 3.41 | NA | Safety | 201585/primar<br>y_02/T3.52 | Summary of Drug-related Subject-level<br>Characteristics of Study Drug Injection Site<br>Reaction Adverse Events (Maintenance<br>Phase) - Overall and Common (RPV) | | W48, W96 |
| 3.37 | 3.42 | NA | Safety | 201585/primar<br>y_02/T3.53 | Summary of Overall and Common Drug-<br>related Study Drug Injection Site Reaction | Footnote may be adjusted for clarifications. | W48, W96 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | | Adverse Events by Visit and Maximum Severity (Maintenance Phase) - RPV | | |
| 3.38 | 3.43 | NA | Safety | 201585/primar<br>y_02/T3.54 | Summary of Maximum Drug-related Study<br>Drug Injection Site Reaction Adverse Event<br>Grade by Needle Length (Maintenance<br>Phase) – Common (RPV) | Update the needle length in column header to be "<=1.5 inches', '>1.5 to < 2 inches' and '>=2 inches' respectively. Change the first footnote to 'Note: Common ISR includes pain, induration, nodules and any other ISR with >=5% subjects in either treatment arm.'. Remove the second footnote. | W48, W96 |
| Laborat | ory: Chem | nistry and | Hematology | | | | |
| 3.39 | 3.44 | 3.14 | Safety | 201585/primar<br>y_02/T3.55 | Summary of Chemistry Changes from<br>Baseline by Visit (Maintenance + Extension<br>Phase) | Present GFR, lipids and glucose in both conventional and standard units. Change 'Post Baseline' to 'Postbaseline' in the footnote. | W48, W96,<br>EOS |
| 3.40 | 3.45 | 3.15 | Safety | 201585/primar<br>y_02/T3.59 | Summary of Chemistry Values by Visit (Maintenance + Extension Phase) | Present GFR, lipids and glucose in both conventional and standard units. Change 'Post Baseline' to 'Postbaseline' in the footnote. | W48, W96,<br>EOS |
| 3.41 | 3.46 | 3.16 | Safety | 201585/primar<br>y_02/T3.60 | Summary of Hematology Changes from Baseline by Visit (Maintenance + Extension Phase) | Change 'Post Baseline' to 'Post-baseline' in the footnote. | W48, W96,<br>EOS |
| 3.42 | 3.47 | 3.17 | Safety | 201585/primar<br>y_02/T3.59 | Summary of Hematology Values by Visit (Maintenance + Extension Phase) | Remove the first footnote. Change 'Post Baseline' to 'Post-baseline' in the footnote. | W48, W96,<br>EOS |
| 3.43 | 3.48 | NA | Safety | 201585/primar | Summary of Maximum Post-Baseline | Add "Emergent is relative to last | W48, W96 |

| Safety 1 | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | y_02/T3.61 | Emergent Chemistry Toxicities (Maintenance Phase) | toxicity up to and including baseline." to the end of the second footnote. | |
| NA | 3.49 | 3.18 | Safety | 201585/primar<br>y_02/T3.61 | Summary of Maximum Post-Baseline<br>Emergent Chemistry Toxicities<br>(Maintenance + Extension Phase) | Adjust the footnote similar to above. | W96, EOS |
| 3.44 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.64 | Summary of Maximum Post-Baseline<br>Emergent Chemistry Toxicities - Oral Lead-<br>in Period during the Maintenance Phase | Display both arms. Adjust the footnote similarly to above. | W48 |
| 3.45 | 3.50 | NA | Safety | 201585/primar<br>y_02/T3.65 | Summary of Maximum Post-Baseline<br>Emergent Hematology Toxicities<br>(Maintenance Phase) | Adjust the footnote similarly to above. | W48, W96 |
| NA | 3.51 | 3.19 | Safety | 201585/primar<br>y_02/T3.65 | Summary of Maximum Post-Baseline<br>Emergent Hematology Toxicities<br>(Maintenance + Extension Phase) | Adjust the footnote similarly to above. | W96, EOS |
| 3.46 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.68 | Summary of Maximum Post-Baseline<br>Emergent Hematology Toxicities - Oral<br>Lead-in Period during the Maintenance<br>Phase | Display both arms. Adjust the footnote similarly to above. | W48 |
| NA | 3.114 | NA | Safety | Shell SAF_T2 | Summary of Expected and Missed Visits (Maintenance Phase) - Hematology and Chemistry | | W96 |
| Laborat | ory: Urina | lysis | | | | | |
| 3.47 | 3.52 | 3.20 | Safety | 201585/primar<br>y_02/T3.69 | Summary of Urinalysis Dipstick Results by Visit (Maintenance Phase) | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96 |
| 3.48 | 3.53 | 3.21 | Safety | 201585/primar<br>y_02/T3.70 | Summary of Urine Concentrations<br>Changes from Baseline by Visit<br>(Maintenance Phase) | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.49 | 3.54 | NA | Safety | 201585/primar<br>y_02/T3.71 | Summary of Changes in Proteinuria Baseline Laboratory Result to Maximum Post-Baseline Laboratory Result (Maintenance Phase) | Change 'Post Baseline' to 'Post-<br>Baseline' in the footnote. | W48, W96 |
| Laborat | ory: Lipid | | | | | | |
| 3.50 | 3.55 | NA | Safety | 201585/primar<br>y_02/T3.72 | Summary of Changes in Baseline NCEP<br>Fasting Lipid Category to Maximum Post-<br>Baseline Category – Triglycerides<br>(Maintenance Phase) | For WK96, update the title to be " Category (Triglycerides, Lipids LOCF) – Maintenance Phase". | W48, W96 |
| 3.51 | 3.56 | NA | Safety | 201585/primar<br>y_02/T3.73 | Summary of Changes in Baseline NCEP<br>Fasting Lipid Category to Maximum Post-<br>Baseline Category – Total Cholesterol<br>(Maintenance Phase) | For WK96, update the title to be " Category (Total Cholesterol, Lipids LOCF) – Maintenance Phase". | W48, W96 |
| 3.52 | 3.57 | NA | Safety | 201585/primar<br>y_02/T3.74 | Summary of Changes in Baseline NCEP<br>Fasting Lipid Category to Minimum Post-<br>Baseline Category – HDL Cholesterol<br>(Maintenance Phase) | For WK96, update the title to be " Category (HDL Cholesterol, Lipids LOCF) – Maintenance Phase". | W48, W96 |
| 3.53 | 3.58 | NA | Safety | 201585/primar<br>y_02/T3.75 | Summary of Changes in Baseline NCEP<br>Fasting Lipid Category to Maximum Post-<br>Baseline Category – LDL Cholesterol<br>(Maintenance Phase) | For WK96, update the title to be "<br>Category (LDL Cholesterol, Lipids<br>LOCF) – Maintenance Phase". | W48, W96 |
| 3.54 | 3.59 | NA | Safety | 201585/primar<br>y_02/T3.58 | Summary of Fasting Lipids Percentage<br>Changes from Baseline by Visit<br>(Maintenance Phase) - Lipids LOCF | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96 |
| 3.55 | 3.60 | NA | Safety | 201585/primar<br>y_02/T3.76 | Summary of Fasting TC/HDL ratio<br>Changes from Baseline (Maintenance<br>Phase) – Lipids LOCF | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Laborat | ory: Hepa | tobiliary ( | Liver) | | | | |
| 3.56 | 3.61 | NA | Safety | 201585/primar<br>y_02/T3.80 | Summary of Liver Monitoring/Stopping<br>Event Reporting (Maintenance Phase) | For WK96: Remove "Monitoring/" from the title, remove liver monitoring related text, footnote and section in the table. | W48, W96 |
| 3.57 | 3.62 | NA | Safety | 201585/primar<br>y_02/T3.81 | Summary of Subjects Meeting Hepatobiliary Abnormality Criteria (Maintenance Phase) | | W48, W96 |
| NA | 3.63 | 3.22 | Safety | 201585/primar<br>y_02/T3.81 | Summary of Subjects Meeting<br>Hepatobiliary Abnormality Criteria<br>(Maintenance +Extension Phase) | | W96, EOS |
| 3.58 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.84 | Summary of Subjects Meeting Hepatobiliary Abnormality Criteria – Oral Lead-in Period during the Maintenance Phase | Display both arms. | W48 |
| ECG | | | | | | | |
| 3.59 | 3.64 | 3.23 | Safety | 201585/primar<br>y_02/T3.85 | Summary of ECG Findings (Maintenance Phase) | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96 |
| 3.60 | 3.65 | 3.24 | Safety | 201585/primar<br>y_02/T3.88 | Summary of Change from Baseline in ECG values by Visit (Maintenance Phase) | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96 |
| 3.61 | 3.66 | 3.25 | Safety | 201585/primar<br>y_02/T3.91 | Summary of QTc Values by Category (Maintenance Phase) | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96 |
| 3.62 | 3.67 | 3.26 | Safety | 201585/primar<br>y_02/T3.94 | Summary of Change from Baseline QTc<br>Values by Category (Maintenance Phase) | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96 |
| Vital Sig | ns and e | C-SSRS | | | | | |
| 3.63 | 3.68 | NA | Safety | 201585/primar | Summary of Change from Baseline in Vital | Change 'Post Baseline' to 'Post- | W48, W96 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | y_02/T3.97 | Signs by Visit (Maintenance Phase) | Baseline' in the footnote. | |
| 3.64 | 3.69 | NA | Safety | SAFE_T1 | Summary of BMI Shift from Baseline by Visit (Maintenance Phase) | For WK96: Add "Sex and" before "Visit" in the title. | W48, W96 |
| NA | 3.70 | NA | Safety | 207966/primar<br>y_02/T3.64 | Summary of BMI Shift from Baseline by Strata and Visit (Maintenance Phase) | Display by strata instead of sex (i.e. prior exposure to CAB + RPV: All, 0, 1-24, >24 weeks) and visit, add a footnote for strata. | W96 |
| NA | 3.71 | NA | Safety | 207966/primar<br>y_02/T3.63 | Summary of Change from Baseline in<br>Weight and BMI by Strata and Visit<br>(Maintenance Phase) | Display by strata (i.e. prior exposure to CAB + RPV: All, 0, 1-24, >24 weeks) and parameter, add a footnote for strata. | W96 |
| 3.65 | 3.72 | NA | Safety | 201585/primar<br>y_02/T3.99 | Summary of Subjects with eC-SSRS<br>Suicidal Ideation or Behaviour<br>(Maintenance Phase) | Change 'post baseline' to 'post-<br>baseline' in the row header. | W48, W96 |
| Adverse | Event of | Special In | nterest (AESI) | | | | |
| 3.66 | 3.73 | NA | Safety | 201585/primar<br>y_02/T3.100 | Summary of Depression, Anxiety and Suicidal Ideation/Behaviour Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and Prior History of Depression, Anxiety and Suicidal Ideation at Screening (Maintenance Phase) | For WK96, follow display 207966/primary_13/T3.98. | W48, W96 |
| NA | 3.74 | 3.27 | Safety | 207966/primar<br>y_13/T3.98 | Summary of Depression, Anxiety and Suicidal Ideation/Behaviour Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and Prior History of Depression, Anxiety and Suicidal Ideation at Screening (Maintenance + Extension | | W96, EOS |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | | Phase) | | |
| 3.67-<br>3.83 | 3.75-<br>3.91 | NA | Safety | 209522/iss_01/<br>T3.38-3.49,<br>T3.51-3.55 | Summary of XXX Adverse Events of<br>Special Interest by System Organ Class<br>and Preferred Term (Number of Subjects<br>and Occurrence) – Maintenance Phase | Only display data from this study, no need for showing study number. For 'XXX', refer to Table 4. | W48, W96 |
| NA | 3.92-<br>3.108 | 3.28-<br>3.44 | Safety | 207966/primar<br>y_02T3.67-<br>3.83 | Summary of XXX Adverse Events of<br>Special Interest by System Organ Class<br>and Preferred Term (Number of Subjects<br>and Occurrence) – Maintenance +<br>Extension Phase | | W96, EOS |
| 3.84 | 3.109 | NA | Safety | 209522/iss_01/<br>T3.62 | Summary of Characteristics of Common<br>Adverse Events of Special Interest –<br>Maintenance Phase | Only display data from this study, no need for showing study number. Present by individual common AESI. For WK96, add a footnote, "Note: Percentages are based on the Number of subjects with Event. For Event Characteristics, Outcome and Action Taken sections, a subject can be counted in more than one category." | W48, W96 |
| NA | 3.110 | 3.45 | Safety | 207966/primar<br>y_02/T3.84 | Summary of Characteristics of Common<br>Adverse Events of Special Interest –<br>Maintenance + Extension Phase | For WK96, add a similar footnote to Table 3.109. | W96, EOS |
| NA | 3.111 | 3.46 | Safety | 207966/regqry<br>_2019_01/T3.2<br>07 | Summary of Syncope and Presyncope<br>Adverse Events - Maintenance + Extension<br>Phase | Replace row label "Syncope or Presyncope" with "Number of Subjects with Syncope or Presyncope". | W96, EOS |
| NA | 3.112 | 3.47 | Safety | 207966/regqry | Summary of Syncope and Presyncope | Row labels and footnotes may be | W96, EOS |

| Safety 7 | Safety Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | _2019_01/T3.2<br>08 | Adverse Events and Injection Visits -<br>Maintenance + Extension Phase | adjusted as appropriate. | |
| COVID- | 19 Advers | e Event | | | | | |
| NA | 3.113 | 3.48 | Safety | 207966/primar<br>y_02/T3.6 | Summary of COVID-19 Adverse Events by<br>System Organ Class and Maximum<br>Toxicity (Maintenance + Extension Phase) | | W96, EOS |
| NA | 3.115 | 3.49 | Safety | Shell SAF_T3 | Summary of COVID-19 Assessments (Maintenance + Extension Phase) | | W96, EOS |

# 15.15.5.5. Safety Figures

**Note:** Unless otherwise specified, display both arms.

| Safety I | Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.1 | 3.1 | NA | Safety | 201585/primar<br>y_02/F3.1 | Plot of Common Adverse Events and Relative Risk - Q8W vs. Q4W (Maintenance Phase) – Excluding Study Drug ISRs | Remove the second footnote. | HL, W48, W96 |
| NA | NA | 3.1 | Safety | 207966/primar<br>y_02/F3.1 | Plot of Common Adverse Events and Relative Risk - Q8W vs. Q4W (Maintenance + Extension Phase) - Excluding Study Drug ISRs | | EOS |
| 3.2 | 3.2 NA Safety 201585/prima y_02/F3.1 | | 201585/primar<br>y_02/F3.1 | Plot of Common Study Drug Injection Site Reaction<br>Adverse Events and Relative Risk - Q8W vs. Q4W<br>(Maintenance Phase) | Remove the second footnote. | HL, W48, W96 | |
| NA | NA | 3.2 | Safety | 207966/primar<br>y_02/F3.2 | Plot of Common Study Drug Injection Site Reaction<br>Adverse Events and Relative Risk - Q8W vs. Q4W<br>(Maintenance +Extension Phase) | | EOS |
| 3.3 | 3.3 | NA | Safety | 201585/primar<br>y_02/F3.5 | Plot of Onset, Duration, and Severity of Overall and Common Study Drug Injection Site Reaction AEs by Maximum Grade — CAB and/or RPV (Maintenance Phase) | | W48, W96 |
| 3.4 | 3.4 | NA | Safety | 201585/primar<br>y_02/F3.6 | Plot of Onset, Duration, and Severity of Overall and Common Drug-related Study Drug Injection Site Reaction AEs by Maximum Grade — CAB (Maintenance Phase) | | W48, W96 |
| 3.5 | 3.5 | NA | Safety | 201585/primar<br>y_02/F3.7 | Plot of Onset, Duration, and Severity of Overall and Common Drug-related Study Drug Injection Site Reaction AEs by Maximum Grade — RPV (Maintenance Phase) | | W48, W96 |
| 3.6 | 3.6 | NA | Safety | 201585/primar | Plot of Incidence of Maintenance Phase Study | Footnote may be adjusted for | W48, W96 |

| Safety I | Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | y_02/F3.8 | Drug Injection Site Reaction Adverse Events by Visit (Overall and Common) – CAB and/or RPV | clarifications. | |
| NA | NA | 3.3 | Safety | 207966/primar<br>y_02/F3.6 | Plot of Incidence of Maintenance and Extension<br>Phase Study Drug Injection Site Reaction Adverse<br>Events by Visit (Overall and Common) – CAB<br>and/or RPV | | EOS |
| 3.7 | 3.7 | NA | Safety | 201585/primar<br>y_02/F3.9 | Plot of Incidence of Maintenance Phase Drug-<br>Related Study Drug Injection Site Reaction<br>Adverse Events by Visit (Overall and Common) –<br>CAB | Footnote may be adjusted for clarifications. | W48, W96 |
| NA | NA | 3.4 | Safety | 207966/primar<br>y_02/F3.7 | Plot of Incidence of Maintenance and Extension<br>Phase Drug-Related Study Drug Injection Site<br>Reaction Adverse Events by Visit (Overall and<br>Common) – CAB | | EOS |
| 3.8 | 3.8 | NA | Safety | 201585/primar<br>y_02/F3.10 | Plot of Incidence of Maintenance Phase Drug-<br>Related Study Drug Injection Site Reaction<br>Adverse Events by Visit (Overall and Common) –<br>RPV | Footnote may be adjusted for clarifications. | W48, W96 |
| NA | NA | 3.5 | Safety | 207966/primar<br>y_02/F3.8 | Plot of Incidence of Maintenance and Extension<br>Phase Drug-Related Study Drug Injection Site<br>Reaction Adverse Events by Visit (Overall and<br>Common) – RPV | | EOS |
| 3.9 | 3.9 | NA | Safety | 201585/primar<br>y_02/F3.11 | Plot of Incidence of Grade 3-5 Maintenance Phase<br>Study Drug Injection Site Reaction Adverse Events<br>by Visit (Overall and Common) - CAB and/or RPV | Footnote may be adjusted for clarifications. | W48, W96 |
| 3.10 | 3.10 | NA | Safety | 201585/primar<br>y_02/F3.12 | Plot of Incidence of Grade 3-5 Maintenance Phase<br>Drug-related Study Drug Injection Site Reaction | Footnote may be adjusted for clarifications. | W48, W96 |

| Safety I | Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | | Adverse Events by Visit (Overall and Common) - CAB | | |
| 3.11 | 3.11 | NA | Safety | 201585/primar<br>y_02/F3.13 | Plot of Incidence of Grade 3-5 Maintenance Phase<br>Drug-related Study Drug Injection Site Reaction<br>Adverse Events by Visit (Overall and Common) -<br>RPV | Footnote may be adjusted for clarifications. | W48, W96 |
| 3.12 | 3.12 | NA | Safety | 201585/primar<br>y_02/F3.2 | Scatter Plot of Maximum vs. Baseline for ALT (Maintenance Phase) | Display at log10 scale. | HL, W48, W96 |
| NA | 3.13 | 3.6 | Safety | 207966/primar<br>y_02/F3.12 | Scatter Plot of Maximum vs. Baseline for ALT (Maintenance + Extension Phase) | | W96, EOS |
| 3.13 | 3.14 | NA | Safety | 201585/primar<br>y_02/F3.3 | Scatter Plot of Maximum Total Bilirubin vs.<br>Maximum ALT (Maintenance Phase) | | HL, W48, W96 |
| NA | 3.15 | 3.7 | Safety | 207966/primar<br>y_02/F3.13 | Scatter Plot of Maximum Total Bilirubin vs. Maximum ALT (Maintenance + Extension Phase) | | W96, EOS |
| 3.14 | 3.16 | NA | Safety | 201585/primar<br>y_02/F3.4 | Matrix Plot of Maximum Liver Chemistries during the Maintenance Phase | | HL, W48, W96 |
| NA | 3.17 | 3.8 | Safety | 207966/primar<br>y_02/F3.14 | Matrix Plot of Maximum Liver Chemistries during the Maintenance and Extension Phase | | W96, EOS |
| 3.15 | 3.18 | NA | Safety | 201585/primar<br>y_02/F3.14 | Bar Chart of Lipid NCEP Categories at Week 48 vs. Baseline – Triglycerides, Total Cholesterol, LDL Cholesterol | For WK96, replace 'Week 48' with 'Week 96' and add "(Lipids LOCF)" to the end of the title | W48, W96 |
| 3.16 | 3.19 | NA | Safety | 201585/primar<br>y_02/F3.15 | Bar Chart of Lipid NCEP Categories at Week 48 vs. Baseline - HDL Cholesterol | For WK96, replace 'Week 48' with 'Week 96' and add "(Lipids LOCF)" to the end of the title. | W48, W96 |

| Safety I | Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.17 | 3.20 | NA | Safety | SAFE_F1 | Histogram of Timeliness of Injections (Maintenance Phase) | | W48, W96 |
| 3.18 | 3.21 | NA | Safety | 207966/primar<br>y_02/F3.18 | Plot of Incidence of Maintenance Phase Study<br>Drug Injection Site Reaction Adverse Events by<br>Strata and Visit (Overall and Common) - CAB<br>and/or RPV | | W48, W96 |
| NA | NA | 3.9 | Safety | 207966/primar<br>y_02/F3.18 | Plot of Incidence of Maintenance and Extension<br>Phase Study Drug Injection Site Reaction Adverse<br>Events by Strata and Visit (Overall and Common) -<br>CAB and/or RPV | | EOS |
| NA | 3.22 | 3.10 | Safety | 207966/regqry<br>_2019_01/F3.2<br>03 | Patient Profile for Subjects with Syncope or<br>Presyncope Adverse Events (Maintenance +<br>Extension Phase) | Footnotes may be adjusted as appropriate. | WK96, EOS |

#### 15.15.5.6. Pharmacokinetic Tables

**Note:** For WK48 deliverable, data from visits up to Week 48 are included. For WK96 deliverable, except for Table 4.8- Table 4.9, add "(Maintenance Phase)" after visit in the title. Table 4.8- Table 4.9 will only be produced if additional LTFU PK storage samples since the last analysis data cut are planned to be analysed.

| Pharma | cokinetic | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.1 | 4.1 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.1 | Summary of Plasma CAB PK Concentration (ug/mL) -Time Data by Treatment and Visit – Including Log-transformed Statistics | Remove the first footnote. | W48, W96 |
| 4.2 | 4.2 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.2 | Summary of Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit – Including Log-<br>transformed Statistics | Remove the first footnote. | W48, W96 |
| 4.3 | 4.3 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.3 | Summary of Evaluable Plasma CAB PK<br>Concentration (ug/mL) -Time Data by Treatment<br>and Visit – Including Log-transformed Statistics | Remove the first footnote. | W48, W96 |
| 4.4 | 4.4 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.4 | Summary of Evaluable Plasma RPV PK<br>Concentration (ng/mL) -Time Data by Treatment<br>and Visit – Including Log-transformed Statistics | Remove the first footnote. | W48, W96 |
| 4.5 | 4.5 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.3 | Summary of Evaluable Plasma CAB PK Concentration (ug/mL) -Time Data by Strata and Treatment and Visit – Including Log-transformed Statistics | Display by rederived randomization strata and add footnote for strata. | W48, W96 |
| 4.6 | 4.6 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.4 | Summary of Evaluable Plasma RPV PK Concentration (ng/mL) -Time Data by Strata and Treatment and Visit – Including Log-transformed Statistics | Display by rederived randomization strata and add footnote for strata. | W48, W96 |

| Pharma | cokinetic | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.7 | NA | NA | Pharmacokinetic | 201585/primary_<br>02/T4.6 | Summary of Results of Steady State Assessment by Strata for Q8W Arm- Evaluable Concentration | Display by rederived randomization strata and add footnote for strata. For Q8W arm only. | W48 |
| NA | 4.7 | NA | Pharmacokinetic | Shell PK_T1 | Summary of Expected and Missed Visits by Strata and Treatment (Maintenance Phase) – Plasma CAB PK Concentration | | W96 |
| NA | 4.8 | NA | Pharmacokinetic | Shell PK_T1 | Summary of Expected and Missed Visits by Strata and Treatment (Maintenance Phase) – Plasma RPV PK Concentration | | W96 |
| NA | 4.9 | 4.1 | Long-term<br>Follow-up | 207966/primary_<br>02/T4.1 | Summary of Plasma CAB PK Concentration (ug/mL) -Time Data by Treatment and Visit (Long-term Follow-up Phase) - Including Log-transformed Statistics | Remove the column 'Pl.<br>Time' and the second<br>footnote. Produce only if<br>we have additional LTFU<br>storage samples planned<br>to be analysed since last<br>analysis data cut. | W96, EOS |
| NA | 4.10 | 4.2 | Long-term<br>Follow-up | 207966/primary_<br>02/T4.2 | Summary of Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit (Long-term Follow-up Phase) - Including Log-transformed Statistics | Remove the column 'Pl.<br>Time' and the second<br>footnote. Produce only if<br>we have additional LTFU<br>samples planned to be<br>analysed since last<br>analysis data cut. | W96, EOS |

### 15.15.5.7. Pharmacokinetic Figures

**Note:** Unless otherwise specified, display both arms. For WK96 deliverable, add "- Maintenance Phase" to the end of the title except for Figure 4.17; display Week 96 visit next to Week 48 visit in the mean and median summary figures and add a footnote as appropriate.

| Pharma | cokinetic | Figures | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.1 | 4.1 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.1 | Individual Plasma CAB Concentration-<br>Time Plots (Linear and Semi-Log) | Also include prior exposure to CAB+RPV (e.g. 0, 1-24, >24 weeks) for each subject. | W48, W96 |
| 4.2 | 4.2 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.2 | Individual Plasma RPV Concentration-<br>Time Plots (Linear and Semi-Log) | Also include prior exposure to CAB+RPV (e.g. 0, 1-24, >24 weeks) for each subject. | W48, W96 |
| 4.3 | 4.3 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.3 | Mean (SD) Plasma CAB Concentration-<br>Time Plots (Linear and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.4 | 4.4 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.5 | Mean (SD) Plasma RPV Concentration-<br>Time Plots (Linear and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.5 | 4.5 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.7 | Mean (SD) Evaluable Plasma CAB<br>Concentration-Time Plots (Linear and<br>Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.6 | 4.6 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.9 | Mean (SD) Evaluable Plasma RPV<br>Concentration-Time Plots (Linear and<br>Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.7 | 4.7 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.7 | Mean (SD) Evaluable Plasma CAB<br>Concentration-Time Plots by Strata<br>(Linear and Semi-Log) | Display by rederived randomization strata and add footnote for strata. For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.8 | 4.8 | NA | Pharmacokinetic | 201585/primary_02/ | Mean (SD) Evaluable Plasma RPV | Display by rederived | W48, W96 |

| Pharma | cokinetic | Figures | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| | | | | F4.9 | Concentration-Time Plots by Strata (Linear and Semi-Log) | randomization strata and add footnote for strata. For WK48, data from visits up to Week 48 are included. | |
| 4.9 | 4.9 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.4 | Median (5th and 95th Percentile) Plasma<br>CAB Concentration-Time Plots (Linear<br>and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.10 | 4.10 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.6 | Median (5th and 95th Percentile) Plasma<br>RPV Concentration-Time Plots (Linear<br>and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.11 | 4.11 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.8 | Median (5th and 95th Percentile) Evaluable Plasma CAB Concentration- Time Plots (Linear and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.12 | 4.12 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.10 | Median (5th and 95th Percentile) Evaluable Plasma RPV Concentration- Time Plots (Linear and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.13 | 4.13 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.8 | Median (5th and 95th Percentile) Evaluable Plasma CAB Concentration- Time Plots by Strata (Linear and Semi- Log) | Display by rederived randomization strata and add footnote for strata. For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.14 | 4.14 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.10 | Median (5th and 95th Percentile) Evaluable Plasma RPV Concentration- Time Plots by Strata (Linear and Semi- Log) | Display by rederived randomization strata and add footnote for strata. For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.15 | 4.17 | 4.1 | Long-term | 207966/primary_02/ | Plasma PK Concentration-Time since | For W96 and EOS: Plot by | W48, W96, |

| Pharma | cokinetic | Figures | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| | | | Follow-up | F4.15 | Last Injection Plots by Strata | treatment instead of by strata and change "Strata" to be "Treatment" in the title; Colorcode different strata of prior exposure; exclude RPV concentrations on/after the start of LTFU oral RPV and add footnote for this exclusion; will only be produced if additional LTFU PK storage samples since the last analysis data cut are planned to be analysed. | EOS |
| 4.16 | 4.15 | NA | Pharmacokinetic | 207966/primary_06/<br>F4.16 | Median Evaluable Plasma CAB Trough PK Concentration (ug/mL) - Time Plots by Treatment and Strata (Linear and Semi-Log) | | W48, W96 |
| 4.17 | 4.16 | NA | Pharmacokinetic | 207966/primary_06/<br>F4.17 | Median Evaluable Plasma RPV Trough PK Concentration (ng/mL) - Time Plots by Treatment and Strata (Linear and Semi-Log) | | W48, W96 |

## 15.15.5.8. Pharmacokinetic / Pharmacodynamic Tables

**Note:** Unless otherwise specified, display by treatment arm.

| Pharma | cokinetic | : / Pharma | acodynamic Tables | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| PK / PD | Efficacy | | | | | | |
| 5.1 | NA | NA | Pharmacokinetic | 201584/primary_0<br>1/T5.1 | Univariable Logistic Regression Analysis of Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 by Trough PK Concentration and Subgroup for Subjects without Prior Exposure to CAB + RPV | | W48 |
| 5.2 | NA | NA | Pharmacokinetic | 201584/primary_0<br>1/T5.2 | Multivariable Logistic Regression Analysis of Predictors of Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 for Subjects without Prior Exposure to CAB + RPV | | W48 |
| 5.3 | NA | NA | Pharmacokinetic | 201584/primary_0<br>1/T5.5 | Summary of Week 8 Trough CAB PK concentration by Snapshot 'HIV-1 RNA ≥50 c/mL' (Yes vs. No) at Week 48 for Subjects without Prior Exposure to CAB + RPV – Including Log-transformed Statistics | | W48 |
| 5.4 | NA | NA | Pharmacokinetic | 201584/primary_0<br>1/T5.6 | Summary of Week 8 Trough RPV PK concentration by Snapshot 'HIV-1 RNA ≥50 c/mL' (Yes vs. No) at Week 48 for Subjects without Prior Exposure to CAB + RPV – Including Log-transformed Statistics | | W48 |

## 15.15.5.9. Pharmacokinetic / Pharmacodynamic Figures

| Pharma | Pharmacokinetic / Pharmacodynamic Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| PK / PD | Efficacy / | Analyses | | | | | |
| 5.1 | NA | NA | Pharmacokinetic | 201585/primary_<br>02/F5.3 | Scatter Plot of Week 8 Trough CAB PK Concentration by Snapshot 'HIV-1 RNA ≥50 c/mL' (Yes vs. No) at Week 48 for Subjects without Prior Exposure to CAB + RPV | | W48 |
| 5.2 | NA | NA | Pharmacokinetic | 201585/primary_<br>02/F5.4 | Scatter Plot of Week 8 Trough RPV PK Concentration by Snapshot 'HIV-1 RNA ≥50 c/mL' (Yes vs. No) at Week 48 for Subjects without Prior Exposure to CAB + RPV | | W48 |
| 5.3 | 5.1 | NA | Pharmacokinetic | 207966/internal_<br>01/F5.1 | Individual CAB Trough Concentration-time Profiles for Subjects with Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 and Median, 5th & 95th Percentile of CAB Conc-Time Profiles for Other Subjects (Semi-Log) | For WK96, replace 'Week 48' with 'Week 96' and add "-Maintenance Phase" to the end of the title. Display by treatment arm. | W48, W96 |
| 5.4 | 5.2 | NA | Pharmacokinetic | 207966/internal_<br>01/F5.2 | Individual RPV Trough Concentration-time Profiles for Subjects with Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 and Median, 5th & 95th Percentile of RPV Conc-Time Profiles for Other Subjects (Semi-Log) | For WK96, replace 'Week 48' with 'Week 96' and add "-Maintenance Phase" to the end of the title. Display by treatment arm. | W48, W96 |
| 5.5 | NA | NA | Pharmacokinetic | 201585/primary_<br>02/F5.10 | Scatter Plot of Week 8 Trough Concentration of CAB and RPV in Relation to Occurrence of Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 for Subjects without Prior Exposure to CAB + RPV | | W48 |

| Pharma | cokinetic | / Pharma | codynamic Figure | S | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| PK / PD | Safety Ar | nalyses | | | | | |
| 5.6 | NA | NA | Pharmacokinetic | 201585/primary_<br>02/F5.13 | Scatter Plot of Maximum Change from Baseline in ALT versus Last Trough CAB PK Concentrations by Strata and Treatment during the Maintenance Phase | Display by strata and treatment arm. Add footnote for rederived randomization strata. | W48 |
| 5.7 | NA | NA | Pharmacokinetic | 201585/primary_<br>02/F5.14 | Scatter Plot of Maximum Change from Baseline in ALT versus Last Trough RPV PK Concentrations by Strata and Treatment during the Maintenance Phase | Display by strata and treatment arm. Add footnote for rederived randomization strata. | W48 |
| 5.8 | NA | NA | Pharmacokinetic | 201585/primary_<br>02/F5.15 | Scatter Plot of Maximum Change from Baseline in Total Bilirubin versus Last Trough CAB PK Concentrations by Strata and Treatment during the Maintenance Phase | Display by strata and treatment arm. Add footnote for rederived randomization strata. | W48 |
| 5.9 | NA | NA | Pharmacokinetic | 201585/primary_<br>02/F5.16 | Scatter Plot of Maximum Change from Baseline in Total Bilirubin versus Last Trough RPV PK Concentrations by Strata and Treatment during the Maintenance Phase | Display by strata and treatment arm. Add footnote for rederived randomization strata. | W48 |
| 5.10 | NA | NA | Pharmacokinetic | 201585/primary_<br>02/F5.17 | Box Plot of Maximum Toxicity Grades of<br>Most Frequently Reported Study Drug ISR<br>Adverse Events versus Last Trough CAB<br>PK Concentrations during the Maintenance<br>Phase by Strata and Treatment | Display by strata and treatment arm. Add footnote for rederived randomization strata. Adjust the footnotes as appropriate. | W48 |

| Pharma | Pharmacokinetic / Pharmacodynamic Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 5.11 | NA | NA | Pharmacokinetic | 201585/primary_<br>02/F5.18 | Box Plot of Maximum Toxicity Grades of<br>Most Frequently Reported Study Drug ISR<br>Adverse Events versus Last Trough RPV<br>PK Concentrations during the Maintenance<br>Phase by Strata and Treatment | Display by treatment arm. Adjust the footnotes as appropriate. | W48 |

#### 15.15.5.10. Health Outcomes Tables

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Percept | ion of Inje | ection (PI | N) | | | | |
| 6.1 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.1 | Proportion of Subjects with Each Individual Item Score in PIN by Visit –LOCF (Maintenance Phase) | Display both arms. | W48 |
| 6.2 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.2 | Summary of PIN in Domain Scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness) by Visit (Maintenance Phase) | Display both arms. | W48 |
| 6.3 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.3 | Summary and Statistical Analysis of PIN in Domain Scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness) by Visit - LOCF (Maintenance Phase) | Display both arms. Adjust the first half of the footnote to "[1] Week 24/48 was compared with the 1st visit (Week 8) based on Wilcoxon signed-rank test, respectively." | W48 |
| 6.4 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.4 | Summary of PIN Change from Week 8 in Domain Scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness) by Visit (Maintenance Phase) | Display both arms. Adjust the footnote to "Note: Actual values are shown at Week 8." | W48 |

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.5 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.5 | Summary of PIN Change from Week 8 in Domain Scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness) by Visit – LOCF (Maintenance Phase) | Display both arms. Adjust the footnote to "Note: Actual values are shown at Week 8." | W48 |
| 6.6 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.11 | Statistical Analysis of PIN Change from Week 8 in<br>Domain Scores (Bother of ISRs, Leg Movement,<br>Sleep, and Acceptance) and Individual Items<br>Scores (Anxiety before, Pain, Satisfaction, Anxiety<br>After, Willingness) by Visit – LOCF (Maintenance<br>Phase) | Adjust the column header and the footnote as appropriate. | W48 |
| Health-r | related Qu | uality of L | ife (HAT-QoL) | ) | | | |
| 6.7 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.6 | Proportion of Subjects with Each Individual<br>Questionnaire Item Score in HAT-QoL by Visit -<br>LOCF (Maintenance Phase) | | W48 |
| 6.8 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.7 | Summary of Quality of Life (HAT-QoL) Score in Life Satisfaction, HIV Medication, and Disclosure worries by Visit (Maintenance phase) | | W48 |
| 6.9 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.8 | Summary of Quality of Life (HAT-QoL) Score in Life Satisfaction, HIV Medication, and Disclosure worries by Visit - LOCF (Maintenance phase) | | W48 |
| 6.10 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.9 | Summary of Quality of Life Score (HAT-QoL)-<br>Change from Baseline in Life Satisfaction, HIV<br>Medication, and Disclosure Worries by Prior<br>Exposure to CAB+RPV (0 vs. >=1 Weeks) and<br>Visit (Maintenance Phase) | | W48 |

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.11 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.10 | Summary of Quality of Life Score (HAT-QoL)-<br>Change from Baseline in Life Satisfaction, HIV<br>Medication, and Disclosure Worries by Prior<br>Exposure to CAB+RPV (0 vs. >=1 Weeks) and<br>Visit – LOCF (Maintenance Phase) | | W48 |
| 6.12 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.11 | Statistical Analysis of Quality of Life Score (HAT-QoL)- Change from Baseline in Life Satisfaction, HIV Medication, and Disclosure Worries by Visit for Subjects without Prior Exposure to CAB+RPV – LOCF (Maintenance Phase) | Adjust the column header and the footnote as appropriate. | W48 |
| 6.13 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.11 | Statistical Analysis of Quality of Life Score (HAT-QoL)- Change from Baseline in Life Satisfaction, HIV Medication, and Disclosure Worries by Visit for Subjects with Prior Exposure to CAB+RPV – LOCF (Maintenance Phase) | Adjust the column header and the footnote as appropriate. | W48 |
| HIV Trea | atment Sa | atisfaction | n Questionnai | re Status Versior | n (HIVTSQs) | | |
| 6.14 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.18 | Proportion of Subjects with HIVTSQs - Individual Item Scores by Visit - LOCF (Maintenance Phase) | | W48 |
| 6.15 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.19 | Proportion of Subjects with HIVTSQs - Individual Item Scores by Visit and Subgroup - LOCF (Maintenance Phase) | The subgroup includes: prior exposure to CAB+RPV (0, 1-24, >=24 weeks), sex at birth, age (<35, 35 - <50, >=50), race (white, non-white), Baseline CD4+ cell count (<350, 350 - <500, >=500) | W48 |

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.16 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.20 | Summary of HIVTSQs - Total Treatment<br>Satisfaction Score by Visit (Maintenance Phase) | | W48 |
| 6.17 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.21 | Summary of HIVTSQs - Total Treatment<br>Satisfaction Score by Visit – LOCF (Maintenance<br>Phase) | | W48 |
| 6.18 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.22 | Summary of HIVTSQs - Change from Baseline in Total Treatment Satisfaction Score by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit (Maintenance Phase) | | W48 |
| 6.19 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.23 | Summary of HIVTSQs - Change from Baseline in Total Treatment Satisfaction Score by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit – LOCF (Maintenance Phase) | | W48 |
| 6.20 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_03/T7.41 | Summary of HIVTSQs - Change from Baseline in Individual Item Score by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit – LOCF (Maintenance Phase) | | W48 |
| 6.21 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.24 | Statistical Analysis of HIVTSQs - Change from<br>Baseline in Total Treatment Satisfaction Score by<br>Visit for Subjects without Prior Exposure to<br>CAB+RPV - LOCF (Maintenance Phase) | Adjust column header and footnote as appropriate. | W48 |
| 6.22 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.24 | Statistical Analysis of HIVTSQs - Change from<br>Baseline in Total Treatment Satisfaction Score by<br>Visit for Subjects with Prior Exposure to<br>CAB+RPV - LOCF (Maintenance Phase) | Adjust column header and footnote as appropriate. | W48 |

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| HIV Trea | atment Sa | atisfaction | n Questionnai | re Change Version | on (HIVTSQc) | | |
| 6.23 | NA | NA | Q4W<br>ATLAS | 201584/primar<br>y_01/T6.25 | Proportion of Subjects with HIVTSQc - Individual Item Change Score at Week 48 (Maintenance Phase) for Subjects from Q4W ATLAS | | W48 |
| 6.24 | NA | NA | SOC | 201584/primar<br>y_01/T6.25 | Proportion of Subjects with HIVTSQc - Individual Item Change Score at Week 48 (Maintenance Phase) for Subjects from SOC | | W48 |
| 6.25 | NA | NA | Q4W<br>ATLAS | 201584/primar<br>y_01/T6.26 | Summary of HIVTSQc – Total Treatment<br>Satisfaction Change Score at Week 48<br>(Maintenance Phase) for Subjects from Q4W<br>ATLAS | | W48 |
| 6.26 | NA | NA | SOC | 201584/primar<br>y_01/T6.26 | Summary of HIVTSQc – Total Treatment Satisfaction Change Score at Week 48 (Maintenance Phase) for Subjects from SOC | | W48 |
| 6.27 | NA | NA | Q4W<br>ATLAS | 201584/primar<br>y_02/T6.41 | Summary of HIVTSQc – Individual Item Change<br>Score at Week 48 (Maintenance Phase) for<br>Subjects from Q4W ATLAS | | W48 |
| 6.28 | NA | NA | SOC | 201584/primar<br>y_02/T6.41 | Summary of HIVTSQc – Individual Item Change<br>Score at Week 48 (Maintenance Phase) for<br>Subjects from SOC | | W48 |
| 6.29 | NA | NA | Q4W<br>ATLAS | 201584/primar<br>y_01/T6.27 | Statistical Analysis of HIVTSQc – Total Treatment<br>Satisfaction Change Score at Week 48<br>(Maintenance Phase) for Subjects from Q4W<br>ATLAS | Adjust column header and footnote as appropriate. | W48 |
| 6.30 | NA | NA | SOC | 201584/primar<br>y_01/T6.27 | Statistical Analysis of HIVTSQc – Total Treatment<br>Satisfaction Change Score at Week 48<br>(Maintenance Phase) for Subjects from SOC | Adjust column header and footnote as appropriate. | W48 |

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Treatme | ent Accep | tance (A | CCEPT) | | | | |
| 6.31 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.28 | Proportion of Subjects with ACCEPT - Individual Item Score by Visit - LOCF (Maintenance Phase) | | W48 |
| 6.32 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.29 | Summary of Acceptance/General Dimension<br>Score (ACCEPT Questionnaire) by Visit<br>(Maintenance Phase) | | W48 |
| 6.33 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.30 | Summary of Acceptance/General Dimension<br>Score (ACCEPT Questionnaire) by Visit - LOCF<br>(Maintenance Phase) | | W48 |
| 6.34 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.31 | Summary of Change from Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit (Maintenance Phase) | | W48 |
| 6.35 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.32 | Summary of Change from Baseline in<br>Acceptance/General Dimension Score (ACCEPT<br>Questionnaire) by Prior Exposure to CAB+RPV (0<br>vs. >=1 Weeks) and Visit - LOCF (Maintenance<br>Phase) | | W48 |
| 6.36 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.33 | Statistical Analysis of Change from Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit for Subjects without Prior Exposure to CAB+RPV – LOCF (Maintenance Phase) | Adjust column header and footnote as appropriate. | W48 |

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.37 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.33 | Statistical Analysis of Change from Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit for Subjects with Prior Exposure to CAB+RPV – LOCF (Maintenance Phase) | Adjust column header and footnote as appropriate. | W48 |
| Prefere | nce | | | | | | |
| 6.38 | NA | NA | Q4W<br>ATLAS | Shell HO_T1 | Proportion of Subjects with Response to Each Individual Question in Preference Questionnaire at Week 48 (Maintenance Phase) for Subjects from Q4W ATLAS to Q8W ATLAS-2M | Only display Q8W arm. | HL, W48 |
| 6.39 | NA | NA | Intent-to-<br>Treat<br>Exposed | Shell HO_T1 | Proportion of Subjects with Response to Each Individual Question in Preference Questionnaire by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) at Week 48 for Subjects in Q8W ATLAS-2M (Maintenance Phase) | Only display Q8W arm. | W48 |
| 6.40 | NA | NA | Intent-to-<br>Treat<br>Exposed | Shell HO_T1 | Proportion of Subjects with Response to Each Individual Question in Preference Questionnaire at Week 48 for Subjects in Q4W ATLAS-2M (Maintenance Phase) | Only display Q4W arm. | W48 |
| Reason | s for Swit | ch/Conti | nuation | | | | |
| 6.41 | NA | NA | SOC | 201585/primar<br>y_02/T7.40 | Reasons for Switch at Baseline for Subjects from SOC | Remove columns 'Analysis Visit' and 'Total'. For percentages, use the format 'xx / xx (xx%)' where the denominator is the number of subjects with available valid data from the questionnaire. | W48 |
| Health ( | Health Outcomes Tables | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|--|--|--|--|--|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable | | | | | |
| 6.42 | NA | NA | Q4W<br>ATLAS | 201585/primar<br>y_02/T7.40 | Reasons for Continuation at Baseline for Subjects from Q4W ATLAS | Remove columns 'Analysis Visit' and 'Total'. For percentages, use the format 'xx / xx (xx%)' where the denominator is the number of subjects with available valid data from the questionnaire. | W48 | | | | | |

## 15.15.5.11. Health Outcomes Figures

| Health ( | Outcomes | Figures | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.1 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.1 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in HIVTSQs Total Treatment Satisfaction Score over Time(ANCOVA) for Subjects without Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.2 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.1 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in HIVTSQs Total Treatment Satisfaction Score over Time(ANCOVA) for Subjects with Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.3 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.2 | Line Plot of Difference (95% CI) in Adjusted Mean<br>Change from Baseline in HIVTSQs Total Treatment<br>Satisfaction Score over Time (ANCOVA) for<br>Subjects without Prior Exposure to CAB+RPV -<br>LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.4 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.2 | Line Plot of Difference (95% CI) in Adjusted Mean<br>Change from Baseline in HIVTSQs Total Treatment<br>Satisfaction Score over Time (ANCOVA) for<br>Subjects with Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.5 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.5 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in HAT-QoL (Life Satisfaction, HIV medication, and Disclosure Worries) by Visit (ANCOVA) for Subjects without Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |

| Health ( | Outcomes | Figures | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | | | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable | |
| 6.6 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.5 | Line Plot of Adjusted Mean (95% CI) Change from<br>Baseline in HAT-QoL (Life Satisfaction, HIV<br>medication, and Disclosure Worries) by Visit<br>(ANCOVA) for Subjects with Prior Exposure to<br>CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.7 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.6 | Line Plot of Difference in Adjusted Mean (95% CI) Change from Baseline in HAT-QoL (Life Satisfaction, HIV Medication, and Disclosure Worries) by Visit (ANCOVA) for Subjects without Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.8 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.6 | Line Plot of Difference in Adjusted Mean (95% CI) Change from Baseline in HAT-QoL (Life Satisfaction, HIV Medication, and Disclosure Worries) by Visit (ANCOVA) for Subjects with Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |

### **15.15.5.12. Virology Tables**

**Note:** If there is one or more CVFs during the Extension Phase, the tables included in "Genotype" and "Phenotype" below will also be produced for Maintenance and Extension Phase for Week 96 analysis.

| Virolog | Virology Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Genoty | ре | | | | | | |
| 7.1 | 7.1 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.1 | Summary of the Prevalence of Known INI<br>Resistance Mutations at time of CVF (Maintenance<br>Phase) – Plasma Sample | | W48, W96 |
| 7.2 | 7.2 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.2 | Summary of the Prevalence of Major Resistance<br>Mutations of NRTI, NNRTI and PI Class at time of<br>CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| 7.3 | 7.3 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.4 | Summary of Genotypic Susceptibility at time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| Phenot | уре | | | | | | • |
| 7.4 | 7.4 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.3 | Summary of Phenotype Susceptibility at time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| 7.5 | 7.5 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.6 | Summary of Phenotype: Number of Drugs to Which Subject is Phenotypic Resistant or Partial Sensitive or Sensitive at Time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| 7.6 | 7.6 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.7 | Summary of Fold Change to CAB and RPV at Time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |

| Virolog | y Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 7.7 | 7.7 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.5 | Summary of Net Assessment at time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| Miscella | Miscellaneousness | | | | | | |
| 7.8 | 7.8 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.8 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria during the Maintenance Phase | Remove columns for 'ARTs', 'FC for ARTs'. Adjust the footnotes as appropriate. For W96: Include baseline genotypic data from ATLAS PBMC samples; label sample as appropriate. | HL, W48,<br>W96 |
| NA | 7.9 | 7.1 | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.8 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria during the Maintenance and Extension Phase | Remove columns for 'ARTs', 'FC for ARTs'. Adjust the footnotes as appropriate. For W96 and EOS: Include baseline genotypic data from ATLAS PBMC samples; label sample as appropriate. | W96, EOS |
| 7.9 | 7.10 | 7.2 | Safety | 201585/primar<br>y_02/T8.8 | Summary of Viral load, Genotypic and Phenotypic data for Non-CVF Subjects with Genotypic and/or Phenotypic Data | Remove columns for 'ARTs', 'FC for ARTs'. Adjust the footnotes as appropriate. For W96 and EOS: Include baseline genotypic data from ATLAS PBMC samples; label sample as appropriate; remove the last footnote from the same table in WK48 analysis. | W48, W96,<br>EOS |

### 15.15.5.13. ICH Listings

**Note:** Unless otherwise specified, both unique subject ID and latest subject ID for a subject will be included in the listings; display by prior exposure to CAB+RPV (0, 1-24, >24 weeks, refer to Section 15.6.2 for calculation details) for all listings except for study population listings.

| ICH List | tings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Study Population | | | | | | | |
| 1 | 1 | 1 | Randomized | 201585/prima<br>ry_02/L1 | Listing of Subjects Randomized but Not Treated | | W48, W96 |
| 2 | 2 | 2 | Randomized | 201585/prima<br>ry_02/L2 | Listing of Randomized and Actual<br>Strata and Treatment Assignment | Randomized and Actual Treatments will include oral lead-in information (e.g. Oral followed by Q4W). Change the footnote # for column 'Dev.' to be [2]. Add a footnote for actual strata: [1] Actual strata are derived using the prior exposure to CAB+RPV in Study 201585, collected from eCRF. | W48, W96 |
| 3 | 3 | 3 | Screened | 201585/prima<br>ry_02/L3 | Listing of Reasons for Screen Failure | | W48, W96 |
| 4 | 4 | 4 | Intent-to-<br>Treat<br>Exposed | ES2 | Listing of Reasons for Study<br>Withdrawal | For WK96 and EOS: Add a footnote: "Note: This listing includes withdrawals per the data collected from the Study Conclusion eCRF form. It includes withdrawals from Maintenance or Extension Phase, and withdrawals from subjects who completed Maintenance phase and did not enter Extension phase with reasons beyond the | HL, W48, W96,<br>EOS |

| ICH List | ings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| | | | | | | completion of the study commitment." | |
| 5 | 5 | 5 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L5 | Listing of Reasons for Study Drug<br>Discontinuation | | W48, W96, EOS |
| 6 | 6 | 6 | Intent-to-<br>Treat<br>Exposed | DV2 | Listing of Important Protocol<br>Deviations | For W96 and EOS: add a column on the right "COVID-19 Related". The possible values in this column are Y and N, where Y indicates the deviation is COVID-19 related and N indicates the deviation is non-COVID-19 related. | W48, W96, EOS |
| 7 | 7 | 7 | Intent-to-<br>Treat<br>Exposed | DV2 | Listing of Protocol Deviations<br>Leading to Exclusion from the Per-<br>Protocol Population | Remove the last column on the right. | HL, W48, W96 |
| 8 | 8 | 8 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L8 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | W48, W96 |
| 9 | 9 | 9 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L9 | Listing of Demographic<br>Characteristics | | W48, W96, EOS |
| 10 | 10 | 10 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L10 | Listing of Race | | W48, W96, EOS |
| Efficacy | 1 | | | | | | |
| 11 | 11 | 11 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L11 | Listing of Study Outcome (50 c/mL<br>Threshold) at Week 48 – Snapshot<br>Analysis | For WK96: replace "48" with "96" in the title. Add a column "COVID-19 Relatedness" between Columns "Study | HL, W48, W96 |

| ICH List | ings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| | | | | | | Outcome" and "Subreason". Add a footnote "Note: Subjects XXXXX, XXXXX, and XXXXX took SOC oral bridging prior to/during Week 96 and their SOC oral bridging medications are considered part of the study treatment for the purpose of the snapshot. No snapshot penalty is applied to the temporary permitted switch to SOC oral bridging due to COVID-19." | |
| Safety: | Exposure | 9 | | | | | |
| 12 | 12 | 12 | Safety | 201585/prima<br>ry_02/L12 | Listing of Investigational Product Exposure Data | | W48, W96, EOS |
| Safety: | Adverse | Events | | | | | |
| 13 | 13 | 13 | Safety | 201585/prima<br>ry_02/L13 | Listing of Subject Numbers for Individual Adverse Events (Maintenance + Extension Phase) | For WK96 and EOS: Remove "(Maintenance + Extension Phase)" from the title (i.e. no phase restriction); display by Phase and prior exposure to CAB+RPV; adjust the column lengths for a better presentation. | W48, W96, EOS |
| 14 | 14 | 14 | Safety | 201585/prima<br>ry_02/L14 | Listing of Reasons for Considering as a Serious Adverse Event (Maintenance + Extension Phase) | For WK96 and EOS: Remove "(Maintenance + Extension Phase)" from the title (i.e. no phase restriction). | W48, W96, EOS |
| 15 | 15 | 15 | Safety | 201585/prima<br>ry_02/L15 | Listing of Fatal Adverse Events<br>(Maintenance + Extension Phase) | Add Study Period to the 5th Column from the left. For WK96 and EOS: Remove "(Maintenance + Extension Phase)" from the title (i.e. no phase restriction). | W48, W96, EOS |

| ICH List | ings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 16 | 16 | 16 | Safety | 201585/prima<br>ry_02/L16 | Listing of Non-Fatal Serious<br>Adverse Events (Maintenance +<br>Extension Phase) | Add Study Period to the 5 <sup>th</sup> Column from the left. For WK96 and EOS: Remove "(Maintenance + Extension Phase)" from the title (i.e. no phase restriction). | W48, W96, EOS |
| 17 | 17 | 17 | Safety | 201585/prima<br>ry_02/L17 | Listing of Adverse Events Leading<br>to Withdrawal/Permanent<br>Discontinuation of Investigational<br>Product (Maintenance + Extension<br>Phase) | Add Study Period to the 5 <sup>th</sup> Column from the left. | HL, W48, W96,<br>EOS |
| 18 | 18 | 18 | Safety | 201585/prima<br>ry_02/L18 | Listing of Changes in Intensity/Grades of Study Drug Injection Site Adverse Events (Maintenance + Extension Phase) | For WK96 and EOS: Remove "(Maintenance + Extension Phase)" from the title (i.e. no phase restriction). | W48, W96, EOS |
| 19 | 19 | 19 | Safety | 201585/prima<br>ry_03/L30 | Listing of All Adverse Events<br>(Maintenance + Extension Phase) | Add Study Period to the 5 <sup>th</sup> Column from the left. For WK96 and EOS: Remove "(Maintenance + Extension Phase)" from the title (i.e. no phase restriction). | W48, W96, EOS |
| NA | 66 | 66 | Safety | 207966/prima<br>ry_02/L19 | Listing of COVID-19 Adverse<br>Events | | W96, EOS |
| NA | 67 | 67 | Safety | SAF_L1 | Listing of COVID-19 Assessments | | W96, EOS |
| NA | 68 | 68 | Safety | SAF_L2 | Listing of COVID-19 Symptoms | | W96, EOS |
| Safety: | Pregnand | су | | | | | |
| 20 | 20 | 20 | Safety | 201585/prima<br>ry_02/L19 | Listing of Subjects Who Became<br>Pregnant during the Study<br>(Maintenance + Extension Phase) | For EOS, remove "(Maintenance + Extension Phase)" from the title. | W48, W96, EOS |

| ICH List | ings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Safety: | Hepatobi | liary (Liv | ver) | | | | |
| 21 | 21 | 21 | Safety | 201585/prima<br>ry_02/L20 | Listing of Medical Conditions for<br>Subjects with Liver stopping Events | | W48, W96, EOS |
| 22 | 22 | 22 | Safety | 201585/prima<br>ry_02/L21 | Listing of Substance Use for<br>Subjects with Liver Stopping<br>Events | | W48, W96, EOS |
| Safety: | ECG | | | | | | |
| 23 | 23 | 23 | Safety | 201584/prima<br>ry_01/L24 | Listing of ECG Values for Subjects with a Value of Potential Clinical Importance | Remove Phase Treatment from the column header. Add change from baseline values for each of QTc assessment. Adjust the footnote as appropriate. A footnote may be added to clarify the classification of PCI values. | W48, W96 |
| 24 | 24 | 24 | Safety | 201584/prima<br>ry_01/L25 | Listing of ECG Findings | Remove the 'Phase Treatment' from the third column on the left. | W48, W96 |
| Safety: | eC-SSRS | | | | | | |
| 25 | 25 | 25 | Safety | 201585/prima<br>ry_02/L24 | Listing of Possible Suicidality-<br>Related Adverse Event Data: Event<br>and Description (Section 1-Section<br>2) | | W48, W96 |
| 26 | 26 | 26 | Safety | 201585/prima<br>ry_02/L25 | Listing of Possible Suicidality-<br>Related Adverse Event Data:<br>Possible Cause(s) (Section 3) | | W48, W96 |
| 27 | 27 | 27 | Safety | 201585/prima<br>ry_02/L26 | Listing of Possible Suicidality-<br>Related Adverse Event Data | | W48, W96 |

| ICH List | tings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| | | | | | (Section 4) | | |
| 28 | 28 | 28 | Safety | 201585/prima<br>ry_02/L27 | Listing of Possible Suicidality-<br>Related Adverse Event Data<br>(Section 5-Section 8) | | W48, W96 |
| PK | | | | | | | |
| 29 | 29 | 29 | Pharmacoki<br>netic | 201584/prima<br>ry_01/L30 | Listing of Plasma CAB PK<br>Concentration-Time Data | Remove 'Phase Treatment' from the column header. Add a column "Excluded". | W48, W96, EOS |
| 30 | 30 | 30 | Pharmacoki<br>netic | 201584/prima<br>ry_01/L31 | Listing of Plasma RPV PK<br>Concentration-Time Data | Remove 'Phase Treatment' from the column header. Add a column "Excluded". | W48, W96, EOS |

### 15.15.5.14. Non-ICH Listings

**Note:** Unless otherwise specified, both unique subject ID and latest subject ID for a subject will be included in the listings; display by prior exposure to CAB+RPV (0, 1-24, >24 weeks, refer to calculation details in Section 15.6.2) for all listings except for study population listings.

| Non-IC | l Listings | 6 | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Study P | opulation | n | | | | | |
| 31 | 31 | 31 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/L30 | Listing of Reasons for Maintenance Phase Withdrawal | | W48, W96 |
| 32 | 32 | 32 | Oral Lead-<br>in | 201585/primar<br>y_02/L31 | Listing of Reasons for Oral Lead-in Period Withdrawal | | W48, W96 |
| NA | 33 | 33 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/L32 | Listing of Reasons for Extension Phase Withdrawal | | W96, EOS |
| 33 | 34 | 34 | Long-term<br>Follow-up | 201585/primar<br>y_02/L33 | Listing of Reasons for Long-term Follow-up Phase Withdrawal | | W48, W96, EOS |
| 34 | 35 | 35 | Screened | Shell POP_L2 | Listing of Subjects Who were Rescreened | | W48, W96 |
| 35 | 36 | 36 | Intent-to-<br>Treat<br>Exposed | Shell POP_L1 | Listing of Prior ART Medications | Remove the column 'Phase during Which Concomitant' | W48, W96 |
| 36 | 37 | 37 | Intent-to-<br>Treat<br>Exposed | Shell POP_L1 | Listing of Concomitant ART Medications | In case the same medication is concomitant during both maintenance and extension phases, list each of them in two separate rows. For W96 and EOS: add a column "SOC Oral | W48, W96, EOS |

| Non-ICH | l Listings | 3 | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | | | Bridging?" which has values of "Yes" and "No". | |
| 37 | 38 | 38 | Intent-to-<br>Treat<br>Exposed | Shell POP_L1 | Listing of ART Medications Received during Long-term Follow-up Phase | Remove the column 'Phase during Which Concomitant'. For W96 and EOS: add a column "Start Date of the Long-term Follow-up ART/Study Day". | W48, W96, EOS |
| 38 | 39 | 39 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/L39 | Listing of Investigational Product<br>Accountability - Oral Regimens | | W48, W96, EOS |
| 39 | 40 | 40 | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/L43 | Listing of Medical History of Seizure | | W48, W96 |
| NA | 65 | 65 | Intent-to-<br>Treat<br>Exposed | DV2 | Listing of COVID-19 Related Missed Visits and Missed Assessments Protocol Deviations | | W96 |
| Efficacy | 1 | | | | | | |
| 40 | 41 | 41 | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/L40 | Listing of All Plasma HIV-1 RNA Data for Subjects with Confirmed Virologic Failure | In column headers, replace 'Period' with 'Phase', replace 'Sample Day' with 'Study Day'. | W48, W96, EOS |
| 41 | 42 | 42 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/L41 | Listing of All Plasma HIV-1 RNA Data for Subjects with Viral load >=50 c/mL during the Maintenance Phase | In column headers, replace 'Period' with 'Phase', replace 'Sample Day' with 'Study Day'. | HL, W48, W96,<br>EOS |
| 42 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/L41 | Listing of All Plasma HIV-1 RNA Data for Subjects with Viral load >=50 c/mL during the Maintenance Oral Lead-in Period | In column headers, replace 'Period' with 'Phase', replace 'Sample Day' with 'Study Day'. | W48 |
| NA | 64 | 64 | Intent-to- | 207966/primar | Listing of All Plasma HIV-1 RNA Data | | W96, EOS |

| Non-IC | l Listings | 3 | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | Treat<br>Exposed | y_02/L41 | | | |
| 43 | 43 | 43 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/L43 | Listing of HIV-1 Associated Conditions (Maintenance + Extension Phase) | For WK96 and EOS: Do not restrict phases, i.e. remove "(Maintenance + Extension Phase" from the title; add "Phase" to the original "Treatment State" column header and present it as third column on the right. | W48, W96, EOS |
| Safety | | | | | | | |
| 44 | 44 | 44 | Safety | ABC_HSR_EX<br>PO2 | Listing of Abacavir Hypersensitivity Reaction Record - Exposure to Abacavir | | W48, W96 |
| 45 | 45 | 45 | Safety | ABC_HSR_DR<br>UG2 | Listing of Abacavir Hypersensitivity Reaction<br>Record - Subject History of Drug Allergies | | W48, W96 |
| 46 | 46 | 46 | Safety | ABC_HSR_CO<br>ND2 | Listing of Abacavir Hypersensitivity Reaction Record - Subject and Family Conditions | | W48, W96 |
| 47 | 47 | 47 | Safety | ABC_HSR_RA<br>SH2 | Listing of Abacavir Hypersensitivity Reaction Record - Skin Rash Details | | W48, W96 |
| 48 | 48 | 48 | Safety | ABC_HSR_SY<br>MP4 | Listing of Abacavir Hypersensitivity Reaction Record - Symptoms | | W48, W96 |
| 49 | 49 | 49 | Safety | VS4 | Listing of Abacavir Hypersensitivity Reaction<br>Record - Vital Signs | | W48, W96 |
| 50 | 50 | 50 | Safety | ABC_HSR<br>_SYMP6 | Listing of Abacavir Hypersensitivity Reaction<br>Record - Individual Symptoms and Diagnostic<br>Category Assignments (Excluding Other<br>Symptoms) | | W48, W96 |

| Non-ICH | l Listings | 3 | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 51 | 51 | 51 | Safety | ABC_HSR_SY<br>MP7 | Listing of Abacavir Hypersensitivity Reaction<br>Record - Individual Symptoms and Diagnostic<br>Category Assignments (Other Symptoms) | | W48, W96 |
| 52 | 52 | 52 | Safety | 201585/primar<br>y_02/L52 | Listing of Liver Monitoring/Stopping Event Reporting | For WK96, remove "Monitoring/" from the title. | W48, W96, EOS |
| 53 | 53 | 53 | Safety | 201585/primar<br>y_02/L53 | Listing of Liver Event Information for RUCAM Score | | W48, W96, EOS |
| 54 | 54 | 54 | Safety | 201585/primar<br>y_02/L54 | Listing of Liver Biopsy Details | | W48, W96, EOS |
| 55 | 55 | 55 | Safety | 201585/primar<br>y_02/L55 | Listing of Liver Imaging Details | | W48, W96, EOS |
| 56 | 56 | 56 | Safety | 201585/primar<br>y_02/L59 | Listing of Subjects Meeting Hepatobiliary Lab<br>Criteria | For WK96 and EOS: Follow 207966/primary_11/L1; display by phase and prior exposure to CAB+RPV. Screening and LTFU phases are not included. | W48, W96, EOS |
| 57 | 57 | 57 | Safety | 201585/primar<br>y_02/L57 | Listing of Potential QTc Interval Prolonging<br>Events of Interest | Add Study Period to the 5 <sup>th</sup> Column from the left. | W48, W96, EOS |
| 58 | 58 | 58 | Safety | 201585/primar<br>y_02/L58 | Listing of ECG values for Subjects with<br>Potential QTc Interval Prolonging Events of<br>Interest | | W48, W96, EOS |
| 59 | 59 | 59 | Safety | 201584/primar<br>y_01/L64 | Listing of ALT, AST, Bilirubin (including Total<br>and Direct Bilirubin), INR, and ALP for<br>Subjects Meeting Hepatobiliary Lab<br>Abnormality Criteria | Remove 'Only Q4W IM Subjects are presented in this listing.' from the footnote. | HL, W48, W96,<br>EOS |
| 60 | 60 | 60 | Safety | 201585/primar | Listing of Investigational Product Exposure | | W48, W96, EOS |

| Non-ICH | l Listings | 3 | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | y_02/L63 | Data for Subject Receiving Oral Bridging | | |
| 61 | 61 | 61 | Safety | 201584/primar<br>y_01/L66 | Listing of Dosing Errors and IP Device Malfunctions | | W48, W96, EOS |
| Virology | / | | | | | | |
| 62 | 62 | 62 | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/L64 | Listing of Replication Capacity in IN and PR/RT Region | Remove 'of Maintenance Phase' from the column header 'Study Day of Maintenance Phase'. | W48, W96, EOS |
| NA | 63 | 63 | Safety | 207966/primar<br>y_03/L1 | Listing of Resistance Associated Mutations (Pre-specified INSTI and IAS-USA NNRTI) | Remove "Excluded from PRC (Yes/No) from the first left column; remove the second left column; remove Study Day; mutations are per definition in Section 15.6.7. | W96, EOS |
| PK | | | | | | | |
| 63 | 69 | 69 | Long-term<br>Follow-up | 207966/primar<br>y_02/L63 | Listing of Plasma PK Concentration-Time Data since Last Injection | For WK96 and EOS: Remove age and add LTFU oral RPV start date; add asterisk to RPV concentration taken on/after the start of LTFU oral RPV and add a footnote explaining the asterisk, will be produced only if additional LTFU PK storage samples since last analysis data cut are planned to be analysed. | W48, W96, EOS |

# 15.15.6. List of Data Displays for Week 152 Planned Analyses

## 15.15.6.1. Study Population Tables

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Subject | Disposition | | | | |
| 1.1 | Randomized | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | 'No Treatment' column is not needed. | W152 |
| 1.2 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T1.3 | Summary of Subject Accountability: Study Conclusion Record | Add section for "COVID-19 Relatedness of the Withdrawal" with "Yes", "No" and "Unknown" categories. | W152 |
| 1.3 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T1.4 | Summary of Subject Accountability:<br>Extension Phase Conclusion Record | Add section for "COVID-19 Relatedness of the Withdrawal" with "Yes", "No" and "Unknown" categories. | W152 |
| 1.4 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T1.5 | Summary of Subject Accountability: Maintenance + Extension Phase Conclusion Record | Add section for "COVID-19 Relatedness of the Withdrawal" with "Yes", "No" and "Unknown" categories. | W152 |
| 1.5 | Long-term<br>Follow-up | 207966/primary_15/T1.6 | Summary of Subject Accountability: Long-<br>term Follow-up Phase Conclusion Record | Add section for "COVID-19 Relatedness of the Withdrawal" with "Yes", "No" and "Unknown" categories. If there are AEs leading to withdrawal, add sections for outcome and types similarly to 207966/primary_15/T1.5. | W152 |
| 1.6 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T1.7 | Summary of Subject Disposition at Each Study Phase | | W152 |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 1.7 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T1.8 | Summary of Reasons for Withdrawal at Each Study Phase | Remove the last footnote in example shell. | W152 |
| 1.8 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T1.9 | Summary of Subject Accountability: Withdrawals by Visit (Maintenance + Extension Phase) | | W152 |
| 1.9 | Intent-to-<br>Treat<br>Exposed | 201584/primary_15/T1.10 | Summary of Study Drug Discontinuation | Add section for "COVID-19 Relatedness of the Study Drug Discontinuation" with "Yes", "No" and "Unknown" categories. | W152 |
| 1.10 | Screened | 207966/primary_15/T1.14 | Summary of Study Populations | | W152 |
| 1.11 | Intent-to-<br>Treat<br>Exposed | DV1a | Summary of Important Protocol Deviations | | W152 |
| 1.12 | Intent-to-<br>Treat<br>Exposed | DV1a | Summary of Important Protocol Deviations (Maintenance + Extension Phase) | | W152 |
| 1.13 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T1.15 | Summary of Protocol Deviations Leading to Exclusion from the Per-Protocol Population | | W152 |
| 1.14 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T1.36 | Summary of Important COVID-19 Related Protocol Deviations | | W152 |
| 1.15 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T1.37 | Summary of Important Non-COVID-19<br>Related Protocol Deviations | | W152 |

| Study P | opulation Tab | les | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 1.16 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T1.16 | Summary of Demographic Characteristics | | W152 |
| 1.17 | Intent-to-<br>Treat<br>Exposed | DM5 | Summary of Race and Racial Combinations | | W152 |
| 1.18 | Intent-to-<br>Treat<br>Exposed | DM6 | Summary of Race and Racial<br>Combinations Details | | W152 |
| Medical | Conditions an | d Medications | | | |
| 1.19 | Intent-to-<br>Treat<br>Exposed | MH1 | Summary of Current Medical Conditions | | W152 |
| 1.20 | Intent-to-<br>Treat<br>Exposed | MH1 | Summary of Past Medical Conditions | | W152 |
| 1.21 | Intent-to-<br>Treat<br>Exposed | MH4 | Summary of Current Cardiac,<br>Gastrointestinal, Metabolism and Nutrition,<br>Psychiatric, Renal and Urinary, Nervous<br>System Conditions, and Hepatobiliary<br>Disorders | | W152 |
| 1.22 | Intent-to-<br>Treat<br>Exposed | MH4 | Summary of Past Cardiac,<br>Gastrointestinal, Metabolism and Nutrition,<br>Psychiatric, Renal and Urinary, Nervous<br>System Conditions, and Hepatobiliary<br>Disorders | | W152 |

| Study P | opulation Tab | les | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 1.23 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T1.30 | Summary of Prior ART Medications | Use "TENOFOVIR" for TDF and "TENOFOVIR ALAFENAMIDE" for TAF. Add a footnote "Note: TENOFOVIR refers to tenofovir disoproxil fumarate in the table.". | W152 |
| 1.24 | Intent-to-<br>Treat<br>Exposed | CM8 | Summary of Concomitant Non-ART<br>Medication Ingredient Combinations<br>(Maintenance + Extension Phase) | | W152 |
| 1.25 | Intent-to-<br>Treat<br>Exposed | 201585/primary_02/T1.33 | Summary of Lipid Modifying Agent Use at Baseline | | W152 |
| 1.26 | Intent-to-<br>Treat<br>Exposed | 201585/primary_02/T1.34 | Summary of Lipid Modifying Agent Use<br>Started during the Maintenance and<br>Extension Phase | | W152 |
| Visits In | npacted by CO | VID-19 Pandemic | | | |
| 1.27 | Intent-to-<br>Treat<br>Exposed | PAN4 | Summary of COVID-19 Pandemic Visit Impacts | | W152 |

### 15.15.6.2. Efficacy Tables

**Note:** For subgroup analyses, include rederived randomization strata (i.e. prior exposure to CAB+RPV: 0, 1-24, >24 weeks), all demographic and baseline characteristic subgroups as mentioned in EMA Subgroup Category 2 in Section 5.4.2, unless otherwise specified. Not all subjects on Q8W arm are planned to have viral load data collected at Week 4 (Week 4A or 4B), so leave Week 4 data blank for Q8W arm in by-visit snapshot analysis.

| Efficacy | / Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.1 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 152 – Snapshot Analysis – ITT-E | | W152 |
| 2.2 | Per-<br>Protocol | 207966/primary_15/T2.2 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 152 – Snapshot Analysis – Per-Protocol | | W152 |
| 2.3 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.3 | Summary of Study Outcomes (50 c/mL Threshold) at Week 152 – Snapshot Analysis | | W152 |
| 2.4 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.4 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 152 - Snapshot Analysis | | W152 |
| 2.5 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.5 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 152 by Subgroup - Snapshot Analysis | | W152 |
| 2.6 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.6 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 152 among Subjects with >=1 Weeks Prior Exposure to CAB+RPV - Snapshot Analysis | | W152 |

| Efficacy | / Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.7 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.7 | Summary of Study Outcomes (50 c/mL Threshold) at Week 152 by Subgroup – Snapshot Analysis | | W152 |
| 2.8 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.8 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 152 – Snapshot Analysis – ITT-E | | W152 |
| 2.9 | Per-<br>Protocol | 207966/primary_15/T2.9 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 152 – Snapshot Analysis – Per-Protocol | | W152 |
| 2.10 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.10 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 152 - Snapshot Analysis | | W152 |
| 2.11 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.11 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 152 by Subgroup - Snapshot Analysis | | W152 |
| 2.12 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.12 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 152 among Subjects with >=1 Weeks Prior Exposure to CAB+RPV - Snapshot Analysis | | W152 |
| 2.13 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.13 | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Visit (Up to Week 152, Maintenance + Extension Phase) – Snapshot Analysis | | W152 |
| 2.14 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.14 | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Subgroup and Visit (Up to Week 152, Maintenance + Extension Phase) – Snapshot Analysis | | W152 |

| Efficacy | / Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.15 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.15 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit (Up to Week 152, Maintenance + Extension Phase) – Snapshot Analysis | | W152 |
| 2.16 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.16 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Subgroup and Visit (Up to Week 152, Maintenance + Extension Phase) – Snapshot Analysis | | W152 |
| 2.17 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.17 | Proportion of Subjects with Plasma HIV-1 RNA <200 c/mL by Visit (Up to Week 152, Maintenance + Extension Phase) – Snapshot Analysis | | W152 |
| 2.18 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.18 | Proportion of Subjects with Plasma HIV-1 RNA >=200 c/mL by Visit (Up to Week 152, Maintenance + Extension Phase) – Snapshot Analysis | | W152 |
| 2.19 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.27 | Summary of Study Outcomes (200 c/mL Threshold) at Week 152 – Snapshot Analysis | | W152 |
| 2.20 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.19 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Failure at Week 152 - Treatment Related Discontinuation = Failure | Replace "Week 96" with "Week 152" in row labels. Change the upper bound in the second footnote to be "study day 1092". | W152 |
| 2.21 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.20 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Failure at Week 152 - Efficacy Related Discontinuation = Failure | Replace "Week 96" with "Week 152" in row labels. Change the upper bound in the first footnote to be "study day 1092". | W152 |

| Efficacy | / Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.22 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.21 | Proportion of Subjects with HIV-1 RNA >=50 c/mL at Week 152 (Snapshot) by Last Delay in IP Injection | Replace 'Week 96' with 'Week 152', and replace "(i.e. missing visit or withdrawal)" with "(e.g. missing visit, remote visit or withdrawal) in the footnote. | W152 |
| 2.23 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.38 | Summary of Change from Baseline in Plasma HIV-1 RNA (log10 c/mL) by Visit (Maintenance + Extension Phase) | | W152 |
| 2.24 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.22 | Summary of Plasma HIV-1 RNA (log10 c/mL) by Visit (Maintenance + Extension Phase) | | W152 |
| 2.25 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.23 | Cumulative Proportion of Subjects Meeting Confirmed Virology Failure Criteria by Visit (Up to Week 152, Maintenance + Extension Phase) | | W152 |
| 2.26 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.24 | Cumulative Proportion of Subjects Meeting Confirmed Virology Failure Criteria (Maintenance + Extension Phase) | | W152 |
| 2.27 | Confirmed<br>Virologic<br>Failure | 207966/primary_15/T2.25 | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmation of Confirmed Virologic Failure (Maintenance + Extension Phase) | | W152 |
| 2.28 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.26 | Proportion of Subjects with Plasma HIV-1 RNA <2 c/mL by Visit (Maintenance + Extension Phase) | | W152 |
| 2.29 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.28 | Summary of Subjects per Viral Load Category by Visit (Up to Week 152, Maintenance + Extension Phase) | | W152 |

| Efficacy | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.30 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.29 | Summary of Change from Baseline in CD4+ Cell Count (cells/mm^3) by Visit (Maintenance + Extension Phase) | | W152 |
| 2.31 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.30 | Summary of Change from Baseline in CD4+ Cell Count (cells/mm^3) at Week 152 by Subgroup (Extension Phase) | | W152 |
| 2.32 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.31 | Summary of CD4+ Cell Count (cells/mm^3) by Visit (Maintenance + Extension Phase) | | W152 |
| 2.33 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.32 | Summary of Change from Baseline in CD8+ Cell Count (cells/mm^3) by Visit (Maintenance + Extension Phase) | | W152 |
| 2.34 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.33 | Summary of CD8+ Cell Count (cells/mm^3) by Visit (Maintenance + Extension Phase) | | W152 |
| 2.35 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.34 | Summary of CD4+/CD8+ Ratio Cell Count (cells/mm^3) by Visit (Maintenance + Extension Phase) | | W152 |
| 2.36 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.35 | Summary of HIV-1 Associated Conditions Including Recurrences (Maintenance + Extension Phase) | | W152 |
| 2.37 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.36 | Summary of HIV-1 Associated Conditions Excluding Recurrences (Maintenance + Extension Phase) | | W152 |
| 2.38 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/T2.37 | Summary of HIV-1 Disease Progression and/or Deaths (Maintenance + Extension Phase) | Replace "maintenance" with<br>"maintenance and extension" in<br>the second footnote. | W152 |

### 15.15.6.3. Efficacy Figures

**Note:** For subgroup analyses, include rederived randomization strata (i.e. prior exposure to CAB+RPV: 0, 1-24, >24 weeks), all demographic and baseline characteristic subgroups as mentioned in EMA Subgroup Category 2 in Section 5.4.2, unless otherwise specified. Not all subjects on Q8W arm are planned to have viral load data collected at Week 4 (Week 4A or 4B), so leave Week 4 data blank for Q8W arm in by-visit snapshot analysis.

| Efficacy | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.1 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/F2.1 | Proportion (95% CI) of Subjects with HIV-1 RNA ≥50 c/mL by Visit (Up to Week 152, Maintenance + Extension Phase) – Snapshot Analysis | | W152 |
| 2.2 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/F2.2 | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA ≥50 c/mL at Week 152 by Subgroup – Snapshot Analysis | | W152 |
| 2.3 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/F2.3 | Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL by Visit (Up to Week 152, Maintenance + Extension Phase) – Snapshot Analysis | | W152 |
| 2.4 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/F2.4 | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL at Week 152 by Subgroup – Snapshot Analysis | | W152 |
| 2.5 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/F2.5 | Proportion (95% CI) of Subjects with HIV-1 RNA >=200 c/mL by Visit (Up to Week 152, Maintenance + Extension Phase) – Snapshot Analysis | | W152 |
| 2.6 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/F2.6 | Proportion (95% CI) of Subjects with HIV-1 RNA <200 c/mL by Visit (Up to Week 152, Maintenance + Extension Phase) – Snapshot Analysis | | W152 |
| 2.7 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/F2.7 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit – for CVF Subjects | | W152 |

| Efficacy Figures | | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.8 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/F2.8 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit for subjects Who are in the Category of 'HIV-1 RNA >=50 c/mL' at Week 152 per Snapshot Algorithm | | W152 |

## 15.15.6.4. Safety Tables

| Safety 7 | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Exposu | re | | | | |
| 3.1 | Safety | 207966/primary_15/T3.2 | Summary of Extent of Exposure to Study<br>Treatment including SOC Oral Bridging<br>(Maintenance + Extension Phase) | The levels for categorical summaries except for oral lead-in will be selected as appropriate. | W152 |
| 3.2 | Safety | 207966/primary_15/T3.3 | Summary of Needle Length and Gauge for CAB Injection (Maintenance + Extension Phase) | | W152 |
| 3.3 | Safety | 207966/primary_15/T3.4 | Summary of Needle Length and Gauge for RPV Injection (Maintenance + Extension Phase) | | W152 |
| 3.4 | Safety | 207966/primary_15/T3.5 | Summary of Adherence to CAB/RPV Injection<br>Dosing Schedule (Maintenance + Extension<br>Phase) | Replace rows for missed Injection with those specified in Section 15.6.4. Adjust the footnote as appropriate. For missed reloading rows, leave blank for Q4W. | W152 |
| Adverse | e Events | | | | |
| 3.5 | Safety | 207966/primary_15/T3.6 | Summary of All Adverse Events by System<br>Organ Class (Maintenance + Extension Phase) | | W152 |
| 3.6 | Safety | 207966/primary_15/T3.8 | Summary of All Adverse Events by System<br>Organ Class and Maximum Toxicity<br>(Maintenance + Extension Phase) | | W152 |
| 3.7 | Safety | 207966/primary_15/T3.8 | Summary of All Adverse Events by System<br>Organ Class and Maximum Toxicity (Extension<br>Phase) | | W152 |
| 3.8 | Safety | 207966/primary_15/T3.9 | Summary of All Adverse Events Excluding<br>Study Drug Injection Site Reactions by System<br>Organ Class and Maximum Toxicity | | W152 |

| Safety Tables | | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | (Maintenance + Extension Phase) | | |
| 3.9 | Safety | 207966/primary_15/T3.10 | Summary of All On-treatment Adverse Events by System Organ Class and Maximum Toxicity (Maintenance + Extension Phase) | | W152 |
| 3.10 | Safety | 207966/primary_15/T3.11 | Summary of Common Adverse Events (>=5%) by Overall Frequency (Maintenance + Extension Phase) | | W152 |
| 3.11 | Safety | 207966/primary_15/T3.12 | Summary of Common Grade 2-5 Adverse<br>Events (>=1%) by Overall Frequency<br>(Maintenance + Extension Phase) | | W152 |
| 3.12 | Safety | 207966/primary_15/T3.13 | Summary of All Drug-related Adverse Events by System Organ Class (Maintenance + Extension Phase) | | W152 |
| 3.13 | Safety | 207966/primary_15/T3.15 | Summary of All Drug-related Adverse Events by<br>System Organ Class and Maximum Toxicity<br>(Maintenance + Extension Phase) | | W152 |
| 3.14 | Safety | 207966/primary_15/T3.15 | Summary of All Drug-related Adverse Events by<br>System Organ Class and Maximum Toxicity<br>(Extension Phase) | | W152 |
| 3.15 | Safety | 207966/primary_15/T3.16 | Summary of All Drug-related Adverse Events<br>Excluding Study Drug Injection Site Reactions<br>by System Organ Class and Maximum Toxicity<br>(Maintenance + Extension Phase) | | W152 |
| 3.16 | Safety | 207966/primary_15/T3.17 | Summary of All Drug-Related Grade 2-5<br>Adverse Events by Overall Frequency<br>(Maintenance + Extension Phase) | | W152 |
| Serious | and Other Sig | gnificant Adverse Events | | | |

| Safety 7 | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.17 | Safety | 207966/primary_15/T3.19 | Summary of Serious Adverse Events by System Organ Class (Maintenance + Extension Phase) | | W152 |
| 3.18 | Long-term<br>Follow-up | 207966/primary_15/T3.20 | Summary of Serious Adverse Events by System Organ Class (Long-term Follow-up Phase) | | W152 |
| 3.19 | Safety | 207966/primary_15/T3.22 | Summary of Drug-related Serious Adverse<br>Events by System Organ Class (Maintenance +<br>Extension Phase) | | W152 |
| 3.20 | Safety | 207966/primary_15/T3.23 | Summary of Non-Fatal Serious Adverse Events by Overall Frequency (Maintenance + Extension Phase) | | W152 |
| 3.21 | Safety | 207966/primary_15/T3.24 | Summary of Drug-related Non-Fatal Serious<br>Adverse Events by Overall Frequency<br>(Maintenance + Extension Phase) | | W152 |
| 3.22 | Safety | 207966/primary_15/T3.26 | Summary of Adverse Events Leading to<br>Withdrawal/Permanent Discontinuation of<br>Investigational Product by System Organ Class<br>(Maintenance + Extension Phase) | Adjust the footnote as needed, depending on the given data. | W152 |
| 3.23 | Safety | 207966/primary_15/T3.25 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class (Extension Phase) | | W152 |
| 3.24 | Safety | 207966/primary_15/T3.27 | Summary of Common (>=5%) Non-Serious<br>Adverse Events (Maintenance + Extension<br>Phase) | | W152 |
| 3.25 | Safety | 207966/primary_15/T3.28 | Summary of Subjects and Number of<br>Occurrences of Common (>=5%) Non-Serious<br>Adverse Events by System Organ Class | | W152 |

| Safety 7 | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | (Maintenance + Extension Phase) | | |
| 3.26 | Safety | 207966/primary_15/T3.29 | Summary of Subjects and Number of occurrences of SAEs, Fatal SAEs, and Drugrelated SAEs (Maintenance + Extension Phase) | | W152 |
| Study D | rug Injection | Site Reaction Adverse Even | ts | | |
| 3.27 | Safety | 207966/primary_15/T3.32 | Summary of Study Drug Injection Site Reaction<br>Adverse Events (Event-level Summary) –<br>(Maintenance + Extension Phase) | | W152 |
| 3.28 | Safety | 207966/primary_15/T3.34 | Summary of Subject-level Characteristics of<br>Study Drug Injection Site Reaction Adverse<br>Events – Overall and Common (Maintenance +<br>Extension Phase) | | W152 |
| 3.29 | Safety | 207966/primary_15/T3.35 | Summary of Study Drug Injection Site Reaction<br>Adverse Events by Visit and Maximum Severity<br>– Overall and Common (Maintenance +<br>Extension Phase) | | W152 |
| 3.30 | Safety | 207966/primary_15/T3.36 | Summary of Drug-related Study Drug Injection<br>Site Reaction Adverse Events (Event-level<br>Summary) - CAB (Maintenance + Extension<br>Phase) | | W152 |
| 3.31 | Safety | 207966/primary_15/T3.37 | Summary of Drug-related Subject-level<br>Characteristics of Study Drug Injection Site<br>Reaction Adverse Events (Maintenance +<br>Extension Phase) - Overall and Common (CAB) | | W152 |
| 3.32 | Safety | 207966/primary_15/T3.38 | Summary of Overall and Common Drug-related<br>Study Drug Injection Site Reaction Adverse<br>Events by Visit and Maximum Severity | | W152 |

| Safety 1 | <b>Tables</b> | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | (Maintenance + Extension Phase) - CAB | | |
| 3.33 | Safety | 207966/primary_15/T3.39 | Summary of Maximum Drug-related Study Drug<br>Injection Site Reaction Adverse Event Grade by<br>Needle Length (Maintenance + Extension<br>Phase) – Common (CAB) | Replace "maintenance" with "maintenance and extension" in the footnote. | W152 |
| 3.34 | Safety | 207966/primary_15/T3.40 | Summary of Drug-related Study Drug Injection<br>Site Reaction Adverse Events (Event-level<br>Summary) - RPV (Maintenance + Extension<br>Phase) | | W152 |
| 3.35 | Safety | 207966/primary_15/T3.41 | Summary of Drug-related Subject-level<br>Characteristics of Study Drug Injection Site<br>Reaction Adverse Events (Maintenance +<br>Extension Phase) - Overall and Common (RPV) | | W152 |
| 3.36 | Safety | 207966/primary_15/T3.42 | Summary of Overall and Common Drug-related<br>Study Drug Injection Site Reaction Adverse<br>Events by Visit and Maximum Severity<br>(Maintenance + Extension Phase) - RPV | | W152 |
| 3.37 | Safety | 207966/primary_15/T3.43 | Summary of Maximum Drug-related Study Drug<br>Injection Site Reaction Adverse Event Grade by<br>Needle Length (Maintenance + Extension<br>Phase) – Common (RPV) | Replace "maintenance" with<br>"maintenance and extension" in the footnote. | W152 |
| Laborat | ory: Chemistr | y and Hematology | | | · |
| 3.38 | Safety | 207966/primary_15/T3.44 | Summary of Chemistry Changes from Baseline by Visit (Maintenance + Extension Phase) | | W152 |
| 3.39 | Safety | 207966/primary_15/T3.45 | Summary of Chemistry Values by Visit (Maintenance + Extension Phase) | | W152 |
| 3.40 | Safety | 207966/primary_15/T3.46 | Summary of Hematology Changes from | | W152 |

| Safety 7 | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | Baseline by Visit (Maintenance + Extension Phase) | | |
| 3.41 | Safety | 207966/primary_15/T3.47 | Summary of Hematology Values by Visit (Maintenance + Extension Phase) | | W152 |
| 3.42 | Safety | 207966/primary_15/T3.49 | Summary of Maximum Post-Baseline Emergent Chemistry Toxicities (Maintenance + Extension Phase) | | W152 |
| 3.43 | Safety | 207966/primary_15/T3.51 | Summary of Maximum Post-Baseline Emergent<br>Hematology Toxicities (Maintenance +<br>Extension Phase) | | W152 |
| Laborat | ory: Urinalysis | S | | | |
| 3.44 | Safety | 207966/primary_15/T3.52 | Summary of Urinalysis Dipstick Results by Visit (Maintenance + Extension Phase) | | W152 |
| 3.45 | Safety | 207966/primary_15/T3.53 | Summary of Urine Concentrations Changes from Baseline by Visit (Maintenance + Extension Phase) | | W152 |
| 3.46 | Safety | 207966/primary_15/T3.54 | Summary of Changes in Proteinuria Baseline<br>Laboratory Result to Maximum Post-Baseline<br>Laboratory Result (Maintenance + Extension<br>Phase) | | W152 |
| Laborat | ory: Lipid | | | | |
| 3.47 | Safety | 207966/primary_15/T3.55 | Summary of Changes in Baseline NCEP Fasting<br>Lipid Category to Maximum Post-Baseline<br>Category (Triglycerides, Lipids LOCF) -<br>Maintenance + Extension Phase | Replace "Maintenance" with<br>"Maintenance and Extension" in the<br>second footnote. | W152 |
| 3.48 | Safety | 207966/primary_15/T3.56 | Summary of Changes in Baseline NCEP Fasting | Replace "Maintenance" with | W152 |

| Safety 7 | <b>Tables</b> | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | Lipid Category to Maximum Post-Baseline<br>Category (Total Cholesterol, Lipids LOCF) -<br>Maintenance + Extension Phase | "Maintenance and Extension" in the second footnote. | |
| 3.49 | Safety | 207966/primary_15/T3.57 | Summary of Changes in Baseline NCEP Fasting<br>Lipid Category to Minimum Post-Baseline<br>Category (HDL Cholesterol, Lipids LOCF) -<br>Maintenance + Extension Phase | Replace "Maintenance" with<br>"Maintenance and Extension" in the<br>second footnote. | W152 |
| 3.50 | Safety | 207966/primary_15/T3.58 | Summary of Changes in Baseline NCEP Fasting<br>Lipid Category to Maximum Post-Baseline<br>Category (LDL Cholesterol, Lipids LOCF) -<br>Maintenance + Extension Phase | Replace "Maintenance" with<br>"Maintenance and Extension" in the<br>second footnote. | W152 |
| 3.51 | Safety | 207966/primary_15/T3.59 | Summary of Fasting Lipids Percentage<br>Changes from Baseline by Visit (Maintenance +<br>Extension Phase) - Lipids LOCF | | W152 |
| 3.52 | Safety | 207966/primary_15/T3.60 | Summary of Fasting TC/HDL ratio Changes from Baseline (Maintenance + Extension Phase) – Lipids LOCF | | W152 |
| Laborat | ory: Hepatobi | liary (Liver) | | | |
| 3.53 | Safety | 207966/primary_15/T3.61 | Summary of Liver Stopping Event Reporting (Maintenance + Extension Phase) | | W152 |
| 3.54 | Safety | 207966/primary_15/T3.63 | Summary of Subjects Meeting Hepatobiliary<br>Abnormality Criteria (Maintenance +Extension<br>Phase) | | W152 |
| ECG | | | | | |
| 3.55 | Safety | 207966/primary_15/T3.64 | Summary of ECG Findings (Maintenance + Extension Phase) | | W152 |

| Safety 7 | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.56 | Safety | 207966/primary_15/T3.65 | Summary of Change from Baseline in ECG values by Visit (Maintenance + Extension Phase) | | W152 |
| 3.57 | Safety | 207966/primary_15/T3.66 | Summary of QTc Values by Category (Maintenance + Extension Phase) | | W152 |
| 3.58 | Safety | 207966/primary_15/T3.67 | Summary of Change from Baseline QTc Values by Category (Maintenance + Extension Phase) | | W152 |
| Vital Sig | gns | | | | |
| 3.59 | Safety | 207966/primary_15/T3.68 | Summary of Change from Baseline in Vital Signs by Visit (Maintenance + Extension Phase) | | W152 |
| 3.60 | Safety | 207966/primary_15/T3.69 | Summary of BMI Shift from Baseline by Sex and Visit (Maintenance + Extension Phase) | | W152 |
| 3.61 | Safety | 207966/primary_15/T3.70 | Summary of BMI Shift from Baseline by Strata and Visit (Maintenance + Extension Phase) | | W152 |
| 3.62 | Safety | 207966/primary_15/T3.71 | Summary of Change from Baseline in Weight and BMI by Strata and Visit (Maintenance + Extension Phase) | | W152 |
| Adverse | Event of Spe | cial Interest (AESI) | | | |
| 3.63 | Safety | 207966/primary_15/T3.74 | Summary of Depression, Anxiety and Suicidal Ideation/Behaviour Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and Prior History of Depression, Anxiety and Suicidal Ideation at Screening (Maintenance + Extension Phase) | May need to adjust the footnote given the data. | W152 |
| 3.64-<br>3.80 | Safety | 207966/primary_15/T3.92-<br>3.108 | Summary of XXX Adverse Events of Special<br>Interest by System Organ Class and Preferred<br>Term (Number of Subjects and Occurrence) – | | W152 |

| Safety 7 | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | Maintenance + Extension Phase | | |
| 3.81 | Safety | 207966/primary_15/T3.110 | Summary of Characteristics of Common<br>Adverse Events of Special Interest –<br>Maintenance + Extension Phase | | W152 |
| 3.82 | Safety | 207966/primary_15/T3.111 | Summary of Syncope and Presyncope Adverse Events - Maintenance + Extension Phase | | W152 |
| 3.83 | Safety | 207966/primary_15/T3.112 | Summary of Syncope and Presyncope Adverse<br>Events and Injection Visits - Maintenance +<br>Extension Phase | | W152 |
| COVID- | 19 Adverse Ev | rent | | | |
| 3.84 | Safety | 207966/primary_15/T3.113 | Summary of COVID-19 Adverse Events by<br>System Organ Class and Maximum Toxicity<br>(Maintenance + Extension Phase) | | W152 |
| 3.85 | Safety | 207966/primary_15/T3.115 | Summary of COVID-19 Assessments (Maintenance + Extension Phase) | Place "Within" in front of "14" in the first footnote. If COVID-19 assessments are collected multiple times during the study, a combination of standard displays PAN1A and PAN2A with appropriate adjustments may be used. | W152 |
# 15.15.6.5. Safety Figures

| Safety Figures | | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.1 | Safety | 207966/primary_15/F3.1 | Plot of Common Adverse Events and Relative Risk - Q8W vs. Q4W (Maintenance + Extension Phase) – Excluding Study Drug ISRs | | W152 |
| 3.2 | Safety | 207966/primary_15/F3.2 | Plot of Common Study Drug Injection Site Reaction<br>Adverse Events and Relative Risk - Q8W vs. Q4W<br>(Maintenance +Extension Phase) | | W152 |
| 3.3 | Safety | 207966/primary_02/F3.6 | Plot of Incidence of Maintenance and Extension Phase<br>Study Drug Injection Site Reaction Adverse Events by<br>Visit (Overall and Common) – CAB and/or RPV | | W152 |
| 3.4 | Safety | 207966/primary_15/F3.7 | Plot of Incidence of Maintenance and Extension Phase<br>Drug-Related Study Drug Injection Site Reaction<br>Adverse Events by Visit (Overall and Common) – CAB | | W152 |
| 3.5 | Safety | 207966/primary_15/F3.8 | Plot of Incidence of Maintenance and Extension Phase<br>Drug-Related Study Drug Injection Site Reaction<br>Adverse Events by Visit (Overall and Common) – RPV | | W152 |
| 3.6 | Safety | 207966/primary_15/F3.21 | Plot of Incidence of Maintenance and Extension Phase<br>Study Drug Injection Site Reaction Adverse Events by<br>Strata and Visit (Overall and Common) - CAB and/or<br>RPV | | W152 |
| 3.7 | Safety | 207966/primary_15/F3.13 | Scatter Plot of Maximum vs. Baseline for ALT (Maintenance + Extension Phase) | | W152 |
| 3.8 | Safety | 207966/primary_15/F3.15 | Scatter Plot of Maximum Total Bilirubin vs. Maximum ALT (Maintenance + Extension Phase) | | W152 |
| 3.9 | Safety | 207966/primary_15/F3.18 | Bar Chart of Lipid NCEP Categories at Week 152 vs. Baseline – Triglycerides, Total Cholesterol, LDL | | W152 |

| Safety F | Safety Figures | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | Cholesterol (Lipids LOCF) | | |
| 3.10 | Safety | 207966/primary_15/F3.19 | Bar Chart of Lipid NCEP Categories at Week 152 vs. Baseline - HDL Cholesterol (Lipids LOCF) | | W152 |
| 3.11 | Safety | 207966/primary_15/F3.20 | Histogram of Timeliness of Injections (Maintenance + Extension Phase) | | W152 |
| 3.12 | Safety | 207966/primary_15/F3.22 | Patient Profile for Subjects with Syncope or Presyncope Adverse Events (Maintenance + Extension Phase) | | W152 |

#### 15.15.6.6. Pharmacokinetic Tables

| Pharmac | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.1 | Pharmacokinetic | 207966/primary_15/T4.1 | Summary of Plasma CAB PK Concentration (ug/mL) -<br>Time Data by Treatment and Visit (Maintenance +<br>Extension Phase) – Including Log-transformed Statistics | Add Week 156 for Q4W, Week 160 for Q8W. Add following to the second footnote: PK samples were collected at Week 156 (for Q4W subjects) or Week 160 (for Q8W subjects) if Week 152 PK samples were missed (e.g. due to the delays in protocol amendment approvals or site errors). | W152 |
| 4.2 | Pharmacokinetic | 207966/primary_15/T4.2 | Summary of Plasma RPV PK Concentration (ng/mL) -<br>Time Data by Treatment and Visit (Maintenance +<br>Extension Phase) – Including Log-transformed Statistics | Similar notes to above. | W152 |
| 4.3 | Pharmacokinetic | 207966/primary_15/T4.3 | Summary of Evaluable Plasma CAB PK Concentration (ug/mL) -Time Data by Treatment and Visit (Maintenance + Extension Phase) – Including Log-transformed Statistics | Similar notes to above. | W152 |
| 4.4 | Pharmacokinetic | 207966/primary_15/T4.4 | Summary of Evaluable Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit (Maintenance + Extension Phase) – Including Log-transformed Statistics | Similar notes to above. | W152 |
| 4.5 | Pharmacokinetic | 207966/primary_15/T4.5 | Summary of Evaluable Plasma CAB PK Concentration (ug/mL) -Time Data by Strata and Treatment and Visit (Maintenance + Extension Phase) – Including Log-transformed Statistics | Similar notes to above. | W152 |

| Pharmacokinetic Tables | | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.6 | Pharmacokinetic | 207966/primary_15/T4.6 | Summary of Evaluable Plasma RPV PK Concentration (ng/mL) -Time Data by Strata and Treatment and Visit (Maintenance + Extension Phase) – Including Log-transformed Statistics | Similar notes to above. | W152 |
| 4.7 | Long-term Follow-<br>up | 207966/primary_15/T4.1 | Summary of Plasma CAB PK Concentration (ug/mL) -<br>Time Data by Treatment and Visit (Long-term Follow-up<br>Phase) - Including Log-transformed Statistics | Remove the column 'Pl.<br>Time' and the second<br>footnote. | W152 |
| 4.8 | Long-term Follow-<br>up | 207966/primary_15/T4.2 | Summary of Plasma RPV PK Concentration (ng/mL) -<br>Time Data by Treatment and Visit (Long-term Follow-up<br>Phase) - Including Log-transformed Statistics | Remove the column 'Pl.<br>Time' and the second<br>footnote. | W152 |

## 15.15.6.7. Pharmacokinetic Figures

| Pharmaco | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.1 | Pharmacokinetic | 207966/primary_15/F4.1 | Individual Plasma CAB Concentration-Time<br>Plots (Linear and Semi-Log) – Maintenance +<br>Extension Phase | | W152 |
| 4.2 | Pharmacokinetic | 207966/primary_15/F4.2 | Individual Plasma RPV Concentration-Time<br>Plots (Linear and Semi-Log) – Maintenance +<br>Extension Phase | | W152 |
| 4.3 | Pharmacokinetic | 207966/primary_15/F4.3 | Mean (SD) Plasma CAB Concentration-Time<br>Plots (Linear and Semi-Log) – Maintenance +<br>Extension Phase | Treat Week 152 similarly to Week 96 on X axis and update the relevant footnote as "To save the plotting space, Week 96 is displayed next to Week 48 and Week 152 is displayed next to Week 152, with hashes to indicate the X axis break." | W152 |
| 4.4 | Pharmacokinetic | 207966/primary_15/F4.4 | Mean (SD) Plasma RPV Concentration-Time<br>Plots (Linear and Semi-Log) – Maintenance +<br>Extension Phase | Similar notes to above. | W152 |
| 4.5 | Pharmacokinetic | 207966/primary_15/F4.5 | Mean (SD) Evaluable Plasma CAB Concentration-Time Plots (Linear and Semi-<br>Log) – Maintenance + Extension Phase | Similar notes to above. | W152 |
| 4.6 | Pharmacokinetic | 207966/primary_15/F4.6 | Mean (SD) Evaluable Plasma RPV Concentration-Time Plots (Linear and Semi-<br>Log) – Maintenance + Extension Phase | Similar notes to above. | W152 |
| 4.7 | Pharmacokinetic | 207966/primary_15/F4.7 | Mean (SD) Evaluable Plasma CAB Concentration-Time Plots by Strata (Linear and Semi-Log) – Maintenance + Extension | Similar notes to above. | W152 |

| Pharmaco | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | Phase | | |
| 4.8 | Pharmacokinetic | 207966/primary_15/F4.8 | Mean (SD) Evaluable Plasma RPV<br>Concentration-Time Plots by Strata (Linear<br>and Semi-Log) – Maintenance + Extension<br>Phase | Similar notes to above. | W152 |
| 4.9 | Pharmacokinetic | 207966/primary_15/F4.9 | Median (5th and 95th Percentile) Plasma CAB<br>Concentration-Time Plots (Linear and Semi-<br>Log) – Maintenance + Extension Phase | Similar notes to above. | W152 |
| 4.10 | Pharmacokinetic | 207966/primary_15/F4.10 | Median (5th and 95th Percentile) Plasma RPV<br>Concentration-Time Plots (Linear and Semi-<br>Log) – Maintenance + Extension Phase | Similar notes to above. | W152 |
| 4.11 | Pharmacokinetic | 207966/primary_15/F4.11 | Median (5th and 95th Percentile) Evaluable<br>Plasma CAB Concentration-Time Plots (Linear<br>and Semi-Log) – Maintenance + Extension<br>Phase | Similar notes to above. | W152 |
| 4.12 | Pharmacokinetic | 207966/primary_15/F4.12 | Median (5th and 95th Percentile) Evaluable<br>Plasma RPV Concentration-Time Plots (Linear<br>and Semi-Log) – Maintenance + Extension<br>Phase | Similar notes to above. | W152 |
| 4.13 | Pharmacokinetic | 207966/primary_15/F4.13 | Median (5th and 95th Percentile) Evaluable<br>Plasma CAB Concentration-Time Plots by<br>Strata (Linear and Semi-Log) – Maintenance +<br>Extension Phase | Similar notes to above. | W152 |
| 4.14 | Pharmacokinetic | 207966/primary_15/F4.14 | Median (5th and 95th Percentile) Evaluable<br>Plasma RPV Concentration-Time Plots by<br>Strata (Linear and Semi-Log) – Maintenance +<br>Extension Phase | Similar notes to above. | W152 |

| Pharmaco | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.15 | Pharmacokinetic | 207966/primary_15/F4.15 | Median Evaluable Plasma CAB Trough PK<br>Concentration (ug/mL) - Time Plots by<br>Treatment and Strata (Linear and Semi-Log) –<br>Maintenance + Extension Phase | Similar notes to above. | W152 |
| 4.16 | Pharmacokinetic | 207966/primary_15/F4.16 | Median Evaluable Plasma RPV Trough PK<br>Concentration (ng/mL) - Time Plots by<br>Treatment and Strata (Linear and Semi-Log) –<br>Maintenance + Extension Phase | Similar notes to above. | W152 |
| 4.17 | Long-term Follow-<br>up | 207966/primary_02/F4.15 | Plasma PK Concentration-Time since Last Injection Plots by Overall and Strata | Add plot for overall. Exclude RPV concentrations on/after the start of oral RPV that was received after the last injection. Add a footnote: "Note: For subjects who received oral RPV after the last injection, the RPV concentrations taken on or after the start of such oral RPV are excluded from the plot." | W152 |

## 15.15.6.8. Pharmacokinetic / Pharmacodynamic Figures

| Pharmac | Pharmacokinetic / Pharmacodynamic Figures | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| PK / PD E | PK / PD Efficacy Analyses | | | | |
| 5.1 | Pharmacokinetic | 207966/primary_15/F5.1 | Individual CAB Trough Concentration-time Profiles for Subjects with Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 152 and Median, 5th & 95th Percentile of CAB Conc-Time Profiles for Other Subjects (Semi-Log) – Maintenance + Extension Phase | | W152 |
| 5.2 | Pharmacokinetic | 207966/primary_15/F5.2 | Individual RPV Trough Concentration-time Profiles for Subjects with Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 152 and Median, 5th & 95th Percentile of RPV Conc-Time Profiles for Other Subjects (Semi-Log) – Maintenance + Extension Phase | | W152 |
| PK / PD S | Safety Analyses | | | | |
| 5.3 | Pharmacokinetic | 207966/primary_02/F5.6 | Scatter Plot of Maximum Change from Baseline in ALT versus Last Trough CAB PK Concentrations by Strata and Treatment during the Maintenance and Extension Phase | Replace "Maintenance" with<br>"Maintenance and Extension" in<br>the first footnote. | W152 |
| 5.4 | Pharmacokinetic | 207966/primary_02/F5.7 | Scatter Plot of Maximum Change from Baseline in ALT versus Last Trough RPV PK Concentrations by Strata and Treatment during the Maintenance and Extension Phase | Replace "Maintenance" with<br>"Maintenance and Extension" in<br>the first footnote. | W152 |
| 5.5 | Pharmacokinetic | 207966/primary_02/F5.8 | Scatter Plot of Maximum Change from Baseline in Total Bilirubin versus Last Trough CAB PK Concentrations by Strata and Treatment during the Maintenance and Extension Phase | Replace "Maintenance" with<br>"Maintenance and Extension" in<br>the first footnote. | W152 |

| Pharmac | Pharmacokinetic / Pharmacodynamic Figures | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 5.6 | Pharmacokinetic | 207966/primary_02/F5.9 | Scatter Plot of Maximum Change from Baseline in Total Bilirubin versus Last Trough RPV PK Concentrations by Strata and Treatment during the Maintenance and Extension Phase | Replace "Maintenance" with<br>"Maintenance and Extension" in<br>the first footnote. | W152 |
| 5.7 | Pharmacokinetic | 207966/primary_02/F5.13 | Scatter Plot of Change from Baseline in Predose QTcF versus CAB Trough PK Concentration at Week 152 by Treatment | Adjust the alignment of the footnote. | W152 |
| 5.8 | Pharmacokinetic | 207966/primary_02/F5.14 | Scatter Plot of Change from Baseline in Predose QTcF versus RPV Trough PK Concentration at Week 152 by Treatment | Adjust the alignment of the footnote. | W152 |

#### 15.15.6.9. Health Outcomes Tables

| Health ( | Health Outcomes Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Percept | Perception of Injection (PIN) | | | | |
| 6.1 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.1 | Proportion of Subjects with Each Individual Item<br>Score in PIN by Visit - LOCF (Maintenance +<br>Extension Phase) | | W152 |
| 6.2 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.2 | Summary of PIN in Domain Scores (Bother of ISRs, Leg Movement, Sleep and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety after and Willingness) by Visit (Maintenance + Extension Phase) | | W152 |
| 6.3 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.3 | Summary and Statistical Analysis of PIN in Domain Scores (Bother of ISRs, Leg Movement, Sleep and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety after and Willingness) by Visit - LOCF (Maintenance + Extension Phase) | Adjust the first half of the footnote to "[1] Week 24/48/152 was compared with the 1st visit (Week 8) based on Wilcoxon signed-rank test, respectively." | W152 |
| 6.4 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.4 | Summary of PIN Change from Week 8 in Domain<br>Scores (Bother of ISRs, Leg Movement, Sleep and<br>Acceptance) and Individual Items Scores (Anxiety<br>before, Pain, Satisfaction, Anxiety after and<br>Willingness) by Visit (Maintenance + Extension<br>Phase) | | W152 |

| Health C | Health Outcomes Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 6.5 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.5 | Summary of PIN Change from Week 8 in Domain<br>Scores (Bother of ISRs, Leg Movement, Sleep and<br>Acceptance) and Individual Items Scores (Anxiety<br>before, Pain, Satisfaction, Anxiety after and<br>Willingness) by Visit - LOCF (Maintenance +<br>Extension Phase) | | W152 |
| 6.6 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.6 | Statistical Analysis of PIN Change from Week 8 in<br>Domain Scores (Bother of ISRs, Leg Movement,<br>Sleep and Acceptance) and Individual Items<br>Scores (Anxiety before, Pain, Satisfaction, Anxiety<br>after and Willingness) by Visit - LOCF<br>(Maintenance + Extension Phase) | Adjust second the footnote per modelling result. | W152 |
| HIV Trea | atment Satisfa | ction Questionnaire Status V | ersion (HIVTSQs) | | |
| 6.7 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.14 | Proportion of Subjects with HIVTSQs - Individual Item Scores by Visit - LOCF (Maintenance + Extension Phase) | | W152 |
| 6.8 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.15 | Proportion of Subjects with HIVTSQs - Individual Item Scores by Visit and Subgroup - LOCF (Maintenance + Extension Phase) | The subgroup includes: prior exposure to CAB+RPV (0, 1-24, >=24 weeks), sex at birth, age (<35, 35 - <50, >=50), race (white, non-white), Baseline CD4+ cell count (<350, 350 - <500, >=500) | W152 |
| 6.9 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.16 | Summary of HIVTSQs - Total Treatment<br>Satisfaction Score by Visit (Maintenance +<br>Extension Phase) | | W152 |

| Health Outcomes Tables | | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 6.10 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.17 | Summary of HIVTSQs - Total Treatment Satisfaction Score by Visit - LOCF (Maintenance + Extension Phase) | | W152 |
| 6.11 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.18 | Summary of HIVTSQs - Change from Baseline in Total Treatment Satisfaction Score by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit (Maintenance + Extension Phase) | | W152 |
| 6.12 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.19 | Summary of HIVTSQs - Change from Baseline in Total Treatment Satisfaction Score by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit - LOCF (Maintenance + Extension Phase) | | W152 |
| 6.13 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.20 | Summary of HIVTSQs - Change from Baseline in Individual Item Score by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit - LOCF (Maintenance + Extension Phase) | | W152 |
| 6.14 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.21 | Statistical Analysis of HIVTSQs - Change from Baseline in Total Treatment Satisfaction Score by Visit for Subjects without Prior Exposure to CAB+RPV - LOCF (Maintenance + Extension Phase) | Adjust the second footnote based on the modelling result. | W152 |
| 6.15 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.22 | Statistical Analysis of HIVTSQs - Change from Baseline in Total Treatment Satisfaction Score by Visit for Subjects with Prior Exposure to CAB+RPV - LOCF (Maintenance + Extension Phase) | Adjust the second footnote based on the modelling result. | W152 |
| Treatme | ent Acceptance | e (ACCEPT) | | | |

| Health C | Health Outcomes Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 6.16 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.31 | Proportion of Subjects with ACCEPT - Individual Item Score by Visit - LOCF (Maintenance + Extension Phase) | | W152 |
| 6.17 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.32 | Summary of Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit (Maintenance + Extension Phase) | | W152 |
| 6.18 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.33 | Summary of Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit - LOCF (Maintenance + Extension Phase) | | W152 |
| 6.19 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.34 | Summary of Change from Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit (Maintenance + Extension Phase) | | W152 |
| 6.20 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.35 | Summary of Change from Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit - LOCF (Maintenance + Extension Phase) | | W152 |
| 6.21 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.36 | Statistical Analysis of Change from Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit for Subjects without Prior Exposure to CAB+RPV - LOCF (Maintenance + Extension Phase) | Adjust the second footnote based on the modelling result. | W152 |

| Health Outcomes Tables | | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 6.22 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/T6.37 | Statistical Analysis of Change from Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit for Subjects with Prior Exposure to CAB+RPV - LOCF (Maintenance + Extension Phase) | Adjust the second footnote based on the modelling result. | W152 |
| Reason | s for Oral Brid | ging and Preference | | | |
| 6.23 | Oral<br>Bridging | Shell HO_T2 | Proportion of Subjects with Response to Each Individual Question in Reasons for Oral Bridging and Preference Questionnaire at Week 152 (Extension Phase) | | W152 |

## 15.15.6.10. Health Outcomes Figures

| Health C | Health Outcomes Figures | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 6.1 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/F6.1 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in HIVTSQs Total Treatment Satisfaction Score over Time (ANCOVA) for Subjects without Prior Exposure to CAB+RPV - LOCF | | W152 |
| 6.2 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/F6.2 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in HIVTSQs Total Treatment Satisfaction Score over Time (ANCOVA) for Subjects with Prior Exposure to CAB+RPV - LOCF | | W152 |
| 6.3 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/F6.3 | Line Plot of Difference (95% CI) in Adjusted Mean<br>Change from Baseline in HIVTSQs Total Treatment<br>Satisfaction Score over Time (ANCOVA) for Subjects<br>without Prior Exposure to CAB+RPV - LOCF | | W152 |
| 6.4 | Intent-to-<br>Treat<br>Exposed | 207966/primary_02/F6.4 | Line Plot of Difference (95% CI) in Adjusted Mean<br>Change from Baseline in HIVTSQs Total Treatment<br>Satisfaction Score over Time (ANCOVA) for Subjects with<br>Prior Exposure to CAB+RPV - LOCF | | W152 |

## 15.15.6.11. Virology Tables

| Virology | Virology Tables | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Genoty | ре | | | | |
| 7.1 | Confirmed<br>Virologic<br>Failure | 207966/primary_15/T7.1 | Summary of the Prevalence of Known INI Resistance<br>Mutations at time of CVF (Maintenance + Extension<br>Phase) – Plasma Sample | | W152 |
| 7.2 | Confirmed<br>Virologic<br>Failure | 207966/primary_15/T7.2 | Summary of the Prevalence of Major Resistance<br>Mutations of NRTI, NNRTI and PI Class at time of CVF<br>(Maintenance + Extension Phase) - Plasma Sample | | W152 |
| 7.3 | Confirmed<br>Virologic<br>Failure | 207966/primary_15/T7.3 | Summary of Genotypic Susceptibility at time of CVF (Maintenance + Extension Phase) - Plasma Sample | | W152 |
| Phenoty | /pe | | | | |
| 7.4 | Confirmed<br>Virologic<br>Failure | 207966/primary_15/T7.4 | Summary of Phenotype Susceptibility at time of CVF (Maintenance + Extension Phase) - Plasma Sample | | W152 |
| 7.5 | Confirmed<br>Virologic<br>Failure | 207966/primary_15/T7.5 | Summary of Phenotype: Number of Drugs to Which<br>Subject is Phenotypic Resistant or Partial Sensitive or<br>Sensitive at Time of CVF (Maintenance + Extension<br>Phase) - Plasma Sample | | W152 |
| 7.6 | Confirmed<br>Virologic<br>Failure | 207966/primary_15/T7.6 | Summary of Fold Change to CAB and RPV at Time of CVF (Maintenance + Extension Phase) - Plasma Sample | | W152 |
| 7.7 | Confirmed<br>Virologic<br>Failure | 207966/primary_15/T7.7 | Summary of Net Assessment at time of CVF (Maintenance + Extension Phase) - Plasma Sample | | W152 |

| Virology Tables | | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Other | | | | | |
| 7.8 | Confirmed<br>Virologic<br>Failure | 207966/primary_15/T7.9 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria during the Maintenance and Extension Phase | | W152 |
| 7.9 | Safety | 207966/primary_15/T7.10 | Summary of Viral load, Genotypic and Phenotypic data for Non-CVF Subjects with Genotypic and/or Phenotypic Data | | W152 |

#### 15.15.6.12. ICH Listings

**Note:** Unless otherwise specified, both unique subject ID and latest subject ID for a subject will be included in the listings; display by prior exposure to CAB+RPV (0, 1-24, >24 weeks, refer to Section 15.6.2 for calculation details) for all listings except for study population listings.

| ICH List | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Study P | opulation | | | | |
| 1 | Intent-to-Treat<br>Exposed | 207966/primary_15/L4 | Listing of Reasons for Study<br>Withdrawal | | W152 |
| 2 | Intent-to-Treat<br>Exposed | 207966/primary_15/L5 | Listing of Reasons for Study Drug Discontinuation | | W152 |
| 3 | Intent-to-Treat<br>Exposed | 207966/primary_15/L6 | Listing of Important Protocol Deviations | | W152 |
| 4 | Intent-to-Treat<br>Exposed | 207966/primary_15/L7 | Listing of Protocol Deviations<br>Leading to Exclusion from the Per-<br>Protocol Population | | W152 |
| 5 | Intent-to-Treat<br>Exposed | 207966/primary_15/L9 | Listing of Demographic Characteristics | | W152 |
| 6 | Intent-to-Treat<br>Exposed | 207966/primary_15/L10 | Listing of Race | | W152 |
| 7 | Intent-to-Treat<br>Exposed | 207966/primary_15/L8 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | W152 |
| Efficacy | | | | | |
| 8 | Intent-to-Treat<br>Exposed | 207966/primary_15/L11 | Listing of Study Outcome (50 c/mL<br>Threshold) at Week 152 – Snapshot | Update the footnote per given data. | W152 |

| ICH List | ings | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | Analysis | | |
| Safety | | | | | |
| 9 | Safety | 207966/primary_15/L12 | Listing of Investigational Product Exposure Data | | W152 |
| 10 | Safety | 207966/primary_15/L13 | Listing of Subject Numbers for Individual Adverse Events | | W152 |
| 11 | Safety | 207966/primary_15/L14 | Listing of Reasons for Considering as a Serious Adverse Event | | W152 |
| 12 | Safety | 207966/primary_15/L15 | Listing of Fatal Adverse Events | | W152 |
| 13 | Safety | 207966/primary_15/L16 | Listing of Non-Fatal Serious Adverse Events | | W152 |
| 14 | Safety | 207966/primary_15/L17 | Listing of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product (Maintenance + Extension Phase) | | W152 |
| 15 | Safety | 207966/primary_15/L18 | Listing of Changes in<br>Intensity/Grades of Study Drug<br>Injection Site Adverse Events | | W152 |
| 16 | Safety | 207966/primary_15/L19 | Listing of All Adverse Events | | W152 |
| 17 | Safety | 207966/primary_15/L66 | Listing of COVID-19 Adverse Events | | W152 |
| 18 | Safety | 207966/primary_15/L67 | Listing of COVID-19 Assessments | | W152 |
| 19 | Safety | 207966/primary_15/L68 | Listing of COVID-19 Symptoms | | W152 |
| 20 | Safety | 207966/primary_15/L20 | Listing of Subjects Who Became Pregnant during the Study | | W152 |

| ICH List | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 21 | Safety | 207966/primary_15/L21 | Listing of Medical Conditions for<br>Subjects with Liver stopping Events | | W152 |
| 22 | Safety | 207966/primary_15/L22 | Listing of Substance Use for<br>Subjects with Liver Stopping Events | | W152 |
| 23 | Safety | 207966/primary_15/L23 | Listing of ECG Values for Subjects with a Value of Potential Clinical Importance | | W152 |
| 24 | Safety | 207966/primary_15/L24 | Listing of ECG Findings | | W152 |
| PK | | | | | |
| 25 | Pharmacokinetic | 207966/primary_15/L29 | Listing of Plasma CAB PK<br>Concentration-Time Data | | W152 |
| 26 | Pharmacokinetic | 207966/primary_15/L30 | Listing of Plasma RPV PK<br>Concentration-Time Data | | W152 |

#### 15.15.6.13. Non-ICH Listings

**Note:** Unless otherwise specified, both unique subject ID and latest subject ID for a subject will be included in the listings; display by prior exposure to CAB+RPV (0, 1-24, >24 weeks, refer to calculation details in Section 15.6.2) for all listings except for study population listings.

| Non-ICH | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Study P | opulation | | | | |
| 27 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/L33 | Listing of Reasons for Extension Phase Withdrawal | | W152 |
| 28 | Long-term<br>Follow-up | 207966/primary_15/L34 | Listing of Reasons for Long-term Follow-up Phase Withdrawal | | W152 |
| 29 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/L36 | Listing of Prior ART Medications | | W152 |
| 30 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/L37 | Listing of Concomitant ART Medications | In case the same medication is concomitant during both maintenance and extension phases, list each of them in two separate rows. | W152 |
| 31 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/L38 | Listing of ART Medications Received during Long-<br>term Follow-up Phase | | W152 |
| 32 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/L39 | Listing of Investigational Product Accountability - Oral Regimens | | W152 |
| 33 | Intent-to- | 207966/primary_15/L6 | Listing of Non-important COVID-19 Related | Remove the column, "COVID-19 | W152 |

| Non-ICH | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | Treat<br>Exposed | | Protocol Deviations | Related". | |
| 34 | Intent-to-<br>Treat<br>Exposed | PAN5A | Country Level Listing of Dates of Waves of COVID-<br>19 Pandemic Measures | Only include countries that are applicable to the study. The covidimt dataset from arenv/arcomn/covid uses the IMT alerts to determine when pandemic measures began. Use this dataset as source to obtain the start and end dates of pandemic measures. Follow the instructions available in the same location for appropriate data use. | W152 |
| Efficacy | 1 | | | | |
| 35 | Confirmed<br>Virologic<br>Failure | 207966/primary_15/L41 | Listing of All Plasma HIV-1 RNA Data for Subjects with Confirmed Virologic Failure | | W152 |
| 36 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/L42 | Listing of All Plasma HIV-1 RNA Data for Subjects with Viral load >=50 c/mL during the Maintenance and Extension Phase | | W152 |
| 37 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/L64 | Listing of All Plasma HIV-1 RNA Data | | W152 |
| 38 | Intent-to-<br>Treat<br>Exposed | 207966/primary_15/L43 | Listing of HIV-1 Associated Conditions | | W152 |
| Safety | | | | | |
| 39 | Safety | 207966/primary_15/L52 | Listing of Liver Stopping Event Reporting | | W152 |

| Non-ICH | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 40 | Safety | 207966/primary_15/L53 | Listing of Liver Event Information for RUCAM Score | | W152 |
| 41 | Safety | 207966/primary_15/L54 | Listing of Liver Biopsy Details | | W152 |
| 42 | Safety | 207966/primary_15/L55 | Listing of Liver Imaging Details | | W152 |
| 43 | Safety | 207966/primary_15/L56 | Listing of Subjects Meeting Hepatobiliary Lab<br>Criteria | Only Maintenance and Extension phases are included. | W152 |
| 44 | Safety | 207966/primary_15/L57 | Listing of Potential QTc Interval Prolonging Events of Interest | | W152 |
| 45 | Safety | 207966/primary_15/L58 | Listing of ECG values for Subjects with Potential QTc Interval Prolonging Events of Interest | | W152 |
| 46 | Safety | 207966/primary_15/L59 | Listing of ALT, AST, Bilirubin (including Total and Direct Bilirubin), INR, and ALP for Subjects Meeting Hepatobiliary Lab Abnormality Criteria | | W152 |
| 47 | Safety | 207966/primary_15/L61 | Listing of Dosing Errors and IP Device Malfunctions | | W152 |
| 48 | Safety | SAF_L3 | Listing of Selected Study Treatment Data for Subjects Who Had Planned Reloading Injections | | W152 |
| Virology | / | | | | |
| 49 | Confirmed<br>Virologic<br>Failure | 207966/primary_15/L62 | Listing of Replication Capacity in IN and PR/RT Region | | W152 |
| 50 | Safety | 207966/primary_15/L63 | Listing of Resistance Associated Mutations (Prespecified INSTI and IAS-USA NNRTI) | | W152 |
| PK | | | | | |
| 51 | Long-term<br>Follow-up | 207966/primary_02/L63 | Listing of Plasma PK Concentration-Time Data since Last Injection | Remove age and add "Start Date of Oral RPV after Last Injection" after "Baseline BMI (kg/m^2)" in the | W152 |

| Non-ICH | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. in<br>W152 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | | second column from the left; add asterisk to RPV concentration taken on/after the start of such oral RPV. and add a footnote, "Note: the RPV concentrations marked with an asterisk were taken on/after the start date of the oral RPV." | |

#### 15.15.7. List of Data Displays for Sub-study Analysis

Unless otherwise specified, in sub-study analysis, age refers to the age at the sub-study screening, Baseline weight and Baseline BMI refer to the weight and BMI at the sub-study baseline respectively, and the listings will not be presented by prior exposure to CAB + RPV as the shell.

#### 15.15.7.1. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Subje | ct Disposition | | | | |
| 1.1 | Sub-study ITT-E | 207966/primary_34/T1.1 | Summary of Number of Sub-study<br>Subjects Enrolled by Country and Site ID | | Sub-study |
| 1.2 | Sub-study<br>Screened | 207966/primary_15/T1.2 | Summary of Screening Status and Reasons for Sub-study Screening Failures | | Sub-study |
| 1.3 | Sub-study ITT-E | 207966/primary_34/T1.2 | Summary of Subject Accountability: Substudy Conclusion Record | Remove the first footnote. Re-number the footnotes and the corresponding numbers in the display. | Sub-study |
| 1.4 | Sub-study ITT-E | 207966/primary_34/T1.3 | Summary of Subject Accountability: Thigh Injection Phase Conclusion Record | | Sub-study |
| 1.5 | Sub-study ITT-E | 207966/primary_34/T1.3 | Summary of Subject Accountability:<br>Return to Gluteal Injection Phase<br>Conclusion Record | | Sub-study |
| 1.6 | Sub-study ITT-E | 207966/primary_34/T1.6 | Summary of Subject Disposition at Each Study Phase | Present following phases in order: Thigh Injection Phase, Extension Phase (after withdrawal from the Thigh Injection phase), Long-term Follow-up Phase (after withdrawal from the Thigh Injection phase), Return to Gluteal Injection Phase, | Sub-study |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | | Extension Phase (after withdrawal from the Return to Gluteal Injection phase or substudy completion), Long-term Follow-up Phase (after withdrawal from the Return to Gluteal Injection phase or sub-study completion). | |
| 1.7 | Sub-study ITT-E | 207966/primary_34/T1.9 | Summary of Study Drug Discontinuation | | Sub-study |
| 1.8 | Sub-study<br>Screened | 207966/primary_34/T1.10 | Summary of Study Populations | Only include analysis populations used in the sub-study analysis. | Sub-study |
| 1.9 | Sub-study ITT-E | 207966/primary_34/T1.11 | Summary of Important Protocol Deviations in Sub-study | | Sub-study |
| 1.10 | Sub-study ITT-E | 207966/primary_34/T1.11 | Summary of Important Protocol Deviations (Thigh Injection Phase) | | Sub-study |
| 1.11 | Sub-study ITT-E | 207966/primary_15/T1.13 | Summary of Inclusion/Exclusion Criteria Deviations in Sub-study | | Sub-study |
| 1.12 | Sub-study ITT-E | 207966/primary_34/T1.14 | Summary of Important COVID-19 Related Protocol Deviations in Sub-study | | Sub-study |
| 1.13 | Sub-study ITT-E | 207966/primary_34/T1.15 | Summary of Important Non-COVID-19<br>Related Protocol Deviations in Sub-study | | Sub-study |
| Demo | graphic and Baseli | ine Characteristics | | | |
| 1.14 | Sub-study ITT-E | 207966/primary_34/T1.16 | Summary of Demographic Characteristics | Add [1] after "Age (y)" and "Age group (y)"; add the footnote "[1] Age is calculated with respect to the first sub-study screening visit."; for Weight and BMI, change the label to be "Weight (kg) at Sub-study Baseline" and "BMI (kg/m^2) at Sub-study Baseline" respectively. | Sub-study |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 1.15 | Sub-study ITT-E | 207966/primary_34/T1.17 | Summary of Race and Racial Combinations | | Sub-study |
| 1.16 | Sub-study ITT-E | 207966/primary_34/T1.18 | Summary of Race and Racial Combinations Details | | Sub-study |
| Medic | ations and Smokin | g Status | | | |
| 1.17 | Sub-study ITT-E | Shell POP_T2 | Summary of Extent of Exposure to Study<br>Treatment including SOC Oral Bridging<br>Prior to the First Thigh Injection | | Sub-study |
| 1.18 | Sub-study ITT-E | 207966/primary_34/T1.24 | Summary of Concomitant Non-ART<br>Medication Ingredient Combinations<br>(Thigh Injection Phase) | | Sub-study |
| 1.19 | Sub-study ITT-E | SU1 | Summary of Smoking Status at Sub-study Baseline | Only include "History of smoking use" section. | Sub-study |
| Visits | Visits Impacted by COVID-19 Pandemic | | | | |
| 1.20 | Sub-study ITT-E | 207966/primary_34/T1.27 | Summary of COVID-19 Pandemic Visit Impacts in Sub-study | Only include visits in sub-study. Remove the last footnote. | Sub-study |

#### 15.15.7.2. Efficacy Tables

Note: The following subgroups will be included in the subgroup analysis: Age (<50 vs >=50), Race (White vs Non-white), Sex at Birth (Female vs Male), Sub-study Baseline BMI (<30, >=30).

| Efficac | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.1 | Sub-study ITT-E | 207966/primary_34/T2.3 | Summary of Study Outcomes (50 c/mL Threshold) at Sub-study Week 16 – Snapshot Analysis | | Sub-study |
| 2.2 | Sub-study ITT-E | 207966/primary_34/T2.7 | Summary of Study Outcomes (50 c/mL Threshold) at Sub-study Week 16 by Subgroup – Snapshot Analysis | | Sub-study |
| 2.3 | Sub-study ITT-E | 207966/primary_34/T2.13 | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Visit (Thigh Injection Phase) – Snapshot Analysis | | Sub-study |
| 2.4 | Sub-study ITT-E | 207966/primary_34/T2.14 | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Subgroup and Visit (Thigh Injection Phase) – Snapshot Analysis | | Sub-study |
| 2.5 | Sub-study ITT-E | 207966/primary_34/T2.15 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit (Thigh Injection Phase) – Snapshot Analysis | | Sub-study |
| 2.6 | Sub-study ITT-E | 207966/primary_34/T2.16 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Subgroup and Visit (Thigh Injection Phase) – Snapshot Analysis | | Sub-study |
| 2.7 | Sub-study ITT-E | 207966/primary_34/T2.23 | Summary of Change from Sub-study Baseline in Plasma HIV-1 RNA (log10 c/mL) by Visit (Thigh Injection + Return to Gluteal Injection Phase) | | Sub-study |
| 2.8 | Sub-study ITT-E | 207966/primary_34/T2.24 | Summary of Plasma HIV-1 RNA (log10 c/mL) by Visit (Thigh Injection + Return to Gluteal Injection Phase) | | Sub-study |

| Efficac | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.9 | Sub-study ITT-E | 207966/primary_34/T2.25 | Cumulative Proportion of Subjects Meeting Confirmed Virology Failure Criteria by Visit (Thigh Injection + Return to Gluteal Injection Phase) | | Sub-study |
| 2.10 | Sub-study CVF | 207966/primary_34/T2.27 | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmation of Confirmed Virologic Failure (Thigh Injection + Return to Gluteal Injection Phase) | Produce only when data available for the population of interest. | Sub-study |
| 2.11 | Sub-study ITT-E | 207966/primary_34/T2.29 | Summary of Subjects per Viral Load Category by Visit (Thigh Injection Phase) | | Sub-study |
| 2.12 | Sub-study ITT-E | 207966/primary_34/T2.30 | Summary of Change from Sub-study Baseline in CD4+<br>Cell Count (cells/mm^3) by Visit (Thigh Injection +<br>Return to Gluteal Injection Phase) | | Sub-study |
| 2.13 | Sub-study ITT-E | 207966/primary_34/T2.31 | Summary of Change from Sub-study Baseline in CD4+<br>Cell Count (cells/mm^3) at Sub-study Week 16 by<br>Subgroup | Replace "Baseline" with "Substudy baseline" in the footnote. | |
| 2.14 | Sub-study ITT-E | 207966/primary_34/T2.32 | Summary of CD4+ Cell Count (cells/mm^3) by Visit (Thigh Injection + Return to Gluteal Injection Phase) | | Sub-study |
| 2.15 | Sub-study ITT-E | 207966/primary_34/T2.33 | Summary of Change from Sub-study Baseline in CD8+Cell Count (cells/mm^3) by Visit (Thigh Injection Phase) | Replace "Baseline" with "Substudy baseline" in the footnote. | Sub-study |
| 2.16 | Sub-study ITT-E | 207966/primary_34/T2.34 | Summary of CD8+ Cell Count (cells/mm^3) by Visit (Thigh Injection Phase) | | Sub-study |
| 2.17 | Sub-study ITT-E | 207966/primary_34/T2.35 | Summary of CD4+/CD8+ Ratio Cell Count (cells/mm^3) by Visit (Thigh Injection Phase) | | Sub-study |
| 2.18 | Sub-study ITT-E | 207966/primary_34/T2.36 | Summary of HIV-1 Associated Conditions Including Recurrences (Thigh Injection + Return to Gluteal Injection Phase) | Produce only when data available for the population of interest. | Sub-study |

| Efficac | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.19 | Sub-study ITT-E | 207966/primary_34/T2.37 | Summary of HIV-1 Associated Conditions Excluding<br>Recurrences (Thigh Injection + Return to Gluteal<br>Injection Phase) | Produce only when data available for the population of interest. | Sub-study |
| 2.20 | Sub-study ITT-E | 207966/primary_34/T2.38 | Summary of HIV-1 Disease Progression from Sub-study Baseline and/or Deaths (Thigh Injection + Return to Gluteal Injection Phase) | Replace "maintenance and extension phase" in the second footnote with "thigh injection or return to gluteal injection phase". | Sub-study |

## 15.15.7.3. Efficacy Figures

| Efficac | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.1 | Sub-study ITT-E | 207966/primary_34/F2.1 | Proportion (95% CI) of Subjects with HIV-1 RNA ≥50 c/mL by Visit (Thigh Injection Phase) – Snapshot Analysis | | Sub-study |
| 2.2 | Sub-study ITT-E | 207966/primary_34/F2.3 | Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL by Visit (Thigh Injection Phase) – Snapshot Analysis | | Sub-study |
| 2.3 | Sub-study CVF | 207966/primary_34/F2.7 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit – for CVF Subjects | Produce only when data available for the population of interest. Replace the first footnote with "First vertical reference line corresponds to the date of first thigh injection." | Sub-study |
| 2.4 | Sub-study ITT-E | 207966/primary_34/F2.8 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit for subjects Who are in the Category of 'HIV-1 RNA >=50 c/mL' at Sub-study Week 16 per Snapshot Algorithm | Produce only when data available for the population of interest. Replace the first footnote with "First vertical reference line corresponds to the date of first thigh injection." | Sub-study |

# 15.15.7.4. Safety Tables

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Expos | ure | | | | |
| 3.1 | Sub-study<br>Safety | 207966/primary_34/T3.1 | Summary of Extent of Exposure to Study<br>Treatment (Thigh Injection + Return to Gluteal<br>Injection Phase) | Include both continuous and categorical summaries for Exposure (No. of Thigh Injection Visits), Exposure (No. of Return to Gluteal Injection Visits), Exposure (No. of Injection Visits), Overall Exposure to Study Treatment during the Thigh Injection Phase, Overall Exposure to Study Treatment during the Thigh Injection + Return to Gluteal Injection Phase. The levels for categorical summaries will be selected as appropriate. Remove the footnote. | Sub-study |
| 3.2 | Sub-study<br>Safety | 207966/primary_34/T3.2 | Summary of Needle Length and Gauge for CAB Injection (Thigh Injection Phase) | Replace the "at Maintenance + Extension Phase" in footnote with "during the Thigh Injection phase". | Sub-study |
| 3.3 | Sub-study<br>Safety | 207966/primary_34/T3.3 | Summary of Needle Length and Gauge for RPV Injection (Thigh Injection Phase) | Replace the "at Maintenance + Extension Phase" in footnote with "during the Thigh Injection phase". | Sub-study |
| 3.4 | Sub-study<br>Safety | 207966/primary_34/T3.4 | Summary of Adherence to CAB/RPV Injection Dosing Schedule (Thigh Injection Phase) | Remove the missed Injection related rows from shell. Add "Missed Injection" row. Replace the footnote with "[1] The total number of expected thigh injection visits following the first thigh injection." Add a footnote "Note: Oral bridging is not allowed in the sub-study.". | Sub-study |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.5 | Sub-study<br>Safety | 207966/primary_34/T3.4 | Summary of Adherence to CAB/RPV Injection<br>Dosing Schedule (Thigh Injection + Return to<br>Gluteal Injection Phase) | Remove the missed Injection related rows from shell. Add "Missed Injection" row. Replace the footnote with "[1] The total number of expected injection visits in sub-study following the first thigh injection." Add a footnote "Note: Oral bridging is not allowed in the substudy.". | Sub-study |
| Advers | se Events | | | | • |
| 3.6 | Sub-study<br>Safety | 207966/primary_34/T3.6 | Summary of All Adverse Events by System<br>Organ Class and Maximum Toxicity (Thigh<br>Injection Phase) | | Sub-study |
| 3.7 | Sub-study<br>Safety | 207966/primary_34/T3.6 | Summary of All Adverse Events by System<br>Organ Class and Maximum Toxicity (Thigh<br>Injection + Return to Gluteal Injection Phase) | | Sub-study |
| 3.8 | Sub-study<br>Safety | 207966/primary_34/T3.8 | Summary of All Adverse Events Excluding<br>Study Drug Injection Site Reactions by System<br>Organ Class and Maximum Toxicity (Thigh<br>Injection Phase) | | Sub-study |
| 3.9 | Sub-study<br>Safety | 207966/primary_34/T3.10 | Summary of Common Adverse Events (>=5%) by Overall Frequency (Thigh Injection Phase) | | Sub-study |
| 3.10 | Sub-study<br>Safety | 207966/primary_34/T3.11 | Summary of Common Grade 2-5 Adverse<br>Events (>=1%) by Overall Frequency (Thigh<br>Injection Phase) | | Sub-study |
| 3.11 | Sub-study<br>Safety | 207966/primary_34/T3.13 | Summary of All Drug-related Adverse Events<br>by System Organ Class and Maximum Toxicity<br>(Thigh Injection Phase) | | Sub-study |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.12 | Sub-study<br>Safety | 207966/primary_34/T3.15 | Summary of All Drug-related Adverse Events<br>Excluding Study Drug Injection Site Reactions<br>by System Organ Class and Maximum Toxicity<br>(Thigh Injection Phase) | | Sub-study |
| 3.13 | Sub-study<br>Safety | 207966/primary_34/T3.16 | Summary of All Drug-Related Grade 2-5<br>Adverse Events by Overall Frequency (Thigh<br>Injection Phase) | | Sub-study |
| Seriou | s and Other Sigi | nificant Adverse Events | | | |
| 3.14 | Sub-study<br>Safety | 207966/primary_34/T3.17 | Summary of Serious Adverse Events by<br>System Organ Class (Thigh Injection Phase) | | Sub-study |
| 3.15 | Sub-study<br>Safety | 207966/primary_34/T3.17 | Summary of Serious Adverse Events by<br>System Organ Class (Thigh Injection +Return<br>to Gluteal Injection Phase) | | Sub-study |
| 3.16 | Sub-study<br>Safety | 207966/primary_34/T3.19 | Summary of Drug-related Serious Adverse<br>Events by System Organ Class (Thigh<br>Injection Phase) | | Sub-study |
| 3.17 | Sub-study<br>Safety | 207966/primary_34/T3.22 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product or Withdrawal from Study by System Organ Class (Thigh Injection Phase) | Remove the footnote. | Sub-study |
| 3.18 | Sub-study<br>Safety | 207966/primary_34/T3.22 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class (Thigh Injection + Return to Gluteal Injection Phase) | Remove the footnote. | Sub-study |
| 3.19 | Sub-study | 207966/primary_34/T3.25 | Summary of Subjects and Number of | | Sub-study |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | Safety | | Occurrences of Common (>=5%) Non-Serious<br>Adverse Events by System Organ Class<br>(Thigh Injection Phase) | | |
| 3.20 | Sub-study<br>Safety | 207966/primary_34/T3.26 | Summary of Subjects and Number of occurrences of SAEs, Fatal SAEs, and Drugrelated SAEs (Thigh Injection Phase) | | Sub-study |
| Study | Drug Injection S | ite Reaction Adverse Events | | | |
| 3.21 | Sub-study<br>Safety | 207966/primary_34/T3.27 | Summary of Study Drug Injection Site<br>Reaction Adverse Events (Event-level<br>Summary) – (Thigh Injection Phase) | | Sub-study |
| 3.22 | Sub-study<br>Safety | 207966/primary_34/T3.28 | Summary of Subject-level Characteristics of<br>Study Drug Injection Site Reaction Adverse<br>Events – Overall and Common (Thigh Injection<br>Phase) | | Sub-study |
| 3.23 | Sub-study<br>Safety | 207966/primary_34/T3.29 | Summary of Study Drug Injection Site<br>Reaction Adverse Events by Visit and<br>Maximum Severity – Overall and Common in<br>Sub-study | | Sub-study |
| 3.24 | Sub-study<br>Safety | 207966/primary_34/T3.30 | Summary of Drug-related Study Drug Injection<br>Site Reaction Adverse Events (Event-level<br>Summary) - CAB (Thigh Injection Phase) | | Sub-study |
| 3.25 | Sub-study<br>Safety | 207966/primary_34/T3.31 | Summary of Drug-related Subject-level<br>Characteristics of Study Drug Injection Site<br>Reaction Adverse Events (Thigh Injection<br>Phase) - Overall and Common (CAB) | | Sub-study |
| 3.26 | Sub-study<br>Safety | 207966/primary_34/T3.32 | Summary of Overall and Common Drug-<br>related Study Drug Injection Site Reaction | | Sub-study |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | Adverse Events by Visit and Maximum<br>Severity in Sub-study - CAB | | |
| 3.27 | Sub-study<br>Safety | 207966/primary_34/T3.33 | Summary of Maximum Drug-related Study<br>Drug Injection Site Reaction Adverse Event<br>Grade by Needle Length (Thigh Injection<br>Phase) – Common (CAB) | Replace "Mnt + Ext" with "Thigh Injection" in the footnote. | Sub-study |
| 3.28 | Sub-study<br>Safety | 207966/primary_34/T3.34 | Summary of Drug-related Study Drug Injection<br>Site Reaction Adverse Events (Event-level<br>Summary) - RPV (Thigh Injection Phase) | | Sub-study |
| 3.29 | Sub-study<br>Safety | 207966/primary_34/T3.35 | Summary of Drug-related Subject-level<br>Characteristics of Study Drug Injection Site<br>Reaction Adverse Events (Thigh Injection<br>Phase) - Overall and Common (RPV) | | Sub-study |
| 3.30 | Sub-study<br>Safety | 207966/primary_34/T3.36 | Summary of Overall and Common Drug-<br>related Study Drug Injection Site Reaction<br>Adverse Events by Visit and Maximum<br>Severity in Sub-study - RPV | | Sub-study |
| 3.31 | Sub-study<br>Safety | 207966/primary_34/T3.37 | Summary of Maximum Drug-related Study<br>Drug Injection Site Reaction Adverse Event<br>Grade by Needle Length (Thigh Injection<br>Phase) – Common (RPV) | Replace "Mnt + Ext" with "Thigh Injection" in the footnote. | Sub-study |
| Labora | atory: Chemistry | and Hematology | | | |
| 3.32 | Sub-study<br>Safety | 207966/primary_34/T3.38 | Summary of Chemistry Changes from Substudy Baseline by Visit (Thigh Injection + Return to Gluteal Injection Phase) | | Sub-study |
| 3.33 | Sub-study<br>Safety | 207966/primary_34/T3.39 | Summary of Chemistry Values by Visit (Thigh Injection + Return to Gluteal Injection Phase) | | Sub-study |
| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.34 | Sub-study<br>Safety | 207966/primary_34/T3.40 | Summary of Hematology Changes from Substudy Baseline by Visit (Thigh Injection + Return to Gluteal Injection Phase) | | Sub-study |
| 3.35 | Sub-study<br>Safety | 207966/primary_34/T3.41 | Summary of Hematology Values by Visit (Thigh Injection + Return to Gluteal Injection Phase) | | Sub-study |
| 3.36 | Sub-study<br>Safety | 207966/primary_34/T3.42 | Summary of Maximum Post Sub-study<br>Baseline Emergent Chemistry Toxicities (Thigh<br>Injection Phase) | Add "sub-study" before "baseline" in the second footnote. | Sub-study |
| 3.37 | Sub-study<br>Safety | 207966/primary_34/T3.43 | Summary of Maximum Post Sub-study<br>Baseline Emergent Hematology Toxicities<br>(Thigh Injection Phase) | Add "sub-study" before "baseline" in the footnote. | Sub-study |
| Labora | tory: Urinalysis | | | | |
| 3.38 | Sub-study<br>Safety | 207966/primary_34/T3.44 | Summary of Urinalysis Dipstick Results by Visit (Thigh Injection Phase) | | Sub-study |
| 3.39 | Sub-study<br>Safety | 207966/primary_34/T3.45 | Summary of Urine Concentrations Changes from Sub-study Baseline by Visit (Thigh Injection Phase) | Add "sub-study" before "baseline" in the second footnote. | Sub-study |
| 3.40 | Sub-study<br>Safety | 207966/primary_34/T3.46 | Summary of Changes in Proteinuria Baseline<br>Laboratory Result to Maximum Post Sub-study<br>Baseline Laboratory Result (Thigh Injection<br>Phase) | | Sub-study |
| Labora | tory: Hepatobili | ary (Liver) | | | |
| 3.41 | Sub-study<br>Safety | 207966/primary_34/T3.53 | Summary of Liver Stopping Event Reporting (Thigh Injection Phase) | | Sub-study |
| 3.42 | Sub-study | 207966/primary_34/T3.54 | Summary of Subjects Meeting Hepatobiliary | | Sub-study |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | Safety | | Abnormality Criteria (Thigh Injection Phase) | | |
| ECG | | | | | |
| 3.43 | Sub-study<br>Safety | 207966/primary_34/T3.55 | Summary of ECG Findings (Thigh Injection Phase) | | Sub-study |
| 3.44 | Sub-study<br>Safety | 207966/primary_34/T3.56 | Summary of Change from Sub-study Baseline in ECG values by Visit (Thigh Injection Phase) | Add "sub-study" before "baseline" in the first footnote. | Sub-study |
| 3.45 | Sub-study<br>Safety | 207966/primary_34/T3.57 | Summary of QTc Values by Category (Thigh Injection Phase) | | Sub-study |
| 3.46 | Sub-study<br>Safety | 207966/primary_34/T3.58 | Summary of Change from Sub-study Baseline QTc Values by Category (Thigh Injection Phase) | | Sub-study |
| Vital S | igns | | | | |
| 3.47 | Sub-study<br>Safety | 207966/primary_34/T3.59 | Summary of Change from Sub-study Baseline in Vital Signs by Visit (Thigh Injection Phase) | Add "sub-study" before "baseline" in the first footnote. | Sub-study |
| Advers | se Event of Spec | ial Interest (AESI) | | | |
| 3.48 | Sub-study<br>Safety | 207966/primary_34/T3.63 | Summary of Depression, Anxiety and Suicidal Ideation/Behaviour Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and Prior History of Depression, Anxiety and Suicidal Ideation at Screening (Thigh Injection Phase) | May need to adjust the first footnote given the data. Add a footnote: "Note: The prior history of depression, anxiety and suicidal ideation was collected at the main study screening". | Sub-study |
| 3.49-<br>3.66 | Sub-study<br>Safety | 207966/primary_34/T3.64-<br>3.80 | Summary of XXX Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrence) – Thigh Injection Phase | | Sub-study |
| 3.67 | Sub-study | 207966/primary_34/T3.81 | Summary of Characteristics of Common | | Sub-study |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | Safety | | Adverse Events of Special Interest – Thigh Injection Phase | | |
| COVID | )-19 Adverse Eve | ent | | | |
| 3.68 | Sub-study<br>Safety | 207966/primary_34/T3.84 | Summary of COVID-19 Adverse Events by<br>System Organ Class and Maximum Toxicity<br>(Thigh Injection Phase) | | Sub-study |
| 3.69 | Sub-study<br>Safety | PAN1A | Summary of COVID-19 Assessments for<br>Subjects with Suspected, Probable or<br>Confirmed COVID-19 Case Diagnosis in Sub-<br>study | Replace the first footnote with "[1] COVID-19 case diagnosis is based on WHO definition that was in effect at the time of diagnosis.". Add a footnote "Note: only the assessments with the associated COVID-19 adverse event (as recorded in the COVID-19 Coronavirus Infection Assessment eCRF form) started in the sub-study are included.". | Sub-study |
| 3.70 | Sub-study<br>Safety | PAN2A | Summary of COVID-19 Additional<br>Assessments for Subjects with Suspected,<br>Probable or Confirmed COVID-19 Case<br>Diagnosis in Sub-study | Add a footnote "Note: only the assessments with the associated COVID-19 adverse event (as recorded in the COVID-19 Coronavirus Infection Assessment eCRF form) started in the sub-study are included.". | Sub-study |

# 15.15.7.5. Safety Figures

| Safety F | Safety Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.1 | Sub-study<br>Safety | 213500/primary_03/F3.2 | Plot of Incidence of Sub-study Study Drug Injection Site<br>Reaction Adverse Events by Visit (Overall and<br>Common) | Within each page, display CAB<br>LA and/or RPV LA, CAB LA-<br>Drug- Related, RPV LA-Drug-<br>Related | Sub-study |
| 3.2 | Sub-study<br>Safety | 207966/primary_34/F3.7 | Scatter Plot of Maximum vs. Sub-study Baseline for ALT (Thigh Injection Phase) | Add "Sub-study" to the front of "Baseline" in the x axis label. | Sub-study |
| 3.3 | Sub-study<br>Safety | 207966/primary_34/F3.8 | Scatter Plot of Maximum Total Bilirubin vs. Maximum ALT (Thigh Injection Phase) | | Sub-study |
| 3.4 | Sub-study<br>Safety | 207966/primary_34/F3.11 | Histogram of Timeliness of Injections (Thigh Injection Phase) | | Sub-study |

#### 15.15.7.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.1 | Sub-study PK<br>Concentration | 207966/primary_34/T4.1 | Summary of Plasma CAB PK Concentration (ug/mL) - Time Data by Treatment and Visit in Sub-study - Including Log-transformed Statistics | Remove the last two footnotes. | Sub-study |
| 4.2 | Sub-study PK<br>Concentration | 207966/primary_34/T4.2 | Summary of Plasma RPV PK Concentration (ng/mL) -<br>Time Data by Treatment and Visit in Sub-study -<br>Including Log-transformed Statistics | Remove the last two footnotes. | Sub-study |
| 4.3 | Sub-study PK<br>Concentration | 207966/primary_34/T4.3 | Summary of Evaluable Plasma CAB PK Concentration (ug/mL) - Time Data by Treatment and Visit in Sub-study - Including Log-transformed Statistics | Remove the last footnote. | Sub-study |
| 4.4 | Sub-study PK<br>Concentration | 207966/primary_34/T4.4 | Summary of Evaluable Plasma RPV PK Concentration (ng/mL) - Time Data by Treatment and Visit in Sub-study - Including Log-transformed Statistics | Remove the last footnote. | Sub-study |
| 4.5 | Sub-study PK<br>Parameter | PK06 | Summary of Plasma CAB PK Parameters (non-transformed and log-transformed) by Treatment and Dosing Interval in Sub-study | Remove Column "{Additional time variable}". Replace treatment columns with columns for dosing intervals as specified in Section 15.6.5. Add Min and Max after %CVb for log-transformed data. Add %CV after SD for non-transformed data. Add Q1 and Q3 after Median to both types of data. | Sub-study |

| Pharmac | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.6 | Sub-study PK<br>Parameter | PK06 | Summary of Plasma RPV PK Parameters (non-<br>transformed and log-transformed) by Treatment and<br>Dosing Interval in Sub-study | Similar notes to above. | Sub-study |
| 4.7 | Sub-study PK<br>Parameter | Shell PK_T2 | Statistical Analysis of Plasma CAB PK Parameters by Treatment in Sub-study | | Sub-study |
| 4.8 | Sub-study PK<br>Parameter | Shell PK_T2 | Statistical Analysis of Plasma RPV PK Parameters by Treatment in Sub-study | | Sub-study |

# 15.15.7.7. Pharmacokinetic Figures

| Pharmacokinetic Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.1 | Sub-study PK<br>Concentration | 207966/primary_34/F4.1 | Individual Plasma CAB Concentration-Time Plots (Linear and Semi-Log) in Sub-study | Remove the second footnote. | Sub-study |
| 4.2 | Sub-study PK<br>Concentration | 207966/primary_34/F4.2 | Individual Plasma RPV Concentration-Time Plots (Linear and Semi-Log) in Sub-study | Remove the second footnote. | Sub-study |
| 4.3 | Sub-study PK<br>Concentration | 207966/primary_34/F4.5 | Mean (SD) Evaluable Plasma CAB<br>Concentration-Time Plots (Linear and Semi-<br>Log) in Sub-study | Remove the first footnote. | Sub-study |
| 4.4 | Sub-study PK<br>Concentration | 207966/primary_34/F4.6 | Mean (SD) Evaluable Plasma RPV<br>Concentration-Time Plots (Linear and Semi-<br>Log) in Sub-study | Remove the first footnote. | Sub-study |
| 4.5 | Sub-study PK<br>Concentration | 207966/primary_34/F4.11 | Median (5th and 95th Percentile) Evaluable Plasma CAB Concentration-Time Plots (Linear and Semi-Log) in Sub-study | Remove the first footnote. | Sub-study |
| 4.6 | Sub-study PK<br>Concentration | 207966/primary_34/F4.12 | Median (5th and 95th Percentile) Evaluable<br>Plasma RPV Concentration-Time Plots (Linear<br>and Semi-Log) in Sub-study | Remove the first footnote. | Sub-study |
| 4.7 | Sub-study PK<br>Parameter | 205696/final/F3.6 | Geometric Mean Ratios and 90% Cls of<br>Plasma CAB PK Parameters in Sub-study by<br>Treatment and Comparison Type | Use "PK parameter name (n=xx)" for y axis label, add "Geometric Mean Ratio with 90% CI" for x axis label. Remove the footnotes from shell. Add Footnote: Note: The geometric mean ratios and 90% CIs come from the statistical analysis of the PK parameters using a mixed effects model as specified in the analysis plan. | Sub-study |

| Pharmacokinetic Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | | Page by Treatment and Parameter. The parameters include Ctau, Cmax and AUC(0- tau). Each page contains comparison types First Thigh vs. Gluteal and Last Thigh vs. Gluteal. | |
| 4.8 | Sub-study PK<br>Parameter | 205696/final/F3.6 | Geometric Mean Ratios and 90% CIs of RPV PK Parameters in Sub-study by Treatment and Comparison Type | Similar notes to above. | Sub-study |

#### 15.15.7.8. Health Outcomes Tables

| Health C | Health Outcomes Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| HIV Trea | atment Satisfac | tion Questionnaire Status o | or Change Version (HIVTSQs, HIVTSQc) | | |
| 6.1 | Sub-study<br>ITT-E | 207966/primary_34/T6.7 | Proportion of Subjects with HIVTSQs - Individual Item Scores by Visit in Sub-study | | Sub-study |
| 6.2 | Sub-study<br>ITT-E | 207966/primary_34/T6.9 | Summary of HIVTSQs - Total Treatment Satisfaction Score by Visit in Sub-study | Add a column "P Value [1]" to the right of the Column "Max." Add the footnote: [1] Sub-study Week 16, Sub-study Week 24 (for Q8W arm) or 20 (for Q4W arm) are compared with the Substudy Baseline using Wilcoxon signed-rank test." | Sub-study |
| 6.3 | Sub-study<br>ITT-E | 207966/primary_34/T6.11 | Summary of HIVTSQs - Change in Total Treatment Satisfaction Score in Sub-study | Remove the column 'Prior Exposure to CAB+RPV (weeks)'. Replace "Act. Rel. Time" With "Change", the new "Change" column includes "Change from Baseline to Week 16" for both arms, "Change from Baseline to Week 20" for Q4W and "Change from Baseline to Week 24" for Q8W, "Change from Week 16 to Week 20" for Q4W arm and "Change from Week 16 to Week 20" for Q8W. Remove the footnote. | Sub-study |
| 6.4 | Sub-study<br>ITT-E | 207966/primary_34/T6.13 | Summary of HIVTSQs - Change in Individual Item Score in Sub-study | Similar notes to above. | Sub-study |

| Health C | Health Outcomes Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 6.5 | Sub-study<br>ITT-E | 207966/primary_02/T6.23 | Proportion of Subjects with HIVTSQc - Individual Item Change Score at Sub-study Week 16 (Thigh Injection Phase) | | Sub-study |
| 6.6 | Sub-study<br>ITT-E | 207966/primary_02/T6.27 | Summary of HIVTSQc - Individual Item Change<br>Score at Sub-study Week 16 (Thigh Injection<br>Phase) | | Sub-study |
| 6.7 | Sub-study<br>ITT-E | 207966/primary_02/T6.25 | Summary of HIVTSQc - Total Treatment Satisfaction Change Score at Sub-study Week 16 (Thigh Injection Phase) | | Sub-study |
| Tolerabi | ility of Injection | (NRS) | | | |
| 6.8 | Sub-study<br>ITT-E | Shell HO_T3 | Proportion of Subjects with Each Tolerability of Injection (NRS) Score by Visit in Sub-study | | Sub-study |
| 6.9 | Sub-study<br>ITT-E | 201584/primary_01/T6.35 | Summary of Tolerability of Injection (NRS) Score by Visit in Sub-study | | Sub-study |

| Health C | Health Outcomes Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 6.10 | Sub-study<br>ITT-E | 201584/primary_01/T6.37 | Summary of Change in Tolerability of Injection (NRS) Score in Sub-study | Replace "Actual Relative Time" with "Change". In this column, for Q4W: "Change from Week -4 to Day 1", "Change from Week -3 to Week 1", "Change from Day 1 to Week 12", "Change from Week 1 to Week 13", Change from Week 12 to Week 16", "Change from Week 13 to Week 17", for Q8W: "Change from Week -8 to Day 1", "Change from Week -7 to Week 1", "Change from Day 1 to Week 8", "Change from Week 1 to Week 9", "Change from Week 8 to Week 16", "Change from Week 9 to Week 17". | Sub-study |
| Preferer | псе | | | | |
| 6.11 | Sub-study<br>ITT-E | Shell HO_T4 | Proportion of Subjects with Response to Each Individual Question in Preference Thigh Injection vs Gluteal Injection Questionnaire by Visit in Substudy | | Sub-study |

### 15.15.7.9. Virology Tables

Tables 7.1-7.6 will only be produced when at least one treatment group has >5 subjects in Sub-study CVF population. Tables 7.8-7.9 will only be produced when data are available.

| Virology | Virology Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Genoty | ре | | | | |
| 7.1 | Sub-study<br>CVF | 207966/primary_34/T7.1 | Summary of the Prevalence of Known INI Resistance<br>Mutations at time of CVF (Thigh Injection + Return to<br>Gluteal Injection Phase) – Plasma Sample | | Sub-study |
| 7.2 | Sub-study<br>CVF | 207966/primary_34/T7.2 | Summary of the Prevalence of Major Resistance<br>Mutations of NRTI, NNRTI and PI Class at time of CVF<br>(Thigh Injection + Return to Gluteal Injection Phase) -<br>Plasma Sample | | Sub-study |
| 7.3 | Sub-study<br>CVF | 207966/primary_34/T7.3 | Summary of Genotypic Susceptibility at time of CVF (Thigh Injection + Return to Gluteal Injection Phase) - Plasma Sample | | Sub-study |
| Phenoty | /pe | | | | |
| 7.4 | Sub-study<br>CVF | 207966/primary_34/T7.4 | Summary of Phenotype Susceptibility at time of CVF (Thigh Injection + Return to Gluteal Injection Phase) - Plasma Sample | | Sub-study |
| 7.5 | Sub-study<br>CVF | 207966/primary_34/T7.5 | Summary of Phenotype: Number of Drugs to Which<br>Subject is Phenotypic Resistant or Partial Sensitive or<br>Sensitive at Time of CVF (Thigh Injection + Return to<br>Gluteal Injection Phase) - Plasma Sample | | Sub-study |
| 7.6 | Sub-study<br>CVF | 207966/primary_34/T7.6 | Summary of Fold Change to CAB and RPV at Time of CVF (Thigh Injection + Return to Gluteal Injection Phase) - Plasma Sample | | Sub-study |

| Virology | Virology Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 7.7 | Sub-study<br>CVF | 207966/primary_34/T7.7 | Summary of Net Assessment at time of CVF (Thigh Injection + Return to Gluteal Injection Phase) - Plasma Sample | | Sub-study |
| Other | Other | | | | |
| 7.8 | Sub-study<br>CVF | 207966/primary_34/T7.8 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria during the Thigh Injection or Return to Gluteal Injection Phase | | Sub-study |
| 7.9 | Sub-study<br>Safety | 207966/primary_34/T7.9 | Summary of Viral load, Genotypic and Phenotypic data for Non-CVF Subjects with Genotypic and/or Phenotypic Data in Sub-study | | Sub-study |

# 15.15.7.10. ICH Listings

| ICH Lis | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Study F | opulation | | | | |
| 1 | Sub-study<br>Screened | 207966/primary_15/L3 | Listing of Reasons for Screen Failure in Sub-study | | Sub-study |
| 2 | Sub-study ITT-E | 207966/primary_34/L1 | Listing of Reasons for Sub-study<br>Withdrawal | | Sub-study |
| 3 | Sub-study ITT-E | 207966/primary_34/L2 | Listing of Reasons for Study Drug<br>Discontinuation | | Sub-study |
| 4 | Sub-study ITT-E | 207966/primary_34/L3 | Listing of Important Protocol Deviations | | Sub-study |
| 5 | Sub-study ITT-E | 207966/primary_34/L7 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | Sub-study |
| 6 | Sub-study ITT-E | 207966/primary_34/L5 | Listing of Demographic<br>Characteristics | Add "BMI (kg/m^2)" to the right of "Weight (kg)". Add the following sentence to footnote [1]: Age is calculated with respect to the subject's first sub-study screening visit. Add a footnote for BMI and Weight: [2] BMI and Weight are derived at Sub-study Baseline. | Sub-study |
| Efficacy | | | | | |
| 7 | Sub-study ITT-E | 207966/primary_34/L8 | Listing of Study Outcome (50 c/mL<br>Threshold) at Sub-study Week 16 –<br>Snapshot Analysis | Remove the footnote. | Sub-study |
| Safety | | | | | |
| 8 | Sub-study | 207966/primary_34/L9 | Listing of Investigational Product | | Sub-study |

| ICH List | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | Safety | | Exposure Data | | |
| 9 | Sub-study<br>Safety | 207966/primary_34/L10 | Listing of Subject Numbers for<br>Individual Adverse Events | | Sub-study |
| 10 | Sub-study<br>Safety | 207966/primary_34/L11 | Listing of Reasons for Considering as a Serious Adverse Event | | Sub-study |
| 11 | Sub-study<br>Safety | 207966/primary_34/L12 | Listing of Fatal Adverse Events | | Sub-study |
| 12 | Sub-study<br>Safety | 207966/primary_34/L13 | Listing of Non-Fatal Serious Adverse Events | | Sub-study |
| 13 | Sub-study<br>Safety | 207966/primary_34/L14 | Listing of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product or Withdrawal from Study | | Sub-study |
| 14 | Sub-study<br>Safety | 207966/primary_34/L15 | Listing of Changes in<br>Intensity/Grades of Study Drug<br>Injection Site Adverse Events | | Sub-study |
| 15 | Sub-study<br>Safety | 207966/primary_34/L16 | Listing of All Adverse Events | | Sub-study |
| 16 | Sub-study<br>Safety | 207966/primary_34/L17 | Listing of COVID-19 Adverse Events | | Sub-study |
| 17 | Sub-study<br>Safety | 207966/primary_34/L18 | Listing of COVID-19 Assessments | | Sub-study |
| 18 | Sub-study<br>Safety | 207966/primary_34/L19 | Listing of COVID-19 Symptoms | | Sub-study |
| 19 | Sub-study<br>Safety | 207966/primary_34/L20 | Listing of Subjects Who Became Pregnant during the Study | Add a footnote: "Note: As pregnancy status is not collected in eCRF for the long-term follow- | Sub-study |

| ICH List | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | | up phase, this listing does not include subjects who became pregnant during the long-term follow-up phase." | |
| 20 | Sub-study<br>Safety | 207966/primary_34/L23 | Listing of ECG Values for Subjects with a Value of Potential Clinical Importance in Sub-study | In footnote, add "sub-study" before the "baseline". Add following to the footnote, "The changes from baseline provided in this listing are with respect to the sub-study baseline." | Sub-study |
| PK | РК | | | | |
| 21 | Sub-study PK<br>Concentration | 207966/primary_34/L25 | Listing of Plasma CAB PK<br>Concentration-Time Data | Remove the Column "Excluded" and remove the first footnote. Present nominal visit before the analysis visit. Replace "Race Detail" with "Sub-study Baseline BMI (kg/m^2)" in the second column on the left. | Sub-study |
| 22 | Sub-study PK<br>Concentration | 207966/primary_34/L26 | Listing of Plasma RPV PK<br>Concentration-Time Data | Similar notes to above. | Sub-study |

# 15.15.7.11. Non-ICH Listings

| Non-ICI | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Study F | Population | | | | |
| 23 | Sub-study ITT-E | 207966/primary_3<br>4/L27 | Listing of Reasons for Thigh Injection Phase Withdrawal | | Sub-study |
| 24 | Sub-study ITT-E | 207966/primary_3<br>4/L27 | Listing of Reasons for Return to Gluteal Injection Phase Withdrawal | | Sub-study |
| 25 | Sub-study LTFU | 207966/primary_3<br>4/L28 | Listing of Reasons for Long-term Follow-up Phase Withdrawal | | Sub-study |
| 26 | Sub-study ITT-E | Shell POP_L2 | Listing of Exposure to Study Treatment including SOC Oral Bridging Prior to the First Thigh Injection | | Sub-study |
| 27 | Sub-study ITT-E | 207966/primary_3<br>4/L30 | Listing of Concomitant ART Medications | | Sub-study |
| 28 | Sub-study ITT-E | 207966/primary_3<br>4/L31 | Listing of ART Medications Received during Long-<br>term Follow-up Phase | | Sub-study |
| 29 | Sub-study ITT-E | 207966/primary_3<br>4/L34 | Country Level Listing of Dates of Waves of COVID-<br>19 Pandemic Measures for Countries Participating<br>in Sub-study | | Sub-study |
| 30 | Sub-study ITT-E | 209493/final_02/L<br>52 | Listing of Transition to CAB + RPV LA Marketed Product Status | Replace "Subject Id." with "Latest Subject Id." in the column header. | Sub-study |
| Efficacy | у | | | | |
| 31 | Sub-study CVF | 207966/primary_3<br>4/L35 | Listing of All Plasma HIV-1 RNA Data for Subjects with Confirmed Virologic Failure | Produce only when data are available. | Sub-study |
| 32 | Sub-study ITT-E | 207966/primary_3<br>4/L36 | Listing of All Plasma HIV-1 RNA Data for Subjects with Viral load >=50 c/mL during the Thigh Injection or Return to Gluteal Injection Phase | | Sub-study |

| Non-ICH | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 33 | Sub-study ITT-E | 207966/primary_3<br>4/L37 | Listing of All Plasma HIV-1 RNA Data | | Sub-study |
| 34 | Sub-study ITT-E | 207966/primary_3<br>4/L38 | Listing of HIV-1 Associated Conditions | Produce only when data are available. | Sub-study |
| Safety | | | | | |
| 35 | Sub-study<br>Safety | 207966/primary_3<br>4/L43 | Listing of Subjects Meeting Hepatobiliary Lab<br>Criteria (Thigh Injection + Return to Gluteal<br>Injection Phase) | Present by phase. | Sub-study |
| 36 | Sub-study<br>Safety | 207966/primary_3<br>4/L45 | Listing of ECG values for Subjects with Potential QTc Interval Prolonging Events of Interest in Substudy | | Sub-study |
| 37 | Sub-study<br>Safety | 207966/primary_3<br>4/L47 | Listing of Dosing Errors and IP Device Malfunctions in Substudy | | Sub-study |
| PK | | | | | |
| 38 | Sub-study PK<br>Parameter | Shell PK_L1 | Listing of Plasma PK Parameters in Sub-study | | Sub-study |

# 15.16. Appendix 16: Example Mock Shells for Data Displays

Available upon request

# Signature Page for $\,207966\ TMF\text{-}15024301\ v1.0$

| Reason for signing: Approved | Name: PPD<br>Role: A<br>Date of signature: 23-Sep-2022 14:42:03 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: PPD<br>Role: A<br>Date of signature: 23-Sep-2022 14:48:11 GMT+0000 |

Signature Page for TMF-15024301 v1.0